Official Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo- and Active-controlled

Trial of Brexpiprazole (1 - 3 mg/day) as Monotherapy or as Combination Therapy in

the Treatment of Adults with Post-traumatic Stress Disorder

NCT Number: NCT03033069

**Document Date:** SAP Version Final: 07 November 2018

# Documentation of Statistical Methods Table of Contents

| Table of Conte | nts | 1 |
|---|---|---|
| Statistical Ana | lysis Plan; Final: 07 Nov 2018 | 4 |
| STAT-1.1 | Adjusted Mean Change in | |
| | CAPS-5 Line Items - MMRM (Intent to Treat | |
| | Sample) | 56 |
| STAT-1.2 | Adjusted Mean Change from Baeline (Day 0) in SOTS Line | |
| | Items at Week 12 - MMRM (Intent to Treat Sample) | 69 |
| STAT-1.3 | Adjusted Mean Change in | |
| | PCL-5 Line Items - MMRM (Intent to Treat | |
| | Sample) | 74 |
| STAT-1.4 | Adjusted Mean Change in | |
| | HADS Line Items - MMRM (Intent to Treat | |
| | Sample) | 83 |
| STAT-3.1 | MMRM Output for Test on Treatment by Gender Interaction | |
| | (Intent to Treat Sample) | 89 |
| STAT-3.2 | MMRM Output for Test on Treatment by Race Interaction | |
| | (Intent to Treat Sample) | 128 |
| STAT-3.3 | MMRM Output for Test on Treatment by Age | |
| 21111 0.0 | (< 55 vs >= 55) Interaction (Intent to Treat | |
| | Sample) | 167 |
| STAT-3.4.1 | MMRM Output for Test on Treatment by | 10, |
| 51711 5.1.1 | 20 Percent Improvement Subgroup Interaction | |
| | (Intent to Treat Sample) | 206 |
| STAT-3.4.2 | MMRM Output for Test on Treatment by | 200 |
| 51711 5.4.2 | 25 Percent Improvement Subgroup Interaction | |
| | (Intent to Treat Sample) | 248 |
| STAT-3.4.3 | MMRM Output for Test on Treatment by | 240 |
| SIAI-3.4.3 | 30 Percent Improvement Subgroup Interaction | |
| | (Intent to Treat Sample) | 290 |
| STAT-3.5 | MMRM Output for Test on Treatment by Type of Trauma | 290 |
| S1A1-3.3 | Interaction (Intent to Treat Sample) | 329 |
| STAT-3.6 | MMRM Output for Test on Treatment by Psychosocial | 329 |
| 31A1-3.0 | | |
| | Support at Baseline Interaction (Intent to Treat Sample) | 366 |
| STAT-3.7 | MMRM Output for Test on Treatment by Previous | 300 |
| 31A1-3./ | • | |
| | Pharmacological Treatment Intervention for PTSD | 405 |
| CTAT 2 0 | Interaction (Intent to Treat Sample) | 403 |
| STAT-3.8 | MMRM Output for Test on Treatment by Use of Wearable | 111 |
| CTAT 2 O | Device Interaction (Intent to Treat Sample) | 444 |
| STAT-3.9 | MMRM Output for Test on Treatment by Years Since Index | |
| | Traumatic Event Interaction (Intent to Treat | 403 |
| | Sample) | 483 |

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.

| STAT-3.10 | MMRM Output for Test on Treatment by Age | |
|---|---|---|
| | (< 30 vs 30-40 vs >= 40) Interaction (Intent to | |
| | Treat Sample) | 531 |
| STAT-4.1.1 | Proc Mixed Output for Change | |
| | in CAPS-5 Total Score, MMRM (UN), | |
| | DDFM = KENWARDROGER (Intent to Treat Sample) | 579 |
| STAT-4.1.2 | Proc Mixed Output for Change | |
| | in CAPS-5 Total Score, MMRM (UN), | |
| | DDFM = SATTERTHWAITE (Intent to Treat Sample) | 593 |
| STAT-4.2 | Proc GLM Output for Change | |
| | in CAPS-5 Total Score, LOCF (Intent | |
| | | 605 |
| STAT-4.3 | to Treat Sample) | 000 |
| 511115 | in CAPS-5 Total Score, OC (Intent to | |
| | Treat Sample) | 611 |
| STAT-4.4 | Proc GLM Output for Treatment by Center Interaction | 011 |
| 51711 4.4 | in CAPS-5 Total Score, LOCF (Intent to Treat | |
| | | 617 |
| STAT-4.5.1 | Sample) Summary of Mean Change | 017 |
| S1A1-4.5.1 | in CAPS-5 Total Score By Center - LOCF (Intent | |
| | | 619 |
| CTAT 452 | to Treat Sample) | 019 |
| STAT-4.5.2 | | |
| | Score Among Treatment Groups By | 622 |
| CTAT 4.6 | Center - LOCF (Intent to Treat Sample) | 622 |
| STAT-4.6 | Unadjusted Mean Change to | |
| | Phase B by Study Week CAPS-5 Total Score, LOCF (Intent | (00 |
| CTAT AT | to Treat Sample) | 623 |
| STAT-4.7 | Unadjusted Mean Change to | |
| | Phase B by Study Week CAPS-5 Total Score, OC (Intent to | 6.60 |
| GT 4 T 4 G | Treat Sample) | 663 |
| STAT-4.8 | Non-Parametric Stratified by Center and Type of Trauma | |
| | Analysis of Mean Change to | |
| | Phase B by Study Week in CAPS-5 Total (Intent to Treat | |
| | Sample) | 703 |
| STAT-4.9 | Residual from Proc Mixed for Change from | |
| | Baseline in CAPS-5 Total Score, Primary Efficacy Analysis | |
| | Model (Intent to Treat Sample) | 707 |
| STAT-4.10 | Proc Mixed Output Using Heterogeneous Variance Structure | |
| | for Treatment Groups (Intent to Treat Sample) | 716 |
| STAT-5.1 | Proc Mixed Output for Change | |
| | in CGI-S Scale, MMRM (UN) (Intent to Treat | |
| | Sample) | 736 |
| STAT-5.2 | Proc GLM Output for Change | |
| | in CGI-S Scale, LOCF (Intent to Treat | |
| | Sample) | 750 |

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.

| STAT-5.3 | Proc GLM Output for Change | |
|------------|---------------------------------------------------------|-----|
| | in CGI-S Scale, OC (Intent to Treat Sample) | 756 |
| STAT-6.1.1 | Shapiro-Wilk Test for Residual by Week from Proc Mixed | |
| | for in CAPS-5 Total | |
| | Score, Primary Efficacy Analysis Mode (Intent to Treat | |
| | Sample) | 762 |
| STAT-6.1.2 | Residual by Week from Proc Mixed for Change | |
| | in CAPS-5 Total Score, Primary Efficacy | |
| | Analysis Model (Intent to Treat Sample) | 763 |
| STAT1-1.1 | Adjusted Mean Change in | |
| | CAPS-5 Line Items - MMRM (Modified Intent | |
| | to Treat Sample) | 795 |
| STAT1-1.2 | Adjusted Mean Change from Baseline (Day 0) in SOTS Line | |
| | Items at Week 12 - MMRM (Modified Intent to Treat | |
| | Sample) | 808 |
| STAT1-1.3 | Adjusted Mean Change in | |
| | PCL-5 Line Items - MMRM (Modified Intent to | |
| | Treat Sample) | 813 |
| STAT1-1.4 | Adjusted Mean Change in | |
| | HADS Line Items - MMRM (Modified Intent to | |
| | Treat Sample) | 822 |

# Otsuka Pharmaceutical Development & Commercialization, Inc.

Investigational New Drug

Brexpiprazole (OPC-34712)

A Phase 2, Multicenter, Randomized, Double-blind, Placebo- and Active-controlled Trial of Brexpiprazole (1 - 3 mg/day) as Monotherapy or as Combination Therapy in the Treatment of Adults with Post-traumatic Stress Disorder

Protocol No. 331-201-00061 IND No. 117,549

# Statistical Analysis Plan

Version: Final

Date: November 07, 2018


Confidential
May not be used, divulged, published or otherwise disclosed
without the consent of Otsuka Pharmaceutical Development & Commercialization, Inc.


1

# **Table of Contents**

| Tabl | le of Contents | <u>2</u> |
|---|---|---|
| 1 | Introduction5 | |
| 2 | Study Objectives5 | |
| 3 | Trial Details | 5 |
| 3.1 | Study Design | 5 |
| 3.2 | Trial Treatments | 7 |
| 3.2.1 | Trial Treatment Administration | 8 |
| 3.2.2 | Brexpiprazole Administration | 8 |
| 3.2.3 | Combination of Brexpiprazole plus Zoloft (Sertraline) | 8 |
| 3.2.4 | Zoloft (Sertraline) Administration | 9 |
| 3.2.5 | Placebo Administration | 10 |
| 4 | Sample Size and Power Justification | 10 |
| 5 | Data Sets for Analysis and Missing Data | 11 |
| 5.1 | Data Sets for Analysis | 11 |
| 5.2 | Handling of Missing Data | 11 |
| 6 | Study Conduct | 13 |
| 6.1 | Subject Disposition, Completion Rate and Reasons for Discontinua | ation 13 |
| 6.2 | Treatment Compliance | |
| 6.3 | Protocol Deviation | |
| 7 | Baseline Characteristics | 13 |
| 7.1 | Baseline Definition | 13 |
| 7.2 | Demographic Characteristics | 14 |
| 7.3 | Medical and Psychiatric History and Treatment for PTSD | |
| 7.4 | Neuropsychiatric Diagnosis | |
| 7.5 | Baseline PTSD Evaluation | 14 |
| 8 | Efficacy Analysis | 15 |
| 8.1 | Primary Efficacy Endpoint | 15 |
| 8.1.1 | Primary Efficacy Analysis | 15 |
| 8.1.2 | Technical Computation Details for Primary Efficacy Analysis | 17 |
| Confid | dential - Proprietary Information 2 | 07 November 2018 |

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.

| 8.1.3 | Sensitivity Analyses | 17 |
|---|---|---|
| 8.1.3.1 | Sensitivity Analyses for Missing at Random (MAR) Assur | nption 17 |
| 8.1.3.2 | Sensitivity Analyses for Violation of Normality Assumption | on 19 |
| 8.1.4 | Subgroup Analyses | 19 |
| 8.2 | Other Efficacy Endpoints | 20 |
| 8.3 | Analyses for Sleep-related Endpoints | 21 |
| 8.4 | Exploratory Analysis | 23 |
| | | 24 |
| 9 S | afety Analysis | 24 |
| 9.1 | Adverse Events | 24 |
| 9.2 | Clinical Laboratory Tests | 25 |
| 9.2.1 | Clinical Laboratory Tests in Phase B | 26 |
| 9.2.2 | Drug Induced Liver Injury (DILI) | 26 |
| 9.2.3 | Metabolic Change | 26 |
| 9.3 | Vital Signs | 27 |
| 9.4 | 12-Lead ECG | 27 |
| 9.5 | Physical Examinations | 28 |
| 9.5.1 | Body Weight, Waist Circumference and BMI | 29 |
| 9.6 | SAS, AIMS, and BARS | 29 |
| 9.7 | Suicidality Data | 29 |
| 9.8 | Concomitant Medications | 30 |
| 9.9 | Extent of Exposure | 30 |
| 10 C | onventions | 31 |
| 10.1 | Study Visit Windows | 31 |
| 10.2 | Pooling of small centers | 32 |
| 10.3 | Scales: Rules for Scoring and Handling of Missing Data | 32 |
| 10.3.1 | CAPS-5 | 32 |
| 10.3.2 | SOTS | 33 |
| 10.3.3 | CGI-S | 33 |
| 10.3.4 | PCL-5 | 33 |
| 10.3.5 | HADS | 34 |
| Confident | ial - Proprietary Information 3 | 07 November 20 |

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.

| 13 | Proposed List of Summary Tables | 40 |
|--------|-----------------------------------------------------|----|
| 12 | Potential Clinical Relevance Criteria from Protocol | 37 |
| 11 | References | 36 |
| 10.3.9 | C-SSRS | 35 |
| 10.3.8 | BARS | 35 |
| 10.3.7 | 7 AIMS | 34 |
| 10.3.6 | SAS | 34 |

## 1 Introduction

This statistical analysis plan (SAP) documents the statistical methodology and data analysis algorithms and conventions to be applied for statistical analysis and reporting of efficacy and safety data of study 331-201-00061. All amendments to the protocol and Addendum to protocol amendment are taken into consideration in developing this SAP.

# 2 Study Objectives

Primary: To evaluate the efficacy of brexpiprazole as monotherapy or as combination treatment therapy with Zoloft (sertraline) in adult subjects with post-traumatic stress disorder (PTSD).

Secondary: To evaluate the safety and tolerability of brexpiprazole 1 to 3 mg/day as monotherapy or as combination treatment with Zoloft (sertraline) in adult subjects with PTSD.

#### 3 Trial Details

# 3.1 Study Design

This is a phase 2, randomized, double-blind, placebo- and active-controlled, 4-arm trial to evaluate the efficacy, safety and tolerability of brexpiprazole (1 - 3 mg/day) as monotherapy or as combination therapy with Zoloft (sertraline) in adult subjects with PTSD. See Figure 3.1-1 for a schematic of the trial design.



Figure 3.1-1 Unblinded Trial Design Schematic


6

The trial will be organized as follows:

Screening Phase: The screening period will be 14 days and will begin when informed consent is signed. An extension can be requested from the medical monitor, if needed to meet eligibility requirements. The purpose of the screening period is to assess eligibility criteria at 1 or more visits (as necessary to complete screening assessments) and to washout prohibited concomitant pharmacotherapy, if applicable. An interactive response technology (IRT) or equivalent will be used to obtain an identification (ID) number for each subject with documented consent. Subjects will be between 18 and 65 years of age, inclusive, at the time of screening and will have a diagnosis of PTSD as defined by Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria.

All subjects must agree to discontinue all prohibited medications during the screening period in order to meet the protocol-specified washout periods.

Blinded Phase B (Treatment Phase): At Week 1, subjects will be randomly assigned in a 1:1:1:1 ratio to one of one of the following double-blind treatment regimens:

- brexpiprazole monotherapy
- brexpiprazole and Zoloft (sertraline) combination therapy
- Zoloft (sertraline) monotherapy
- placebo

Subjects will attend visits at Baseline (Day 0) and Weeks 1, 2, 3, 4, 6, 8, 10, and 12 during the treatment phase.

Follow-up: If any subject discontinues the trial early, every effort should be made to complete the Week 12/early termination (ET) evaluations as soon as possible and whenever possible prior to starting any new medication or treatment. All subjects (completers and early withdrawals) will be contacted to monitor for safety events via telephone or clinic visit for 14 (+2) days after the last dose of investigational medicinal product (IMP). Any subject who withdraws because of a serious adverse event (SAE) should be seen in the clinic, if possible.

#### 3.2 Trial Treatments

During Phase B, all subjects receive daily: one tablet (active or placebo-matched brexpiprazole) and two Zoloft (sertraline) capsules (active or placebo-matched).


7

#### 3.2.1 Trial Treatment Administration

During Phase B (treatment phase), subjects will receive IMP, consisting of brexpiprazole monotherapy, brexpiprazole + Zoloft (sertraline), Zoloft (sertraline) monotherapy, or placebo, depending on the subject's treatment assignment.

All doses of IMP should be taken together at the same time each day, if possible. All doses of IMP can be taken without regard to meals. If tolerability issues arise, the timing of administration of the IMP may be adjusted at the investigator's discretion in order to achieve optimum tolerability and compliance.

## 3.2.2 Brexpiprazole Administration




8








#### 3.2.5 Placebo Administration

As shown in Table 3.2.5-1, subjects assigned to placebo for both treatments (sertraline and brexpiprazole).



# 4 Sample Size and Power Justification

The primary efficacy endpoint is defined as change from baseline (Week 1 visit) in the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) total score.

Sixty-eight subjects per arm will provide at least 80% power at a 2-sided alpha level of 0.05 to detect the treatment difference of -6.5 points in primary efficacy endpoint for active arm vs placebo with a standard deviation (SD) of 13. Adjusting for 10% non-evaluable subjects, the total number of subjects to be randomized is 75 per treatment arm.


10

Further adjusting for 10% dropout between Baseline (Day 0) Visit and randomization, approximately 332 subjects are expected to be enrolled in the trial.

# 5 Data Sets for Analysis and Missing Data

## 5.1 Data Sets for Analysis

The following analysis samples are defined for this trial:

Enrolled Sample: comprises all subjects enrolled

Randomized Sample: comprises all subjects randomized into this trial

**Safety Sample**: comprises all subjects in the Randomized Sample who were administered at least one dose of double-blind IMP

**Intent to Treat (ITT) Sample**: comprises of all subjects in the Randomized Sample who took at least one dose of double-blind IMP and have a baseline and at least one post baseline evaluation for the CAPS-5 total score

To evaluate the efficacy of the study drug on the placebo non-responders, the following analysis sample is added.

The modified ITT Sample (mITT): comprises those subjects in the ITT Sample who meet the following two criteria:

- 1) CAPS-5 total score is at least 27 at the randomization visit (Week 1).
- 2) Improvement (in terms of reduction in CAPS-5 total score) in CAPS-5 total score is less than 30% at end of the placebo run-in phase (from Baseline (Day 0) to randomization visit (Week 1)).

In general, baseline of an efficacy endpoint is defined as the last available measurement before the first dose of double-blind IMP.

#### 5.2 Handling of Missing Data

The CAPS-5 is a clinician-rated, structured interview designed to assess PTSD diagnostic status and symptoms severity as defined by the DSM-5. This trial will use the CAPS-5 Past Month and CAPS-5 Past Week versions of the scale. The CAPS-5 comprises questions that target the onset and duration of symptoms, subjective distress, impact of symptoms on social and occupational functioning, improvement in symptoms since a previous CAPS-5 administration, overall response validity, overall PTSD severity, and specifications for the dissociative subtype (depersonalization and derealization).


11

The CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms (items 1-20) from the following categories:

Category B: Intrusion symptoms (5 items);

Category C: Avoidance symptoms (2 items);

Category D: Cognition and mood symptoms (7 items); and

Category E: Arousal and reactivity symptoms (6 items)

If there are more than 1 item in each of categories B, D and E with a missing score, or any item in Category C with a missing score, the CAPS-5 total score is set to missing. For each category (B, D or E) with a missing score, the imputed subscores for that category is the average of the existing scores in the category multiplied by the total number of questions in the category. The CAPS-5 total score will then be imputed by adding all the subscores from categories B, C, D and E.

In general, missing data will be handled by analysis of mixed-effect model repeated measures (MMRM) methodology based on observed-case (OC) data from protocol-specified visits under the assumption of missing at random.

MMRM assumes data are missing at random (MAR), which is a reasonable assumption in longitudinal clinical trials in PTSD<sup>1</sup>. However, the possibility of "missing not at random" (MNAR) data can never be ruled out. As sensitivity analyses, selection model<sup>2</sup>, pattern-mixture model<sup>3,4,5,6</sup>, and/or shared parameter model<sup>7</sup> will be used to explore data missing mechanisms of MNAR and investigate the response profile of dropout reason. Details are provided in Section 8.1.3 Sensitivity Analysis.

The Observed Cases (OC) data set will consist of actual observations recorded at each visit during Phase B and no missing data will be imputed. MMRM, Wu-Bailey, and pattern-mixture model will be performed on the OC dataset.

The Last Observation Carried Forward (LOCF) data set will include data recorded at a scheduled Phase B visit or, if no observation is recorded at that visit, data carried forward from the previous scheduled Phase B visit. Baseline (Week 1 visit) data will not be carried forward to impute missing values for the LOCF data set. The analysis of covariance (ANCOVA) analysis will be performed for the change from baseline in blinded phase B (LOCF) in CAPS-5 total score as sensitivity analysis. The ANCOVA\_LOCF model includes treatment and study center as main effects, and baseline value as a covariate.

For categorical response/remission variables, OC analyses will be performed in addition to LOCF analyses. Study center will not be included in the models for OC analyses.

# 6 Study Conduct

## 6.1 Subject Disposition, Completion Rate and Reasons for Discontinuation

Subject disposition will be summarized for the Randomized Sample by treatment group, and by center.

Subject completion rate and reasons for discontinuation will be summarized for the Randomized Sample by treatment group. Subject completion rate for Phase B will also be summarized by treatment group and week for the Randomized Sample.

## 6.2 Treatment Compliance

Based on the Investigational medicinal product (IMP) panel of the CRF, compliance in taking IMP is calculated by dividing the number of tablets/capsules taken by the total number of tablets/capsules the patients were scheduled to take during the study period. Compliance is calculated on double-blind IMP for Phase B. For lost-to-follow up patients, last IMP end date record will be used as the treatment end date.

#### 6.3 Protocol Deviation

7.1

Protocol deviations will be summarized by center and type of deviation for randomized subjects by treatment group. A listing of protocol deviations will be provided.

#### 7 Baseline Characteristics

**Baseline Definition** 

# 7.2 Demographic Characteristics

Baseline demographic characteristics include age, sex, race, ethnicity, height, weight, waist circumference, and body mass index (BMI). For the Randomized Sample, demographic characteristics will be summarized by treatment group.

Mean, range and standard deviation will be used to describe continuous variables such as age. Frequency distributions will be tabulated for categorical variables such as race.

#### 7.3 Medical and Psychiatric History and Treatment for PTSD

A summary of medical and psychiatric history will be presented for the Randomized Sample (by treatment group and overall). Summarized data will include the number of years since index traumatic event that led to development of PTSD and the number of years since onset of first symptoms leading to the diagnosis of PTSD based on data collected in CRF page "Medical - Psychiatric History and Concomitant Medications Review". A summary of PTSD treatment based on the Emory Treatment Resistance Interview (E-TRIP) will also be presented for the Randomized Sample (by treatment group and overall). Psychiatric medication taken prior to the start of IMP will be listed.

## 7.4 Neuropsychiatric Diagnosis

A summary of the MINI International Neuropsychiatric Interview (M.I.N.I.) will be presented for the Randomized Sample (by treatment group and overall). Summarized will be the number and percentage of patients who meet each diagnosis criteria, and number and percentage of patients with each primary diagnosis.

A summary of the Life Events Checklist (LEC-5) extended version will also be presented for the Randomized Sample (by treatment group and overall). Summarized will be the number and percentage of patients with each response to each question in Part 1.

In addition, a summary of the Ohio State University Traumatic Brain Injury Identification (OSU TBI-ID) method will be presented for the Randomized Sample (by treatment group and overall). Summarized will be the number and percentage of patients' answers (yes/no) to each question in Part 1 and the first question in Part 3.

#### 7.5 Baseline PTSD Evaluation

For the Randomized Sample, baseline PTSD scale evaluation will be summarized by treatment group and overall. The mean, median, range and standard deviation will be used to


14

summarize the assessments of: CAPS-5 total score, Symptoms of Trauma Scale (SOTS) total score, Clinical Global Impression – Severity (CGI-S) Score, PTSD Checklist for DSM-5 (PCL-5) total score, and Hospital Anxiety and Depression Scale (HADS) subscale scores (depression and anxiety).

# 8 Efficacy Analysis

All efficacy analyses will be performed on the Intent to Treat Sample, and patients will be included in the treatment group as randomized. All efficacy analyses will also be performed on the mITT Sample unless specified otherwise. The sensitivity analyses and analyses for sleep-related endpoints will not be performed on the mITT Sample.

For analysis of Phase B data, the baseline measurement, which is defined in Section 7.1, is considered as "baseline" for Phase B. Statistical comparisons are based on 2-sided, .05 significance levels.

## 8.1 Primary Efficacy Endpoint

The primary efficacy endpoint is the change from baseline in the CAPS- 5 total score.

# 8.1.1 Primary Efficacy Analysis

The objective of the primary analysis is to evaluate the efficacy of brexpiprazole as monotherapy or as combination treatment with Zoloft (sertraline) in adult subjects with PTSD.

The estimand for the primary efficacy analysis is the difference in outcome improvement if all subjects tolerated and adhered to their treatment. This approach is Estimand #3 recommended by the 2010 National Academy of Sciences' National Research Council report on prevention and treatment of missing data and ICH E9 (R1) "Addendum to Statistical Principles for Clinical Trials on Choosing Appropriate Estimands and Defining Sensitivity Analyses in Clinical Trials".

This estimand focuses on the efficacy of brexpiprazole as monotherapy or as combination treatment with Zoloft (sertraline) in change from the baseline in CAPS-5 total score. The objective of this trial is consistent with the election of an efficacy rather than effectiveness estimand.

The primary analysis will be performed on the Intent to Treat Sample. Change from baseline in CAPS-5 total score will be analyzed using a Mixed Model Repeated Measures (MMRM) analysis with an unstructured (UN) variance covariance structure. The model will include fixed class-effect terms for treatment, trial site, type of trauma (combat related Yes/No), visit week, and an interaction term of treatment by visit week and include the interaction term of baseline values of CAPS-5 total score by visit week as a covariate. All scheduled visits during double-blind treatment will be included in the model but primary comparison will be performed.

In case there is a convergence problem with MMRM model with the UN variance covariance matrix, the following structures other than unstructured will be used in order of 1) heterogeneous toeplitz (TOEPH), 2) heterogeneous autoregressive of order 1 (ARH1), and 3) heterogeneous compound symmetry (CSH) and the first (co)variance structure converging to the best fit will be used as the primary analysis. If a structured covariance has to be used, the empirical "sandwich" estimator of the standard error of the fixed effects parameters will be used in order to deal with possible model misspecification of the covariance matrix.

Small centers will be defined as centers that do not have at least one evaluable subject (evaluable with regard to the primary efficacy variable) in each treatment arm and each type of trauma (combat related Yes/No) in Phase B. All small centers will be pooled to form "pseudo centers" for the purpose of analysis according to the following algorithm. Small centers will be ordered from the largest to the smallest based on the number of evaluable subjects (i.e., subjects who have baseline and at least one post-baseline value for the primary endpoint in Phase B). The process will start by pooling the largest of the small centers with the smallest of the small centers until a non-small center is formed. This process will be repeated using the centers left out of the previous pass. In case of ties in center size among the largest centers, the center with the smallest center code will be selected. In case of ties in center size among the smallest centers, the center with the largest center code will be selected. If any centers are left out at the end of this process, they will be pooled with the smallest pseudo centers, or if no pseudo centers exist, they will be pooled with the smallest non-small center.

The following 5 comparisons after randomization will be estimated as the difference between Least Squares means utilizing the computing software SAS procedure PROC MIXED.

- Brexpiprazole plus Sertraline vs Placebo
- Brexpiprazole plus Sertraline vs Sertraline


16

- Brexpiprazole plus Sertraline vs Brexpiprazole
- Brexpiprazole vs Placebo
- Sertraline vs Placebo (as assay sensitivity analysis)

The hierarchical testing procedure that was planned in the protocol will not be performed due to the exploratory nature of the PoC (Proof of Concept) study.

#### 8.1.2 Technical Computation Details for Primary Efficacy Analysis

The SAS code for the PROC MIXED procedure to carry out the above MMRM analysis with an unstructured variance covariance structure is illustrated as follows:

```
proc mixed;
class treatment center visit subjid traumatype;
model change=treatment traumatype center visit treatment*visit baseline*visit /s cl
ddfm=kenwardroger;
repeated visit /type=un subject=subjid r rcorr;
lsmeans treament*visit / pdiff cl alpha=0.05 slice=visit;
run;
```

## 8.1.3 Sensitivity Analyses

## 8.1.3.1 Sensitivity Analyses for Missing at Random (MAR) Assumption

Traditionally the dropout mechanisms are divided into three types (Little, 1995): (1) Missing Completely at Random (MCAR), in which the probability of dropout doesn't depend on the observed data and the missing data; (2) Missing at Random (MAR), in which the probability of dropout depends on the observed data, and (3) Missing Not at Random (MNAR), where the probability of dropout depends on the missing data and possibly the observed data.

Most of MNAR methods (Diggle P, Kenward MG, 1994) have treated all observations with dropout as if they fall within the same dropout type. In practice, we would find that different dropout reasons may be related to the outcomes in different ways, for example, detailed dropout reasons for this study are: adverse events (AE), lack of efficacy (LOE), lost to follow-up, protocol deviation, sponsor discontinued study, subject met (protocol specified) withdrawal criteria, subject was withdrawn from participation by the investigator, and subject withdrew consent to participate. Dropout due to an AE and LOE may lead to MNAR dropout. Subject withdrew consent may also lead to MNAR dropout. However, it is debatable whether a dropout caused by subjects withdrew consent is MAR or MNAR. Except AE, LOE, and subject withdrew consent, all the other dropout reasons may be assumed as either MCAR or MAR dropout.


17

As sensitivity analyses for missing at random (MAR) assumption, analyses for missing not at random (MNAR) will be carried out. Pattern Mixture Models (PMM) based on Multiple Imputation (MI) with mixed missing data mechanisms will be used to investigate the response profile of dropout patients by last dropout reason under MNAR mechanism for the following three scenarios:

- 1) Dropout reasons due to either AE or LOE as MNAR
- 2) Dropout reasons due to either AE or LOE or subject withdrew consent as MNAR
- 3) All dropouts as MNAR

#### **Delta Adjustment Imputation Methods**

This MNAR sensitivity analysis is to departure from MAR assumption by progressively increasing the delta until conclusion from the primary analysis is overturned. The delta is 0%, 10%, 20%, 30%, .., 100% of the expected treatment difference of 6.5 points and/or the observed treatment difference between the active arm and Placebo from the primary analysis of MMRM model until conclusion of the primary analysis is overturned. When delta=0 it is MAR. When delta > 0 it is MNAR.

- 1) Using Monte Carlo Markov Chain (MCMC) methodology from PROC MI to impute the intermittent missing data to a monotone missing pattern;
- Using a standard MAR-based multiple imputation approach from PROC MI to impute the monotone missingness data
- 3) For patients in the treated group and with a dropout reason of AE or LOE or subject withdrew consent, a delta will be added for all the values after the dropout time.
- 4) Using MMRM model in the primary analysis to analyzed the completed data using PROC MIXED on the multiple imputed data
- 5) Obtaining the overall results using PROC MIANALYZE.

#### **Placebo Based Imputation Methods**

Similar to "Standard" multiple imputations, except parameters for imputation model obtained from only the placebo (control) group. Missing data for both placebo and drug group are imputed based on the imputation model derived from placebo data. If drug improved outcomes prior to dropout, this benefit is carried into subsequent imputed values, but will diminish over time in accordance with the correlation structure.

In addition, model based MNAR methods such as the shared parameter model (Wu and Baily, 1989) and random coefficient pattern mixture model (Hedeker D, Gibbons RD, 1997) will be also performed.


18

#### **LOCF and OC Analyses**

Change from baseline for the CAPS-5 total score will be evaluated using ANCOVA treatment and, in LOCF analyses, study center and type of trauma as main effects. For the OC analyses, study center and type of trauma will not be included in the model.

## 8.1.3.2 Sensitivity Analyses for Violation of Normality Assumption

The primary endpoint MMRM analysis is a maximum likelihood method that relies on normality assumption. Residual analyses will be carried out to examine model assumption.

In the case of gross violations of the normality assumptions, nonparametric van Elteren test<sup>8</sup> (van Elteren, 1960) will be performed to compare treatment effect on both LOCF dataset and Multiple Imputation (MI) data. The van Elteren test is a generalized Cochran-Mantel-Haenszel (CMH) procedure useful for stratified continuous data in non-normal setting. It belongs to a general family of Mantel-Haenszel mean score tests. The test is performed via SAS procedure PROC FREQ, by including CMH2 and SCORES=MODRIDIT options in the TABLE statement. The stratification factor is trial center and type of trauma.

In addition, other methods that are robust to distributional assumption will also be performed to provide different views on the primary efficacy result, these include generalized estimating equations (GEE), weighted GEE (WGEE), and MI-robust regression<sup>9</sup>.

For MI-van Elteren test and MI-robust regression, imputation datasets will be generated with SAS MI procedure, each dataset will be analyzed, then an overall estimate is derived with SAS MIANALYZE procedure.

#### 8.1.4 Subgroup Analyses

Subgroup analyses of change from baseline (Week 1 visit) in CAPS-5 total score to every study week in Phase B will be performed by the following factors:

- Sex (Based on the biological status at birth)
- Race (White and All Other Races)
- Age (Age<55, and Age $\geq$ 55)




19



- Type of trauma (combat related Yes/No)
- Presence/Absence of psychosocial support at baseline
- Previous pharmacological treatment intervention for PTSD (Yes/No)
- Use of the wearable device (Yes/No). Subjects who have actigraphy data are considered as using the wearable device.
- Years since the index traumatic event ( $<5, \ge 5$  <10, and  $\ge 10$  years)
- Age group (Age $\leq$ 30, Age $\geq$ 30  $\leq$ 40, and Age $\geq$ 40)

All subgroup analyses will be conducted using the same MMRM analysis as for the primary efficacy analysis except that the fixed class effect term for trial center and type of trauma will not be included in the model.

Interaction effects of treatment-by-subgroup will be assessed for the subgroups identified in the previous paragraph. MMRM analyses will be performed by adding addition of terms for subgroup-by-week and treatment-by-subgroup-by-week. These treatment-by subgroup interaction analyses will be presented in statistical documentation.

## 8.2 Other Efficacy Endpoints

Other efficacy variables are as follows:

- 1) Change from baseline in CAPS-5 for every trial week visit in Phase B;
- 2) Change from baseline for every trial week visit in Phase B in PTSD behavior cluster sub scores of CAPS-5:
  - re-experiencing cluster sub score
  - avoidance cluster sub score
  - negative cognitions and mood cluster sub score
  - arousal cluster sub score
- 3) Change from baseline for every trial week visit in Phase B in CGI-S score;
- 4) Response at each visit in Phase B as defined by:
  - decrease from baseline  $\geq$  30% in CAPS-5 total score
  - decrease from baseline by > 11 points in CAPS-5 total score


20

- 5) Shift in CAPS-5 PTSD severity category (moderate, severe or extreme at baseline to asymptomatic, mild, moderate, severe or extreme at each visit). The following categories are based on CAPS-5 total score.
  - 0 19 = asymptomatic/few symptoms,
  - 20 39 = mild PTSD/subthreshold,
  - 40 59 = moderate PTSD/threshold
  - 60 79 = severe PTSD symptomatology
  - $\geq$  80 = extreme PTSD symptomatology
- 6) Change from baseline in SOTS total score for every trial week visit in Phase B;
- 7) Change from baseline in HADS subscale score (anxiety and depression) for every trial week visit in Phase B;
- 8) Change from baseline in PCL-5 total score for every trial week visit in Phase B;
- 9) Sleep related endpoints (see Section 8.3 for details)

The continuous efficacy endpoints will be analyzed using MMRM model similar to that of pre-specified for change from baseline in CAPS-5 total score, correcting for the relevant values at randomization.

The response in variables will be evaluated by the Cochran-Mantel-Haenszel (CMH) General Association Test controlling, in LOCF analysis, for study center and type of trauma.

LOCF and OC analyses using ANCOVA will also be conducted for the continuous efficacy endpoints. The LOCF analysis model includes baseline value as covariate, and, treatment trial center and type of trauma as main effects. For the OC analyses, the model includes terms for baseline value as covariate, and treatment as main effect; trial center and type of trauma will not be included in the model.

Statistical significance for analysis of all other efficacy variables (1) through (4) and (6) through (9) will be evaluated at a nominal 0.05 level (two-sided).

As assay sensitivity analysis, a comparison of sertraline versus placebo will be performed for other efficacy endpoints.

## 8.3 Analyses for Sleep-related Endpoints

The sleep-related endpoints are derived from the data downloaded from the wearable device. Use of the wearable device is optional. The analyses for sleep-related endpoints will include only subjects who agree to the use of the wearable device.

The sleep-related endpoints are as follows:

- Change from baseline in sleep parameters (Sleep Efficiency, Wake after Sleep Onset, Total Sleep Time, and Sleep Latency) for every week in Phase B;
- Proportion of subjects within the normal range of each sleep parameter for every week in Phase B. The normal range of each sleep parameter is defined as follows:
  - Sleep Efficiency: 85% or greater
  - o Wake after Sleep Onset: less than 40 minutes
  - o Total Sleep Time: greater than 370 minutes
  - o Sleep Latency: 10-20 minutes
- Shift in status (within or out of the normal range at baseline to within or out of the normal range at each week) for each sleep parameter

Change from baseline in sleep parameters will be analyzed similarly to other continuous efficacy endpoints. Proportion of subjects within the normal range of each sleep parameter will be analyzed similarly to the response in other efficacy endpoints.

Subgroup analyses of change from baseline in CAPS-5 total score and CGI-S score to every study week in Phase B will be performed by the status (within or out of the normal range) of sleep parameters (Sleep Efficiency, Wake after Sleep Onset, Total Sleep Time, and Sleep Latency) at baseline. Summary statistics will be provided.

Additionally, subgroup analyses of change from baseline (Week 1 visit) in sleep parameters to every study week in Phase B will be performed based on the following baseline characteristics. Summary statistics will be provided.

- Type of trauma (combat related Yes/No)
- History of TBI (Question 1 Yes/No in Step 1 of the OSU TBI-ID)
- Use (current, former or never) of tobacco, alcohol and drug substance based on Tobacco-Alcohol-Substance Use Review form. The use of current, former or never is defined as follows.
  - If subjects used any types of tobacco/alcohol/drug currently then the use at baseline is current; if subjects did not use any types of tobacco/alcohol/drug currently and used any types formerly then the use at baseline is former; otherwise the use at baseline is never.

Relationships between sleep parameters and the following scales will be explored using Pearson correlation coefficient.

- CAPS-5 total score
- CGI-S score

- HADS subscale score (anxiety and depression)
- E6 'Sleep disturbance severity' (score ranging from 0 to 4) from CAPS-5
- Item 2 'Repeated, disturbing dreams of the stressful experience' (score ranging from 0 to 4) from PCL-5
- Item 20 'Trouble falling or staying asleep' (score ranging from 0 to 4) from PCL-5
- Item 1 'Re-experiencing' (score ranging from 1 to 7) from SOTS

Relationships between sleep parameters and the following binary scales will be explored using Chi-square test for independence between sleep parameters (within or out of normal range) and the clinical scales (yes or no) if data allow.

- E6 'Sleep disturbance symptom' (Yes/No) from CAPS-5
- Suicidality from C-SSRS. Suicidality is defined as report of at least one occurrence of any type of suicidal ideation or at least one occurrence of any type of suicidal behavior during assessment period (count each person only once).

The mean daily values of sleep parameters per patient per week will be calculated as the mean of the available daily values in 7 days interval prior to the week. Baseline (Week 1) value is the mean of the available daily values from 7 days prior to Day 1 (relative to the first day of double-blind IMP in Phase B). Week 2 value is the mean of the available daily values from Day 1 to Day 7, Week 3 value is the mean of the available daily values from Day 8 to Day 14, ... etc.

#### 8.4 Exploratory Analysis

Exploratory efficacy analyses will be presented in Statistical Documentation.

Treatment-by-center interaction will be assessed by including the treatment-by-center-by-visit interaction in the model. Results for study centers will be displayed from largest center to smallest center.

Line Item score will be performed for CAPS-5, HADS and PCL-5 on change from baseline and for SOTS on change from baseline to Week 12 using the MMRM model for CAPS-5, SOTS, HADS and PCL-5, where Cohen's D Effect Size is the difference between the two means divided by their standard deviation [as defined by Cohen's D and reviewed on pages 4-6 from the Sage book "Effect Size for ANOVA Designs" (Vol 129) by Cortina and Nouri]. For MMRM (using SAS PROC MIXED), LSMean difference of treatment effects for the between brexpiprazole + sertraline vs placebo, brexpiprazole vs placebo, and brexpiprazole + sertraline vs sertraline, separately, and the corresponding standard error of the difference (Stderr) will be obtained with an Estimate statement. Let n1 and n2 denote the


23

respective sample sizes of the two groups to compare, Effect Size = d = (LSMean1 - LSMean2) / Sigma, where Sigma = Stderr / SQRT( 1/n1 + 1/n2).



# 9 Safety Analysis

Standard safety variables to be analyzed include Adverse Events (AEs), clinical laboratory tests, vital signs, body weight, waist circumference, BMI, 12-lead electrocardiograms (ECGs), and physical examinations. In addition, data from the following safety scales will be evaluated: Abnormal Involuntary Movement Scale (AIMS), Simpson-Angus Scale (SAS), Barnes Akathisia Rating Scale (BARS) and Columbia-Suicide Severity Rating Scale (C-SSRS).

Analyses of Phase B safety data will be performed on the Safety Sample unless indicated otherwise. In general, baseline of a safety variable is defined as the last observation of the variable before taking the first dose of IMP, unless specified otherwise. Prospectively defined criteria will be used to identify potentially clinically relevant abnormal values for clinical laboratory tests, vital signs, ECGs, and body weight.

#### 9.1 Adverse Events

All adverse events will be coded by System Organ Class (SOC) and Preferred Term (PT) according to the Medical Dictionary for Regulatory Activities (MedDRA). AEs that are sexspecific, e.g., ovarian cancer, will have their incidence rates evaluated for the specific sex.

Treatment-emergent AEs (TEAEs) in Phase B are defined as AEs with an onset date on or after the start of double-blind IMP (Week 1). In more detail, TEAEs are all adverse events which started after start of double blind IMP;

Adverse events occurring up to 30 days after the last day of IMP will be included in the summary tables.

The incidence of the following events in Phase B will be tabulated by treatment group and overall using the Safety Sample:

- a) TEAEs
- b) TEAEs by severity


24

- c) TEAEs potentially causally related to the IMP as assessed by the investigator
- d) TEAEs with an outcome of death
- e) Serious TEAEs
- f) TEAEs leading to discontinuations of the IMP

The above summaries (b), (e) and (f) will also be prepared for TEAEs potentially causally related to the IMP.

In addition, incidence of TEAE during Phase B of at least 5% in any treatment group other than placebo group, and also greater than placebo by SOC and PT will be provided.

Incidence of TEAEs by SOC and PT will be summarized for sex, race and age subgroups.

EPS-related AEs will be grouped into five categories.

- 1) Dystonic Events, which include cervical spasm, dystonia, emprosthotonos, muscle contractions involuntary, muscle rigidity, muscle spasms, muscle spasticity, myotonia, nuchal rigidity, oculogyration, opisthotonos, pleurothotonus, risus sardonicus, torticollis, and trismus;
- 2) Parkinsonian Events, which include akinesia, asterixis, athetosis, bradykinesia, cogwheel rigidity, essential tremor, extrapyramidal disorder, freezing phenomenon, gait festinating, hypertonia, hypokinesia, hypokinesia neonatal, intention tremor, masked facies, parkinson's disease, parkinsonian crisis, parkinsonian gait, parkinsonian rest tremor, parkinsonism, tremor, and tremor neonatal;
- 3) Akathisia Events, which include akathisia, hyperkinesia, and psychomotor hyperactivity;
- 4) Dyskinetic Events, which include ballismus, buccoglossal syndrome, choreoathetosis, clumsiness, dyskinesia, dyskinesia neonatal, dyskinesia oesophageal, fumbling, nodding of head, on and off phenomenon, and tardive dyskinesia;
- 5) Residual Events, which include chorea, huntington's chorea, muscle twitching, and myoclonus.

Unless otherwise specified, in general, analysis of safety data will be performed on observed case and for last visit.

#### 9.2 Clinical Laboratory Tests

Summary statistics for routine clinical laboratory measurements and prolactin concentrations will be provided. For Phase B laboratory tests, change from baseline will be summarized by

treatment group. Potentially clinically relevant (PCR) results in laboratory tests will also be summarized.

# 9.2.1 Clinical Laboratory Tests in Phase B

Potentially clinically relevant laboratory measurement test results in Phase B will be identified for the Safety Sample and will be summarized by treatment group and listed. Criteria for identifying laboratory values of potential clinical relevance are provided in Appendix 2.

# 9.2.2 Drug Induced Liver Injury (DILI)

Total bilirubin level should be checked for any subject with increased ALT or AST levels  $\geq$  three times the upper normal limits (ULN) or baseline.

- Reporting all DILI as SAE to the FDA based on Hy's Law:
  - $\square$  AST or ALT  $\geq$  3 x ULN or baseline and
  - $\Box$  T Bili  $\geq 2$  x ULN or baseline

A separate incidence table will be provided for DILI cases, and the corresponding listing will be provided for the Safety Sample during Phase B.

## 9.2.3 Metabolic Change

In addition to mean change from baseline, incidence of treatment emergent significant changes in fasting lipids, fasting glucose, and metabolic syndrome will be summarized by treatment group using the following criteria.

| Criteria for Treatment-Emergent Significant Change in Lipids and Glucose | | |
|---|---|---|
| LAB PARAMETER | BASELINE <sup>1</sup> | ANYTIME POST BASELINE |
| LDL Direct, Fasting | Borderline 100-<160 | High >=160 |
| (MG/DL) | Normal/Borderline <160 | High >=160 |
| | Normal <100 | Borderline/High >=100 |
| | Any Value | Increased >=30 |
| HDL Cholesterol, Fasting | Normal >=40 | Low <40 |
| (MG/DL) | Any Value | Decreased >=20 |
| Triglycerides, Fasting | Normal <150 | High 200-<500 |
| (MG/DL) | Borderline 150-<200 | High 200-<500 |
| | Normal/Borderline <200 | High 200-<500 |
| | Normal <150 | Borderline/High/Very High >=150 |


26

| Criteria for Treatment-Emergent Significant Change in Lipids and Glucose | | |
|---|---|---|
| LAB PARAMETER | BASELINE <sup>1</sup> | ANYTIME POST BASELINE |
| | Any Value | Increased >=50 |
| Glucose Fasting, Serum | Normal <100 | High >=126 |
| (MG/DL) | Impaired 100-<126 | High >=126 |
| | Normal/Impaired <126 | High >=126 |
| | Any Value | Increased >=10 |

BASELINE IS CALCULATED FROM WEEK 1

| Criteria for Treatment-Emergent Metabolic Syndrome | |
|---|---|
| DESCRIPTION | ANYTIME POST BASELINE <sup>1</sup> |
| Central Obesity | Waist Circumference >=102cm(MALE), >=88cm (FEMALE) |
| Dyslipidemia | Triglycerides >= 150mg/dl |
| Dyslipidemia | HDL < 40mg/dl (MALE), <50mg/dl (FEMALE) |
| Supine Blood Pressure | Systolic>=130mmHg and Diastolic>=85mmHg |
| Glucose Fasting, Serum | >=100mg/dl |
| Metabolic Syndrome | Met 3 Or More of the Above Criteria at a Visit |

BASELINE IS CALCULATED FROM WEEK 1

# 9.3 Vital Signs

Summary statistics for vital signs will be provided. For Phase B vital signs, change from baseline (Week 1 visit) will be summarized for the Safety Sample by treatment group.

Potentially clinically relevant vital signs measurements identified in Phase B for the Safety Sample will be summarized by treatment group. Criteria for identifying vital signs of potential clinical relevance are provided in Appendix 1. All potentially clinically relevant events or changes will be listed and included in summary tables.

#### 9.4 12-Lead ECG

Summary statistics and incidence of potentially clinically relevant changes will be provided for ECG parameters.


27

For the analysis of QT and QTc, data from three consecutive complexes (representing three consecutive heart beats) will be measured to determine average values. The following QT corrections will be used for reporting purposes in the clinical study report:

- 1) QTcB is the length of the QT interval corrected for heart rate by the Bazett formula: QTcB=QT/(RR)<sup>0.5</sup> and
- 2) QTcF is the length of the QT interval corrected for heart rate by the Fridericia formula:  $QTcF=QT/(RR)^{0.33}$
- 3) QTcN is the length of the QT interval corrected for heart rate by the FDA Neuropharm Division formula: QTcN=QT/(RR)<sup>0.37</sup>

Potentially clinically relevant changes in the 12-lead ECG identified in Phase B for the Safety Sample will be listed and summarized by treatment group. Criteria for identifying ECG measurements of potential clinical relevance are provided in Appendix 3.

Categorical changes in ECG parameters during Phase B will be summarized based on the following criteria:

| Categorical Change Criteria in QT/QTc Parameters | | |
|---|---|---|
| Classification | Category | Criteria |
| QT | New Onset (> 450 Msec) | New onset (>450 msec) in QT means a subject who |
| | | attains a value > 450 msec during treatment period |
| | | but not at baseline. |
| QTc * | New Onset (≥ 450 Msec | New onset ( $\geq 450$ Msec for men and ( $\geq 470$ Msec |
| | for men and $\geq$ 470 Msec | for women) in QTc means a subject who attains a |
| | for women) | value $\geq 450$ Msec for men or $\geq 470$ Msec for |
| | | women during treatment period but not at baseline. |
| | New Onset (≥ 450 Msec | New onset ( $\geq 450$ Msec for men and $\geq 470$ Msec for |
| | for men and $\geq$ 470 Msec | women) and |
| | for women) | > 10% increase in QTc means a subject who attains |
| | And > 10% Increase | a value $\geq 450$ Msec for men or $\geq 470$ Msec for |
| | | women, and > 10% increase during treatment period |
| | | but not at baseline |
| | New Onset (> 500 Msec) | New onset (> 500 msec) in QTc means a subject |
| | | who attains a value > 500 msec during treatment |
| | | period but not at baseline. |
| | Increase 30 - 60 Msec | Increase from baseline value $> 30$ and $\le 60$ msec in |
| | | QTc |
| | Increase > 60 Msec | Increase from baseline value > 60 msec in QTc |

<sup>\*</sup> QTc categorical change criteria apply to QTcB, QTcF and QTcN.

#### 9.5 Physical Examinations

By-patient listings will be provided for physical examination.


28

# 9.5.1 Body Weight, Waist Circumference and BMI

| Analyses of body weight, waist circumference and BMI will be performed for the Safety |
|---|
| Sample. |
| Dody moss index is defined as visight in hill around divided by the agreement height in material |
| Body mass index is defined as weight in kilograms divided by the square of height in meters. |
| 9.6 SAS, AIMS, and BARS |
| The mean change from baseline to every study week in Phase B obtained from the SAS total score, AIMS total score (total of the first 7 item scores), and the BARS Global Clinical Results will be presented for every scheduled visit, including Week 12. |
| Assessment will be tabulated and analyzed using ANCOVA. Analyses will be performed on the OC data set. In addition, analyses will be performed using the maximum (i.e. the worst) value observed during Phase B |
| The same analyses will be performed on the AIMS individual item scores 8, 9, and 10. In addition, incidence of BARS Global Clinical Assessment of Akathisia during Phase B by severity category will be provided. Analyses of these EPS rating scales will be performed for the Safety Sample. |
| 9.7 Suicidality Data |
| Suicidality will be monitored during the study using the C-SSRS and will be summarized as |
| number and percentage of subjects reporting any suicidal behavior, ideation, behavior by type |
| (4 types), ideation by type (5 types) and treatment emergent suicidal behavior and ideation. |
| Summary will be provided for Phase B. |


29

Suicidality is defined as report of at least one occurrence of any type of suicidal ideation or at least one occurrence of any type of suicidal behavior during assessment period (count each person only once).

Treatment emergent suicidal behavior and ideation is summarized by four types: Emergence of suicidal ideation, Emergence of serious suicidal ideation, Worsening of suicidal ideation, Emergence of suicidal behavior.

Emergence of suicidal behavior/ideation is defined as report of any type of suicidal behavior/ideation during treatment when there was no baseline suicidal behavior/ideation.

Emergence of serious suicidal ideation is defined as observation of suicidal ideation severity rating of 4 or 5 during treatment when there was no baseline suicidal ideation.

Worsening of suicidal ideation is defined as a suicidal ideation severity rating that is more severe than it was at baseline.

#### 9.8 Concomitant Medications

Number and proportion of patients taking concomitant medications prior to Phase B, during Phase B, and after study therapy are tabulated by drug classification using the WHO drug dictionary. For Phase B Randomized Sample, data will be presented by treatment group and overall.

#### 9.9 Extent of Exposure

The start date of double-blind IMP will be the first day of double-blind dosing. The number and percentage of patients who receive double-blind IMP (brexpiprazole or sertraline), will be presented by week and by treatment group. Each dosing week will be based on the actual week; i.e., Day 1-7 in Week 1, Day 8-14 in Week 2, etc. This summary will be performed on the Safety Sample.

The mean daily dosage will be summarized by week and treatment group using descriptive statistics. The mean daily dosage per patient per week will be determined for each week of the study. This will be calculated by dividing the sum of individual total doses by the number of days in the week interval. The summary will contain for each treatment group the number of

patients receiving double-blind IMP, and the mean and range of the mean daily dose for each week.

All the exposure analyses will be done for brexpiprazole or sertraline, separately.

#### 10 Conventions

## 10.1 Study Visit Windows

Study visit windows will be used to map visits using study day intervals. This visit window convention applies to tables and listings for all efficacy and safety scales (CAPS-5, SOTS, CGI-S, PCL-5, HADS, SAS, AIMS, and BARS). This derived study window variable will be named as WEEK and will be footnoted. In listings it will be listed along with the CRF study visit.

Table 10.1A shows classifications for study day intervals in Phase B. The variable "target day" is defined using the number of days since the start of double-blind dosing in Phase B. The first day of double-blind dosing is defined as "Day 1".

If more than one observation falls within a particular study day interval, then the last observation within that interval is used. Evaluations occurring more than 7 days after the last double-blind dosing date will not be mapped into study visit windows, and will be excluded from the analysis.

Table 10.1A: Study Day and Visit Windows in Phase B

| Week | Target Day <sup>a</sup> | Study Day Interval <sup>a</sup> |
|------|-------------------------|---------------------------------|
| 2 | 7 | 2-10 |
| 3 | 14 | 11-17 |
| 4 | 21 | 18-24 |
| 6 | 35 | 25-38 |
| 8 | 49 | 39-52 |
| 10 | 63 | 53-66 |
| 12 | 77 | 67-84 <sup>b</sup> |

a Relative to the first day of double-blind IMP in Phase B.


31

b Evaluations occurring more than seven days after the last double-blind dosing date will be excluded from the Phase B analyses.

## 10.2 Pooling of small centers

Primary efficacy analysis will be performed on the Intent to Treat Sample which comprises those subjects in the Randomized Sample who have a baseline value and at least one post-baseline value for CAPS-5 total score in Phase B. Small centers will be defined as centers that do not have at least one evaluable subject (evaluable with regard to the primary efficacy variable) in each treatment arm and each type of trauma (combat related Yes/No) in Phase B. All small centers will be pooled to form "pseudo centers" for the purpose of analysis according to the following algorithm. Small centers will be ordered from the largest to the smallest based on the number of evaluable subjects

at least one post-randomization value for CAPS-5 total score in Phase B). The process will start by pooling the largest of the small centers with the smallest of the small centers until a non-small center is formed. This process will be repeated using the centers left out of the previous pass. In case of ties in center size among the largest centers, the center with the smallest center code will be selected. In case of ties in center size among the smallest centers, the center with the largest center code will be selected. If any centers are left out at the end of this process, they will be pooled with the smallest pseudo centers, or if no pseudo centers exist, they will be pooled with the smallest non-small center.

Primary efficacy analysis will also be performed on the mITT Sample. The process of pooling of small centers for the analysis based on the mITT Sample is similar to the process for ITT Sample.

#### 10.3 Scales: Rules for Scoring and Handling of Missing Data

#### 10.3.1 CAPS-5

The CAPS-5 is a clinician-rated, structured interview designed to assess PTSD diagnostic status and symptoms severity as defined by the DSM-5. This trial will use the CAPS-5 Past Month and CAPS-5 Past Week versions of the scale. The CAPS-5 comprises questions that target the onset and duration of symptoms, subjective distress, impact of symptoms on social and occupational functioning, improvement in symptoms since a previous CAPS-5 administration, overall response validity, overall PTSD severity, and specifications for the dissociative subtype (depersonalization and derealization).

The CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms (items 1-20) from the following categories:

Category B: Intrusion symptoms (5 items);


32
Category C: Avoidance symptoms (2 items);

Category D: Cognition and mood symptoms (7 items); and

Category E: Arousal and reactivity symptoms (6 items)

If there are more than 1 item in each of categories B, D and E with a missing score, or any item in Category C with a missing score, the CAPS-5 total score is set to missing. For each category (B, D or E) with a missing score, the imputed subscores for that category is the average of the existing scores in the category multiplied by the total number of questions in the category. The CAPS-5 total score will then be imputed by adding all the subscores from categories B, C, D and E.

### 10.3.2 SOTS

The SOTS is a 12-item 7-point symptom severity rating scale designed to measure change. Ratings for each of the 12 symptoms can range from 1 = Absent to 7 = Extreme. Because the SOTS provides a means of rating of symptoms at 7 levels of severity (absent, minimal, mild, moderate, moderate severe, severe, and extreme), it can assess changes in trauma symptoms, which will become increasingly important as new interventions, both psychosocial and pharmacological, emerge.

The SOTS total score is calculated by summing scores from all 12 items. The SOTS total score will be un-evaluable if fewer than 10 of the 12 items are recorded. If 10 or 11 of the 12 items are recorded, the SOTS score will be the mean of the recorded items multiplied by 12 and then rounded to the first decimal place.

#### 10.3.3 CGI-S

The severity of illness for each subject will be rated using the CGI-S. CGI-S items are: 0 = not assessed, 1 = normal, not at all ill, 2 = borderline mentally ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill patients. The score 0 = not assessed) will be set to missing. The CGI-S is therefore a 7-point scale from 1 through 7.

#### 10.3.4 PCL-5

The PCL-5 is a checklist of problems that people sometimes have in response to a very stressful experience. Subjects need to indicate a number to the right of each problem to indicate how much they have been bothered by that problem in the past month. The scale rates items from 0 (not at all), 1 (a little bit), 2 (moderately), 3 (quite a bit), and 4 (extremely).


33

The PCL-5 total score is calculated by summing severity scores for scores from all 20 items. The PCL-5 total score will be un-evaluable if fewer than 16 of the 20 items are recorded. If 16 to 19 of the 20 items are recorded, the PCL-5 total score will be the mean of the recorded items multiplied by 20 and then rounded to the first decimal place.

#### 10.3.5 HADS

The HADS is a subject-rated scale designed to screen for anxiety and depressive states in medical subjects. The HADS consists of 2 subscales: The D-scale measures depression and the A-scale measures anxiety. Each subscale contains 7 items, and each item is rated from 0 (absent) to 3 (maximum severity). The score of each subscale is the sum of scores from each item in the subscale. Each subscale ranges from 0 to 21, The subscales will be analyzed separately. If there are more than 1 item with missing score for a give subscale, the score of the subscale is set to be missing. If 6 of the 7 items are recorded, the score of the subscale will be the mean of the recorded items multiplied by 7 and then rounded to the first decimal place.

#### 10.3.6 SAS

The SAS will be used to evaluate extrapyramidal symptoms (EPS). It consists of a list of 10 symptoms of Parkinsonism (gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, head rotation, glabella tap, tremor, salivation, and akathisia). Each item will be rated on a 5-point scale, with a score of zero representing absence of symptoms, and a score of 4 representing a severe condition. The SAS Total score is the sum of ratings for all 10 items, with possible Total scores from 0 to 40. The SAS Total score will be un-evaluable if less than 8 of the 10 items are recorded. If 8 or 9 of the 10 items are recorded, the Total score will be the mean of the recorded items multiplied by 10 and then rounded to the first decimal place.

#### 10.3.7 AIMS

The AIMS is a 12-item scale. The first 10 items are rated from 0 to 4 (0=best, 4=worst). An item score of 0, depending on the item, either means: no abnormal involuntary movement (AIM), or no incapacitation due to AIM, or no awareness of AIM. An item score of 4 either means: severe AIM, or severe incapacitation due to AIM, or being aware of, and severe distress caused by AIM. Items 11 and 12, related to dental status, have dichotomous responses, 0=no and 1=yes. The AIMS Total Score is the sum of the ratings for the first seven items. The possible total scores are from 0 to 28. The AIMS Total Score will be un-evaluable if less than 6 of the first 7 items are recorded. If 6 of the items are recorded, then the total

score will be the mean of the recorded items multiplied by 7 and then rounded to the first decimal place.

#### 10.3.8 BARS

The BARS consists of 4 items related to akathisia: objective observation of akathisia by the investigator, subjective feelings of restlessness by the subject, subjective distress due to akathisia, and global clinical assessment of akathisia. The first 3 items will be rated on a 4-point scale, with a score of zero representing absence of symptoms and a score of 3 representing a severe condition. The global clinical evaluation will be made on a 6-point scale, with zero representing absence of symptoms and a score of 5 representing severe akathisia.

#### 10.3.9 C-SSRS

Suicidality will be monitored during the trial using the C-SSRS. This trial will use the "baseline/screening" and "Since Last Visit" versions of the scale. The "baseline/screening" version, which assesses the lifetime experience of the subject with suicide events and suicidal ideation and the occurrence of suicide events and/or ideation within a specified time period prior to entry into the trial, will be completed for all subjects at screening to determine eligibility. Any subject with active suicidal ideation within the last 6 months, suicidal behaviors within the last 2 years, or who in the clinical judgment of the investigator presents a serious risk of suicide should be excluded from the trial. The "Since Last Visit" C-SSRS form will also be completed at all visits after screening.

## 11 References

- Siddiqui O, Hung JHM, O'Neill R. MMRM vs. LOCF: A comprehensive comparison based on simulation study and 25 NDA datasets. J Biopharmaceutical Stats. 2009; 19(2):227-46.
- Diggle P, Kenward MG. Informative drop-out in longitudinal data analysis. Applied Statistics. 1994;43:49-93.
- Little RJA. Pattern-mixture models for multivariate incomplete data. J Am Stat Assoc. 1993;88:125-34.
- <sup>4</sup> Little RJA. Modeling the drop-out mechanism in repeated measures studies. J Am Stat Assoc. 1995;90:1112-21.
- Hedeker D, Gibbons RD. Application of random effects pattern-mixture models for missing data in longitudinal studies. Psychological Methods. 1997;2:64-78.
- Ali MW, Siddiqui O. Multiple imputation compared with some information dropout procedures in the estimation and comparison of rates of change in longitudinal clinical trials with dropouts. J Biopharmaceutical Stats. 2000;10(2):165-81.
- Wu MC, Bailey KR. Estimation and comparison of changes in the presence of informative right censoring: Conditional linear model. Biometrics. 1989;45:939-55.
- van Elteren, PH. On the combination of independent two sample tests of Wilcoxon. Bull Int Stat Inst. 1960;37:351-61.
- Mehrotra D, Li X, Liu J, Lu K. Analysis of Longitudinal Clinical Trials with Missing Data Using Multiple Imputation in Conjunction with Robust Regression. Biometrics 2012;68:1250-1259.
- Cortina, J. M., & Nouri, H. (2000). *Effect size for ANOVA designs*. Thousand Oaks, Calif.: Sage Publications.

## 12 Potential Clinical Relevance Criteria from Protocol

## **Appendix 1** Criteria for Identifying Vital Signs of Potential Clinical Relevance

| Variable | Criterion Value <sup>a</sup> | Change Relative to Baseline <sup>a</sup> |
|---|---|---|
| Heart Rate <sup>b</sup> | > 120 bpm<br>< 50 bpm | ≥ 15 bpm increase<br>≥ 15 bpm decrease |
| Systolic Blood Pressure <sup>b</sup> | > 180 mmHg<br>< 90 mmHg | ≥ 20 mmHg increase<br>≥ 20 mmHg decrease |
| Diastolic Blood Pressure <sup>b</sup> | > 105 mmHg<br>< 50 mmHg | ≥ 15 mmHg increase<br>≥ 15 mmHg decrease |
| Orthostatic Hypotension | ≥ 20 mmHg decrease in systolic blood<br>pressure and a ≥ 25 bpm increase in<br>heart rate from supine to<br>sitting/standing | Not Applicable (baseline status not considered) |
| Weight | - | ≥ 7% increase<br>≥ 7% decrease |

<sup>&</sup>lt;sup>a</sup> In order to be identified as potentially clinically relevant, an on-treatment value must meet the "Criterion Value" and also represent a change from the subject's baseline value of at least the magnitude shown in the "Change Relative to Baseline" column.

<sup>&</sup>lt;sup>b</sup> As defined in "Supplementary Suggestions for Preparing an Integrated Summary of Safety Information in an Original NDA Submission and for Organizing Information in Periodic Safety Updates," FDA Division of Neuropharmacological Drug Products draft (2/27/87).

Appendix 2 Criteria for Identifying Laboratory Values of Potential Clinical Relevance

| <b>Laboratory Tests</b> | Criteria |
|---|---|
| Chemistry | |
| AST (SGOT) | $\geq$ 3 x upper limit of normal (ULN) |
| ALT (SGPT) | $\geq 3 \times ULN$ |
| Alkaline phosphatase | $\geq 3 \times ULN$ |
| Lactate dehydrogenase (LDH) | $\geq 3 \times ULN$ |
| Blood urea nitrogen (BUN) | $\geq 30 \text{ mg/dL}$ |
| Creatinine | $\geq 2.0 \text{ mg/dL}$ |
| Uric Acid | |
| Men | $\geq 10.5 \text{ mg/dL}$ |
| Women | $\geq$ 8.5 mg/dL |
| Bilirubin (total) | $\geq 2.0 \text{ mg/dL}$ |
| Creatine phosphokinase (CPK) | $\geq 3 \times ULN$ |
| Prolactin | > ULN |
| Hematology | |
| Hematocrit | |
| Men | $\leq$ 37 % and decrease of $\geq$ 3 percentage points from Baseline |
| Women | $\leq$ 32 % and decrease of $\geq$ 3 percentage points from Baseline |
| Hemoglobin | |
| Men | $\leq 11.5 \text{ g/dL}$ |
| Women | $\leq 9.5 \text{ g/dL}$ |
| White blood count | $\leq 2,800/ \text{ mm}^3 \text{ or } \geq 16,000/ \text{ mm}^3$ |
| Eosinophils | ≥ 10% |
| Neutrophils | ≤ 15% |
| Absolute neutrophil count | $\leq 1,000/\mathrm{mm}^3$ |
| Platelet count | $\leq 75,000/ \text{ mm}^3 \text{ or } \geq 700,000/ \text{ mm}^3$ |
| Urinalysis | |
| Protein | Increase of $\geq 2$ units |
| Glucose | Increase of $\geq 2$ units |
| Casts | Increase of $\geq 2$ units |
| Additional Criteria | |
| Chloride | $\leq$ 90 mEq/L or $\geq$ 118 mEq/L |
| Potassium | $\leq 2.5 \text{ mEq/L or} \geq 6.5 \text{ mEq/L}$ |
| Sodium | $\leq$ 126 mEq/L or $\geq$ 156 mEq/L |
| Calcium | $\leq 8.2 \text{ mg/dL or} \geq 12 \text{ mg/dL}$ |
| Glucose | |
| Fasting | $\geq 100 \text{ mg/dL}$ |
| Non-Fasting | $\geq 200 \text{ mg/dL}$ |
| Total Cholesterol, Fasting | $\geq 240 \text{ mg/dL}$ |
| LDL Cholesterol, Fasting | $\geq 160 \text{ mg/dL}$ |
| HDL Cholesterol, Fasting | |
| Men | < 40 mg/dL |
| Women | < 50 mg/dL |
| Triglycerides, Fasting | ≥ 150 mg/dL |


38

Appendix 3 Criteria for Identifying ECG Measurements of Potential Clinical Relevance

| Variable | Criterion Value <sup>a</sup> | Change Relative to Baseline <sup>a</sup> |
|---|---|---|
| Rate | | |
| Tachycardia | ≥ 120 bpm | increase of $\geq 15$ bpm |
| Bradycardia | ≤ 50 bpm | decrease of $\geq 15$ bpm |
| Rhythm | | |
| Sinus tachycardia <sup>b</sup> | ≥ 120 bpm | increase of $\geq 15$ bpm |
| Sinus bradycardia <sup>c</sup> | ≤ 50 bpm | decrease of $\geq 15$ bpm |
| Supraventricular premature beat | all | not present → present |
| Ventricular premature beat | all | not present → present |
| Supraventricular tachycardia | all | not present → present |
| Ventricular tachycardia | all | not present → present |
| Atrial fibrillation | all | not present → present |
| Atrial flutter | all | not present $\rightarrow$ present |
| Conduction | | |
| 1° atrioventricular block | $PR \ge 200 \text{ msec}$ | increase of $\geq 50$ msec |
| 2° atrioventricular block | all | not present $\rightarrow$ present |
| 3° atrioventricular block | all | not present $\rightarrow$ present |
| Left bundle-branch block | all | not present $\rightarrow$ present |
| Right bundle-branch block | all | not present $\rightarrow$ present |
| Pre-excitation syndrome | all | not present $\rightarrow$ present |
| Other intraventricular conduction block <sup>d</sup> | QRS $\geq$ 120 msec | increase of $\geq 20$ msec |
| Infarction | | |
| Acute or subacute | all | not present → present |
| Old | all | not present → present |
| | | ≥ 12 weeks post study entry |
| ST/T Morphological | | |
| Myocardial Ischemia | all | not present $\rightarrow$ present |
| Symmetrical T-wave inversion | all | not present $\rightarrow$ present |
| Increase in QTc | QTcF $\geq$ 450 msec | |
| | (men) $QTcF \ge 470 \text{ msec}$ | |
| | (women) | |

<sup>&</sup>lt;sup>a</sup> In order to be identified as potentially clinically relevant, an on-treatment value must meet the "Criterion Value" and also represent a change from the subject's baseline value of at least the magnitude shown in the "Change Relative to Baseline" column.


39

<sup>&</sup>lt;sup>b</sup> No current diagnosis of supraventricular tachycardia, ventricular tachycardia, atrial fibrillation, atrial flutter, or other rhythm abnormality.

<sup>&</sup>lt;sup>c</sup> No current diagnosis of atrial fibrillation, atrial flutter, or other rhythm abnormality.

<sup>&</sup>lt;sup>d</sup> No current diagnosis of left bundle branch block or right bundle branch block.

# 13 Proposed List of Summary Tables

- CT-1.1 Subject Disposition (Randomized Sample)
- CT-1.2 Subject Disposition by Center (Randomized Sample)
- CT-1.3 Subject Completion Rates by Week During Phase B (Randomized Sample)
- CT-1.4.1 Enrollment by Country (Randomized Sample)
- CT-1.4.2 Enrollment by Country by Age Group (Randomized Sample)
- CT-2.1 Reasons for Discontinuation in Phase B (Randomized Sample)
- CT-3.1.1 Demographic and Baseline Characteristics (Randomized Sample)
- CT-3.1.2 Demographic and Baseline Characteristics by Trauma Type (Randomized Sample)
- CT-3.1.3 Demographic and Baseline Characteristics by Use of Wearable Device (Randomized Sample)
- CT-3.1.4 Demographic and Baseline Characteristics by Placebo 20% Non-Responder Status (Randomized Sample)
- CT-3.1.5 Demographic and Baseline Characteristics by Placebo 25% Non-Responder Status (Randomized Sample)
- CT-3.1.6 Demographic and Baseline Characteristics by Placebo 30% Non-Responder Status (Randomized Sample)
- CT-3.2.1 Medical History (Randomized Sample)
- CT-3.2.2 Psychiatric History (Randomized Sample)
- CT-3.2.3 PTSD Treatment History Based on Emory Treatment Resistance Interview (E-TRIP) (Randomized Sample)
- CT-3.2.4 PTSD Disease History (Randomized Sample)
- CT-3.3.1 MINI International Neuropsychiatric Interview (M.I.N.I.) (Randomized Sample)
- CT-3.3.2 Summary on Life Events Checklist for DSM-5 (LEC-5) (Randomized Sample)
- CT-3.3.3 Summary on Ohio State University Traumatic Brain Injury Identification (OSU TBI-ID) Method (Randomized Sample)
- CT-3.4 Baseline Psychiatric Scale Evaluations (Randomized Sample)
- CT-4.1 Concomitant Medications: Medications Taken Prior to Start of Study Therapy (Safety Sample)
- CT-4.2 Concomitant Medications: Medications Taken During Phase B (Safety Sample)
- CT-4.3 Concomitant Medications: Medications Taken Post Study Therapy (Safety Sample)
- CT-5.1 Summary of Efficacy Results (Intent to Treat Sample)
- CT-5.2.1 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score MMRM, UN (Intent to Treat Sample)
- CT-5.2.2 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score MMRM, TOEPH Empirical (Intent to Treat Sample)
- CT-5.2.3 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score MMRM, ARH1 Empirical (Intent to Treat Sample)


40



- CT-5.7.1 Summary of Mean Change from Baseline (Day 0) to Phase B by Study Week in Symptoms of Trauma Scale (SOTS) Total Score MMRM, UN (Intent to Treat Sample)
- CT-5.7.2 Summary of Mean Change from Baseline (Day 0) to Phase B by Study Week in Symptoms of Trauma Scale (SOTS) Total Score LOCF (Intent to Treat Sample)
- CT-5.7.3 Summary of Mean Change from Baseline (Day 0) to Phase B by Study Week in Symptoms of Trauma Scale (SOTS) Total Score OC (Intent to Treat Sample)


41




42

- CT-5.10.5.5 Summary of Mean Change
  Parameters by Use of Tobacco OC (Intent to Treat Sample)
- CT-5.10.6 Correlations between Sleep Parameters and Clinical Scales
- CT-5.10.7 Relationship between Sleep Parameters and Categorical Clinical Scales
- CT-5.11.1 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score MI, VAN ELTEREN TEST (Intent to Treat Sample)
- CT-5.11.2 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score GEE (Intent to Treat Sample)
- CT-5.11.3 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score WGEE (Intent to Treat Sample)
- CT-5.12.1 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 1) in CAPS-5 Total Score Assume All Dropouts as MNAR (Intent to Treat Sample)
- CT-5.12.2 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 2) in CAPS-5 Total Score Assume All Dropouts as MNAR (Intent to Treat Sample)
- CT-5.12.3 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 1) in CAPS-5 Total Score Dropout due to AE or LOE or Withdrew Consent as MNAR (Intent to Treat Sample)
- CT-5.12.4 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 2) in CAPS-5 Total Score Dropout due to AE or LOE or Withdrew Consent as MNAR (Intent to Treat Sample)
- CT-5.12.5 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 1) in CAPS-5 Total Score Dropouts due to AE or Lack of Efficacy (LOE) as MNAR (Intent to Treat Sample)
- CT-5.12.6 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 2) in CAPS-5 Total Score Dropouts due to AE or Lack of Efficacy (LOE) as MNAR (Intent to Treat Sample)
- CT-5.12.7 Sensitivity Analysis of MNAR using Placebo Based Imputation in CAPS-5 Total Score (Intent to Treat Sample)
- CT-5.12.8 Sensitivity Analysis of MNAR Using Model Based Methods: Shared Parameter Model and Random Coefficient Pattern Mixture Model –OC (Intent to Treat Sample)
- CT1-5.1 Summary of Efficacy Results (Modified Intent to Treat Sample)
- CT1-5.2.1 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score MMRM, UN (Modified Intent to Treat Sample)
- CT1-5.2.2 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score MMRM, TOEPH Empirical (Modified Intent to Treat Sample)
- CT1-5.2.3 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score MMRM, ARH1 Empirical (Modified Intent to Treat Sample)
- CT1-5.2.4 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score MMRM, CSH Empirical (Modified Intent to Treat Sample)


43



- CT1-5.7.2 Summary of Mean Change from Baseline (Day 0) to Phase B by Study Week in Symptoms of Trauma Scale (SOTS) Total Score - LOCF (Modified Intent to Treat Sample)
- CT1-5.7.3 Summary of Mean Change from Baseline (Day 0) to Phase B by Study Week in Symptoms of Trauma Scale (SOTS) Total Score - OC (Modified Intent to Treat Sample)


44




45



CT-6.9.2 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in the Subgroup with >=5-<10 Years Since Index Traumatic Event – MMRM (Intent to Treat Sample)

CT-6.9.3 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in the Subgroup with >=10 Years Since Index Traumatic Event – MMRM (Intent to Treat Sample)

CT-6.10.1 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in Subjects <30 Years of Age – MMRM (Intent to Treat Sample)

CT-6.10.2 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in Subjects >=30-<40 Years of Age or Older – MMRM (Intent to Treat Sample)

CT-6.10.3 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in Subjects 40 Years of Age or Older – MMRM (Intent to Treat Sample)


46

- CT1-6.1.1 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in the Subgroup of Females MMRM (Modified Intent to Treat Sample)
- CT1-6.1.2 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in the Subgroup of Males MMRM (Modified Intent to Treat Sample)
- CT1-6.2.1 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in the Subgroup of Whites MMRM (Modified Intent to Treat Sample)
- CT1-6.2.2 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in the Subgroup of All Other Races MMRM (Modified Intent to Treat Sample)
- CT1-6.3.1 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in SubjeCT1s <55 Years of Age MMRM (Modified Intent to Treat Sample)
- CT1-6.3.2 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in SubjeCT1s >=55 Years of Age or Older MMRM (Modified Intent to Treat Sample)
- CT1-6.4.1.1 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in SubjeCT1s with <20% Improvement and CAPS-5 Total Score at Least 27 at Week 1 MMRM (Modified Intent to Treat Sample)
- CT1-6.4.1.2 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in Subjects with >=20% Improvement or CAPS-5 Total Score <27 at Week 1 MMRM (Modified Intent to Treat Sample)
- CT1-6.4.2.1 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in Subjects with <25% Improvement and CAPS-5 Total Score at Least 27 at Week 1 MMRM (Modified Intent to Treat Sample)
- CT1-6.4.2.2 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in Subjects with >=25% Improvement or CAPS-5 Total Score <27 at Week 1 MMRM (Modified Intent to Treat Sample)
- CT1-6.5.1 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in the Subgroup with Combat-related Trauma MMRM (Modified Intent to Treat Sample)
- CT1-6.5.2 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in the Subgroup without Combat-related Trauma MMRM (Modified Intent to Treat Sample)
- CT1-6.6.1 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in the Subgroup with Psychosocial Support at Baseline MMRM (Modified Intent to Treat Sample)
- CT1-6.6.2 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in the Subgroup without Psychosocial Support at Baseline MMRM (Modified Intent to Treat Sample)
- CT1-6.7.1 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in the Subgroup with Previous Pharmacological Treatment Intervention for PTSD MMRM (Modified Intent to Treat Sample)
- CT1-6.7.2 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in the Subgroup without Previous Pharmacological Treatment Intervention for PTSD MMRM (Modified Intent to Treat Sample)


47

- CT1-6.8.1 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in the Subgroup with Use of Wearable Device MMRM (Modified Intent to Treat Sample)
- CT1-6.8.2 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in the Subgroup without Use of Wearable Device MMRM (Modified Intent to Treat Sample)
- CT1-6.9.1 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in the Subgroup with <5 Years Since Index Traumatic Event MMRM (Modified Intent to Treat Sample)
- CT1-6.9.2 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in the Subgroup with >=5-<10 Years Since Index Traumatic Event MMRM (Modified Intent to Treat Sample)
- CT1-6.9.3 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in the Subgroup with >=10 Years Since Index Traumatic Event MMRM (Modified Intent to Treat Sample)
- CT1-6.10.1 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in Subjects <30 Years of Age MMRM (Modified Intent to Treat Sample)
- CT1-6.10.2 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in Subjects >=30-<40 Years of Age or Older MMRM (Modified Intent to Treat Sample)
- CT1-6.10.3 Summary of Mean Change to Phase B by Study Week in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score in Subjects 40 Years of Age or Older MMRM (Modified Intent to Treat Sample)
- CT-7.1 Extent of Exposure to Study Medication During Phase B (Safety Sample)
- CT-7.2.1 Number and Percentage of Subjects Receiving Brexpiprazole and Mean and Range of Average Daily Dose in Phase B (Safety Sample)
- CT-7.2.2 Number and Percentage of Subjects Receiving Sertraline and Mean and Range of Average Daily Dose in Phase B (Safety Sample)
- CT-8.1 Adverse Events (Safety Sample)
- CT-8.2.1 Incidence of TEAEs During Phase B by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.2.2 Incidence of TEAEs During Phase B by System Organ Class, MedDRA Preferred Term and Severity (Safety Sample)
- CT-8.2.3 Incidence of TEAE During Phase B of at Least 5% in Any Brexipiprozole or Sertraline Group and Greater Than Placebo by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.2.4 Incidence of TEAEs During Phase B by System Organ Class and MedDRA Preferred Term, by Sex (Safety Sample)
- CT-8.2.5 Incidence of TEAEs During Phase B by System Organ Class and MedDRA Preferred Term, by Race (Safety Sample)
- CT-8.2.6 Incidence of TEAEs During Phase B by System Organ Class and MedDRA Preferred Term, by Age (Safety Sample)
- CT-8.2.7 Incidence of Non-Serious TEAE During Phase B of at Least 5% in Any Brexipiprozole or Sertraline Group and Greater Than Placebo by System Organ Class and MedDRA Preferred Term (Safety Sample)


48

- CT-8.2.8 Incidence of TEAE During Phase B of at Least 2% in Any Brexipiprozole or Sertraline Group and Greater Than Placebo by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.2.9 Occurrence (Number of Events) of Serious Treatment-Emergent Adverse Events by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.2.10 Incidence and Occurrence (Number of Events) of All Treatment-Emergent Adverse Events Greater Than or Equal To 5% in Any Treatment Group by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.2.11 Incidence and Occurrence (Number of Events) of Non-Serious Treatment-Emergent Adverse Events Greater Than or Equal To 5% in Any Treatment Group by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.3.1 Incidence of Potentially Drug-Related TEAEs During Phase B by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.3.2 Incidence of Potentially Drug-Related TEAEs During Phase B by System Organ Class, MedDRA Preferred Term and Severity (Safety Sample)
- CT-8.4 Incidence of Deaths Due to TEAEs During Phase B by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.5.1 Incidence of Serious TEAEs During Phase B by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.5.2 Incidence of Serious TEAEs During Phase B by System Organ Class, MedDRA Preferred Term and Severity (Safety Sample)
- CT-8.6.1 Incidence of TEAEs Resulting in Discontinuation from Study Medication During Phase B by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.6.2 Incidence of TEAEs Resulting in Discontinuation from Study Medication During Phase B by System Organ Class, MedDRA Preferred Term and Severity (Safety Sample)
- CT-8.7.1 Incidence of TE EPS-related AEs During Phase B by EPS Category and MedDRA Preferred Term (Safety Sample)
- CT-8.7.2 Incidence of Onset of Akathisia Adverse Event by Week During Phase B (Safety Sample)
- CT-9.1 Listing of Deaths

(Safety Sample)

- CT-9.2 Listing of Serious Adverse Events
- CT-9.3.1 Listing of Discontinuations from Study Medication Due to Adverse Events During Phase B
- CT-9.3.2 Listing of Discontinuations from Study Medication Due to Adverse Events
- CT-10.1 Criteria for Laboratory Test Values with Potential Clinical Relevance
- CT-10.2.1 Listing of Laboratory Test Values with Potential Clinical Relevance During Phase B by Subject (Safety Sample)
- CT-10.2.2 Listing of Laboratory Test Values with Potential Clinical Relevance During Phase B by Test (Safety Sample)
- CT-10.2.3 Incidence of Laboratory Test Values with Potential Clinical Relevance During Phase B (Safety Sample)
- CT-10.3.1 Mean Change in Clinical Laboratory Test Results Serum Chemistry (Safety Sample)

  CT-10.3.2 Mean Change in Clinical Laboratory Test Results Hematology
- CT-10.3.3 Mean Change in Clinical Laboratory Test Results Urinalysis (Safety Sample)


49

- CT-10.3.4 Mean Change in Clinical Laboratory Test Results Prolactin, by Sex (Safety Sample)
- CT-10.4.1 Incidence of Laboratory Test Values with Potential Clinical Relevance During Phase B Prolactin (Safety Sample)
- CT-10.4.2 Listing of Laboratory Test Values with Potential Clinical Relevance During Phase B Prolactin (Safety Sample)
- CT-10.5.1.1 Incidence of Treatment-Emergent Significant Change in Lipids During Phase B (Safety Sample)
- CT-10.5.1.2 Listing of Treatment-Emergent Significant Change in Lipids During Phase B (Safety Sample)
- CT-10.5.2.1 Incidence of Treatment-Emergent Significant Change in Glucose During Phase B (Safety Sample)
- CT-10.5.2.2 Listing of Treatment-Emergent Significant Change in Glucose During Phase B (Safety Sample)
- CT-10.5.3.1 Incidence of Treatment-Emergent Metabolic Syndrome During Phase B (Safety Sample)
- CT-10.5.3.2 Listing of Treatment-Emergent Metabolic Syndrome During Phase B (Safety Sample)
- CT-10.6 Incidence of Potentially Liver Injury Related Laboratory Test Abnormalities During Phase B (Safety Sample)
- CT-10.7 Listing of Potentially Liver Injury Related Laboratory Test Abnormalities During Phase B (Safety Sample)
- CT-11.1 Criteria for Potentially Clinically Relevant Abnormalities in Vital Signs
- CT-11.2.1 Listing of Potentially Clinically Relevant Abnormalities in Vital Signs During Phase B (Safety Sample)
- CT-11.2.2 Incidence of Potentially Clinically Relevant Abnormalities in Vital Signs During Phase B (Safety Sample)
- CT-11.2.3 Mean Change from in Vital Signs During Phase B (Safety Sample)
- CT-11.3.1 Listing of Potentially Clinically Relevant Abnormalities in Vital Signs Sample) (Safety
- CT-11.3.2 Incidence of Potentially Clinically Relevant Abnormalities in Vital Signs (Safety Sample)
- CT-11.3.3 Mean Change from Baseline in Vital Signs (Safety Sample)
- CT-12.1.1 Criteria for Potentially Clinically Relevant Abnormalities in ECG Evaluations
- CT-12.1.2 ECG Diagnosis Mapping for Potentially Clinically Relevant Electrocardiogram Abnormalities
- CT-12.2.1 Listing of Potentially Clinically Relevant Abnormalities in ECG Evaluations During Phase B (Safety Sample)
- CT-12.2.2 Incidence of Potentially Clinically Relevant Changes in ECG Evaluations During Phase B (Safety Sample)
- CT-12.2.3 Mean Change in Electrocardiogram Results During Phase B (Safety Sample)
- CT-12.3.1 Listing of Categorical Changes in QT/QTc During Phase B (Safety Sample)
- CT-12.3.2 Incidence of Categorical Changes in QT/QTc During Phase B (Safety Sample)
- CT-13.1 Summary of Mean Change from Baseline (Day 0) to Phase B by Study Week in Simpson-Angus Scale (SAS) Total Score (Safety Sample)
- CT-13.2 Summary of Mean Change from Baseline (Day 0) to Phase B by Study Week in Abnormal Involuntary Movement Scale (AIMS) Total Score and Item Scores 8, 9 and 10 (Safety Sample)


50

- CT-13.3.1 Summary of Mean Change from Baseline (Day 0) to Phase B by Study Week in Barnes Akathisia Rating Scale (BARS) Global Clinical Assessment of Akathisia (Safety Sample)
- CT-13.3.2 Incidence of Barnes Akathisia Rating Scale (BARS) Global Clinical Assessment of Akathisia During Phase B (Safety Sample)
- CT-14.1.1 Columbia-Suicide Severity Rating Scale(C-SSRS) During Phase B, Suicidality (Safety Sample)
- CT-14.1.2 Columbia-Suicide Severity Rating Scale(C-SSRS) During Phase B, Suicidal Behavior by Type (Safety Sample)
- CT-14.1.3 Columbia-Suicide Severity Rating Scale(C-SSRS) During Phase B, Suicidal Ideation by Type (Safety Sample)
- CT-14.1.4 Columbia-Suicide Severity Rating Scale(C-SSRS) During Phase B, Treatment Emergent Suicidal Behavior and Ideation (Safety Sample)
- CT-14.1.5 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Treatment Emergent Suicidal Ideation During Phase B (Safety Sample)
- CT-14.1.6 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Treatment Emergent Suicidal Behavior During Phase B (Safety Sample)
- CT-14.1.7 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Treatment Emergent Serious Suicidal Ideation During Phase B (Safety Sample)
- CT-14.1.8 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Worsening Suicidal Ideation During Phase B (Safety Sample)
- CT-14.2.1 Columbia-Suicide Severity Rating Scale(C-SSRS) Suicidality (Safety Sample)
- CT-14.2.2 Columbia-Suicide Severity Rating Scale(C-SSRS) , Suicidal Behavior by Type (Safety Sample)
- CT-14.2.3 Columbia-Suicide Severity Rating Scale(C-SSRS) Suicidal Ideation by Type (Safety Sample)
- CT-14.2.4 Columbia-Suicide Severity Rating Scale(C-SSRS)

  Behavior and Ideation (Safety Sample)

  Treatment Emergent Suicidal
- CT-14.2.5 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Treatment Emergent Suicidal Ideation (Safety Sample)
- CT-14.2.6 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Treatment Emergent Suicidal Behavior (Safety Sample)
- CT-14.2.7 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Treatment Emergent Serious Suicidal Ideation (Safety Sample)
- CT-14.2.8 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Worsening Suicidal Ideation (Safety Sample)
- CT-15.1.1 Summary of Mean Change Weight (kg) (Safety Sample) to Phase B by Study Week in Body
- CT-15.1.2 Summary of Proportion of Patients with Potentially Clinically Relevant Weight Gain or Weight Loss During Phase B (Safety Sample)
- CT-15.2 Summary of Mean Change to Phase B by Study Week in Waist Circumference (cm) (Safety Sample)
- CT-15.3 Summary of Mean Change (Safety Sample) to Phase B by Study Week in BMI (kg/m2)




# This page is a manifestation of an electronically captured signature

# SIGNATURE PAGE

Document Name: 331-201-00061\_Statistical\_Analysis\_Plan\_Final

Document Number: 1000021467

**Document Version: 3.0** 

| Signed by | Meaning of Signature | Server Date (dd-MMM- yyyyy hh:min) - UTC timezone |
|---|---|---|
| | Clinical Approval | 11-Nov-2018<br>22:04:23 |
| | Biostatistics Approval | 08-Nov-2018<br>22:07:22 |

BREXPIPRAZOLE 1 OF 13
PROTOCOL 331-201-00061

| | | | Adju | sted | Mean | Change | | STAT-1.1 in CAPS-5 Line Items - MMRM (Intent to Treat Sample) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CAPS<br>Line Items | | | ERT <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | | X²<br>LSMean<br>Change¹ | N | SER<br>MEAN<br>Base | T <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
| CAPSW-INTRUSIVE<br>MEMORIES<br>SEVERITY | 77 2 | 2.22 | -1.25 | 69 | 2.03 | -1.03 | 75 | 2.16 | -0.71 | 78 | 2.00 | -0.99 | BREX+SERT VS PLACEBO | -0.26 | 0.2237 | -0.20 |
| SEVERITY | | | | | | | | | | | | | BREX+SERT VS SERT | -0.54 | 0.0137 | -0.40 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.23 | 0.3141 | -0.17 |
| | | | | | | | | | | | | | BREX VS PLACEBO | -0.03 | 0.8871 | -0.02 |
| | | | | | | | | | | | | | SERT VS PLACEBO | 0.28 | 0.1936 | 0.21 |
| CAPSW-DISTRESSI<br>NG DREAMS<br>SEVERITY | 77 | 1.19 | -0.64 | 69 | 1.42 | -0.60 | 75 | 1.63 | -0.48 | 78 | 1.38 | -0.57 | BREX+SERT VS PLACEBO | -0.07 | 0.7364 | -0.05 |
| SEVERIII | | | | | | | | | | | | | BREX+SERT VS SERT | -0.15 | 0.4517 | -0.12 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.03 | 0.8745 | -0.03 |
| | | | | | | | | | | | | | BREX VS PLACEBO | -0.03 | 0.8738 | -0.03 |
| | | | | | | | | | | | | | SERT VS PLACEBO | 0.09 | 0.6670 | 0.07 |
| CAPSW-DISSOCIAT<br>IVE REACTIONS<br>SEVERITY | 77 ( | 0.81 | -0.62 | 69 | 0.67 | -0.38 | 75 | 0.80 | -0.29 | 78 | 0.82 | -0.48 | BREX+SERT VS PLACEBO | -0.14 | 0.3462 | -0.15 |
| SEVERITI | | | | | | | | | | | | | BREX+SERT VS SERT | -0.33 | 0.0335 | -0.35 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.24 | 0.1331 | -0.25 |
| | | | | | | | | | | | | | BREX VS PLACEBO | 0.10 | 0.5279 | 0.10 |
| | | | | | | | | | | | | | VO I DITOUDO | 0.10 | 0.52/5 | 0.10 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

SERT VS PLACEBO

0.19

0.2205

0.20

FILE: caps\_itema.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.1 FINAL

CAPSW-AVOID MEM THGHTS FEELNGS SEVERITY

-0.52

BREX+SERT VS SERT

0.0162 -0.39

BREXPIPRAZOLE 2 OF 13

| | Adjust | ced Mean Change | (Intent to T | in CAPS-5 Lingreat Sample) | e Items - M | MRM | | |
|---|---|---|---|---|---|---|---|---|
| CAPS<br>Line Items | BREX+SERT²<br>MEAN LSMean<br>N Base Change¹ | BREX <sup>2</sup><br>MEAN LSMean<br>N Base Change <sup>1</sup> | SERT <sup>2</sup><br>MEAN LSMean<br>N Base Change <sup>1</sup> | PLACEBO<br>MEAN LSMean<br>N Base Change <sup>1</sup> | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
| CAPSW-CUED PSYCLOGICAL DISTRESS SEVERITY | 77 2.17 -1.14 | 69 1.90 -0.98 | 75 2.15 -0.84 | 78 2.17 -0.86 | BREX+SERT VS PLACEBO | -0.29 | 0.1627 | -0.23 |
| SEVERTT | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.30<br>-0.16<br>-0.13<br>0.02 | 0.1494<br>0.4608<br>0.5654<br>0.9397 | -0.23<br>-0.12<br>-0.10<br>0.01 |
| CAPSW-CUED PSYCLOGICAL REACTION SEVERITY | 77 2.00 -1.26 | 69 1.84 -1.16 | 75 2.07 -0.54 | 78 2.05 -0.62 | BREX+SERT VS PLACEBO | -0.64 | 0.0021 | -0.50 |
| | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.72<br>-0.10<br>-0.55<br>0.08 | 0.0007<br>0.6630<br>0.0125<br>0.7018 | -0.56<br>-0.07<br>-0.42<br>0.06 |

STAT-1.1

77 2.38 -1.17 69 2.12 -0.70 75 2.41 -0.65 78 2.33 -0.86 BREX+SERT VS PLACEBO -0.31 0.1417 -0.24

FILE: caps\_itema.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.1 FINAL

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

BREXPIPRAZOLE 3 OF 13

| | Adjusted Mean Change in CAPS-5 Line Items - MMRM (Intent to Treat Sample) | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| CAPS<br>Line Items | BREX+SERT <sup>2</sup><br>MEAN LSMean<br>N Base Change <sup>1</sup> | BREX <sup>2</sup><br>MEAN LSMean<br>N Base Change <sup>1</sup> | SERT <sup>2</sup><br>MEAN LSMean<br>N Base Change <sup>1</sup> | PLACEBO<br>MEAN LSMean<br>N Base Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
| CAPSW-AVOID<br>MEM THGHTS<br>FEELNGS<br>SEVERITY | | | | | BREX+SERT VS BREX | -0.47 | 0.0377 | -0.35 |
| | | | | | BREX VS PLACEBO<br>SERT VS PLACEBO | 0.16<br>0.21 | 0.4737<br>0.3233 | 0.12<br>0.16 |
| CAPSW-AVOID<br>EXTERNL<br>REMINDRS | 77 2.13 -0.95 | 69 2.03 -0.71 | 75 2.27 -0.65 | 78 2.22 -0.75 | BREX+SERT VS PLACEBO | -0.20 | 0.3393 | -0.15 |
| SEVERITY | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.30<br>-0.24<br>0.04<br>0.10 | 0.1556<br>0.2772<br>0.8505<br>0.6244 | -0.23<br>-0.18<br>0.03<br>0.08 |
| CAPSW-INABLTY RECAL ASPCT | 77 0.71 -0.25 | 69 0.78 -0.21 | 75 0.55 -0.17 | 78 0.55 -0.25 | BREX+SERT VS PLACEBO | -0.00 | 0.9956 | -0.00 |
| EVNT SEVERITY | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.08<br>-0.04<br>0.04<br>0.07 | 0.5116<br>0.7358<br>0.7377<br>0.5087 | -0.11<br>-0.06<br>0.06<br>0.11 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itema.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.1 FINAL

EXPTNS SEVERITY

CAPSW-DIST

COGTNS LEADNG

-0.22 0.2521

-0.30 0.1285

0.0193

0.1639 -0.22

0.8469

-0.48

-0.04

-0.19

-0.39

-0.03

-0.25

BREXPIPRAZOLE 4 OF 13

| | Adjusted | Mean Change | (Intent to Tre | in CAPS-5 Lin<br>at Sample) | e Items - M | - MMRM | |
|---|---|---|---|---|---|---|---|
| CAPS<br>Line Items | BREX+SERT <sup>2</sup><br>MEAN LSMean<br>N Base Change <sup>1</sup> N | BREX <sup>2</sup> MEAN LSMean Base Change <sup>1</sup> | SERT <sup>2</sup><br>MEAN LSMean<br>N Base Change <sup>1</sup> | PLACEBO<br>MEAN LSMean<br>N Base Change <sup>1</sup> | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT 1 P-V | COHEN'S D<br>EFFECT<br>VALUE¹ SIZE |
| CAPSW-EXGGRTD<br>NEG BELIFS | 77 2.30 -1.02 6 | 9 2.13 -0.54 | 75 2.27 -0.79 | 78 2.05 -0.50 | BREX+SERT VS PLACEBO | -0.52 0 | .0074 -0.43 |

BREX+SERT VS SERT

BREX+SERT VS BREX

BREX VS PLACEBO SERT VS PLACEBO

STAT-1 1

| BLAME SEVERITY | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | | BREX+SERT VS SERT | -0.17 | 0.3946 | -0.14 |
| | | | | | BREX+SERT VS BREX | -0.07 | 0.7477 | -0.05 |
| | | | | | BREX VS PLACEBO | -0.21 | 0.3088 | -0.17 |
| | | | | | SERT VS PLACEBO | -0.11 | 0.5918 | -0.09 |
| CAPSW-PRSISTNT<br>NEG EMOTNL | 77 2.09 -0.99 | 69 2.23 -0.84 | 75 2.28 -0.86 | 78 2.10 -0.53 | BREX+SERT VS PLACEBO | -0.46 | 0.0183 | -0.38 |
| STATE SEVERITY | | | | | BREX+SERT VS SERT | -0.13 | 0.5152 | -0.11 |
| | | | | | BREX+SERT VS BREX | -0.14 | 0.4877 | -0.12 |
| | | | | | BREX VS PLACEBO | -0.32 | 0.1222 | -0.26 |
| | | | | | SERT VS PLACEBO | -0.33 | 0.0918 | -0.27 |

77 1.81 -0.86 69 1.41 -0.79 75 1.89 -0.69 78 1.38 -0.59 BREX+SERT VS PLACEBO -0.27

FILE: caps\_itema.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.1 FINAL

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

BREXPIPRAZOLE 5 OF 13

| | | | Adjust: | ed Me | ean Ch | STAT-1.1 In Change in CAPS-5 Line Items - MMRM (Intent to Treat Sample) | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CAPS<br>Line Items | | | ERT <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | | X <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | | T²<br>LSMean<br>Change¹ | N | | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
| CAPSW-DIMISHD<br>INTRST<br>ACTVTIES<br>SEVERITY | 77 2 | 2.01 | -1.09 | 69 | 1.97 | -0.54 | 75 | 2.04 | -0.55 | 78 | 2.05 | -0.62 | BREX+SERT VS PLACEBO | -0.48 | 0.0195 | -0.38 |
| OD V DICE I I | | | | | | | | | | | | | BREX+SERT VS SERT | -0.54 | 0.0087 | -0.43 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.55 | 0.0112 | -0.42 |
| | | | | | | | | | | | | | BREX VS PLACEBO | 0.08 | 0.7236 | 0.06 |
| | | | | | | | | | | | | | SERT VS PLACEBO | 0.07 | 0.7334 | 0.06 |
| CAPSW-DETACHMNT<br>ESTRNGMNT<br>OTHRS SEVERITY | 77 2 | 2.30 | -0.87 | 69 | 2.00 | -0.73 | 75 | 2.25 | -0.63 | 78 | 2.35 | -0.46 | BREX+SERT VS PLACEBO | -0.41 | 0.0519 | -0.31 |
| JINKO SEVEKIII | | | | | | | | | | | | | BREX+SERT VS SERT | -0.25 | 0.2515 | -0.19 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.15 | 0.5203 | -0.11 |
| | | | | | | | | | | | | | BREX VS PLACEBO | -0.27 | 0.2344 | -0.20 |
| | | | | | | | | | | | | | SERT VS PLACEBO | -0.17 | 0.4383 | -0.13 |
| CAPSW-PRSISTNT<br>INAB EXP<br>POSTVE SEVERITY | 77 | 1.83 | -0.91 | 69 | 1.62 | -0.42 | 75 | 1.80 | -0.54 | 78 | 1.78 | -0.38 | BREX+SERT VS PLACEBO | -0.53 | 0.0068 | -0.44 |
| FOSIVE SEVERIII | | | | | | | | | | | | | BREX+SERT VS SERT | -0.38 | 0.0606 | -0.31 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.49 | 0.0185 | -0.39 |
| | | | | | | | | | | | | | BREX VS PLACEBO | -0.04 | 0.8497 | -0.03 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itema.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.1 FINAL

BREXPIPRAZOLE 6 OF 13

| | | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|
| | SERT VS PLACEBO | -0.16 | 0.4225 | -0.13 |
| 78 1.53 -0.37 | BREX+SERT VS PLACEBO | -0.13 | 0.4921 | -0.11 |
| | BREX+SERT VS BREX<br>BREX VS PLACEBO | -0.00<br>0.09<br>-0.22<br>-0.13 | 0.9896<br>0.6777<br>0.2837<br>0.5028 | -0.00<br>0.07<br>-0.18<br>-0.11 |
| 78 0.32 -0.10 | BREX+SERT VS PLACEBO | -0.02 | 0.8469 | -0.03 |
| | BREX+SERT VS BREX<br>BREX VS PLACEBO | 0.06<br>-0.00<br>-0.01<br>-0.07 | 0.5354<br>0.9591<br>0.8960<br>0.4115 | 0.10<br>-0.01<br>-0.02<br>-0.13 |
| | | -0.42<br>-0.11 | 0.0237 | -0.37<br>-0.10 |
| _ | MEAN LSMean N Base Change 78 1.53 -0.37 78 0.32 -0.10 | MEAN LSMean TREATMENT COMPARISON SERT VS PLACEBO REX+SERT VS PLACEBO BREX+SERT VS SERT BREX+SERT VS BREX BREX VS PLACEBO SERT VS PLACEBO BREX+SERT VS BREX BREX VS PLACEBO BREX+SERT VS PLACEBO SERT VS PLACEBO BREX+SERT VS SERT BREX+SERT VS BREX BREX VS PLACEBO SERT VS PLACEBO SERT VS PLACEBO SERT VS PLACEBO SERT VS PLACEBO | MEAN LSMean TREATMENT COMPARISON EFFECT | MEAN LSMean TREATMENT TREATMENT EFFECT P-VALUE |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itema.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.1 FINAL

0.6425

-0.07

BREXPIPRAZOLE 7 OF 13

CAPSW-EXAGGERAT 77 1.30 -0.49 69 1.36 -0.46 75 1.47 -0.47 78 1.23 -0.41 BREX+SERT VS PLACEBO -0.09

| | | | | | | | | (In | tent to T | reat | : Sampl | .e)<br> | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CAPS<br>Line Items | N | BREX+S<br>MEAN<br>Base | LSMean | N | BRE<br>MEAN<br>Base | LSMean | N | SER<br>MEAN<br>Base | T²<br>LSMean<br>Change¹ | N | PLAC<br>MEAN<br>Base | LSMean | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
| CAPSW-HYPERVIGI | | | | | | | | | | | | | BREX+SERT VS BREX | -0.41 | 0.0382 | -0.35 |
| | | | | | | | | | | | | | BREX VS PLACEBO<br>SERT VS PLACEBO | -0.01<br>-0.31 | 0.9537<br>0.0996 | -0.01<br>-0.27 |

| | | | | | | | | | | | | | BREX+SERT VS SERT | -0.02 | 0.9011 | -0.02 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.03 | 0.8656 | -0.03 |
| | | | | | | | | | | | | | BREX VS PLACEBO | -0.05 | 0.7881 | -0.04 |
| | | | | | | | | | | | | | SERT VS PLACEBO | -0.06 | 0.7373 | -0.05 |
| CAPSW-PRBLMS | 77 | 2.00 | -0.73 | 69 | 2.13 | -0.58 | 75 | 1.85 | -0.61 | 78 | 2.01 | -0.55 | BREX+SERT VS PLACEBO | -0.18 | 0.3372 | -0.15 |
| WTH | | | | | | | | | | | | | | | | |
| CONCENTED A RECON | | | | | | | | | | | | | | | | |

CONCENTRATION SEVERITY

D STRTLE RESPNSE SEVERITY

BREX+SERT VS SERT -0.12 0.5197 -0.10
BREX+SERT VS BREX -0.14 0.4690 -0.12
BREX VS PLACEBO -0.03 0.8586 -0.03
SERT VS PLACEBO -0.06 0.7634 -0.05

in CAPS-5 Line Items

FILE: caps\_itema.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.1 FINAL

Adjusted Mean Change

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

BREXPIPRAZOLE 8 OF 13

Adjusted Mean Change In CAPS-5 Line Items — MMRM (Intent to Treat Sample)

| CAPS<br>Line Items | | BREX+S<br>MEAN<br>Base | LSMean<br>Change¹ | | Base | X <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | SER<br>MEAN<br>Base | T <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT 1 | P-VALUE¹ | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CAPSW-SLEEP<br>DISTURBANCE<br>SEVERITY | 77 | 2.18 | -0.69 | 69 | 2.30 | -0.84 | 75 | 2.63 | -0.34 | 78 | 2.55 | -0.33 | BREX+SERT VS PLACEBO | -0.37 | 0.0850 | -0.28 |
| | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.36<br>0.15<br>-0.51<br>-0.01 | 0.1024<br>0.5147<br>0.0212<br>0.9560 | -0.27<br>0.11<br>-0.38<br>-0.01 |
| CAPSW-SUBJECTIV<br>E DISTRESS<br>SEVERITY | 77 | 2.48 | -0.89 | 69 | 2.38 | -0.59 | 75 | 2.51 | -0.59 | 78 | 2.33 | -0.60 | BREX+SERT VS PLACEBO | -0.29 | 0.0306 | -0.35 |
| SEVERITY | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.30<br>-0.30<br>0.01<br>0.02 | 0.0242<br>0.0356<br>0.9468<br>0.9004 | -0.37<br>-0.35<br>0.01<br>0.02 |
| CAPSW-IMPAIRMNT<br>SOCIAL FUNCTNG | 77 | 2.49 | -1.19 | 69 | 2.22 | -0.81 | 75 | 2.45 | -0.81 | 78 | 2.37 | -0.61 | BREX+SERT VS PLACEBO | -0.58 | 0.0003 | -0.58 |
| SEVERITY | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.38<br>-0.37<br>-0.21<br>-0.20 | 0.0213<br>0.0299<br>0.2177<br>0.2102 | -0.38<br>-0.36<br>-0.20<br>-0.20 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itema.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.1 FINAL

BREXPIPRAZOLE 9 OF 13

| STAT-1.1 | <u> </u> |
|----------------------|-----------------------------|
| Adjusted Mean Change | in CAPS-5 Line Items - MMRM |
| (Intent to Treat | t Sample) |

| CAPS<br>Line Items | | BREX+S<br>MEAN<br>Base | ERT <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | BRE<br>MEAN<br>Base | X <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | SER<br>MEAN<br>Base | T <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE 1 | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CAPSW-IMPAIRMNT<br>OCCUP FUNCTNG<br>SEVERITY | 77 | 2.22 | -0.82 | 69 | 1.96 | -0.64 | 75 | 2.21 | -0.69 | 78 | 2.18 | -0.54 | BREX+SERT VS PLACEBO | -0.28 | 0.1021 | -0.26 |
| | | | | | | | | | | | | | BREX+SERT VS SERT | -0.13 | 0.4576 | -0.12 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.19 | 0.3116 | -0.17 |
| | | | | | | | | | | | | | BREX VS PLACEBO | -0.10 | 0.5921 | -0.09 |
| | | | | | | | | | | | | | SERT VS PLACEBO | -0.15 | 0.3823 | -0.14 |
| CAPSW-SEVERITY<br>SUBTOTAL G | 77 | 7.19 | -2.91 | 69 | 6.55 | -1.95 | 75 | 7.17 | -2.09 | 78 | 6.88 | -1.70 | BREX+SERT VS PLACEBO | -1.21 | 0.0015 | -0.52 |
| SOBIOTAL G | | | | | | | | | | | | | BREX+SERT VS SERT | -0.82 | 0.0336 | -0.35 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.96 | 0.0171 | -0.40 |
| | | | | | | | | | | | | | BREX VS PLACEBO | -0.25 | 0.5240 | -0.11 |
| | | | | | | | | | | | | | SERT VS PLACEBO | -0.39 | 0.3037 | -0.17 |
| CAPSW-GLOBAL<br>VALIDITY | 77 | 0.22 | 0.03 | 69 | 0.16 | -0.01 | 75 | 0.17 | -0.08 | 78 | 0.09 | 0.00 | BREX+SERT VS PLACEBO | 0.02 | 0.6452 | 0.07 |
| VALIDITY | | | | | | | | | | | | | BREX+SERT VS SERT | 0.11 | 0.0328 | 0.35 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | 0.04 | 0.4345 | 0.13 |
| | | | | | | | | | | | | | BREX VS PLACEBO | -0.02 | 0.7219 | -0.06 |
| | | | | | | | | | | | | | SERT VS PLACEBO | -0.08 | 0.0850 | -0.28 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itema.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.1 FINAL

BREXPIPRAZOLE 10 OF 13 PROTOCOL 331-201-00061

| Adjusted Mean Change | in CAPS-5 Line Items - MMRM (Intent to Treat Sample) |
|----------------------|------------------------------------------------------|

| CAPS<br>Line Items | | BREX+S<br>MEAN<br>Base | ERT <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | BRE<br>MEAN<br>Base | X <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | SER<br>MEAN<br>Base | T <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CAPSW-GLOBAL<br>SEVERITY | 77 | 2.55 | -0.87 | 69 | 2.41 | -0.69 | 75 | 2.53 | -0.57 | 78 | 2.38 | -0.58 | BREX+SERT VS PLACEBO | -0.29 | 0.0481 | -0.32 |
| DEVENTI | | | | | | | | | | | | | BREX+SERT VS SERT | -0.30 | 0.0417 | -0.33 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.18 | 0.2402 | -0.20 |
| | | | | | | | | | | | | | BREX VS PLACEBO | -0.11 | 0.4809 | -0.12 |
| | | | | | | | | | | | | | SERT VS PLACEBO | 0.01 | 0.9241 | 0.02 |
| CAPSW-GLOBAL<br>IMPROVEMENT | 77 | 3.42 | -1.30 | 69 | 3.25 | -0.99 | 75 | 3.40 | -0.80 | 78 | 3.33 | -0.92 | BREX+SERT VS PLACEBO | -0.38 | 0.0416 | -0.33 |
| 1111110121111 | | | | | | | | | | | | | BREX+SERT VS SERT | -0.50 | 0.0094 | -0.42 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.31 | 0.1261 | -0.25 |
| | | | | | | | | | | | | | BREX VS PLACEBO | -0.08 | 0.7004 | -0.06 |
| | | | | | | | | | | | | | SERT VS PLACEBO | 0.12 | 0.5373 | 0.10 |
| CAPSW-DEPERSONA<br>LIZATION<br>SEVERITY | 77 | 0.27 | -0.27 | 69 | 0.29 | -0.14 | 75 | 0.28 | -0.24 | 78 | 0.24 | -0.22 | BREX+SERT VS PLACEBO | -0.05 | 0.4467 | -0.12 |
| SEVERIII | | | | | | | | | | | | | BREX+SERT VS SERT | -0.03 | 0.6785 | -0.07 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.13 | 0.0561 | -0.32 |
| | | | | | | | | | | | | | BREX VS PLACEBO | 0.08 | 0.2217 | 0.20 |
| | | | | | | | | | | | | | SERT VS PLACEBO | -0.02 | 0.7365 | -0.05 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itema.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.1 FINAL

SUBSCALE B TOTAL SEVERITY

SCORE

-2.06 0.0058

-0.76 0.3235

0.67

-0.63 0.4075

0.3560

-0.45

-0.16

-0.14

0.15

BREXPIPRAZOLE 11 OF 13 PROTOCOL 331-201-00061

| | | | | | | | | (In | tent to T | reat | | e) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CAPS<br>Line Items | | BREX+S<br>MEAN<br>Base | ERT <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | | | | N | SER<br>MEAN<br>Base | T²<br>LSMean<br>Change¹ | N<br> | | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
| CAPSW-DEREALIZA TION SEVERITY | 77 | 0.29 | -0.23 | 69 | 0.29 | 0.12 | 75 | 0.21 | -0.13 | 78 | 0.23 | -0.23 | BREX+SERT VS PLACEBO | 0.00 | 0.9549 | 0.01 |
| | | | | | | | | | | | | | BREX+SERT VS SERT | -0.10 | 0.1687 | -0.22 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.11 | 0.1528 | -0.24 |
| | | | | | | | | | | | | | BREX VS PLACEBO | 0.12 | 0.1337 | 0.25 |
| | | | | | | | | | | | | | SERT VS PLACEBO | 0.11 | 0.1472 | 0.24 |
| CAPSW-SEVERITY<br>SUBTOTAL DISS | 77 | 0.56 | -0.50 | 69 | 0.58 | -0.26 | 75 | 0.49 | -0.37 | 78 | 0.47 | -0.45 | BREX+SERT VS PLACEBO | -0.05 | 0.6680 | -0.07 |
| | | | | | | | | | | | | | BREX+SERT VS SERT | -0.13 | 0.2612 | -0.18 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.24 | 0.0416 | -0.34 |
| | | | | | | | | | | | | | BREX VS PLACEBO | 0.19 | 0.0954 | 0.28 |
| | | | | | | | | | | | | | SERT VS PLACEBO | 0.08 | 0.4740 | 0.12 |
| CAPS-5 | 77 | 8.39 | -4.93 | 69 | 7.86 | -4.17 | 75 | 8.80 | -2.87 | 78 | 8.42 | -3.55 | BREX+SERT VS PLACEBO | -1.38 | 0.0564 | -0.31 |

in CAPS-5 Line Items - MMRM

BREX+SERT VS SERT

BREX+SERT VS BREX

BREX VS PLACEBO

SERT VS PLACEBO

FILE: caps\_itema.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.1 FINAL

Adjusted Mean Change

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

BREXPIPRAZOLE 12 OF 13 PROTOCOL 331-201-00061

| | | justed Mean Change | | in CAPS-5 Lindireat Sample) | e Items – M | MRM | | |
|---|---|---|---|---|---|---|---|---|
| CAPS<br>Line Items | BREX+SERT <sup>2</sup><br>MEAN LSMe<br>N Base Chan | | SERT <sup>2</sup><br>MEAN LSMean<br>N Base Change <sup>1</sup> | PLACEBO<br>MEAN LSMean<br>N Base Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE¹ | COHEN'S D<br>EFFECT<br>SIZE |
| CAPS-5<br>SUBSCALE C<br>TOTAL SEVERITY<br>SCORE | 77 4.51 -2. | 13 69 4.14 -1.37 | 75 4.68 -1.33 | 78 4.55 -1.60 | BREX+SERT VS PLACEBO | -0.52 | 0.1376 | -0.24 |
| | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.79<br>-0.76<br>0.23<br>0.27 | 0.0273<br>0.0440<br>0.5296<br>0.4408 | -0.36<br>-0.34<br>0.10<br>0.12 |
| CAPS-5<br>SUBSCALE D<br>TOTAL SEVERITY<br>SCORE | 77 13.05 -6. | 12 69 12.14 -3.99 | 75 13.08 -4.30 | 78 12.27 -3.32 | BREX+SERT VS PLACEBO | -2.79 | 0.0007 | -0.55 |
| COM | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -1.82<br>-2.13<br>-0.67<br>-0.98 | 0.0285<br>0.0137<br>0.4296<br>0.2317 | -0.36<br>-0.41<br>-0.13<br>-0.19 |
| CAPS-5<br>SUBSCALE E<br>TOTAL SEVERITY<br>SCORE | 77 9.78 -3. | 33 69 9.74 -2.92 | 75 9.95 -2.77 | 78 9.90 -2.14 | BREX+SERT VS PLACEBO | -1.19 | 0.0366 | -0.34 |
| SCORE | | | | | BREX+SERT VS SERT | -0.56 | 0.3325 | -0.16 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itema.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.1 FINAL

BREXPIPRAZOLE 13 OF 13 PROTOCOL 331-201-00061

| | Adjusted Mean | Change | (Intent to Treat | in CAPS-5 Line<br>Sample) | Items | - MMRM | |
|---|---|---|---|---|---|---|---|
| BRE | X+SERT <sup>2</sup> I | SREX 2 | SERT2 | PLACEBO | | ESTIMATED | COHEN'S |

STAT-1 1

| | BREX | +SERT 2 | BRE | EX 2 | SE: | RT² | PLA | CEBO | | ESTIMATED | | COHEN's D |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CAPS | MEA | N LSMean | MEAN | LSMean | MEAN | LSMean | MEAN | I LSMean | TREATMENT | TREATMENT | | EFFECT |
| Line Items | N Bas | e Change¹ | N Base | Change 1 | N Base | Change 1 | N Base | e Change¹ | COMPARISON | EFFECT 1 | P-VALUE 1 | SIZE |
| CAPS-5<br>SUBSCALE E<br>TOTAL SEVERITY<br>SCORE | | | | | | | | | BREX+SERT VS BREX | -0.40 | 0.5043 | -0.11 |
| SCORE | | | | | | | | | BREX VS PLACEBO<br>SERT VS PLACEBO | -0.79<br>-0.63 | 0.1857<br>0.2708 | -0.22<br>-0.18 |
| CAPS-5 TOTAL<br>SEVERITY SCORE | 77 35. | 73 -16.4 | 69 33.88 | 3 -12.2 | 75 36.5 | 1 -11.4 | 78 35.1 | 4 -10.5 | BREX+SERT VS PLACEBO | -5.99 | 0.0021 | -0.50 |
| | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -5.08<br>-4.24<br>-1.74<br>-0.91 | 0.0106<br>0.0384<br>0.3868<br>0.6399 | -0.42<br>-0.35<br>-0.14<br>-0.08 |

FILE: caps\_itema.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.1 FINAL

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

BREXPIPRAZOLE 1 OF 5

STAT-1.2
Adjusted Mean Change from Baeline (Day 0) in SOTS Line Items at Week 12 - MMRM (Intent to Treat Sample)

| SOTS<br>Line Items | | BREX+S<br>MEAN<br>Base | ERT <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N<br> | | X <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | SER<br>MEAN<br>Base | T <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N<br> | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S I<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOTS-RE-EXPERIE | 74 | 4.64 | -2.34 | 67 | 4.61 | -1.71 | 70 | 4.63 | -1.93 | 75 | 4.44 | -1.84 | BREX+SERT VS PLACEBO | -0.50 | 0.0743 | -0.29 |
| | | | | | | | | | | | | | BREX+SERT VS SERT | -0.41 | 0.1485 | -0.24 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.63 | 0.0344 | -0.36 |
| | | | | | | | | | | | | | BREX VS PLACEBO | 0.13 | 0.6549 | 0.08 |
| | | | | | | | | | | | | | SERT VS PLACEBO | -0.09 | 0.7513 | -0.05 |
| SOTS-HYPERAROUS | 74 | 4.53 | -1.15 | 67 | 4.45 | -1.08 | 70 | 4.59 | -1.65 | 75 | 4.48 | -1.04 | BREX+SERT VS PLACEBO | -0.11 | 0.6565 | -0.07 |
| AL | | | | | | | | | | | | | BREX+SERT VS SERT | 0.50 | 0.0601 | 0.32 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.07 | 0.7903 | -0.04 |
| | | | | | | | | | | | | | BREX VS PLACEBO | -0.04 | 0.8779 | -0.03 |
| | | | | | | | | | | | | | SERT VS PLACEBO | -0.61 | 0.0196 | -0.39 |
| SOTS-AFFECTIVE<br>DYSREGULATION | 74 | 3.46 | -1.58 | 67 | 3.79 | -1.49 | 70 | 3.81 | -1.82 | 75 | 3.45 | -1.50 | BREX+SERT VS PLACEBO | -0.08 | 0.7494 | -0.05 |
| DISKEGULATION | | | | | | | | | | | | | BREX+SERT VS SERT | 0.24 | 0.3563 | 0.15 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.09 | 0.7310 | -0.06 |
| | | | | | | | | | | | | | BREX VS PLACEBO | 0.01 | 0.9641 | 0.01 |
| | | | | | | | | | | | | | SERT VS PLACEBO | -0.32 | 0.2122 | -0.21 |
| SOTS-IMPULSIVIT<br>Y | 74 | 1.95 | -0.48 | 67 | 1.69 | -0.53 | 70 | 2.04 | -0.60 | 75 | 2.03 | -0.59 | BREX+SERT VS PLACEBO | 0.11 | 0.4865 | 0.11 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itemb.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.2 FINAL

BREXPIPRAZOLE 2 OF 5

 $$\tt STAT-1.2$$  Adjusted Mean Change from Baeline (Day 0) in SOTS Line Items at Week 12 - MMRM (Intent to Treat Sample)

| SOTS<br>Line Items | N | BREX+S<br>MEAN<br>Base | LSMean<br>Change¹ | | Base | LSMean<br>Change¹ | N<br> | Base | LSMean<br>Change¹ | N<br> | Base | LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE¹ | COHEN'S I<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOTS-IMPULSIVIT | | | | | | | | | | | | | BREX+SERT VS SERT | 0.13 | 0.4422 | 0.13 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | 0.05 | 0.7742 | 0.05 |
| | | | | | | | | | | | | | BREX VS PLACEBO | 0.06 | 0.7127 | 0.06 |
| | | | | | | | | | | | | | SERT VS PLACEBO | -0.01 | 0.9318 | -0.01 |
| SOTS-AVOIDANCE | 74 | 4.84 | -1.75 | 67 | 4.63 | -1.31 | 70 | 4.89 | -1.48 | 75 | 4.71 | -1.47 | BREX+SERT VS PLACEBO | -0.27 | 0.3319 | -0.16 |
| | | | | | | | | | | | | | BREX+SERT VS SERT | -0.27 | 0.3435 | -0.16 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.44 | 0.1441 | -0.25 |
| | | | | | | | | | | | | | BREX VS PLACEBO | 0.16 | 0.5762 | 0.09 |
| | | | | | | | | | | | | | SERT VS PLACEBO | -0.00 | 0.9956 | -0.00 |
| SOTS-NUMBING | 74 | 3.01 | -1.07 | 67 | 2.93 | -0.71 | 70 | 3.00 | -0.90 | 75 | 3.19 | -0.97 | BREX+SERT VS PLACEBO | -0.10 | 0.6892 | -0.07 |
| | | | | | | | | | | | | | BREX+SERT VS SERT | -0.18 | 0.4808 | -0.12 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.37 | 0.1658 | -0.23 |
| | | | | | | | | | | | | | BREX VS PLACEBO | 0.27 | 0.3069 | 0.17 |
| | | | | | | | | | | | | | SERT VS PLACEBO | 0.08 | 0.7529 | 0.05 |
| CONSCIOUSNESS | 74 | 2.08 | -0.75 | 67 | 2.27 | -0.68 | 70 | 1.70 | -0.55 | 75 | 2.01 | -0.40 | BREX+SERT VS PLACEBO | -0.35 | 0.0455 | -0.33 |
| DISSOCIATION | | | | | | | | | | | | | BREX+SERT VS SERT | -0.19 | 0.2806 | -0.18 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.06 | 0.7318 | -0.06 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itemb.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.2 FINAL

BREXPIPRAZOLE 3 OF 5

 $$\tt STAT-1.2$$  Adjusted Mean Change from Baeline (Day 0) in SOTS Line Items at Week 12 - MMRM (Intent to Treat Sample)

| SOTS<br>Line Items | | BREX+S<br>MEAN<br>Base | ERT <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | BRE<br>MEAN<br>Base | X <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | SER<br>MEAN<br>Base | T²<br>LSMean<br>Change¹ | N | | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOTS-ATTENTIN<br>CONSCIOUSNESS<br>DISSOCIATION | | | | | | | | | | | | | BREX VS PLACEBO | -0.29 | 0.1203 | -0.26 |
| | | | | | | | | | | | | | SERT VS PLACEBO | -0.16 | 0.3679 | -0.15 |
| SOTS-SELF<br>PERCEPTION | 74 | 3.93 | -1.69 | 67 | 4.01 | -1.51 | 70 | 4.04 | -1.49 | 75 | 3.91 | -1.63 | BREX+SERT VS PLACEBO | -0.06 | 0.8272 | -0.04 |
| | | | | | | | | | | | | | BREX+SERT VS SERT | -0.20 | 0.4447 | -0.13 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.17 | 0.5223 | -0.11 |
| | | | | | | | | | | | | | BREX VS PLACEBO | 0.12 | 0.6604 | 0.07 |
| | | | | | | | | | | | | | SERT VS PLACEBO | 0.14 | 0.5779 | 0.09 |
| SOTS-INTERPERSO<br>NAL RELATION | 74 | 4.66 | -1.62 | 67 | 4.54 | -1.49 | 70 | 4.61 | -1.77 | 75 | 4.64 | -1.22 | BREX+SERT VS PLACEBO | -0.40 | 0.1589 | -0.23 |
| | | | | | | | | | | | | | BREX+SERT VS SERT | 0.15 | 0.6021 | 0.09 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.13 | 0.6682 | -0.07 |
| | | | | | | | | | | | | | BREX VS PLACEBO | -0.27 | 0.3647 | -0.15 |
| | | | | | | | | | | | | | SERT VS PLACEBO | -0.55 | 0.0547 | -0.32 |
| SOTS-ALTERATION<br>S IN SEXUAL<br>RELATIONS | 74 | 2.88 | -1.05 | 67 | 2.97 | -0.91 | 70 | 2.91 | -0.74 | 75 | 2.39 | -1.04 | BREX+SERT VS PLACEBO | -0.01 | 0.9734 | -0.01 |
| | | | | | | | | | | | | | BREX+SERT VS SERT | -0.30 | 0.2684 | -0.19 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itemb.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.2 FINAL
BREXPIPRAZOLE 4 OF 5

 $$\tt STAT-1.2$$  Adjusted Mean Change from Baeline (Day 0) in SOTS Line Items at Week 12 - MMRM (Intent to Treat Sample)

| SOTS<br>Line Items | N | BREX+S<br>MEAN<br>Base | ERT <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | BRE<br>MEAN<br>Base | X <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | SER<br>MEAN<br>Base | T²<br>LSMean<br>Change¹ | N | PLACI<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOTS-ALTERATION<br>S IN SEXUAL<br>RELATIONS | | | | | | | | | | | | | BREX+SERT VS BREX | -0.14 | 0.6242 | -0.08 |
| RELATIONS | | | | | | | | | | | | | BREX VS PLACEBO<br>SERT VS PLACEBO | 0.13<br>0.29 | 0.6425<br>0.2805 | 0.08<br>0.18 |
| SOTS-SUSTAINING | 7 | 1 2.82 | -1.12 | 67 | 2.48 | -0.80 | 70 | 2.47 | -0.70 | 75 | 2.69 | -0.78 | BREX+SERT VS PLACEBO | -0.34 | 0.1243 | -0.25 |
| BELIEFS | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.43<br>-0.33<br>-0.01<br>0.09 | 0.0599<br>0.1657<br>0.9546<br>0.7017 | -0.32<br>-0.23<br>-0.01<br>0.06 |
| SOTS-SOMATIC | 7 | 1 2.03 | -0.60 | 67 | 1.81 | -0.60 | 70 | 1.86 | -0.52 | 75 | 1.71 | -0.31 | BREX+SERT VS PLACEBO | -0.29 | 0.0980 | -0.27 |
| DYSREGULATION | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.08<br>-0.00<br>-0.29<br>-0.21 | 0.6656<br>0.9965<br>0.1169<br>0.2265 | -0.07<br>-0.00<br>-0.26<br>-0.20 |
| SOTS TOTAL | 7 | 40.82 | -15.2 | 67 | 40.16 | -12.7 | 70 | 40.56 | -14.0 | 75 | 39.64 | -12.8 | BREX+SERT VS PLACEBO | -2.36 | 0.1481 | -0.24 |
| SCORE | | | | | | | | | | | | | BREX+SERT VS SERT | -1.15 | 0.4872 | -0.12 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itemb.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.2 FINAL

BREXPIPRAZOLE 5 OF 5 PROTOCOL 331-201-00061

STAT-1.2

Adjusted Mean Change from Baeline (Day 0) in SOTS Line Items at Week 12 - MMRM (Intent to Treat Sample)

| SOTS<br>Line Items | BREX+SERT <sup>2</sup><br>MEAN LSMea<br>N Base Chang | SERT <sup>2</sup><br>MEAN LSMean<br>N Base Change <sup>1</sup> | PLACEBO<br>MEAN LSMean<br>N Base Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|
| SOTS TOTAL<br>SCORE | | | | BREX+SERT VS BREX BREX VS PLACEBO SERT VS PLACEBO | -2.46<br>0.10<br>-1.21 | 0.1561<br>0.9554<br>0.4624 | -0.24<br>0.01<br>-0.12 |

1 MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itemb.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.2 FINAL

BREXPIPRAZOLE 1 OF 9

| <br>Adjusted Mean Change | STAT-1.3 in PCL-5 Line Items (Intent to Treat Sample) | - MMRM |
|---|---|---|
| <br> | | |

| PCL5 | BREX+SERT <sup>2</sup><br>MEAN LSMean<br>N Base Change <sup>1</sup> | BREX <sup>2</sup> MEAN LSMean N Base Change <sup>1</sup> | SERT <sup>2</sup> MEAN LSMean N Base Change <sup>1</sup> | PLACEBO<br>MEAN LSMean<br>N Base Change¹ | TREATMENT<br>COMPARISON | ESTIMATED TREATMENT EFFECT 1 P-VALU | COHEN'S D<br>EFFECT<br>E¹ SIZE |
|---|---|---|---|---|---|---|---|
| PCL5-REP DISTRB UNWNTD MEMRS STRESS EXP | 77 2.38 -1.16 | 69 2.26 -0.85 | 75 2.60 -0.85 | 78 2.21 -0.85 | BREX+SERT VS PLACEBO | -0.31 0.071 | 5 -0.29 |
| LAF | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.32 0.074<br>-0.31 0.092<br>-0.00 0.983<br>0.00 0.984 | -0.28<br>-0.00 |
| PCL5-REP<br>DISTRB DREAMS<br>STRESS EXP | 77 1.82 -0.89 | 69 2.12 -0.71 | 75 2.21 -0.69 | 78 1.82 -0.67 | BREX+SERT VS PLACEBO | -0.22 0.241 | 7 -0.19 |
| STRESS EXP | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.20 0.283<br>-0.18 0.358<br>-0.04 0.852<br>-0.01 0.944 | 8 -0.15<br>4 -0.03 |
| PCL5-SUDDN<br>FEELNG STRES | 77 1.55 -0.74 | 69 1.71 -0.69 | 75 1.61 -0.59 | 78 1.44 -0.84 | BREX+SERT VS PLACEBO | 0.10 0.548 | 6 0.10 |
| EXP HAPPN AGAIN | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO | -0.15 0.390<br>-0.04 0.812<br>0.15 0.417 | 5 -0.04 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itemc.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.3 FINAL

BREXPIPRAZOLE 2 OF 9 PROTOCOL 331-201-00061

Adjusted Mean Change in PCL-5 Line Items - MMRM (Intent to Treat Sample)

| PCL5<br>Line Items | N | BREX+S<br>MEAN<br>Base | LSMean | N | BRE<br>MEAN<br>Base | X <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | SER<br>MEAN<br>Base | T²<br>LSMean<br>Change¹ | N | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PCL5-SUDDN<br>FEELNG STRES<br>EXP HAPPN AGAIN | | | | | | | | | | | | | SERT VS PLACEBO | 0.25 | 0.1434 | 0.24 |
| PCL5-FEEL UPST<br>SMTHNG REMNDS<br>STRESS EXP | 7 | 7 2.66 | 5 -1.11 | 69 | 2.39 | -0.67 | 75 | 2.52 | -0.70 | 7 | 8 2.38 | -0.68 | BREX+SERT VS PLACEBO | -0.44 | 0.0214 | -0.37 |
| SINESS EXI | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.41<br>-0.44<br>0.01<br>-0.03 | 0.0331<br>0.0269<br>0.9676<br>0.8914 | -0.35<br>-0.37<br>0.01<br>-0.02 |
| PCL5-HAVNG<br>STRNG PHY<br>REACTNS STRESS | 7 | 7 2.39 | -1.06 | 69 | 2.20 | -0.83 | 75 | 2.41 | -0.66 | 78 | 8 2.26 | -0.74 | BREX+SERT VS PLACEBO | -0.32 | 0.0996 | -0.27 |
| EXP | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.40<br>-0.24<br>-0.08<br>0.08 | 0.0409<br>0.2473<br>0.6847<br>0.6614 | -0.33<br>-0.19<br>-0.07<br>0.07 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

PCL5-AVOID

EXTRNL

0.1626

-0 23

BREX+SERT VS PLACEBO -0.30

BREXPIPRAZOLE 3 OF 9

77 2.56 -0.91 69 2.62 -0.82 75 2.75 -0.69 78 2.44 -0.61

Adjusted Mean Change in PCL-5 Line Items (Intent to Treat Sample) BREX+SERT<sup>2</sup> PLACEBO COHEN's D ESTIMATED PCL5 MEAN LSMean MEAN LSMean TREATMENT EFFECT Line Items N Base Change¹ N Base Change¹ N Base Change¹ N Base Change¹ COMPARISON EFFECT 1 P-VALUE1 SIZE PCL5-AVOID 77 2.64 -1.07 69 2.46 -0.61 75 2.57 -0.52 78 2.63 -0.63 BREX+SERT VS PLACEBO -0.44 0.0395 -0.33 MEMRS THOUGTS FEEL STRES EXP BREX+SERT VS SERT -0.56 0.0116 -0.41 BREX+SERT VS BREX -0.47 0.0399 -0.34 BREX VS PLACEBO 0.03 0.9077 0.02 SERT VS PLACEBO 0.11 0.6017 0.08

REMINDRS STRESS EXP BREX+SERT VS SERT -0.22 0.3205 -0.16 BREX+SERT VS BREX -0.09 0.6967 -0.06 -0.21 0.3466 BREX VS PLACEBO -0.16 SERT VS PLACEBO -0.08 0.7043 -0.06 77 1.26 -0.71 69 1.45 -0.40 75 1.21 -0.62 78 1.23 -0.31 PCL5-TROUBLE BREX+SERT VS PLACEBO -0.40 0.0133 -0.40 REMBRNG IMP PRTS STRES EXP BREX+SERT VS SERT -0.09 0.6039 -0.08 0.0704 -0.30 BREX+SERT VS BREX -0.31 BREX VS PLACEBO -0.09 0.5896 -0.09

FILE: caps\_itemc.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.3 FINAL

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

BREXPIPRAZOLE 4 OF 9 PROTOCOL 331-201-00061

| THOTOGOL GOT L | | d Mean Change | STAT- | in PCL-5 Line | e Items | - MMRM | |
|---|---|---|---|---|---|---|---|
| | BREX+SERT <sup>2</sup> | BREX <sup>2</sup> | SERT <sup>2</sup> | PLACEBO | | ESTIMATED | COHEN's I |
| DCT F | MEDAL TOM | MEAN ICM | MEDNI I CM | MEAN TOMPS | MD E 3 MMENIM | MDE 3 MMENIM | BBBBC |

| PCL5 | N | BREX+S<br>MEAN<br>Base | LSMean | N | BRE<br>MEAN<br>Base | LSMean | N | SER<br>MEAN<br>Base | LSMean | N | | EBO<br>LSMean<br>Change <sup>1</sup> | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PCL5-TROUBLE<br>REMBRNG IMP<br>PRTS STRES EXP | | | | | | | | | | | | | SERT VS PLACEBO | -0.32 | 0.0520 | -0.32 |
| PCL5-HAVG<br>STRNG NEG<br>BELFS SELF PPL<br>WRLD | 7 | 7 2.29 | 9 -1.23 | 69 | 2.14 | -0.74 | 75 | 2.20 | -0.84 | 78 | 2.13 | -0.55 | BREX+SERT VS PLACEBO | -0.68 | 0.0003 | -0.59 |
| WKIID | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.39<br>-0.49<br>-0.20<br>-0.29 | 0.0407<br>0.0140<br>0.3099<br>0.1146 | -0.33<br>-0.41<br>-0.17<br>-0.26 |
| PCL5-BLAMNG<br>SELF OTHRS FOR<br>STRESSFL EXP | 7 | 7 2.13 | 3 -0.87 | 69 | 2.22 | -0.79 | 75 | 2.24 | -0.86 | 78 | 2.13 | -0.68 | BREX+SERT VS PLACEBO | -0.19 | 0.3678 | -0.14 |
| STREET BAT | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.01<br>-0.08<br>-0.11<br>-0.18 | 0.9523<br>0.7148<br>0.6233<br>0.4037 | -0.01<br>-0.06<br>-0.08<br>-0.14 |

FILE: caps\_itemc.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.3 FINAL

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

INTRST ACTIVTIES USD TO ENJOY

BREX+SERT VS SERT -0.68 0.0009 -0.55

BREXPIPRAZOLE 5 OF 9 PROTOCOL 331-201-00061

| | Adjust | ced Mean Change | (Intent to T | reat Sample) | Items - MM | | | |
|---|---|---|---|---|---|---|---|---|
| PCL5<br>Line Items | BREX+SERT <sup>2</sup><br>MEAN LSMean<br>N Base Change <sup>1</sup> | BREX <sup>2</sup><br>MEAN LSMean<br>N Base Change <sup>1</sup> | SERT <sup>2</sup><br>MEAN LSMean<br>N Base Change <sup>1</sup> | PLACEBO<br>MEAN LSMean<br>N Base Change <sup>1</sup> | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
| PCL5-HAVNG<br>STRNG NEG<br>FEELNGS | 77 2.44 -1.05 | 69 2.51 -0.74 | 75 2.49 -0.90 | 78 2.32 -0.74 | BREX+SERT VS PLACEBO | -0.31 | 0.1131 | -0.26 |
| 12221100 | | | | | BREX+SERT VS SERT | -0.15 | 0.4469 | -0.12 |
| | | | | | BREX+SERT VS BREX | -0.32 | 0.1280 | -0.25 |
| | | | | | BREX VS PLACEBO | 0.01 | 0.9775 | 0.00 |
| | | | | | SERT VS PLACEBO | -0.16 | 0.4192 | -0.13 |
| PCL5-LOSS | 77 2.61 -1.34 | 69 2.38 -0.78 | 75 2.41 -0.66 | 78 2.33 -0.76 | BREX+SERT VS PLACEBO | -0.57 | 0.0041 | -0.47 |

| | | | | | | | | | | | BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.56<br>-0.01<br>0.10 | 0.0079<br>0.9433<br>0.5991 | -0.44<br>-0.01<br>0.09 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PCL5-FEELNG<br>DISTANT CUT<br>OFF FROM OTHERS | 77 2. | 53 -1.12 | 69 2 | .68 -0.88 | 75 | 2.75 | -0.84 | 78 | 2.50 -0. | . 62 | BREX+SERT VS PLACEBO | -0.50 | 0.0107 | -0.41 |
| 011 111011 01112110 | | | | | | | | | | | BREX+SERT VS SERT | -0.28 | 0.1647 | -0.23 |
| | | | | | | | | | | | BREX+SERT VS BREX | -0.24 | 0.2412 | -0.19 |
| | | | | | | | | | | | BREX VS PLACEBO | -0.26 | 0.2050 | -0.21 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itemc.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.3 FINAL

PCL5-IRRITBLE

BEHAV ANGRY OUTBRST AGRSV

BREXPIPRAZOLE 6 OF 9 PROTOCOL 331-201-00061

| | | | Adjust | ed M | ean Ch | ange | | (In | tent to T | reat | | CL-5 Line<br>e)<br> | 10 - MM | IRM | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PCL5 Line Items | | | EERT <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | | LSMean | N | SER<br>MEAN<br>Base | LSMean | N | PLAC<br>MEAN<br>Base | LSMean | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE | COHEN'S D<br>EFFECT<br>SIZE |
| PCL5-FEELNG<br>DISTANT CUT<br>OFF FROM OTHERS | | | | | | | | | | | | | SERT VS PLACEBO | -0.22 | 0.2564 | -0.18 |
| PCL5-TRBLE<br>EXPERINCNG<br>POSITIVE<br>FEELNGS | 77 | 2.05 | -0.88 | 69 | 2.19 | -0.65 | 75 | 2.16 | -0.66 | 78 | 2.00 | -0.71 | BREX+SERT VS PLACEBO | -0.16 | 0.3492 | -0.15 |

BREX+SERT VS SERT

BREX+SERT VS BREX

BREX VS PLACEBO

BREX+SERT VS SERT BREX+SERT VS BREX

BREX VS PLACEBO

SERT VS PLACEBO

BREX+SERT VS PLACEBO -0.21

SERT VS PLACEBO

-0.22

-0.23

0.2231

0.2235

0.2766

-0.21 0.3047 -0.17

-0.00 0.9982 -0.00

-0.05 0.8090 -0.04

0.06 0.7334

0.05 0.7582

-0.16 0.4060

-0.20

-0.20

0.06

0.05

-0.18

-0.14

FILE: caps itemc.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC STAT/caps item.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.3

77 1.96 -0.79 69 1.84 -0.58 75 1.83 -0.63 78 1.82 -0.58

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

BREXPIPRAZOLE 7 OF 9 PROTOCOL 331-201-00061

| Adjusted Mean Change | in PCL-5 Line Items (Intent to Treat Sample) | - MMRM |
|----------------------|----------------------------------------------|--------|

| PCL5 Line Items | | BREX+S<br>MEAN<br>Base | ERT <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | BRE<br>MEAN<br>Base | X <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N<br> | SER<br>MEAN<br>Base | LSMean | N | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT 1 | P-VALUE <sup>1</sup> | COHEN'S I<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PCL5-TAKNG TOO<br>MNY RISKS THT<br>CAUSE HARM | 77 | 0.78 | -0.30 | 69 | 0.71 | -0.18 | 75 | 0.79 | -0.48 | 78 | 0.72 | -0.21 | BREX+SERT VS PLACEBO | -0.09 | 0.4502 | -0.12 |
| CAUSE HAIM | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | 0.18<br>-0.12<br>0.03<br>-0.27 | 0.1340<br>0.3379<br>0.8022<br>0.0237 | 0.24<br>-0.16<br>0.04<br>-0.37 |
| PCL5-BEING<br>SUPERALERT<br>WATCHFUL ON<br>GUARD | 77 | 2.86 | -0.70 | 69 | 2.78 | -0.62 | 75 | 2.69 | -0.63 | 78 | 2.68 | -0.64 | BREX+SERT VS PLACEBO | -0.07 | 0.7349 | -0.05 |
| GOARD | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.07<br>-0.08<br>0.02<br>0.00 | 0.7235<br>0.6897<br>0.9365<br>0.9823 | -0.06<br>-0.07<br>0.01<br>0.00 |
| PCL5-FEELING<br>JUMPY OR | 77 | 2.26 | -0.84 | 69 | 2.23 | -0.73 | 75 | 1.97 | -0.58 | 78 | 2.24 | -0.83 | BREX+SERT VS PLACEBO | -0.00 | 0.9802 | -0.00 |
| EASILY STARTLED | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO | -0.25<br>-0.11<br>0.10 | 0.1856<br>0.5805<br>0.5919 | -0.22<br>-0.09<br>0.09 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itemc.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.3 FINAL

BREXPIPRAZOLE 8 OF 9 PROTOCOL 331-201-00061

| | Adjusted Mean Change in PCL-5 Line Items - MMRM (Intent to Treat Sample) | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PCL5<br>Line Items | | ERT <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | | LSMean | MEA | ERT <sup>2</sup><br>N LSMean<br>e Change <sup>1</sup> | PLAC<br>MEAN<br>N Base | LSMean | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT 1 | P-VALUE 1 | COHEN'S D<br>EFFECT<br>SIZE |
| PCL5-FEELING<br>JUMPY OR<br>EASILY STARTLED | | | | | | | | | SERT VS PLACEBO | 0.25 | 0.1874 | 0.21 |
| PCL5-HAVNG<br>DIFFICULTY<br>CONCENTRATNG | 77 2.58 | -0.94 | 69 2.57 | -0.75 | 75 2. | 35 -0.69 | 78 2.38 | -0.62 | BREX+SERT VS PLACEBO | -0.32 | 0.0747 | -0.29 |
| 001102211111110 | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.25<br>-0.20<br>-0.12<br>-0.07 | 0.1674<br>0.2991<br>0.5099<br>0.7080 | -0.22<br>-0.17<br>-0.11<br>-0.06 |
| PCL5-TROUBLE<br>FALLING OR<br>STAYING ASLEEP | 77 2.47 | -0.94 | 69 2.74 | -0.90 | 75 2. | 81 -0.53 | 78 2.83 | -0.70 | BREX+SERT VS PLACEBO | -0.24 | 0.2503 | -0.19 |
| STATING ASLEEF | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.41<br>-0.03<br>-0.20<br>0.17 | 0.0509<br>0.8788<br>0.3415<br>0.4001 | -0.32<br>-0.03<br>-0.16<br>0.14 |
| PCL-5 TOTAL<br>SCORE | 77 44.21 | -18.6 | 69 44.20 | -13.8 | 75 44. | 59 -13.7 | 78 42.49 | -12.6 | BREX+SERT VS PLACEBO | | 0.0143 | -0.40 |
| | | | | | | | | | BREX+SERT VS SERT | -4.93 | 0.0487 | -0.32 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itemc.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.3 FINAL

BREXPIPRAZOLE 9 OF 9

Adjusted Mean Change in PCL-5 Line Items - MMRM (Intent to Treat Sample)

| PCL5 Line Items | BREX+SERT <sup>2</sup><br>MEAN LSMean<br>N Base Change <sup>1</sup> | BREX <sup>2</sup><br>MEAN LSMean<br>N Base Change <sup>1</sup> | PLACEBO<br>MEAN LSMean<br>N Base Change <sup>1</sup> | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | COHEN'S D<br>EFFECT<br>P-VALUE¹ SIZE |
|---|---|---|---|---|---|---|
| PCL-5 TOTAL<br>SCORE | | | | BREX+SERT VS BREX | -4.84 | 0.0607 -0.31 |
| 000112 | | | | BREX VS PLACEBO<br>SERT VS PLACEBO | -1.18<br>-1.08 | 0.6433 -0.08<br>0.6586 -0.07 |

FILE: caps\_itemc.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.3 FINAL

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

BREXPIPRAZOLE 1 OF 6 PROTOCOL 331-201-00061

Adjusted Mean Change in HADS Line Items — MMRM

(Intent to Treat Sample)

| HADS<br>Line Items | | BREX+S<br>MEAN<br>Base | LSMean | N | BRE<br>MEAN<br>Base | | N<br> | SER<br>MEAN<br>Base | T <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | | EBO<br>LSMean<br>Change <sup>1</sup> | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S I<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| HADS01-I FEEL<br>TENSE OR WOUND<br>UP | 77 | 1.97 | -0.73 | 68 | 1.79 | -0.23 | 75 | 1.92 | -0.40 | 78 | 1.91 | -0.42 | BREX+SERT VS PLACEBO | -0.31 | 0.0394 | -0.33 |
| | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.33<br>-0.50<br>0.19<br>0.02 | 0.0305<br>0.0019<br>0.2233<br>0.8822 | -0.35<br>-0.52<br>0.20<br>0.02 |
| HADS01-ENJOY<br>THE THINGS I<br>USED TO ENJOY | 77 | 1.74 | -0.56 | 68 | 1.59 | -0.51 | 75 | 1.63 | -0.23 | 78 | 1.55 | -0.54 | BREX+SERT VS PLACEBO | -0.02 | 0.8919 | -0.02 |
| USED TO ENJOY | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.33<br>-0.05<br>0.03<br>0.31 | 0.0386<br>0.7712<br>0.8685<br>0.0494 | -0.34<br>-0.05<br>0.03<br>0.32 |
| HADS01-SOMETHIN<br>G AWFUL ABOUT<br>TO HAPPEN | 77 | 1.94 | -0.72 | 68 | 1.79 | -0.38 | 75 | 1.88 | -0.39 | 78 | 1.94 | -0.58 | BREX+SERT VS PLACEBO | -0.13 | 0.3534 | -0.15 |
| TO HAPPEN | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.33<br>-0.33<br>0.20<br>0.19 | 0.0284<br>0.0323<br>0.1959<br>0.1909 | -0.36<br>-0.36<br>0.22<br>0.21 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itemd.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.4 FINAL

BREXPIPRAZOLE 2 OF 6 PROTOCOL 331-201-00061

| Adjusted Mean Change | STAT-1.4 in HADS Line Items (Intent to Treat Sample) | - MMRM |
|---|---|---|
| <br> | | |

| HADS<br>Line Items | N | Base | LSMean | N | | X <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | SER<br>MEAN<br>Base | LSMean | N | | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| HADS01-I CAN<br>LAUGH AND SEE<br>FUNNY SIDE | | 1.08 | -0.38 | 68 | 1.06 | -0.03 | 75 | 1.01 | -0.13 | 78 | 0.92 | -0.23 | BREX+SERT VS PLACEBO | -0.15 | 0.2374 | -0.19 |
| FORMI SIDE | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.25<br>-0.35<br>0.21<br>0.10 | 0.0541<br>0.0085<br>0.1205<br>0.4355 | -0.31<br>-0.44<br>0.26<br>0.13 |
| HADS01-WORRYING<br>THOUGHTS GO | 77 | 2.06 | -0.71 | 68 | 1.94 | -0.33 | 75 | 2.07 | -0.42 | 78 | 2.12 | -0.43 | BREX+SERT VS PLACEBO | -0.29 | 0.0646 | -0.30 |
| THROUGH MIND | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.29<br>-0.38<br>0.09<br>0.00 | 0.0677<br>0.0227<br>0.5773<br>0.9893 | -0.30<br>-0.38<br>0.09<br>0.00 |
| HADS01-I FEEL<br>CHEERFUL | 77 | 1.47 | -0.56 | 68 | 1.32 | -0.32 | 75 | 1.41 | -0.37 | 78 | 1.24 | -0.31 | BREX+SERT VS PLACEBO | -0.25 | 0.0526 | -0.31 |
| OHBBAC OB | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.19<br>-0.24<br>-0.01<br>-0.06 | 0.1371<br>0.0835<br>0.9180<br>0.6638 | -0.24<br>-0.29<br>-0.02<br>-0.07 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itemd.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.4 FINAL

BREXPIPRAZOLE 3 OF 6 PROTOCOL 331-201-00061

| Adjusted Mean Change | STAT-1.4 in 1 | HADS Line Items e) | - MMRM |
|----------------------|---------------|--------------------|--------|
| <br> | | | |

| HADS<br>Line Items | | BREX+S<br>MEAN<br>Base | | N | BRE<br>MEAN<br>Base | X <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N | SER<br>MEAN<br>Base | LSMean | N | | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| HADS01-SIT AT<br>EASE AND FEEL<br>RELAXED | 77 | 1.79 | -0.49 | 68 | 1.72 | -0.23 | 75 | 1.73 | -0.23 | 78 | 1.76 | -0.35 | BREX+SERT VS PLACEBO | -0.14 | 0.2632 | -0.18 |
| | | | | | | | | | | | | | BREX+SERT VS SERT | -0.26 | 0.0400 | -0.34 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.26 | 0.0476 | -0.33 |
| | | | | | | | | | | | | | BREX VS PLACEBO | 0.12 | 0.3449 | 0.16 |
| | | | | | | | | | | | | | SERT VS PLACEBO | 0.12 | 0.3290 | 0.16 |
| HADS01-I FEEL<br>AS IF I AM<br>SLOWED DOWN | 77 | 1.60 | -0.65 | 68 | 1.43 | -0.37 | 75 | 1.40 | -0.39 | 78 | 1.51 | -0.54 | BREX+SERT VS PLACEBO | -0.10 | 0.4793 | -0.11 |
| SHOWED DOWN | | | | | | | | | | | | | BREX+SERT VS SERT | -0.26 | 0.0805 | -0.28 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.28 | 0.0696 | -0.30 |
| | | | | | | | | | | | | | BREX VS PLACEBO | 0.18 | 0.2403 | 0.20 |
| | | | | | | | | | | | | | SERT VS PLACEBO | 0.16 | 0.2794 | 0.18 |
| HADS01-BUTTERFL<br>IES IN THE | 77 | 1.31 | -0.36 | 68 | 1.29 | -0.19 | 75 | 1.41 | -0.38 | 78 | 1.32 | -0.45 | BREX+SERT VS PLACEBO | 0.08 | 0.5221 | 0.10 |
| STOMACH | | | | | | | | | | | | | BREX+SERT VS SERT | 0.02 | 0.9061 | 0.02 |
| | | | | | | | | | | | | | BREX+SERT VS BREX | -0.18 | 0.2075 | -0.21 |
| | | | | | | | | | | | | | BREX VS PLACEBO | 0.26 | 0.0603 | 0.31 |
| | | | | | | | | | | | | | SERT VS PLACEBO | 0.07 | 0.6053 | 0.08 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itemd.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.4 FINAL

BREXPIPRAZOLE 4 OF 6 PROTOCOL 331-201-00061

| 11010002 002 202 00002 | Adjusted Mean Change | STAT-1.4 in HADS Line Items Intent to Treat Sample) | - MMRM |
|---|---|---|---|

| HADS<br>Line Items | ME<br>N Ba | ase | LSMean<br>Change¹ | N<br> | BRE<br>MEAN<br>Base | X <sup>2</sup><br>LSMean<br>Change <sup>1</sup> | N<br> | SER<br>MEAN<br>Base | LSMean | N<br> | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| HADS01-LOST<br>INTEREST IN MY<br>APPEARANCE | 77 1 | 1.35 | -0.42 | 68 | 1.28 | -0.31 | 75 | 1.40 | -0.16 | 78 | 1.42 | -0.26 | BREX+SERT VS PLACEBO | -0.16 | 0.2080 | -0.20 |
| III I BIRGINOD | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.26<br>-0.11<br>-0.05<br>0.10 | 0.0491<br>0.4299<br>0.6901<br>0.4551 | -0.32<br>-0.13<br>-0.07<br>0.12 |
| HADS01-FEEL<br>RESTLESS BE ON<br>THE MOVE | 77 1 | 1.90 | -0.59 | 68 | 1.75 | -0.20 | 75 | 1.85 | -0.36 | 78 | 1.85 | -0.36 | BREX+SERT VS PLACEBO | -0.23 | 0.1186 | -0.25 |
| THE MOVE | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.23<br>-0.39<br>0.17<br>0.01 | 0.1153<br>0.0113<br>0.2731<br>0.9652 | -0.26<br>-0.42<br>0.18<br>0.01 |
| HADS01-LOOK<br>FORWARD WITH | 77 1 | 1.60 | -0.51 | 68 | 1.53 | -0.17 | 75 | 1.59 | -0.26 | 78 | 1.29 | -0.30 | BREX+SERT VS PLACEBO | -0.21 | 0.1853 | -0.21 |
| ENJOYMENT | | | | | | | | | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.25<br>-0.34<br>0.13<br>0.04 | 0.1197<br>0.0415<br>0.4292<br>0.8053 | -0.25<br>-0.34<br>0.13<br>0.04 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itemd.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.4 FINAL

BREXPIPRAZOLE 5 OF 6 PROTOCOL 331-201-00061

| Adjusted Mean Change | STAT-1.4 in HADS Line Items - MMRM (Intent to Treat Sample) |
|---|---|

| HADS<br>Line Items | BREX+SERT <sup>2</sup> MEAN LSMean N Base Change <sup>1</sup> | BREX²<br>MEAN LSMean<br>N Base Change¹ | SERT <sup>2</sup><br>MEAN LSMean<br>N Base Change <sup>1</sup> | PLACEBO<br>MEAN LSMean<br>N Base Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT 1 | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|
| HADS01-I GET<br>SUDDEN<br>FEELINGS OF<br>PANIC | 77 1.61 -0.43 | 68 1.68 -0.27 | 75 1.71 -0.37 | 78 1.60 -0.34 | BREX+SERT VS PLACEBO | -0.09 | 0.4975 | -0.11 |
| FANTC | | | | | BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO<br>SERT VS PLACEBO | -0.05<br>-0.16<br>0.06<br>-0.04 | 0.7002<br>0.2751<br>0.6444<br>0.7765 | -0.06<br>-0.18<br>0.08<br>-0.05 |
| HADS01-ENJOY<br>GOOD BOOK | 77 1.44 -0.45 | 68 1.18 -0.12 | 75 1.12 -0.25 | 78 1.03 -0.25 | BREX+SERT VS PLACEBO<br>BREX+SERT VS SERT<br>BREX+SERT VS BREX<br>BREX VS PLACEBO | -0.20<br>-0.33<br>0.13 | 0.1530<br>0.1558<br>0.0232<br>0.3444 | -0.23<br>-0.23<br>-0.38<br>0.16 |
| HADS SUBSCALE<br>A TOTAL SCORE | 77 12.58 -4.00 | 68 11.97 -1.60 | 75 12.57 -2.46 | 78 12.49 -2.80 | BREX+SERT VS PLACEBO BREX+SERT VS SERT BREX+SERT VS BREX BREX VS PLACEBO SERT VS PLACEBO | 0.00<br>-1.20<br>-1.55<br>-2.41<br>1.20<br>0.34 | 0.9935<br>0.0793<br>0.0274<br>0.0010<br>0.0930<br>0.6172 | 0.00<br>-0.28<br>-0.36<br>-0.55<br>0.28<br>0.08 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

FILE: caps\_itemd.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_item.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-1.4 FINAL

BREXPIPRAZOLE 6 OF 6 PROTOCOL 331-201-00061

Adjusted Mean Change in HADS Line Items - MMRM (Intent to Treat Sample)

| HADS<br>Line Items | BREX+SERT <sup>2</sup> MEAN LSMean N Base Change | BREX <sup>2</sup><br>MEAN LSMean<br>N Base Change <sup>1</sup> | SERT <sup>2</sup><br>MEAN LSMean<br>N Base Change <sup>1</sup> | PLACEBO<br>MEAN LSMean<br>N Base Change <sup>1</sup> | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE¹ | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|
| HADS SUBSCALE D TOTAL SCORE | 77 10.27 -3.66 | 68 9.38 -1.75 | 75 9.56 -1.72 | 78 8.97 -2.21 | BREX+SERT VS PLACEBO | -1.45 | 0.0249 | -0.36 |
| 5 101112 00012 | | | | | BREX+SERT VS SERT | -1.94 | 0.0033 | -0.48 |
| | | | | | BREX+SERT VS BREX | -1.91 | 0.0053 | -0.47 |
| | | | | | BREX VS PLACEBO | 0.46 | 0.4939 | 0.11 |
| | | | | | SERT VS PLACEBO | 0.49 | 0.4476 | 0.12 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, TYPE OF TRAUMA, VISIT, TREATMENT BY VISIT AND BASELINE BY

BREXPIPRAZOLE 1 OF 39

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction
(Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Model Information

Data Set WORK.INDATA
Dependent Variable CHG
Covariance Structure Unstructured
Subject Effect SUBJID
Estimation Method REML
Residual Variance Method None

Fixed Effects SE Method Kenward-Roger Degrees of Freedom Method Kenward-Roger

Class Level Information

| Class | Levels | Values |
|------------------|--------|------------------------|
| AVISITN<br>TRTPN | 4 | 3 6 10 12<br>1 2 3 900 |
| POOLCNTR | 10 | |
| COMBFL | 2 | N Y |

FILE: stat2a.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.1 FINAL

BREXPIPRAZOLE 2 OF 39 PROTOCOL 331-201-00061

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Class Level Information

Class Levels Values
SUBJID 299

FILE: stat2a.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.1 FINAL

BREXPIPRAZOLE


3 OF 39

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

The Mixed Procedure



FILE: stat2a.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.1 FINAL

BREXPIPRAZOLE 4 OF 39
STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

The Mixed Procedure



FILE: stat2a.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.1 FINAL

BREXPIPRAZOLE 5 OF 39

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

The Mixed Procedure



FILE: stat2a.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.1 FINAL

BREXPIPRAZOLE 6 OF 39 PROTOCOL 331-201-00061 STAT-3.1 MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample) The Mixed Procedure SEX 2 F M Dimensions Covariance Parameters 10 Columns in X 91 Columns in Z 0 299 Subjects Max Obs per Subject Number of Observations 996 Number of Observations Read Number of Observations Used 996 Number of Observations Not Used

FILE: stat2a.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.1 FINAL

BREXPIPRAZOLE 7 OF 39

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

.\_\_\_\_\_

The Mixed Procedure

Iteration History

| Criterion | -2 Res Log Like | Evaluations | Iteration |
|------------|-----------------|-------------|-----------|
| | 7347.61199056 | 1 | 0 |
| 0.00048752 | 6870.77895648 | 2 | 1 |
| 0.00001813 | 6869.39176021 | 1 | 2 |
| 0.0000003 | 6869.34408788 | 1 | 3 |
| 0.00000000 | 6869.34400894 | 1 | 4 |

Convergence criteria  $\operatorname{met}$ .

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | 78.3536 |
| UN(2,1) | SUBJID | 52.5580 |
| UN(2,2) | SUBJID | 113.32 |
| UN(3,1) | SUBJID | 43.5675 |
| UN(3,2) | SUBJID | 89.6909 |
| UN(3,3) | SUBJID | 124.09 |
| UN(4,1) | SUBJID | 48.7794 |

FILE: stat2a.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.1 FINAL

BREXPIPRAZOLE 8 OF 39

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN (4,2) | SUBJID | 90.3794 |
| UN (4,3) | SUBJID | 106.13 |
| UN (4,4) | SUBJID | 148.60 |

Fit Statistics

| -2 Res Log Likelihood | 6869.3 |
|--------------------------|--------|
| AIC (Smaller is Better) | 6889.3 |
| AICC (Smaller is Better) | 6889.6 |
| BIC (Smaller is Better) | 6926.3 |

Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSo |
|----|------------|------------|
| 9 | 478.27 | < . 000 |

BREXPIPRAZOLE 9 OF 39

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|-------------------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| POOLCNTR | 9 | 278 | 1.66 | 0.0986 |
| COMBFL | 1 | 278 | 3.11 | 0.0788 |
| AVISITN | 3 | 226 | 0.79 | 0.5023 |
| TRTPN | 3 | 264 | 2.42 | 0.0665 |
| AVISITN*TRTPN | 9 | 357 | 1.58 | 0.1209 |
| SEX | 1 | 287 | 0.04 | 0.8490 |
| AVISITN*SEX | 3 | 232 | 1.80 | 0.1474 |
| TRTPN*SEX | 3 | 264 | 0.35 | 0.7878 |
| AVISITN*TRTPN*SEX | 9 | 357 | 0.96 | 0.4707 |
| BASE*AVISITN | 4 | 239 | 14.93 | <.0001 |



FILE: stat2a.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.1 FINAL

BREXPIPRAZOLE 11 OF 39 PROTOCOL 331-201-00061

STAT-3.

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

.....

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY SEX AT Phase B

| | Center<br>(Pooled | Combat<br>Related | | Analysis | Planned | |
|---|---|---|---|---|---|---|
| | Center) | Population | | Visit | Treatment | |
| Effect | for ITT | Flag | Sex | (N) | (N) | Row1 |
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |

FILE: stat2a.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.1 FINAL

BREXPIPRAZOLE 12 OF 39 PROTOCOL 331-201-00061

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY SEX AT Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | Sex | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 12 | 900 | |
| SEX | | | F | | | |
| SEX | | | M | | | |
| AVISITN*SEX | | | F | 3 | | |
| AVISITN*SEX | | | M | 3 | | |
| AVISITN*SEX | | | F | 6 | | |
| AVISITN*SEX | | | M | 6 | | |
| AVISITN*SEX | | | F | 10 | | |
| AVISITN*SEX | | | M | 10 | | |
| AVISITN*SEX | | | F | 12 | | |
| AVISITN*SEX | | | M | 12 | | |
| TRTPN*SEX | | | F | | 1 | 1 |
| TRTPN*SEX | | | M | | 1 | -1 |
| TRTPN*SEX | | | F | | 2 | |
| TRTPN*SEX | | | M | | 2 | |
| TRTPN*SEX | | | F | | 3 | |
| TRTPN*SEX | | | M | | 3 | |
| TRTPN*SEX | | | F | | 900 | -1 |

BREXPIPRAZOLE 13 OF 39 PROTOCOL 331-201-00061

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY SEX AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Sex | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*SEX | | | М | | 900 | 1 |
| AVISITN*TRTPN*SEX | | | F | 3 | 1 | |
| AVISITN*TRTPN*SEX | | | M | 3 | 1 | |
| AVISITN*TRTPN*SEX | | | F | 3 | 2 | |
| AVISITN*TRTPN*SEX | | | M | 3 | 2 | |
| AVISITN*TRTPN*SEX | | | F | 3 | 3 | |
| AVISITN*TRTPN*SEX | | | M | 3 | 3 | |
| AVISITN*TRTPN*SEX | | | F | 3 | 900 | |
| AVISITN*TRTPN*SEX | | | M | 3 | 900 | |
| AVISITN*TRTPN*SEX | | | F | 6 | 1 | |
| AVISITN*TRTPN*SEX | | | M | 6 | 1 | |
| AVISITN*TRTPN*SEX | | | F | 6 | 2 | |
| AVISITN*TRTPN*SEX | | | M | 6 | 2 | |
| AVISITN*TRTPN*SEX | | | F | 6 | 3 | |
| AVISITN*TRTPN*SEX | | | M | 6 | 3 | |
| AVISITN*TRTPN*SEX | | | F | 6 | 900 | |
| AVISITN*TRTPN*SEX | | | M | 6 | 900 | |
| AVISITN*TRTPN*SEX | | | F | 10 | 1 | 1 |

BREXPIPRAZOLE 14 OF 39 PROTOCOL 331-201-00061

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY SEX AT Phase B

| | Center | Combat | | | | |
|-------------------|---------|------------|-----|----------|-----------|------|
| | (Pooled | Related | | Analysis | Planned | |
| | Center) | Population | | Visit | Treatment | |
| Effect | for ITT | Flag | Sex | (N) | (N) | Row1 |
| AVISITN*TRTPN*SEX | | | М | 10 | 1 | -1 |
| AVISITN*TRTPN*SEX | | | F | 10 | 2 | |
| AVISITN*TRTPN*SEX | | | M | 10 | 2 | |
| AVISITN*TRTPN*SEX | | | F | 10 | 3 | |
| AVISITN*TRTPN*SEX | | | M | 10 | 3 | |
| AVISITN*TRTPN*SEX | | | F | 10 | 900 | -1 |
| AVISITN*TRTPN*SEX | | | M | 10 | 900 | 1 |
| AVISITN*TRTPN*SEX | | | F | 12 | 1 | |
| AVISITN*TRTPN*SEX | | | M | 12 | 1 | |
| AVISITN*TRTPN*SEX | | | F | 12 | 2 | |
| AVISITN*TRTPN*SEX | | | M | 12 | 2 | |
| AVISITN*TRTPN*SEX | | | F | 12 | 3 | |
| AVISITN*TRTPN*SEX | | | M | 12 | 3 | |
| AVISITN*TRTPN*SEX | | | F | 12 | 900 | |
| AVISITN*TRTPN*SEX | | | M | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |



FILE: stat2a.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.1 FINAL

BREXPIPRAZOLE 16 OF 39 PROTOCOL 331-201-00061

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY SEX AT Phase B

| <b>7</b> 66 . | Center<br>(Pooled<br>Center) | | | Analysis<br>Visit | Treatment | _ 1 |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | Sex | (N) | (N) | Row1 |
| POOLCNTR | | | | | | |
| POOLCNTR | | | | | | |
| POOLCNTR | | | | | | |
| COMBFL | | N | | | | |
| COMBFL | | Y | | | | |
| AVISITN | | | | 3 | | |
| AVISITN | | | | 6 | | |
| AVISITN | | | | 10 | | |
| AVISITN | | | | 12 | | |
| TRTPN | | | | | 1 | |
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |

FILE: stat2a.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.1 FINAL

AVISITN\*TRTPN

BREXPIPRAZOLE 17 OF 39 PROTOCOL 331-201-00061

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY SEX AT Phase B

| | Center<br>(Pooled<br>Center) | Combat<br>Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | Sex | (N) | (N) | Row1 |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |
| AVISITN*TRTPN | | | | 12 | 900 | |
| SEX | | | F | | | |
| SEX | | | M | | | |
| AVISITN*SEX | | | F | 3 | | |
| AVISITN*SEX | | | M | 3 | | |
| AVISITN*SEX | | | F | 6 | | |
| AVISITN*SEX | | | M | 6 | | |
| AVISITN*SEX | | | F | 10 | | |

FILE: stat2a.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.1 FINAL

BREXPIPRAZOLE 18 OF 39 PROTOCOL 331-201-00061

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY SEX AT Phase B

| | Center | Combat | | 2 | D1 1 | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | | Analysis<br>Visit | Planned | |
| | Center) | Population | _ | | Treatment | |
| Effect | for ITT | Flag | Sex | (N) | (N) | Row1 |
| AVISITN*SEX | | | М | 10 | | |
| AVISITN*SEX | | | F | 12 | | |
| | | | _ | | | |
| AVISITN*SEX | | | M | 12 | | |
| TRTPN*SEX | | | F | | 1 | 1 |
| TRTPN*SEX | | | M | | 1 | -1 |
| TRTPN*SEX | | | F | | 2 | |
| TRTPN*SEX | | | M | | 2 | |
| TRTPN*SEX | | | F | | 3 | -1 |
| TRTPN*SEX | | | M | | 3 | 1 |
| TRTPN*SEX | | | F | | 900 | |
| TRTPN*SEX | | | M | | 900 | |
| AVISITN*TRTPN*SEX | | | F | 3 | 1 | |
| AVISITN*TRTPN*SEX | | | M | 3 | 1 | |
| AVISITN*TRTPN*SEX | | | F | 3 | 2 | |
| AVISITN*TRTPN*SEX | | | M | 3 | 2 | |
| AVISITN*TRTPN*SEX | | | F | 3 | 3 | |
| AVISITN*TRTPN*SEX | | | M | 3 | 3 | |
| AVISITN*TRTPN*SEX | | | F | 3 | 900 | |

BREXPIPRAZOLE 19 OF 39 PROTOCOL 331-201-00061

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY SEX AT Phase B

| | Center | Combat | | | | |
|-------------------|---------|------------|-----|----------|-----------|------|
| | (Pooled | Related | | Analysis | Planned | |
| | Center) | Population | | Visit | Treatment | |
| Effect | for ITT | Flag | Sex | (N) | (N) | Row1 |
| AVISITN*TRTPN*SEX | | | M | 3 | 900 | |
| AVISITN*TRTPN*SEX | | | F | 6 | 1 | |
| AVISITN*TRTPN*SEX | | | M | 6 | 1 | |
| AVISITN*TRTPN*SEX | | | F | 6 | 2 | |
| AVISITN*TRTPN*SEX | | | M | 6 | 2 | |
| AVISITN*TRTPN*SEX | | | F | 6 | 3 | |
| AVISITN*TRTPN*SEX | | | M | 6 | 3 | |
| AVISITN*TRTPN*SEX | | | F | 6 | 900 | |
| AVISITN*TRTPN*SEX | | | M | 6 | 900 | |
| AVISITN*TRTPN*SEX | | | F | 10 | 1 | 1 |
| AVISITN*TRTPN*SEX | | | M | 10 | 1 | -1 |
| AVISITN*TRTPN*SEX | | | F | 10 | 2 | |
| AVISITN*TRTPN*SEX | | | M | 10 | 2 | |
| AVISITN*TRTPN*SEX | | | F | 10 | 3 | -1 |
| AVISITN*TRTPN*SEX | | | M | 10 | 3 | 1 |
| AVISITN*TRTPN*SEX | | | F | 10 | 900 | |
| AVISITN*TRTPN*SEX | | | M | 10 | 900 | |
| AVISITN*TRTPN*SEX | | | F | 12 | 1 | |
BREXPIPRAZOLE 20 OF 39 PROTOCOL 331-201-00061

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY SEX AT Phase B

Center Combat Center) Population for ITT Flor Analysis Planned Visit Treatment Effect (N) (N) Row1 AVISITN\*TRTPN\*SEX 12 AVISITN\*TRTPN\*SEX F 12 2 Μ 12 AVISITN\*TRTPN\*SEX AVISITN\*TRTPN\*SEX F 12 3 AVISITN\*TRTPN\*SEX Μ 12 .3 12 AVISITN\*TRTPN\*SEX F 900 AVISITN\*TRTPN\*SEX M 12 900 BASE\*AVISITN 3 6 BASE\*AVISITN 10 BASE\*AVISITN 12 BASE\*AVISITN



FILE: stat2a.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.1 FINAL

BREXPIPRAZOLE 22 OF 39 PROTOCOL 331-201-00061

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY SEX AT Phase B

| | Center | Combat | | | | |
|---------------|---------|------------|-----|----------|-----------|------|
| | (Pooled | Related | | Analysis | | |
| | Center) | Population | | Visit | Treatment | |
| Effect | for ITT | Flag | Sex | (N) | (N) | Row1 |
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| | | | | | 900 | |
| TRTPN | | | | 2 | | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |

BREXPIPRAZOLE 23 OF 39 PROTOCOL 331-201-00061

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

.....

Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY SEX AT Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | Sex | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 12 | 900 | |
| SEX | | | F | | | |
| SEX | | | M | | | |
| AVISITN*SEX | | | F | 3 | | |
| AVISITN*SEX | | | M | 3 | | |
| AVISITN*SEX | | | F | 6 | | |
| AVISITN*SEX | | | M | 6 | | |
| AVISITN*SEX | | | F | 10 | | |
| AVISITN*SEX | | | M | 10 | | |
| AVISITN*SEX | | | F | 12 | | |
| AVISITN*SEX | | | M | 12 | | |
| TRTPN*SEX | | | F | | 1 | 1 |
| TRTPN*SEX | | | M | | 1 | -1 |
| TRTPN*SEX | | | F | | 2 | -1 |
| TRTPN*SEX | | | M | | 2 | 1 |
| TRTPN*SEX | | | F | | 3 | |
| TRTPN*SEX | | | M | | 3 | |
| TRTPN*SEX | | | F | | 900 | |

BREXPIPRAZOLE 24 OF 39


MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY SEX AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Sex | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|
| TRTPN*SEX | | М | | 900 | |
| AVISITN*TRTPN*SEX | | F | 3 | 1 | |
| AVISITN*TRTPN*SEX | | M | 3 | 1 | |
| AVISITN*TRTPN*SEX | | F | 3 | 2 | |
| AVISITN*TRTPN*SEX | | M | 3 | 2 | |
| AVISITN*TRTPN*SEX | | F | 3 | 3 | |
| AVISITN*TRTPN*SEX | | M | 3 | 3 | |
| AVISITN*TRTPN*SEX | | F | 3 | 900 | |
| AVISITN*TRTPN*SEX | | M | 3 | 900 | |
| AVISITN*TRTPN*SEX | | F | 6 | 1 | |
| AVISITN*TRTPN*SEX | | M | 6 | 1 | |
| AVISITN*TRTPN*SEX | | F | 6 | 2 | |
| AVISITN*TRTPN*SEX | | M | 6 | 2 | |
| AVISITN*TRTPN*SEX | | F | 6 | 3 | |
| AVISITN*TRTPN*SEX | | M | 6 | 3 | |
| AVISITN*TRTPN*SEX | | F | 6 | 900 | |
| AVISITN*TRTPN*SEX | | M | 6 | 900 | |
| AVISITN*TRTPN*SEX | | F | 10 | 1 | 1 |

BREXPIPRAZOLE 25 OF 39 PROTOCOL 331-201-00061

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)



The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY SEX AT Phase B Week 10

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | Sex | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AUTOTMN+MDMDN+OEV | | | М | 1.0 | 1 | 1 |
| AVISITN*TRTPN*SEX | | | | 10 | 1 | -1 |
| AVISITN*TRTPN*SEX | | | F | 10 | 2 | -1 |
| AVISITN*TRTPN*SEX | | | M | 10 | 2 | 1 |
| AVISITN*TRTPN*SEX | | | F | 10 | 3 | |
| AVISITN*TRTPN*SEX | | | M | 10 | 3 | |
| AVISITN*TRTPN*SEX | | | F | 10 | 900 | |
| AVISITN*TRTPN*SEX | | | M | 10 | 900 | |
| AVISITN*TRTPN*SEX | | | F | 12 | 1 | |
| AVISITN*TRTPN*SEX | | | M | 12 | 1 | |
| AVISITN*TRTPN*SEX | | | F | 12 | 2 | |
| AVISITN*TRTPN*SEX | | | M | 12 | 2 | |
| AVISITN*TRTPN*SEX | | | F | 12 | 3 | |
| AVISITN*TRTPN*SEX | | | M | 12 | 3 | |
| AVISITN*TRTPN*SEX | | | F | 12 | 900 | |
| AVISITN*TRTPN*SEX | | | M | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |



FILE: stat2a.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.1 FINAL

BREXPIPRAZOLE 27 OF 39 PROTOCOL 331-201-00061

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY SEX AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Sex | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| POOLCNTR | | | | | | |
| POOLCNTR | | | | | | |
| POOLCNTR | | | | | | |
| COMBFL | | N | | | | |
| COMBFL | | Y | | | | |
| AVISITN | | | | 3 | | |
| AVISITN | | | | 6 | | |
| AVISITN | | | | 10 | | |
| AVISITN | | | | 12 | | |
| TRTPN | | | | | 1 | |
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |

FILE: stat2a.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.1 FINAL

AVISITN\*TRTPN

BREXPIPRAZOLE 28 OF 39 PROTOCOL 331-201-00061

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY SEX AT Phase B

| Center) Population Visit Treatment Effect for ITT Flag Sex (N) (N) AVISITN*TRTPN 6 2 | Row1 |
|---|---|
| AVISITN*TRTPN 6 2 | |
| AVISITN*TRTPN 6 3 | |
| AVISITN*TRTPN 6 900 | |
| AVISITN*TRTPN 10 1 | |
| AVISITN*TRTPN 10 2 | |
| AVISITN*TRTPN 10 3 | |
| AVISITN*TRTPN 10 900 | |
| AVISITN*TRTPN 12 1 | |
| AVISITN*TRTPN 12 2 | |
| AVISITN*TRTPN 12 3 | |
| AVISITN*TRTPN 12 900 | |
| SEX F | |
| SEX M | |
| AVISITN*SEX F 3 | |
| AVISITN*SEX M 3 | |
| AVISITN*SEX F 6 | |
| AVISITN*SEX M 6 | |
| AVISITN*SEX F 10 | |

BREXPIPRAZOLE 29 OF 39


MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY SEX AT Phase B

| | Center | Combat | | | <b>D</b> 11 | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | | Analysis | Planned | |
| | Center) | Population | | Visit | Treatment | |
| Effect | for ITT | Flag | Sex | (N) | (N) | Row1 |
| AVISITN*SEX | | | М | 10 | | |
| | | | F | 12 | | |
| AVISITN*SEX | | | _ | | | |
| AVISITN*SEX | | | M | 12 | | |
| TRTPN*SEX | | | F | | 1 | |
| TRTPN*SEX | | | M | | 1 | |
| TRTPN*SEX | | | F | | 2 | 1 |
| TRTPN*SEX | | | M | | 2 | -1 |
| TRTPN*SEX | | | F | | 3 | |
| TRTPN*SEX | | | M | | 3 | |
| TRTPN*SEX | | | F | | 900 | -1 |
| TRTPN*SEX | | | M | | 900 | 1 |
| AVISITN*TRTPN*SEX | | | F | 3 | 1 | |
| AVISITN*TRTPN*SEX | | | M | 3 | 1 | |
| AVISITN*TRTPN*SEX | | | F | 3 | 2 | |
| AVISITN*TRTPN*SEX | | | M | 3 | 2 | |
| AVISITN*TRTPN*SEX | | | F | 3 | 3 | |
| AVISITN*TRTPN*SEX | | | M | 3 | 3 | |
| AVISITN*TRTPN*SEX | | | F | 3 | 900 | |

BREXPIPRAZOLE 30 OF 39 PROTOCOL 331-201-00061

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY SEX AT Phase B

| <b>-</b> 65 | (Pooled<br>Center) | Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | Sex | (N) | (N) | Row1 |
| AVISITN*TRTPN*SEX | | | М | 3 | 900 | |
| AVISITN*TRTPN*SEX | | | F | 6 | 1 | |
| AVISITN*TRTPN*SEX | | | M | 6 | 1 | |
| AVISITN*TRTPN*SEX | | | F | 6 | 2 | |
| AVISITN*TRTPN*SEX | | | M | 6 | 2 | |
| AVISITN*TRTPN*SEX | | | F | 6 | 3 | |
| AVISITN*TRTPN*SEX | | | M | 6 | 3 | |
| AVISITN*TRTPN*SEX | | | F | 6 | 900 | |
| AVISITN*TRTPN*SEX | | | M | 6 | 900 | |
| AVISITN*TRTPN*SEX | | | F | 10 | 1 | |
| AVISITN*TRTPN*SEX | | | M | 10 | 1 | |
| AVISITN*TRTPN*SEX | | | F | 10 | 2 | 1 |
| AVISITN*TRTPN*SEX | | | M | 10 | 2 | -1 |
| AVISITN*TRTPN*SEX | | | F | 10 | 3 | |
| AVISITN*TRTPN*SEX | | | M | 10 | 3 | |
| AVISITN*TRTPN*SEX | | | F | 10 | 900 | -1 |
| AVISITN*TRTPN*SEX | | | M | 10 | 900 | 1 |
| AVISITN*TRTPN*SEX | | | F | 12 | 1 | |

BREXPIPRAZOLE 31 OF 39 PROTOCOL 331-201-00061

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY SEX AT Phase B

Center Combat Center) Population for ITT Flor Analysis Planned Visit Treatment Effect (N) (N) Row1 AVISITN\*TRTPN\*SEX 12 AVISITN\*TRTPN\*SEX F 12 2 Μ 12 AVISITN\*TRTPN\*SEX AVISITN\*TRTPN\*SEX F 12 3 AVISITN\*TRTPN\*SEX Μ 12 .3 F 12 AVISITN\*TRTPN\*SEX 900 AVISITN\*TRTPN\*SEX M 12 900 BASE\*AVISITN 3 6 BASE\*AVISITN 10 BASE\*AVISITN 12 BASE\*AVISITN



FILE: stat2a.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.1 FINAL

BREXPIPRAZOLE 33 OF 39


MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY SEX AT Phase B

| | (Pooled<br>Center) | Combat<br>Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | Sex | (N) | (N) | Row1 |
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |

BREXPIPRAZOLE 34 OF 39 PROTOCOL 331-201-00061

STAT-3.

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY SEX AT Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | Sex | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 12 | 900 | |
| SEX | | | F | 12 | 900 | |
| SEX | | | M | | | |
| AVISITN*SEX | | | F | 3 | | |
| AVISITN*SEX | | | M | 3 | | |
| AVISITN*SEX | | | F | 6 | | |
| AVISITN*SEX | | | M | 6 | | |
| AVISITN*SEX | | | F | 10 | | |
| AVISITN*SEX | | | M | 10 | | |
| AVISITN*SEX | | | F | 12 | | |
| AVISITN*SEX | | | M | 12 | | |
| TRTPN*SEX | | | F | 12 | 1 | |
| TRTPN*SEX | | | M | | 1 | |
| TRTPN*SEX | | | F | | 2 | |
| TRTPN*SEX | | | M | | 2 | |
| TRTPN*SEX | | | F | | 3 | 1 |
| TRTPN*SEX | | | M | | 3 | -1 |
| TRTPN*SEX<br>TRTPN*SEX | | | F F | | 900 | -1<br>-1 |
| TKILN OFY | | | £ | | 900 | -1 |

BREXPIPRAZOLE 35 OF 39 PROTOCOL 331-201-00061

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY SEX AT Phase B

| | Center | Combat | | | | |
|-------------------|---------|------------|-----|----------|-----------|------|
| | (Pooled | Related | | Analysis | Planned | |
| | Center) | Population | | Visit | Treatment | |
| Effect | for ITT | Flag | Sex | (N) | (N) | Row1 |
| TRTPN*SEX | | | М | | 900 | 1 |
| AVISITN*TRTPN*SEX | | | F | 3 | 1 | |
| AVISITN*TRTPN*SEX | | | M | 3 | 1 | |
| AVISITN*TRTPN*SEX | | | F | 3 | 2 | |
| AVISITN*TRTPN*SEX | | | M | 3 | 2 | |
| AVISITN*TRTPN*SEX | | | F | 3 | 3 | |
| AVISITN*TRTPN*SEX | | | M | 3 | 3 | |
| AVISITN*TRTPN*SEX | | | F | 3 | 900 | |
| AVISITN*TRTPN*SEX | | | M | 3 | 900 | |
| AVISITN*TRTPN*SEX | | | F | 6 | 1 | |
| AVISITN*TRTPN*SEX | | | M | 6 | 1 | |
| AVISITN*TRTPN*SEX | | | F | 6 | 2 | |
| AVISITN*TRTPN*SEX | | | M | 6 | 2 | |
| AVISITN*TRTPN*SEX | | | F | 6 | 3 | |
| AVISITN*TRTPN*SEX | | | M | 6 | 3 | |
| AVISITN*TRTPN*SEX | | | F | 6 | 900 | |
| AVISITN*TRTPN*SEX | | | M | 6 | 900 | |
| AVISITN*TRTPN*SEX | | | F | 10 | 1 | |

BREXPIPRAZOLE 36 OF 39 PROTOCOL 331-201-00061

STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY SEX AT Phase B

| | Center | Combat | | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | | Analysis | Planned | |
| | Center) | Population | | Visit | Treatment | |
| Effect | for ITT | Flag | Sex | (N) | (N) | Row1 |
| AVISITN*TRTPN*SEX | | | M | 10 | 1 | |
| AVISITN*TRTPN*SEX | | | F | 10 | 2 | |
| AVISITN*TRTPN*SEX | | | M | 10 | 2 | |
| AVISITN*TRTPN*SEX | | | F | 10 | 3 | 1 |
| AVISITN*TRTPN*SEX | | | M | 10 | 3 | -1 |
| AVISITN*TRTPN*SEX | | | F | 10 | 900 | -1 |
| AVISITN*TRTPN*SEX | | | M | 10 | 900 | 1 |
| AVISITN*TRTPN*SEX | | | F | 12 | 1 | |
| AVISITN*TRTPN*SEX | | | M | 12 | 1 | |
| AVISITN*TRTPN*SEX | | | F | 12 | 2 | |
| AVISITN*TRTPN*SEX | | | M | 12 | 2 | |
| AVISITN*TRTPN*SEX | | | F | 12 | 3 | |
| AVISITN*TRTPN*SEX | | | M | 12 | 3 | |
| AVISITN*TRTPN*SEX | | | F | 12 | 900 | |
| AVISITN*TRTPN*SEX | | | M | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |

BREXPIPRAZOLE 37 OF 39 PROTOCOL 331-201-00061 STAT-3.1 MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy Y vs. Dummy Z BY SEX AT Phase B Center Combat Center) Population for ITT Fice (Pooled Related Analysis Planned Visit Treatment Effect for ITT Flag Sex (N) (N) Row1 BASE\*AVISITN 12 Estimates Standard Label Estimate Error DF t Value Pr > |t|3.9228 Dummy W vs. Dummy Z BY SEX AT Phase B -2.1308 237 -0.54 0.5875 -1.03 Dummy W vs. Dummy Y BY SEX AT Phase B -4.2187 4.0938 238 0.3038 Dummy W vs. Dummy X BY SEX AT Phase B -3.2445 4.2280 243 -0.77 0.4436

1.1137

2.0878

4.1553 241

238

4.0160

0.27 0.7889

0.6036

0.52

FILE: stat2a.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.1 FINAL

Dummy X vs. Dummy Z BY SEX AT Phase B

Dummy Y vs. Dummy Z BY SEX AT Phase B

BREXPIPRAZOLE 38 OF 39 PROTOCOL 331-201-00061

## STAT-3.1



-----

The Mixed Procedure

Least Squares Means

| | | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | Sex | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN*SEX | F | 3 | 1 | -6.7889 | 1.4561 | 289 | -4.66 | <.0001 | 0.05 | -9.6548 | -3.9231 |
| AVISITN*TRTPN*SEX | M | 3 | 1 | -5.9658 | 1.6705 | 281 | -3.57 | 0.0004 | 0.05 | -9.2540 | -2.6776 |
| AVISITN*TRTPN*SEX | F | 3 | 2 | -3.5409 | 1.4928 | 291 | -2.37 | 0.0183 | 0.05 | -6.4789 | -0.6028 |
| AVISITN*TRTPN*SEX | M | 3 | 2 | -6.7014 | 1.8949 | 279 | -3.54 | 0.0005 | 0.05 | -10.4315 | -2.9712 |
| AVISITN*TRTPN*SEX | F | 3 | 3 | -5.8264 | 1.4309 | 285 | -4.07 | <.0001 | 0.05 | -8.6430 | -3.0099 |
| AVISITN*TRTPN*SEX | M | 3 | 3 | -6.9685 | 1.7744 | 280 | -3.93 | 0.0001 | 0.05 | -10.4614 | -3.4756 |
| AVISITN*TRTPN*SEX | F | 3 | 900 | -6.9522 | 1.4980 | 288 | -4.64 | <.0001 | 0.05 | -9.9007 | -4.0038 |
| AVISITN*TRTPN*SEX | M | 3 | 900 | -5.2610 | 1.5640 | 275 | -3.36 | 0.0009 | 0.05 | -8.3399 | -2.1820 |
| AVISITN*TRTPN*SEX | F | 6 | 1 | -12.3592 | 1.7951 | 299 | -6.89 | <.0001 | 0.05 | -15.8918 | -8.8267 |
| AVISITN*TRTPN*SEX | M | 6 | 1 | -12.8657 | 2.0178 | 254 | -6.38 | <.0001 | 0.05 | -16.8393 | -8.8920 |
| AVISITN*TRTPN*SEX | F | 6 | 2 | -7.2561 | 1.7864 | 299 | -4.06 | <.0001 | 0.05 | -10.7716 | -3.7405 |
| AVISITN*TRTPN*SEX | M | 6 | 2 | -9.3923 | 2.3864 | 269 | -3.94 | 0.0001 | 0.05 | -14.0908 | -4.6939 |
| AVISITN*TRTPN*SEX | F | 6 | 3 | -10.5404 | 1.7494 | 297 | -6.03 | <.0001 | 0.05 | -13.9832 | -7.0977 |
| AVISITN*TRTPN*SEX | M | 6 | 3 | -8.1657 | 2.2259 | 270 | -3.67 | 0.0003 | 0.05 | -12.5479 | -3.7834 |
| AVISITN*TRTPN*SEX | F | 6 | 900 | -9.8078 | 1.7951 | 296 | -5.46 | <.0001 | 0.05 | -13.3405 | -6.2750 |
| AVISITN*TRTPN*SEX | M | 6 | 900 | -7.6519 | 1.9070 | 253 | -4.01 | <.0001 | 0.05 | -11.4076 | -3.8962 |
| AVISITN*TRTPN*SEX | F | 10 | 1 | -18.0953 | 1.8948 | 262 | -9.55 | <.0001 | 0.05 | -21.8262 | -14.3644 |
| AVISITN*TRTPN*SEX | M | 10 | 1 | -14.0253 | 2.1856 | 238 | -6.42 | <.0001 | 0.05 | -18.3309 | -9.7197 |
| AVISITN*TRTPN*SEX | F | 10 | 2 | -12.5259 | 1.9553 | 288 | -6.41 | <.0001 | 0.05 | -16.3744 | -8.6774 |

BREXPIPRAZOLE 39 OF 39 PROTOCOL 331-201-00061

## STAT-3.1

MMRM Output for Test on Treatment by Gender Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Least Squares Means

| | | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | Sex | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN*SEX | М | 10 | 2 | -11.7004 | 2.5767 | 246 | -4.54 | <.0001 | 0.05 | -16.7755 | -6.6253 |
| AVISITN*TRTPN*SEX | F | 10 | 3 | -11.3659 | 1.8419 | 261 | -6.17 | <.0001 | 0.05 | -14.9927 | -7.7391 |
| AVISITN*TRTPN*SEX | M | 10 | 3 | -11.5145 | 2.4232 | 248 | -4.75 | <.0001 | 0.05 | -16.2872 | -6.7419 |
| AVISITN*TRTPN*SEX | F | 10 | 900 | -11.3087 | 1.9194 | 275 | -5.89 | <.0001 | 0.05 | -15.0874 | -7.5300 |
| AVISITN*TRTPN*SEX | M | 10 | 900 | -9.3695 | 2.0402 | 232 | -4.59 | <.0001 | 0.05 | -13.3893 | -5.3498 |
| AVISITN*TRTPN*SEX | F | 12 | 1 | -17.5671 | 2.0876 | 271 | -8.41 | <.0001 | 0.05 | -21.6771 | -13.4570 |
| AVISITN*TRTPN*SEX | M | 12 | 1 | -16.8320 | 2.4007 | 238 | -7.01 | <.0001 | 0.05 | -21.5613 | -12.1026 |
| AVISITN*TRTPN*SEX | F | 12 | 2 | -11.4103 | 2.1389 | 287 | -5.33 | <.0001 | 0.05 | -15.6203 | -7.2003 |
| AVISITN*TRTPN*SEX | M | 12 | 2 | -13.9162 | 2.8294 | 246 | -4.92 | <.0001 | 0.05 | -19.4891 | -8.3432 |
| AVISITN*TRTPN*SEX | F | 12 | 3 | -14.9148 | 2.0092 | 267 | -7.42 | <.0001 | 0.05 | -18.8708 | -10.9589 |
| AVISITN*TRTPN*SEX | M | 12 | 3 | -14.9628 | 2.6369 | 243 | -5.67 | <.0001 | 0.05 | -20.1570 | -9.7687 |
| AVISITN*TRTPN*SEX | F | 12 | 900 | -11.1977 | 2.0889 | 275 | -5.36 | <.0001 | 0.05 | -15.3099 | -7.0854 |
| AVISITN*TRTPN*SEX | M | 12 | 900 | -12.2024 | 2.2546 | 238 | -5.41 | <.0001 | 0.05 | -16.6440 | -7.7609 |

BREXPIPRAZOLE 1 OF 39

STAT-3.2

MMRM Output for Test on Treatment by Race Interaction
(Intent to Treat Sample)

The Mixed Procedure

Model Information

Data Set WORK.INDATA
Dependent Variable CHG
Covariance Structure Unstructured
Subject Effect SUBJID
Estimation Method REML
Residual Variance Method None

Fixed Effects SE Method Kenward-Roger Degrees of Freedom Method Kenward-Roger

Class Level Information

| Class | Levels | Values |
|-------------------|---------|-----------|
| AVISITN | 4 | 3 6 10 12 |
| TRTPN<br>POOLCNTR | 4<br>10 | 1 2 3 900 |
| COMBFL | 2 | N Y |

FILE: stat2b.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.2 FINAL

BREXPIPRAZOLE 3 OF 39

STAT-3.2

MMRM Output for Test on Treatment by Race Interaction

(Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure



FILE: stat2b.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.2 FINAL

BREXPIPRAZOLE

STAT-3.2

MMRM Output for Test on Treatment by Race Interaction
(Intent to Treat Sample)

------

The Mixed Procedure



FILE: stat2b.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.2 FINAL

BREXPIPRAZOLE 5 OF 39
STAT-3.2

MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample)

The Mixed Procedure



FILE: stat2b.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.2 FINAL

BREXPIPRAZOLE 6 OF 39 PROTOCOL 331-201-00061 STAT-3.2 MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample) The Mixed Procedure RACEGRP All Other Races White Dimensions Covariance Parameters 10 Columns in X 91 Columns in Z 0 299 Subjects Max Obs per Subject Number of Observations Number of Observations Read 996
Number of Observations Used 996
7 01 -- wattions Not Used 0

FILE: stat2b.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.2 FINAL

BREXPIPRAZOLE 7 OF 39

MMRM Output for Test on Treatment by Race Interaction
(Intent to Treat Sample)

.....

The Mixed Procedure

Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 7344.39769030 | |
| 1 | 2 | 6876.20343728 | 0.00090786 |
| 2 | 1 | 6873.54971090 | 0.00005851 |
| 3 | 1 | 6873.39279538 | 0.0000031 |
| 4 | 1 | 6873.39198966 | 0.00000000 |

Convergence criteria met.

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | 77.5638 |
| UN(2,1) | SUBJID | 52.8666 |
| UN(2,2) | SUBJID | 114.95 |
| UN(3,1) | SUBJID | 42.8865 |
| UN(3,2) | SUBJID | 90.0751 |
| UN(3,3) | SUBJID | 124.37 |
| UN(4,1) | SUBJID | 48.8023 |

BREXPIPRAZOLE 8 OF 39

MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN (4,2) | SUBJID | 91.3636 |
| UN (4,3) | SUBJID | 106.14 |
| UN (4,4) | SUBJID | 149.07 |

Fit Statistics

| -2 Res Log Likelihood | 6873.4 |
|--------------------------|--------|
| AIC (Smaller is Better) | 6893.4 |
| AICC (Smaller is Better) | 6893.6 |
| BIC (Smaller is Better) | 6930.4 |

Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSc |
|----|------------|------------|
| 9 | 471.01 | < .0001 |

BREXPIPRAZOLE 9 OF 39

STAT-3.2

MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|----------------------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| POOLCNTR | 9 | 276 | 1.43 | 0.1759 |
| COMBFL | 1 | 277 | 3.87 | 0.0502 |
| AVISITN | 3 | 226 | 0.80 | 0.4937 |
| TRTPN | 3 | 262 | 2.12 | 0.0978 |
| AVISITN*TRTPN | 9 | 359 | 2.07 | 0.0315 |
| RACEGRP | 1 | 270 | 0.15 | 0.6951 |
| AVISITN*RACEGRP | 3 | 234 | 0.61 | 0.6066 |
| TRTPN*RACEGRP | 3 | 262 | 0.48 | 0.6967 |
| AVISIT*TRTPN*RACEGRP | 9 | 359 | 0.70 | 0.7068 |
| BASE*AVISITN | 4 | 237 | 14.95 | <.0001 |



FILE: stat2b.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.2 FINAL


STAT-3.2

Combat

Center

MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY RACEGRP AT Phase B Week 10

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | RACEGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |

FILE: stat2b.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.2 FINAL


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction

Combat

Center

(Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY RACEGRP AT Phase B Week 10

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | RACEGRP | | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | | 12 | 900 | |
| RACEGRP | | | All Other Ra | aces | | | |
| RACEGRP | | | White | | | | |
| AVISITN*RACEGRP | | | All Other Ra | aces | 3 | | |
| AVISITN*RACEGRP | | | White | | 3 | | |
| AVISITN*RACEGRP | | | All Other Ra | aces | 6 | | |
| AVISITN*RACEGRP | | | White | | 6 | | |
| AVISITN*RACEGRP | | | All Other Ra | aces | 10 | | |
| AVISITN*RACEGRP | | | White | | 10 | | |
| AVISITN*RACEGRP | | | All Other Ra | aces | 12 | | |
| AVISITN*RACEGRP | | | White | | 12 | | |
| TRTPN*RACEGRP | | | All Other Ra | aces | | 1 | 1 |
| TRTPN*RACEGRP | | | White | | | 1 | -1 |
| TRTPN*RACEGRP | | | All Other Ra | aces | | 2 | |
| TRTPN*RACEGRP | | | White | | | 2 | |
| TRTPN*RACEGRP | | | All Other Ra | aces | | 3 | |
| TRTPN*RACEGRP | | | White | | | 3 | |
| TRTPN*RACEGRP | | | All Other Ra | aces | | 900 | -1 |


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY RACEGRP AT Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | RACEGRP | Analysis<br>Visit<br>(N) | | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*RACEGRP | | | White | | 900 | 1 |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 3 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | White | 3 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 3 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | White | 3 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 3 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | White | 3 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 3 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | White | 3 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 6 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | White | 6 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 6 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | White | 6 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 6 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | White | 6 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 6 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | White | 6 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 10 | 1 | 1 |


MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY RACEGRP AT Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | RACEGRP | Analysis<br>Visit<br>(N) | | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*RACEGRP | | | White | 10 | 1 | -1 |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 10 | 2 | - |
| AVISIT*TRTPN*RACEGRP | | | White | 10 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 10 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | White | 10 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 10 | 900 | -1 |
| AVISIT*TRTPN*RACEGRP | | | White | 10 | 900 | 1 |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 12 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | White | 12 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 12 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | White | 12 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 12 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | White | 12 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 12 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | White | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |



FILE: stat2b.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.2 FINAL

BREXPIPRAZOLE 16 OF 39 PROTOCOL 331-201-00061 STAT-3.2 MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy W vs. Dummy Y BY RACEGRP AT Phase B Center Combat (Pooled Related Analysis Planned Center) Population Visit Treatment Effect for ITT Flag RACEGRP (N) (N) Row1 POOLCNTR POOLCNTR POOLCNTR COMBFL Ν COMBFL Y 3 AVISITN AVISITN 6 AVISITN 10 AVISITN 12 1 TRTPN 2 TRTPN 3 TRTPN 900 TRTPN AVISITN\*TRTPN 3 1 AVISITN\*TRTPN 3 2 AVISITN\*TRTPN 3 3 AVISITN\*TRTPN 3 900 AVISITN\*TRTPN 6 1

FILE: stat2b.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.2 FINAL

MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY RACEGRP AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | RACEGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 6<br>6<br>6<br>10<br>10<br>10<br>10<br>12<br>12<br>12 | 2<br>3<br>900<br>1<br>2<br>3<br>900<br>1<br>2<br>3 | |
| AVISITN*TRTPN RACEGRP RACEGRP AVISITN*RACEGRP AVISITN*RACEGRP AVISITN*RACEGRP AVISITN*RACEGRP AVISITN*RACEGRP | | | All Other Races<br>White<br>All Other Races<br>White<br>All Other Races<br>White<br>All Other Races | 3<br>3<br>6<br>6<br>10 | 900 | |

FILE: stat2b.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC STAT/stat2.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.2


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction

Combat

Center

t on Treatment by Race Interaction (Intent to Treat Sample)

------

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY RACEGRP AT Phase B

| Effect | Related<br>Population<br>Flag | RACEGRP | Analysis<br>Visit<br>(N) | | Row1 |
|---|---|---|---|---|---|
| AVISITN*RACEGRP | | White | 10 | | |
| AVISITN*RACEGRP | | All Other Race | s 12 | | |
| AVISITN*RACEGRP | | White | 12 | | |
| TRTPN*RACEGRP | | All Other Race | S | 1 | 1 |
| TRTPN*RACEGRP | | White | | 1 | -1 |
| TRTPN*RACEGRP | | All Other Race | S | 2 | |
| TRTPN*RACEGRP | | White | | 2 | |
| TRTPN*RACEGRP | | All Other Race | S | 3 | -1 |
| TRTPN*RACEGRP | | White | | 3 | 1 |
| TRTPN*RACEGRP | | All Other Race | S | 900 | |
| TRTPN*RACEGRP | | White | | 900 | |
| AVISIT*TRTPN*RACEGRP | | All Other Race | s 3 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | 3 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Race | s 3 | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | 3 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Race | | 3 | |
| AVISIT*TRTPN*RACEGRP | | White | 3 | 3 | |
| AVISIT*TRTPN*RACEGRP | | All Other Race | s 3 | 900 | |


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY RACEGRP AT Phase B

| Center<br>(Pooled | Combat<br>Related | | Analysis | Planned | | |
|---|---|---|---|---|---|---|
| | Center) | Population | | Visit | | |
| Effect | for ITT | Flag | RACEGRP | (N) | (N) | Row1 |
| | | - | | | | |
| AVISIT*TRTPN*RACEGRP | | | White | 3 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 6 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | White | 6 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 6 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | White | 6 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 6 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | White | 6 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 6 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | White | 6 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 10 | 1 | 1 |
| AVISIT*TRTPN*RACEGRP | | | White | 10 | 1 | -1 |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 10 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | White | 10 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 10 | 3 | -1 |
| AVISIT*TRTPN*RACEGRP | | | White | 10 | 3 | 1 |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 10 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | White | 10 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 12 | 1 | |


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY RACEGRP AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | RACEGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*RACEGRP | | | White | 12 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 12 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | White | 12 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 12 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | White | 12 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 12 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | White | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |
| BASE*AVISITN | | | | 12 | | |



FILE: stat2b.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.2 FINAL


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample)

Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY RACEGRP AT Phase B

| | Center<br>(Pooled | Combat<br>Related | | Analysis | Planned | |
|---|---|---|---|---|---|---|
| | Center) | Population | | Visit | Treatment | |
| Effect | for ITT | Flag | RACEGRP | (N) | (N) | Row1 |
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| | | | | | - | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |

BREXPIPRAZOLE 23 OF 39

Center

Combat

STAT-3.2

MMRM Output for Test on Treatment by Race Interaction
(Intent to Treat Sample)

Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY RACEGRP AT Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | RACEGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 12 | 900 | |
| RACEGRP | | | All Other Race | es | | |
| RACEGRP | | | White | | | |
| AVISITN*RACEGRP | | | All Other Race | es 3 | | |
| AVISITN*RACEGRP | | | White | 3 | | |
| AVISITN*RACEGRP | | | All Other Race | es 6 | | |
| AVISITN*RACEGRP | | | White | 6 | | |
| AVISITN*RACEGRP | | | All Other Race | es 10 | | |
| AVISITN*RACEGRP | | | White | 10 | | |
| AVISITN*RACEGRP | | | All Other Race | es 12 | | |
| AVISITN*RACEGRP | | | White | 12 | | |
| TRTPN*RACEGRP | | | All Other Race | es | 1 | 1 |
| TRTPN*RACEGRP | | | White | | 1 | -1 |
| TRTPN*RACEGRP | | | All Other Race | es | 2 | -1 |
| TRTPN*RACEGRP | | | White | | 2 | 1 |
| TRTPN*RACEGRP | | | All Other Race | es | 3 | |
| TRTPN*RACEGRP | | | White | | 3 | |
| TRTPN*RACEGRP | | | All Other Race | es | 900 | |

BREXPIPRAZOLE 24 OF 39 PROTOCOL 331-201-00061

STAT-3.2

MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample)



The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY RACEGRP AT Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | RACEGRP | Analysis<br>Visit<br>(N) | | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*RACEGRP | | | White | | 900 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 3 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | White | 3 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 3 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | White | 3 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 3 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | White | 3 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 3 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | White | 3 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 6 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | White | 6 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 6 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | White | 6 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 6 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | White | 6 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 6 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | White | 6 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 10 | 1 | 1 |


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY RACEGRP AT Phase B

| | Center<br>(Pooled | Combat<br>Related | | Analusia | Planned | |
|---|---|---|---|---|---|---|
| | | Population | | Analysis<br>Visit | Treatment | |
| | Center) | * | | | | |
| Effect | for ITT | Flag | RACEGRP | (N) | (N) | Row1 |
| AVISIT*TRTPN*RACEGRP | | | White | 10 | 1 | -1 |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 10 | 2 | -1 |
| AVISIT*TRTPN*RACEGRP | | | White | 10 | 2 | 1 |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 10 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | White | 10 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 10 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | White | 10 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 12 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | White | 12 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 12 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | White | 12 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 12 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | White | 12 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 12 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | White | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |



FILE: stat2b.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.2 FINAL

BREXPIPRAZOLE 27 OF 39 PROTOCOL 331-201-00061 STAT-3.2 MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy X vs. Dummy Z BY RACEGRP AT Phase B Center Combat (Pooled Related Analysis Planned Center) Population Visit Treatment Effect for ITT Flag RACEGRP (N) (N) Row1 POOLCNTR POOLCNTR POOLCNTR COMBFL Ν COMBFL Υ 3 AVISITN AVISITN 6 AVISITN 10 AVISITN 12 1 TRTPN 2 TRTPN 3 TRTPN 900 TRTPN AVISITN\*TRTPN 3 1 AVISITN\*TRTPN 3 2 AVISITN\*TRTPN 3 3

FILE: stat2b.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.2 FINAL

AVISITN\*TRTPN

AVISITN\*TRTPN

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.

3

6

900

1


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample)

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY RACEGRP AT Phase B

| | Center<br>(Pooled<br>Center) | Combat<br>Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | RACEGRP | (N) | (N) | Row1 |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |
| AVISITN*TRTPN | | | | 12 | 900 | |
| RACEGRP | | | All Other Races | | | |
| RACEGRP | | | White | | | |
| AVISITN*RACEGRP | | | All Other Races | 3 | | |
| AVISITN*RACEGRP | | | White | 3 | | |
| AVISITN*RACEGRP | | | All Other Races | 6 | | |
| AVISITN*RACEGRP | | | White | 6 | | |
| AVISITN*RACEGRP | | | All Other Races | 10 | | |

BREXPIPRAZOLE 29 OF 39 PROTOCOL 331-201-00061

MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY RACEGRP AT Phase B

| Effect | <br>Combat<br>Related<br>Population<br>Flag | RACEGRP | | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*RACEGRP | | White | | 10 | | |
| AVISITN*RACEGRP | | All Other R | aces | 12 | | |
| AVISITN*RACEGRP | | White | | 12 | | |
| TRTPN*RACEGRP | | All Other R | .aces | | 1 | |
| TRTPN*RACEGRP | | White | | | 1 | |
| TRTPN*RACEGRP | | All Other R | aces | | 2 | 1 |
| TRTPN*RACEGRP | | White | | | 2 | -1 |
| TRTPN*RACEGRP | | All Other R | aces | | 3 | |
| TRTPN*RACEGRP | | White | | | 3 | |
| TRTPN*RACEGRP | | All Other R | aces | | 900 | -1 |
| TRTPN*RACEGRP | | White | | | 900 | 1 |
| AVISIT*TRTPN*RACEGRP | | All Other R | aces | 3 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | | 3 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other R | aces | 3 | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | | 3 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other R | aces | 3 | 3 | |
| AVISIT*TRTPN*RACEGRP | | White | | 3 | 3 | |
| AVISIT*TRTPN*RACEGRP | | All Other R | aces. | 3 | 900 | |


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction
(Intent to Treat Sample)

Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY RACEGRP AT Phase B

| (Pooled Related Center) Population Effect for ITT Flag RACEGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|
| AVISIT*TRTPN*RACEGRP White | 3 | 900 | |
| AVISIT*TRTPN*RACEGRP All Other Races | 6 | 1 | |
| AVISIT*TRTPN*RACEGRP White | 6 | 1 | |
| AVISIT*TRTPN*RACEGRP All Other Races | 6 | 2 | |
| AVISIT*TRTPN*RACEGRP White | 6 | 2 | |
| AVISIT*TRTPN*RACEGRP All Other Races | 6 | 3 | |
| AVISIT*TRTPN*RACEGRP White | 6 | 3 | |
| AVISIT*TRTPN*RACEGRP All Other Races | 6 | 900 | |
| AVISIT*TRTPN*RACEGRP White | 6 | 900 | |
| AVISIT*TRTPN*RACEGRP All Other Races | 10 | 1 | |
| AVISIT*TRTPN*RACEGRP White | 10 | 1 | |
| AVISIT*TRTPN*RACEGRP All Other Races | 10 | 2 | 1 |
| AVISIT*TRTPN*RACEGRP White | 10 | 2 | -1 |
| AVISIT*TRTPN*RACEGRP All Other Races | 10 | 3 | |
| AVISIT*TRTPN*RACEGRP White | 10 | 3 | |
| AVISIT*TRTPN*RACEGRP All Other Races | 10 | 900 | -1 |
| AVISIT*TRTPN*RACEGRP White | 10 | 900 | 1 |
| AVISIT*TRTPN*RACEGRP All Other Races | 12 | 1 | |


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample)

------ Parameter Code=CAPSTOT -------

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY RACEGRP AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | RACEGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*RACEGRP | | | White | 12 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 12 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | White | 12 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 12 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | White | 12 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 12 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | White | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |
| BASE*AVISITN | | | | 12 | | |



FILE: stat2b.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.2 FINAL

BREXPIPRAZOLE 33 OF 39 PROTOCOL 331-201-00061

STAT-3.2

MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY RACEGRP AT Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | RACEGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |


MMRM Output for Test on Treatment by Race Interaction

(Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY RACEGRP AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Population | RACEGRP | Analysis<br>Visit<br>(N) | | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 12 | 900 | |
| RACEGRP | | | All Other Races | | | |
| RACEGRP | | | White | | | |
| AVISITN*RACEGRP | | | All Other Races | 3 | | |
| AVISITN*RACEGRP | | | White | 3 | | |
| AVISITN*RACEGRP | | | All Other Races | 6 | | |
| AVISITN*RACEGRP | | | White | 6 | | |
| AVISITN*RACEGRP | | | All Other Races | 10 | | |
| AVISITN*RACEGRP | | | White | 10 | | |
| AVISITN*RACEGRP | | | All Other Races | 12 | | |
| AVISITN*RACEGRP | | | White | 12 | | |
| TRTPN*RACEGRP | | | All Other Races | | 1 | |
| TRTPN*RACEGRP | | | White | | 1 | |
| TRTPN*RACEGRP | | | All Other Races | | 2 | |
| TRTPN*RACEGRP | | | White | | 2 | |
| TRTPN*RACEGRP | | | All Other Races | | 3 | 1 |
| TRTPN*RACEGRP | | | White | | 3 | -1 |
| TRTPN*RACEGRP | | | All Other Races | | 900 | -1 |
| | | | | | | - |


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY RACEGRP AT Phase B

| Effect | • | Related<br>Population<br>Flag | RACEGRP | Analysis<br>Visit<br>(N) | | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*RACEGRP | | | White | | 900 | 1 |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 3 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | White | 3 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 3 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | White | 3 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 3 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | White | 3 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 3 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | White | 3 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 6 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | White | 6 | 1 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 6 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | White | 6 | 2 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 6 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | White | 6 | 3 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 6 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | White | 6 | 900 | |
| AVISIT*TRTPN*RACEGRP | | | All Other Races | 10 | 1 | |


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY RACEGRP AT Phase B

| Effect | Related<br>Population<br>Flag | RACEGRP | Analysis<br>Visit<br>(N) | | Row1 |
|---|---|---|---|---|---|
| AVISIT*TRTPN*RACEGRP | | White | 1.0 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 10 | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | 10 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 10 | 3 | 1 |
| AVISIT*TRTPN*RACEGRP | | White | 10 | 3 | -1 |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 10 | 900 | -1 |
| AVISIT*TRTPN*RACEGRP | | White | 10 | 900 | 1 |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 12 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | 12 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 12 | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | 12 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 12 | 3 | |
| AVISIT*TRTPN*RACEGRP | | White | 12 | 3 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 12 | 900 | |
| AVISIT*TRTPN*RACEGRP | | White | 12 | 900 | |
| BASE*AVISITN | | | 3 | | |
| BASE*AVISITN | | | 6 | | |
| BASE*AVISITN | | | 10 | | |

BREXPIPRAZOLE 37 OF 39 PROTOCOL 331-201-00061 STAT-3.2 MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy Y vs. Dummy Z BY RACEGRP AT Phase B Center Combat Planned (Pooled Related Analysis Center) Population Visit Treatment Effect for ITT Flag RACEGRP (N) (N) Row1 BASE\*AVISITN 12 Estimates Standard Label Estimate Error DF t Value Pr > |t| 3.9796 233 0.56 0.5758 Dummy W vs. Dummy Z BY RACEGRP AT Phase B 2.2296 Dummy W vs. Dummy Y BY RACEGRP AT Phase B 3.8513 4.1388 231 0.93 0.3531 6.0188 4.1825 239 1.44 0.1514 Dummy W vs. Dummy X BY RACEGRP AT Phase B Dummy X vs. Dummy Z BY RACEGRP AT Phase B -3.7892 4.0544 239 -0.93 0.3509 Dummy Y vs. Dummy Z BY RACEGRP AT Phase B -1.6217 4.0225 234 -0.40 0.6872


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Least Squares Means

| | | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Standard | | | | | | |
| ffect | RACEGRP | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| /ISIT*TRTPN*RACEGRP | All Other Races | 3 | 1 | -3.7243 | 1.7733 | 282 | -2.10 | 0.0366 | 0.05 | -7.2149 | -0.2336 |
| /ISIT*TRTPN*RACEGRP | White | 3 | 1 | -7.9456 | 1.3273 | 282 | -5.99 | <.0001 | 0.05 | -10.5584 | -5.3329 |
| /ISIT*TRTPN*RACEGRP | All Other Races | 3 | 2 | -5.4986 | 1.6869 | 282 | -3.26 | 0.0013 | 0.05 | -8.8192 | -2.1780 |
| /ISIT*TRTPN*RACEGRP | White | 3 | 2 | -3.7950 | 1.5221 | 284 | -2.49 | 0.0132 | 0.05 | -6.7910 | -0.7990 |
| /ISIT*TRTPN*RACEGRP | All Other Races | 3 | 3 | -4.8461 | 1.7959 | 277 | -2.70 | 0.0074 | 0.05 | -8.3814 | -1.3108 |
| /ISIT*TRTPN*RACEGRP | White | 3 | 3 | -6.9219 | 1.3452 | 281 | -5.15 | <.0001 | 0.05 | -9.5698 | -4.2739 |
| /ISIT*TRTPN*RACEGRP | All Other Races | 3 | 900 | -6.4012 | 1.5465 | 279 | -4.14 | <.0001 | 0.05 | -9.4456 | -3.3569 |
| /ISIT*TRTPN*RACEGRP | White | 3 | 900 | -6.0820 | 1.4324 | 280 | -4.25 | <.0001 | 0.05 | -8.9017 | -3.2623 |
| /ISIT*TRTPN*RACEGRP | All Other Races | 6 | 1 | -11.7027 | 2.1912 | 261 | -5.34 | <.0001 | 0.05 | -16.0174 | -7.3880 |
| /ISIT*TRTPN*RACEGRP | White | 6 | 1 | -13.0881 | 1.6668 | 276 | -7.85 | <.0001 | 0.05 | -16.3694 | -9.8068 |
| /ISIT*TRTPN*RACEGRP | All Other Races | 6 | 2 | -8.0389 | 2.1519 | 291 | -3.74 | 0.0002 | 0.05 | -12.2741 | -3.8037 |
| /ISIT*TRTPN*RACEGRP | White | 6 | 2 | -7.8701 | 1.8584 | 270 | -4.23 | <.0001 | 0.05 | -11.5289 | -4.2113 |
| /ISIT*TRTPN*RACEGRP | All Other Races | 6 | 3 | -8.9561 | 2.3820 | 296 | -3.76 | 0.0002 | 0.05 | -13.6438 | -4.2683 |
| /ISIT*TRTPN*RACEGRP | White | 6 | 3 | -9.9980 | 1.6551 | 269 | -6.04 | <.0001 | 0.05 | -13.2566 | -6.7394 |
| /ISIT*TRTPN*RACEGRP | All Other Races | 6 | 900 | -8.8865 | 1.9191 | 271 | -4.63 | <.0001 | 0.05 | -12.6648 | -5.1083 |
| /ISIT*TRTPN*RACEGRP | White | 6 | 900 | -8.9195 | 1.7485 | 261 | -5.10 | <.0001 | 0.05 | -12.3624 | -5.4765 |
| /ISIT*TRTPN*RACEGRP | All Other Races | 10 | 1 | -13.9790 | 2.3550 | 238 | -5.94 | <.0001 | 0.05 | -18.6184 | -9.3396 |
| /ISIT*TRTPN*RACEGRP | White | 10 | 1 | -17.7665 | 1.7633 | 241 | -10.08 | <.0001 | 0.05 | -21.2401 | -14.2930 |
| /ISIT*TRTPN*RACEGRP | All Other Races | 10 | 2 | -13.4589 | 2.3418 | 270 | -5.75 | <.0001 | 0.05 | -18.0693 | -8.8484 |
| | VISIT*TRTPN*RACEGRP | VISIT*TRTPN*RACEGRP White VISIT*TRTPN*RACEGRP All Other Races VISIT*TRTPN*RACEGRP White VISIT*TRTPN*RACEGRP All Other Races VISIT*TRTPN*RACEGRP All Other Races VISIT*TRTPN*RACEGRP White | Visit VISIT*TRTPN*RACEGRP All Other Races 3 VISIT*TRTPN*RACEGRP White 3 VISIT*TRTPN*RACEGRP All Other Races 3 VISIT*TRTPN*RACEGRP All Other Races 3 VISIT*TRTPN*RACEGRP White 6 VISIT*TRTPN*RACEGRP White 10 VISIT*TRTPN*RACEGRP White 10 VISIT*TRTPN*RACEGRP WHITE 10 VISIT*TRTPN*RACEGRP WHIT | Visit Treatment Visit Treatment Visit (N) (N) (N) VISIT*TRTPN*RACEGRP All Other Races 3 | Treatment | Visit Treatment Standard | Treatment Standard Color Color | Treatment Standard Color Color | Visit Treatment Standard Error DF t Value Pr > t Value Pr > t Value Pr > t Value Pr > t Value Pr > t Value Value | Treatment Standard From DF t Value Pr > t Alpha Alpha | Treatment Standard February Standard Standard February Standard Standard |


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction
(Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Least Squares Means

| <b>766</b> | | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | RACEGRP | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISIT*TRTPN*RACEGRP | White | 10 | 2 | -11.2275 | 2.0250 | 255 | -5.54 | <.0001 | 0.05 | -15.2154 | -7.2397 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 10 | 3 | -11.3492 | 2.4400 | 241 | -4.65 | <.0001 | 0.05 | -16.1556 | -6.5428 |
| AVISIT*TRTPN*RACEGRP | White | 10 | 3 | -11.2854 | 1.7825 | 247 | -6.33 | <.0001 | 0.05 | -14.7963 | -7.7745 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 10 | 900 | -9.6251 | 2.0179 | 241 | -4.77 | <.0001 | 0.05 | -13.6001 | -5.6502 |
| AVISIT*TRTPN*RACEGRP | White | 10 | 900 | -11.1830 | 1.8892 | 245 | -5.92 | <.0001 | 0.05 | -14.9041 | -7.4619 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 12 | 1 | -16.5991 | 2.6071 | 246 | -6.37 | <.0001 | 0.05 | -21.7342 | -11.4640 |
| AVISIT*TRTPN*RACEGRP | White | 12 | 1 | -17.6900 | 1.9430 | 247 | -9.10 | <.0001 | 0.05 | -21.5169 | -13.8631 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 12 | 2 | -12.6750 | 2.5704 | 269 | -4.93 | <.0001 | 0.05 | -17.7357 | -7.6143 |
| AVISIT*TRTPN*RACEGRP | White | 12 | 2 | -11.8728 | 2.2224 | 256 | -5.34 | <.0001 | 0.05 | -16.2493 | -7.4964 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 12 | 3 | -16.6030 | 2.6362 | 239 | -6.30 | <.0001 | 0.05 | -21.7962 | -11.4099 |
| AVISIT*TRTPN*RACEGRP | White | 12 | 3 | -13.8895 | 1.9603 | 251 | -7.09 | <.0001 | 0.05 | -17.7502 | -10.0289 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 12 | 900 | -11.6305 | 2.2073 | 246 | -5.27 | <.0001 | 0.05 | -15.9782 | -7.2829 |
| AVISIT*TRTPN*RACEGRP | White | 12 | 900 | -11.7595 | 2.0830 | 251 | -5.65 | <.0001 | 0.05 | -15.8618 | -7.6571 |

BREXPIPRAZOLE 1 OF 39

STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

.\_\_\_\_\_

The Mixed Procedure

Model Information

Data Set WORK.INDATA
Dependent Variable CHG
Covariance Structure Unstructured
Subject Effect SUBJID
Estimation Method REML
Residual Variance Method None

Fixed Effects SE Method Kenward-Roger
Degrees of Freedom Method Kenward-Roger

Class Level Information

BREXPIFRAZOLE


STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction
(Intent to Treat Sample)

The Mixed Procedure

Class Level Information

Class Levels Values

SUBJID 299

FILE: stat2c.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.3 FINAL

BREXPIPRAZOLE 3 OF 39

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

.\_\_\_\_\_

The Mixed Procedure



FILE: stat2c.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.3 FINAL

BREXPIPRAZOLE 4 OF 39

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

.\_\_\_\_\_

The Mixed Procedure



FILE: stat2c.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.3 FINAL

BREXPIPRAZOLE 5 OF 39

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

.\_\_\_\_\_

The Mixed Procedure



FILE: stat2c.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.3 FINAL

BREXPIPRAZOLE 6 OF 39 PROTOCOL 331-201-00061 STAT-3.3 MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample) The Mixed Procedure AGEGRP <55 >=55 Dimensions Covariance Parameters 10 Columns in X 91 Columns in Z 0 299 Subjects Max Obs per Subject Number of Observations 996 Number of Observations Read 996 Number of Observations Used Number of Observations Not Used

FILE: stat2c.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.3 FINAL

BREXPIPRAZOLE 7 OF 39

STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

The Mixed Procedure

Iteration History

| Criterion | -2 Res Log Like | Evaluations | Iteration |
|------------|-----------------|-------------|-----------|
| | 7335.56990357 | 1 | 0 |
| 0.00071726 | 6863.74324538 | 2 | 1 |
| 0.00071726 | 6861.67356308 | | 1 |
| | | 1 | 2 |
| 0.00000013 | 6861.57448148 | 1 | 3 |
| 0.00000000 | 6861.57415440 | 1 | 4 |

Convergence criteria  $\operatorname{met}$ .

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | 77.8543 |
| UN(2,1) | SUBJID | 53.5922 |
| UN(2,2) | SUBJID | 114.49 |
| UN(3,1) | SUBJID | 44.6224 |
| UN(3,2) | SUBJID | 90.7193 |
| UN(3,3) | SUBJID | 125.79 |
| UN(4,1) | SUBJID | 48.6619 |

BREXPIPRAZOLE 8 OF 39

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN (4,2) | SUBJID | 90.5499 |
| UN (4,3) | SUBJID | 105.79 |
| UN (4,4) | SUBJID | 147.93 |

Fit Statistics

| -2 Res Log Likelihood | 6861.6 |
|--------------------------|--------|
| AIC (Smaller is Better) | 6881.6 |
| AICC (Smaller is Better) | 6881.8 |
| BIC (Smaller is Better) | 6918.6 |

Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|----|------------|------------|
| 9 | 474.00 | < .0001 |

BREXPIPRAZOLE 9 OF 39

STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction

(Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|----------------------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| POOLCNTR | 9 | 277 | 1.61 | 0.1108 |
| COMBFL | 1 | 278 | 4.63 | 0.0323 |
| AVISITN | 3 | 228 | 0.28 | 0.8367 |
| TRTPN | 3 | 266 | 2.26 | 0.0821 |
| AVISITN*TRTPN | 9 | 358 | 1.29 | 0.2410 |
| AGEGRP | 1 | 271 | 0.19 | 0.6638 |
| AVISITN*AGEGRP | 3 | 235 | 1.16 | 0.3240 |
| TRTPN*AGEGRP | 3 | 265 | 0.98 | 0.4046 |
| AVISITN*TRTPN*AGEGRP | 9 | 359 | 0.73 | 0.6787 |
| BASE*AVISITN | 4 | 239 | 15.02 | <.0001 |



FILE: stat2c.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.3 FINAL


STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY AGEGRP AT Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | AGEGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |


STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction

(Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY AGEGRP AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | AGEGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 12 | 900 | |
| AGEGRP | | | <55 | | | |
| AGEGRP | | | >=55 | | | |
| AVISITN*AGEGRP | | | <55 | 3 | | |
| AVISITN*AGEGRP | | | >=55 | 3 | | |
| AVISITN*AGEGRP | | | <55 | 6 | | |
| AVISITN*AGEGRP | | | >=55 | 6 | | |
| AVISITN*AGEGRP | | | <55 | 10 | | |
| AVISITN*AGEGRP | | | >=55 | 10 | | |
| AVISITN*AGEGRP | | | <55 | 12 | | |
| AVISITN*AGEGRP | | | >=55 | 12 | | |
| TRTPN*AGEGRP | | | <55 | | 1 | 1 |
| TRTPN*AGEGRP | | | >=55 | | 1 | -1 |
| TRTPN*AGEGRP | | | <55 | | 2 | |
| TRTPN*AGEGRP | | | >=55 | | 2 | |
| TRTPN*AGEGRP | | | <55 | | 3 | |
| TRTPN*AGEGRP | | | >=55 | | 3 | |
| TRTPN*AGEGRP | | | <55 | | 900 | -1 |


STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

------

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY AGEGRP AT Phase B

| 755 | (Pooled<br>Center) | Combat<br>Related<br>Population | 10000 | Analysis<br>Visit | Treatment | D. 1 |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | AGEGRP | (N) | (N) | Row1 |
| TRTPN*AGEGRP | | | >=55 | | 900 | 1 |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 1 | 1 |

STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY AGEGRP AT Phase B

| | Center<br>(Pooled<br>Center) | Combat<br>Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | AGEGRP | (N) | (N) | Row1 |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 1 | -1 |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 900 | -1 |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 900 | 1 |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |



BREXPIPRAZOLE 16 OF 39 PROTOCOL 331-201-00061 STAT-3.3 MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy W vs. Dummy Y BY AGEGRP AT Phase B Center Combat Population Analysis Planned (Pooled Related Visit Center) Treatment Effect for ITT Flag AGEGRP (N) (N) Row1 POOLCNTR POOLCNTR POOLCNTR COMBFL Ν COMBFL Υ 3 AVISITN AVISITN 6 AVISITN 10 AVISITN 12 1 TRTPN 2 TRTPN 3 TRTPN 900 TRTPN AVISITN\*TRTPN 3 1 AVISITN\*TRTPN 3 2 AVISITN\*TRTPN 3

FILE: stat2c.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.3 FINAL

AVISITN\*TRTPN

AVISITN\*TRTPN

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.

3

900

1


STAT-3.

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY AGEGRP AT Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | AGEGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| FITECL | 101 111 | riay | AGEGRP | ( IN ) | (14) | KOMI |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |
| AVISITN*TRTPN | | | | 12 | 900 | |
| AGEGRP | | | <55 | | | |
| AGEGRP | | | >=55 | | | |
| AVISITN*AGEGRP | | | <55 | 3 | | |
| AVISITN*AGEGRP | | | >=55 | 3 | | |
| AVISITN*AGEGRP | | | <55 | 6 | | |
| AVISITN*AGEGRP | | | >=55 | 6 | | |
| AVISITN*AGEGRP | | | <55 | 10 | | |


STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY AGEGRP AT Phase B

| | Center<br>(Pooled<br>Center) | Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | AGEGRP | (N) | (N) | Row1 |
| AVISITN*AGEGRP | | | >=55 | 10 | | |
| AVISITN*AGEGRP | | | <55 | 12 | | |
| AVISITN*AGEGRP | | | >=55 | 12 | | |
| TRTPN*AGEGRP | | | <55 | | 1 | 1 |
| TRTPN*AGEGRP | | | >=55 | | 1 | -1 |
| TRTPN*AGEGRP | | | <55 | | 2 | |
| TRTPN*AGEGRP | | | >=55 | | 2 | |
| TRTPN*AGEGRP | | | <55 | | 3 | -1 |
| TRTPN*AGEGRP | | | >=55 | | 3 | 1 |
| TRTPN*AGEGRP | | | <55 | | 900 | |
| TRTPN*AGEGRP | | | >=55 | | 900 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 900 | |


STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

------

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY AGEGRP AT Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | AGEGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| Effect | 101 111 | riag | AGEGILI | (14) | (14) | NOWI |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 1 | 1 |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 1 | -1 |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 3 | -1 |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 3 | 1 |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 1 | |


STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY AGEGRP AT Phase B

| | Center<br>(Pooled<br>Center) | Combat<br>Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | AGEGRP | (N) | (N) | Row1 |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |
| BASE*AVISITN | | | | 12 | | |




STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

.------

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY AGEGRP AT Phase B

| Dec | Center<br>(Pooled<br>Center)<br>for ITT | Related<br>Population | ACHCDD | Analysis<br>Visit | Planned<br>Treatment | D1 |
|---|---|---|---|---|---|---|
| Effect | ior itt | Flag | AGEGRP | (N) | (N) | Row1 |
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |


STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY AGEGRP AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | AGEGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 12 | 900 | |
| AVISIIN"IRIPN<br>AGEGRP | | | <55 | 12 | 900 | |
| AGEGRP | | | >=55 | 2 | | |
| AVISITN*AGEGRP | | | <55 | 3 | | |
| AVISITN*AGEGRP | | | >=55 | 3 | | |
| AVISITN*AGEGRP | | | <55 | 6 | | |
| AVISITN*AGEGRP | | | >=55 | 6 | | |
| AVISITN*AGEGRP | | | <55 | 10 | | |
| AVISITN*AGEGRP | | | >=55 | 10 | | |
| AVISITN*AGEGRP | | | <55 | 12 | | |
| AVISITN*AGEGRP | | | >=55 | 12 | | |
| TRTPN*AGEGRP | | | <55 | | 1 | 1 |
| TRTPN*AGEGRP | | | >=55 | | 1 | -1 |
| TRTPN*AGEGRP | | | <55 | | 2 | -1 |
| TRTPN*AGEGRP | | | >=55 | | 2 | 1 |
| TRTPN*AGEGRP | | | <55 | | 3 | |
| TRTPN*AGEGRP | | | >=55 | | 3 | |
| TRTPN*AGEGRP | | | <55 | | 900 | |


STAT-3.

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

------

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY AGEGRP AT Phase B

| | Center<br>(Pooled<br>Center) | Combat<br>Related<br>Population | | Analysis<br>Visit | Treatment | |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | AGEGRP | (N) | (N) | Row1 |
| TRTPN*AGEGRP | | | >=55 | | 900 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 1 | 1 |


STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

\_\_\_\_\_

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY AGEGRP AT Phase B

| | Center<br>(Pooled<br>Center) | Combat<br>Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|
| Effect | for ITT | | AGEGRP | (N) | (N) | Row1 |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 1 | -1 |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 2 | -1 |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 2 | 1 |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |



BREXPIPRAZOLE 27 OF 39 PROTOCOL 331-201-00061 STAT-3.3 MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy X vs. Dummy Z BY AGEGRP AT Phase B Center Combat Population Analysis Planned (Pooled Related Visit Center) Treatment Effect for ITT Flag AGEGRP (N) (N) Row1 POOLCNTR POOLCNTR POOLCNTR COMBFL Ν COMBFL Υ

3

6

10

12

3

3

3

1

2

3

900

1

2

3

1

900

FILE: stat2c.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.3 FINAL

AVISITN AVISITN

AVISITN

AVISITN

TRTPN

TRTPN

TRTPN

TRTPN AVISITN\*TRTPN

AVISITN\*TRTPN

AVISITN\*TRTPN

AVISITN\*TRTPN

AVISITN\*TRTPN


STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

.------

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY AGEGRP AT Phase B

| | (Pooled<br>Center) | Combat<br>Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | AGEGRP | (N) | (N) | Row1 |
| BIICCC | 101 111 | 1149 | 11000111 | (14) | (14) | 110111 |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |
| AVISITN*TRTPN | | | | 12 | 900 | |
| AGEGRP | | | <55 | | | |
| AGEGRP | | | >=55 | | | |
| AVISITN*AGEGRP | | | <55 | 3 | | |
| AVISITN*AGEGRP | | | >=55 | 3 | | |
| AVISITN*AGEGRP | | | <55 | 6 | | |
| AVISITN*AGEGRP | | | >=55 | 6 | | |
| AVISITN*AGEGRP | | | <55 | 10 | | |

FILE: stat2c.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.3 FINAL


STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY AGEGRP AT Phase B

| <b>7</b> 66 | (Pooled<br>Center) | Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | - 1 |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | AGEGRP | (N) | (N) | Row1 |
| AVISITN*AGEGRP | | | >=55 | 10 | | |
| AVISITN*AGEGRP | | | <55 | 12 | | |
| AVISITN*AGEGRP | | | >=55 | 12 | | |
| TRTPN*AGEGRP | | | <55 | | 1 | |
| TRTPN*AGEGRP | | | >=55 | | 1 | |
| TRTPN*AGEGRP | | | <55 | | 2 | 1 |
| TRTPN*AGEGRP | | | >=55 | | 2 | -1 |
| TRTPN*AGEGRP | | | <55 | | 3 | |
| TRTPN*AGEGRP | | | >=55 | | 3 | |
| TRTPN*AGEGRP | | | <55 | | 900 | -1 |
| TRTPN*AGEGRP | | | >=55 | | 900 | 1 |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 900 | |


STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY AGEGRP AT Phase B

| | Center<br>(Pooled<br>Center) | Combat<br>Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | AGEGRP | (N) | (N) | Row1 |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 2 | 1 |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 2 | -1 |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 900 | -1 |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 900 | 1 |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 1 | |


STAT-3.

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY AGEGRP AT Phase B

| | Center<br>(Pooled<br>Center) | Combat<br>Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | AGEGRP | (N) | (N) | Row1 |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |
| BASE*AVISITN | | | | 12 | | |




STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY AGEGRP AT Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | AGEGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |


STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY AGEGRP AT Phase B

| 766 | (Pooled<br>Center) | Combat<br>Related<br>Population | ACECDD | Analysis<br>Visit | Planned<br>Treatment | D = 1-1 |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | AGEGRP | (N) | (N) | Row1 |
| AVISITN*TRTPN | | | | 12 | 900 | |
| AGEGRP | | | <55 | | | |
| AGEGRP | | | >=55 | | | |
| AVISITN*AGEGRP | | | <55 | 3 | | |
| AVISITN*AGEGRP | | | >=55 | 3 | | |
| AVISITN*AGEGRP | | | <55 | 6 | | |
| AVISITN*AGEGRP | | | >=55 | 6 | | |
| AVISITN*AGEGRP | | | <55 | 10 | | |
| AVISITN*AGEGRP | | | >=55 | 10 | | |
| AVISITN*AGEGRP | | | <55 | 12 | | |
| AVISITN*AGEGRP | | | >=55 | 12 | | |
| TRTPN*AGEGRP | | | <55 | | 1 | |
| TRTPN*AGEGRP | | | >=55 | | 1 | |
| TRTPN*AGEGRP | | | <55 | | 2 | |
| TRTPN*AGEGRP | | | >=55 | | 2 | |
| TRTPN*AGEGRP | | | <55 | | 3 | 1 |
| TRTPN*AGEGRP | | | >=55 | | 3 | -1 |
| TRTPN*AGEGRP | | | <55 | | 900 | -1 |

BREXPIPRAZOLE 35 OF 39

STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY AGEGRP AT Phase B

| | Center<br>(Pooled<br>Center) | Combat<br>Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | AGEGRP | (N) | (N) | Row1 |
| TRTPN*AGEGRP | | | >=55 | | 900 | 1 |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 3 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 3 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 6 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 6 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 1 | |

FILE: stat2c.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.3 FINAL


STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY AGEGRP AT Phase B

| | (Pooled<br>(Center) | Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | AGEGRP | (N) | (N) | Row1 |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 3 | 1 |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 3 | -1 |
| AVISITN*TRTPN*AGEGRP | | | <55 | 10 | 900 | -1 |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 10 | 900 | 1 |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 1 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 2 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 3 | |
| AVISITN*TRTPN*AGEGRP | | | <55 | 12 | 900 | |
| AVISITN*TRTPN*AGEGRP | | | >=55 | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |

BREXPIPRAZOLE 37 OF 39 PROTOCOL 331-201-00061 STAT-3.3 MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy Y vs. Dummy Z BY AGEGRP AT Phase B Center Combat Center) Population for ITT Plant Analysis Planned Visit Treatment Effect for ITT Flag AGEGRP (N) (N) Row1 BASE\*AVISITN 12 Estimates Standard Label Estimate Error DF t Value Pr > |t| 5.4797 234 Dummy W vs. Dummy Z BY AGEGRP AT Phase B -2.3988 -0.44 0.6620 Dummy W vs. Dummy Y BY AGEGRP AT Phase B -4.7484 5.8120 225 -0.82 0.4148 6.3558 238 0.75 0.4566 Dummy W vs. Dummy X BY AGEGRP AT Phase B 4.7390 -7.1378 6.2185 246 -1.15 0.2521 Dummy X vs. Dummy Z BY AGEGRP AT Phase B Dummy Y vs. Dummy Z BY AGEGRP AT Phase B 2.3495 5.6950 233 0.41 0.6803


STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction

(Intent to Treat Sample)

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Least Squares Means

| | | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Visit | Treatment | | Standard | | | | | _ | |
| Effect | AGEGRP | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN*AGEGRP | <55 | 3 | 1 | -6.0540 | 1.1585 | 285 | -5.23 | <.0001 | 0.05 | -8.3343 | -3.7738 |
| AVISITN*TRTPN*AGEGRP | >=55 | 3 | 1 | -9.3081 | 2.7517 | 277 | -3.38 | 0.0008 | 0.05 | -14.7250 | -3.8912 |
| AVISITN*TRTPN*AGEGRP | <55 | 3 | 2 | -4.5801 | 1.2340 | 285 | -3.71 | 0.0002 | 0.05 | -7.0091 | -2.1512 |
| AVISITN*TRTPN*AGEGRP | >=55 | 3 | 2 | -5.9322 | 3.3290 | 290 | -1.78 | 0.0758 | 0.05 | -12.4843 | 0.6198 |
| AVISITN*TRTPN*AGEGRP | <55 | 3 | 3 | -6.1834 | 1.1706 | 282 | -5.28 | <.0001 | 0.05 | -8.4876 | -3.8792 |
| AVISITN*TRTPN*AGEGRP | >=55 | 3 | 3 | -6.9955 | 3.0210 | 276 | -2.32 | 0.0213 | 0.05 | -12.9426 | -1.0484 |
| AVISITN*TRTPN*AGEGRP | <55 | 3 | 900 | -5.5459 | 1.1533 | 281 | -4.81 | <.0001 | 0.05 | -7.8161 | -3.2758 |
| AVISITN*TRTPN*AGEGRP | >=55 | 3 | 900 | -10.3677 | 2.6369 | 277 | -3.93 | 0.0001 | 0.05 | -15.5586 | -5.1767 |
| AVISITN*TRTPN*AGEGRP | <55 | 6 | 1 | -12.4948 | 1.4252 | 269 | -8.77 | <.0001 | 0.05 | -15.3007 | -9.6889 |
| AVISITN*TRTPN*AGEGRP | >=55 | 6 | 1 | -14.0505 | 3.6151 | 285 | -3.89 | 0.0001 | 0.05 | -21.1662 | -6.9348 |
| AVISITN*TRTPN*AGEGRP | <55 | 6 | 2 | -8.7265 | 1.5135 | 288 | -5.77 | <.0001 | 0.05 | -11.7055 | -5.7476 |
| AVISITN*TRTPN*AGEGRP | >=55 | 6 | 2 | -2.1002 | 4.2485 | 274 | -0.49 | 0.6215 | 0.05 | -10.4640 | 6.2637 |
| AVISITN*TRTPN*AGEGRP | <55 | 6 | 3 | -9.3506 | 1.4610 | 282 | -6.40 | <.0001 | 0.05 | -12.2264 | -6.4747 |
| AVISITN*TRTPN*AGEGRP | >=55 | 6 | 3 | -12.8014 | 3.7811 | 260 | -3.39 | 0.0008 | 0.05 | -20.2468 | -5.3560 |
| AVISITN*TRTPN*AGEGRP | <55 | 6 | 900 | -8.9035 | 1.4066 | 265 | -6.33 | <.0001 | 0.05 | -11.6731 | -6.1339 |
| AVISITN*TRTPN*AGEGRP | >=55 | 6 | 900 | -9.0182 | 3.2840 | 272 | -2.75 | 0.0064 | 0.05 | -15.4835 | -2.5530 |
| AVISITN*TRTPN*AGEGRP | <55 | 10 | 1 | -16.4575 | 1.5350 | 244 | -10.72 | <.0001 | 0.05 | -19.4811 | -13.4338 |
| AVISITN*TRTPN*AGEGRP | >=55 | 10 | 1 | -16.8256 | 3.7412 | 232 | -4.50 | <.0001 | 0.05 | -24.1966 | -9.4546 |
| AVISITN*TRTPN*AGEGRP | <55 | 10 | 2 | -12.6899 | 1.6539 | 274 | -7.67 | <.0001 | 0.05 | -15.9459 | -9.4339 |


STAT-3.3

MMRM Output for Test on Treatment by Age (<55 vs >=55) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Least Squares Means

| Effect | : | AGEGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| AVISIT | TN*TRTPN*AGEGRP | >=55 | 10 | 2 | -8.3190 | 4.7195 | 253 | -1.76 | 0.0792 | 0.05 | -17.6136 | 0.9755 |
| AVISIT | "N*TRTPN*AGEGRP | <55 | 10 | 3 | -10.7824 | 1.5611 | 251 | -6.91 | <.0001 | 0.05 | -13.8569 | -7.7078 |
| AVISIT | "N*TRTPN*AGEGRP | >=55 | 10 | 3 | -15.8989 | 3.9845 | 226 | -3.99 | <.0001 | 0.05 | -23.7505 | -8.0473 |
| AVISIT | N*TRTPN*AGEGRP | <55 | 10 | 900 | -10.1139 | 1.5122 | 244 | -6.69 | <.0001 | 0.05 | -13.0926 | -7.1352 |
| AVISIT | N*TRTPN*AGEGRP | >=55 | 10 | 900 | -12.8809 | 3.4993 | 248 | -3.68 | 0.0003 | 0.05 | -19.7729 | -5.9889 |
| AVISIT | N*TRTPN*AGEGRP | <55 | 12 | 1 | -17.3985 | 1.6839 | 252 | -10.33 | <.0001 | 0.05 | -20.7149 | -14.0822 |
| AVISIT | TN*TRTPN*AGEGRP | >=55 | 12 | 1 | -17.2620 | 4.0450 | 234 | -4.27 | <.0001 | 0.05 | -25.2314 | -9.2927 |
| AVISIT | "N*TRTPN*AGEGRP | <55 | 12 | 2 | -13.0650 | 1.7885 | 271 | -7.30 | <.0001 | 0.05 | -16.5862 | -9.5439 |
| AVISIT | "N*TRTPN*AGEGRP | >=55 | 12 | 2 | -4.7770 | 5.4143 | 276 | -0.88 | 0.3784 | 0.05 | -15.4355 | 5.8815 |
| AVISIT | "N*TRTPN*AGEGRP | <55 | 12 | 3 | -14.4569 | 1.6922 | 254 | -8.54 | <.0001 | 0.05 | -17.7894 | -11.1243 |
| AVISIT | "N*TRTPN*AGEGRP | >=55 | 12 | 3 | -18.6102 | 4.3104 | 228 | -4.32 | <.0001 | 0.05 | -27.1036 | -10.1169 |
| AVISIT | "N*TRTPN*AGEGRP | <55 | 12 | 900 | -11.2200 | 1.6606 | 254 | -6.76 | <.0001 | 0.05 | -14.4902 | -7.9497 |
| AVISIT | TN*TRTPN*AGEGRP | >=55 | 12 | 900 | -14.5274 | 3.6625 | 231 | -3.97 | <.0001 | 0.05 | -21.7435 | -7.3113 |

BREXPIPRAZOLE 1 OF 42 PROTOCOL 331-201-00061 MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample) The Mixed Procedure Model Information Data Set
Dependent Variable
Covariance Structure WORK.INDATA CHG Unstructured SUBJID Estimation Method REML Residual Variance Method None Fixed Effects SE Method Kenward-Roger Degrees of Freedom Method Kenward-Roger Class Level Information Class Levels Values 4 AVISITN 3 6 10 12 1 2 3 900 TRTPN 4 POOLCNTR 10 COMBFL 2 NY

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL











BREXPIPRAZOLE 7 OF 42 PROTOCOL 331-201-00061 STAT-3.4.1 MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample) The Mixed Procedure Iteration History Iteration Evaluations -2 Res Log Like Criterion 7332.70126632 0 1 2 6866.76001648 0.00042716 1 6865.55160256 0.00001410 6865.51465725 3 1 0.00000002 1 6865.51460943 0.00000000 Convergence criteria met. Covariance Parameter Estimates Cov Parm Subject Estimate SUBJID 78.6501 UN(1,1) UN(2,1) SUBJID 52.3865 UN(2,2) SUBJID 110.71 UN(3,1) SUBJID 43.4941 UN(3,2) SUBJID 86.9959 UN(3,3) SUBJID 122.56 UN (4,1) SUBJID 49.1894

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL

BREXPIPRAZOLE 8 OF 42 PROTOCOL 331-201-00061 STAT-3.4.1 MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample) The Mixed Procedure Covariance Parameter Estimates Cov Parm Subject Estimate 88.8299 UN(4,2) SUBJID SUBJID UN(4,3) SUBJID UN(4,4) SUBJID 104.30 147.67 Fit Statistics -2 Res Log Likelihood 6865.5 AIC (Smaller is Better) 6885.5 AICC (Smaller is Better) 6885.7 BIC (Smaller is Better) 6922.5 Null Model Likelihood Ratio Test Chi-Square Pr > ChiSq

467.19

<.0001

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL

BREXPIPRAZOLE

STAT-3.4.1

MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

The Mixed Procedure

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|----------------------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| POOLCNTR | 9 | 277 | 1.63 | 0.1060 |
| COMBFL | 1 | 278 | 3.21 | 0.0743 |
| AVISITN | 3 | 227 | 1.52 | 0.2098 |
| TRTPN | 3 | 267 | 2.99 | 0.0316 |
| AVISITN*TRTPN | 9 | 361 | 2.04 | 0.0347 |
| MPLC20FL | 1 | 278 | 0.00 | 0.9560 |
| AVISITN*MPLC20FL | 3 | 238 | 0.71 | 0.5457 |
| TRTPN*MPLC20FL | 3 | 269 | 1.83 | 0.1427 |
| AVISIT*TRTPN*MPLC20F | 9 | 361 | 1.29 | 0.2401 |
| BASE*AVISITN | 4 | 240 | 8.09 | <.0001 |


BREXPIPRAZOLE 11 OF 42 PROTOCOL 331-201-00061 STAT-3.4.1 MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy W vs. Dummy Z BY MPLC20FL AT Phase B Placebo Center Combat 20% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 TRTPN 2 TRTPN TRTPN 3 900 TRTPN 3 AVISITN\*TRTPN 1 AVISITN\*TRTPN 2 AVISITN\*TRTPN 3 AVISITN\*TRTPN 900 6 AVISITN\*TRTPN 1 6 AVISITN\*TRTPN 2 6 AVISITN\*TRTPN 6 900 AVISITN\*TRTPN AVISITN\*TRTPN 10 1 AVISITN\*TRTPN 10 2 AVISITN\*TRTPN 10 AVISITN\*TRTPN 10 900 AVISITN\*TRTPN 12

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL

BREXPIPRAZOLE 12 OF 42 PROTOCOL 331-201-00061 STAT-3.4.1 MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ----- Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy W vs. Dummy Z BY MPLC20FL AT Phase B Placebo Center Combat 20% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 12 2 AVISITN\*TRTPN 12 AVISITN\*TRTPN 900 AVISITN\*TRTPN 12 MPLC20FL N MPLC20FL Y AVISITN\*MPLC20FL N 3 AVISITN\*MPLC20FL AVISITN\*MPLC20FL N AVISITN\*MPLC20FL Y 6 AVISITN\*MPLC20FL N 10 Y 10 AVISITN\*MPLC20FL AVISITN\*MPLC20FL 12 N AVISITN\*MPLC20FL Y 12 TRTPN\*MPLC20FL N

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL

TRTPN\*MPLC20FL

TRTPN\*MPLC20FL

TRTPN\*MPLC20FL

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.

Y

N

BREXPIPRAZOLE 13 OF 42 PROTOCOL 331-201-00061 STAT-3.4.1 MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy W vs. Dummy Z BY MPLC20FL AT Phase B Placebo Center Combat 20% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 TRTPN\*MPLC20FL Υ TRTPN\*MPLC20FL -1 TRTPN\*MPLC20FL N 900 Y 900 TRTPN\*MPLC20FL 1 3 AVISIT\*TRTPN\*MPLC20F N 1 AVISIT\*TRTPN\*MPLC20F 1 AVISIT\*TRTPN\*MPLC20F AVISIT\*TRTPN\*MPLC20F Y AVISIT\*TRTPN\*MPLC20F N 3 3 Y 3 AVISIT\*TRTPN\*MPLC20F

N

Y

N

Y

N

Y

900

900

1

1

2

3

6

6

6

6

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL

AVISIT\*TRTPN\*MPLC20F

AVISIT\*TRTPN\*MPLC20F

AVISIT\*TRTPN\*MPLC20F

AVISIT\*TRTPN\*MPLC20F

AVISIT\*TRTPN\*MPLC20F

AVISIT\*TRTPN\*MPLC20F

AVISIT\*TRTPN\*MPLC20F

BREXPIPRAZOLE 14 OF 42 PROTOCOL 331-201-00061

MMRM Output for Test on Treatment by STAT-3.4.1

Output for Test on Treatment by (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY MPLC20FL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | 20%<br>Responder<br>Population<br>Flag in | | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*MPLC20F | | | Y | 6 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | N | 6 | 900 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 6 | 900 | |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 1 | 1 |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 1 | -1 |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 900 | -1 |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 900 | 1 |
| AVISIT*TRTPN*MPLC20F | | | N | 12 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 12 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | N | 12 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 12 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | N | 12 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 12 | 3 | |

BREXPIPRAZOLE 15 OF 42 PROTOCOL 331-201-00061 STAT-3.4.1 MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ----- Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy W vs. Dummy Z BY MPLC20FL AT Phase B Placebo Center Combat 20% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) (N) Row1 900 12 AVISIT\*TRTPN\*MPLC20F Y 12 900 AVISIT\*TRTPN\*MPLC20F 3 BASE\*AVISITN 6 BASE\*AVISITN 10 BASE\*AVISITN BASE\*AVISITN 12



BREXPIPRAZOLE 17 OF 42 PROTOCOL 331-201-00061 STAT-3.4.1 MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy W vs. Dummy Y BY MPLC20FL AT Phase B Placebo Center Combat 20% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 TRTPN 2 TRTPN TRTPN 900 TRTPN 3 AVISITN\*TRTPN 1 AVISITN\*TRTPN 2 AVISITN\*TRTPN AVISITN\*TRTPN 900 6 AVISITN\*TRTPN 6 AVISITN\*TRTPN 2 6 AVISITN\*TRTPN 6 900 AVISITN\*TRTPN AVISITN\*TRTPN 10 1 AVISITN\*TRTPN 10 2 AVISITN\*TRTPN 10 AVISITN\*TRTPN 10 900 AVISITN\*TRTPN 12

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL



BREXPIPRAZOLE 19 OF 42 PROTOCOL 331-201-00061 STAT-3.4.1 MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy W vs. Dummy Y BY MPLC20FL AT Phase B Placebo Center Combat 20% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 TRTPN\*MPLC20FL N -1 Υ TRTPN\*MPLC20FL 1 TRTPN\*MPLC20FL N 900 Y 900 TRTPN\*MPLC20FL 3 AVISIT\*TRTPN\*MPLC20F N 1 AVISIT\*TRTPN\*MPLC20F 1 AVISIT\*TRTPN\*MPLC20F AVISIT\*TRTPN\*MPLC20F Y N 3 AVISIT\*TRTPN\*MPLC20F Y 3 AVISIT\*TRTPN\*MPLC20F AVISIT\*TRTPN\*MPLC20F N 900 AVISIT\*TRTPN\*MPLC20F Y 3 900 AVISIT\*TRTPN\*MPLC20F N 6 1 AVISIT\*TRTPN\*MPLC20F Y 6 1 AVISIT\*TRTPN\*MPLC20F N 6 2 AVISIT\*TRTPN\*MPLC20F Y 6

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL

AVISIT\*TRTPN\*MPLC20F

BREXPIPRAZOLE
STAT-3.4.1
MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction

(Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY MPLC20FL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Placebo<br>20%<br>Responder<br>Population<br>Flag in | | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*MPLC20F | | | Y | 6 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | N | 6 | 900 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 6 | 900 | |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 1 | 1 |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 1 | -1 |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 3 | -1 |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 3 | 1 |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 900 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 900 | |
| AVISIT*TRTPN*MPLC20F | | | N | 12 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 12 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | N | 12 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 12 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | N | 12 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 12 | 3 | |

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL

BREXPIPRAZOLE 21 OF 42 PROTOCOL 331-201-00061 STAT-3.4.1 MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy W vs. Dummy Y BY MPLC20FL AT Phase B Placebo Center Combat 20% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) (N) Row1 900 12 AVISIT\*TRTPN\*MPLC20F Y 12 900 AVISIT\*TRTPN\*MPLC20F 3 BASE\*AVISITN 6 BASE\*AVISITN 10 BASE\*AVISITN BASE\*AVISITN 12



BREXPIPRAZOLE 23 OF 42 PROTOCOL 331-201-00061 STAT-3.4.1 MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT --------The Mixed Procedure Coefficients for Dummy W vs. Dummy X BY MPLC20FL AT Phase B Placebo Center Combat 20% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 TRTPN 2 TRTPN TRTPN 900 TRTPN 3 AVISITN\*TRTPN 1 AVISITN\*TRTPN 2 AVISITN\*TRTPN AVISITN\*TRTPN 900 6 AVISITN\*TRTPN 6 AVISITN\*TRTPN 6 AVISITN\*TRTPN 6 900 AVISITN\*TRTPN AVISITN\*TRTPN 10 1 AVISITN\*TRTPN 10 2 AVISITN\*TRTPN 10 AVISITN\*TRTPN 10 900 AVISITN\*TRTPN 12

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL

-1

-1

BREXPIPRAZOLE 24 OF 42 PROTOCOL 331-201-00061 STAT-3.4.1 MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT ------------The Mixed Procedure Coefficients for Dummy W vs. Dummy X BY MPLC20FL AT Phase B Placebo Center Combat 20% Responder (Pooled Related Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) (N) Row1 12 2 AVISITN\*TRTPN 12 AVISITN\*TRTPN 900 AVISITN\*TRTPN 12 MPLC20FL N MPLC20FL Y AVISITN\*MPLC20FL N 3 AVISITN\*MPLC20FL AVISITN\*MPLC20FL N AVISITN\*MPLC20FL Y 6 AVISITN\*MPLC20FL N 10 Y 10 AVISITN\*MPLC20FL AVISITN\*MPLC20FL 12 N AVISITN\*MPLC20FL Y 12 TRTPN\*MPLC20FL N

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL

TRTPN\*MPLC20FL

TRTPN\*MPLC20FL

TRTPN\*MPLC20FL

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.

Y

N

BREXPIPRAZOLE 25 OF 42 PROTOCOL 331-201-00061 STAT-3.4.1 MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy W vs. Dummy X BY MPLC20FL AT Phase B Placebo Center Combat 20% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 TRTPN\*MPLC20FL N Υ TRTPN\*MPLC20FL TRTPN\*MPLC20FL N 900 Y 900 TRTPN\*MPLC20FL 3 AVISIT\*TRTPN\*MPLC20F N 1 AVISIT\*TRTPN\*MPLC20F Y 1 AVISIT\*TRTPN\*MPLC20F AVISIT\*TRTPN\*MPLC20F Y N 3 AVISIT\*TRTPN\*MPLC20F Y AVISIT\*TRTPN\*MPLC20F 3 AVISIT\*TRTPN\*MPLC20F N 900

Y

N

Y

N

Y

3

6

6

6

6

900

1

1

2

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL

AVISIT\*TRTPN\*MPLC20F

AVISIT\*TRTPN\*MPLC20F

AVISIT\*TRTPN\*MPLC20F

AVISIT\*TRTPN\*MPLC20F

AVISIT\*TRTPN\*MPLC20F

AVISIT\*TRTPN\*MPLC20F

BREXPIPRAZOLE 26 OF 42 PROTOCOL 331-201-00061

STAT-3.4.1

MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY MPLC20FL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Placebo<br>20%<br>Responder<br>Population<br>Flag in | | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*MPLC20F | | | Y | 6 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | N | 6 | 900 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 6 | 900 | |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 1 | 1 |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 1 | -1 |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 2 | -1 |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 2 | 1 |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 900 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 900 | |
| AVISIT*TRTPN*MPLC20F | | | N | 12 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 12 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | N | 12 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 12 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | N | 12 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 12 | 3 | |

BREXPIPRAZOLE 27 OF 42 PROTOCOL 331-201-00061 STAT-3.4.1 MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy W vs. Dummy X BY MPLC20FL AT Phase B Placebo Center Combat 20% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) (N) Row1 900 12 AVISIT\*TRTPN\*MPLC20F Y 12 900 AVISIT\*TRTPN\*MPLC20F BASE\*AVISITN 3 6 BASE\*AVISITN 10 BASE\*AVISITN BASE\*AVISITN 12

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL



BREXPIPRAZOLE 29 OF 42 PROTOCOL 331-201-00061 STAT-3.4.1 MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy X vs. Dummy Z BY MPLC20FL AT Phase B Placebo Center Combat 20% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 TRTPN 2 TRTPN TRTPN 3 900 TRTPN 3 AVISITN\*TRTPN 1 AVISITN\*TRTPN 2 AVISITN\*TRTPN 3 AVISITN\*TRTPN 900 6 AVISITN\*TRTPN 1 6 AVISITN\*TRTPN 2 6 AVISITN\*TRTPN 6 900 AVISITN\*TRTPN AVISITN\*TRTPN 10 1 AVISITN\*TRTPN 10 2 AVISITN\*TRTPN 10 AVISITN\*TRTPN 10 900 AVISITN\*TRTPN 12

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL

BREXPIPRAZOLE 30 OF 42 PROTOCOL 331-201-00061 STAT-3.4.1 20 Percent Improvement Subgroup Interaction MMRM Output for Test on Treatment by (Intent to Treat Sample) ------ Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy X vs. Dummy Z BY MPLC20FL AT Phase B Placebo Center Combat 20% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 12 2 AVISITN\*TRTPN 12 AVISITN\*TRTPN 900 AVISITN\*TRTPN 12 MPLC20FL N MPLC20FL Y AVISITN\*MPLC20FL N 3

N

Y

N Y

N

Y

N

Y

N

6 10

10

12

12

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL

AVISITN\*MPLC20FL AVISITN\*MPLC20FL

AVISITN\*MPLC20FL

AVISITN\*MPLC20FL

AVISITN\*MPLC20FL AVISITN\*MPLC20FL

AVISITN\*MPLC20FL

TRTPN\*MPLC20FL

TRTPN\*MPLC20FL

TRTPN\*MPLC20FL

TRTPN\*MPLC20FL

BREXPIPRAZOLE

MMRM Output for Test on Treatment by STAT-3.4.1

(Intent to Treat Sample)

31 OF 42

STAT-3.4.1

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY MPLC20FL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Placebo<br>20%<br>Responder<br>Population<br>Flag in | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*MPLC20FL | | | N | | 3 | |
| TRTPN*MPLC20FL | | | Y | | 3 | |
| TRTPN*MPLC20FL | | | N | | 900 | -1 |
| TRTPN*MPLC20FL | | | Y | | 900 | 1 |
| AVISIT*TRTPN*MPLC20F | | | N | 3 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 3 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | N | 3 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 3 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | N | 3 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 3 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | N | 3 | 900 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 3 | 900 | |
| AVISIT*TRTPN*MPLC20F | | | N | 6 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 6 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | N | 6 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 6 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | N | 6 | 3 | |

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL

BREXPIPRAZOLE

32 OF 42

MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY MPLC20FL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Placebo<br>20%<br>Responder<br>Population<br>Flag in | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*MPLC20F | | | Y | 6 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | N | 6 | 900 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 6 | 900 | |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 2 | 1 |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 2 | -1 |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 900 | -1 |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 900 | 1 |
| AVISIT*TRTPN*MPLC20F | | | N | 12 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 12 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | N | 12 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 12 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | N | 12 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 12 | 3 | |

BREXPIPRAZOLE 33 OF 42 PROTOCOL 331-201-00061 MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy X vs. Dummy Z BY MPLC20FL AT Phase B Placebo Center Combat 20% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) (N) Row1 900 12 AVISIT\*TRTPN\*MPLC20F Y 12 900 AVISIT\*TRTPN\*MPLC20F 3 BASE\*AVISITN 6 BASE\*AVISITN 10 BASE\*AVISITN BASE\*AVISITN 12



BREXPIPRAZOLE 35 OF 42 PROTOCOL 331-201-00061 STAT-3.4.1 MMRM Output for Test on Treatment by 20 Percent Improvement Subgroup Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy Y vs. Dummy Z BY MPLC20FL AT Phase B Placebo Center Combat 20% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 TRTPN 2 TRTPN TRTPN 900 TRTPN 3 AVISITN\*TRTPN 1 AVISITN\*TRTPN 2 AVISITN\*TRTPN AVISITN\*TRTPN 900 6 AVISITN\*TRTPN 1 6 AVISITN\*TRTPN 2 6 AVISITN\*TRTPN 6 900 AVISITN\*TRTPN AVISITN\*TRTPN 10 1 AVISITN\*TRTPN 10 2 AVISITN\*TRTPN 10 AVISITN\*TRTPN 10 900 AVISITN\*TRTPN 12

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY MPLC20FL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Placebo<br>20%<br>Responder<br>Population<br>Flag in | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |
| AVISITN*TRTPN | | | | 12 | 900 | |
| MPLC20FL | | | N | | | |
| MPLC20FL | | | Y | | | |
| AVISITN*MPLC20FL | | | N | 3 | | |
| AVISITN*MPLC20FL | | | Y | 3 | | |
| AVISITN*MPLC20FL | | | N | 6 | | |
| AVISITN*MPLC20FL | | | Y | 6 | | |
| AVISITN*MPLC20FL | | | N | 10 | | |
| AVISITN*MPLC20FL | | | Y | 10 | | |
| AVISITN*MPLC20FL | | | N | 12 | | |
| AVISITN*MPLC20FL | | | Y | 12 | | |
| TRTPN*MPLC20FL | | | N | | 1 | |
| TRTPN*MPLC20FL | | | Y | | 1 | |
| TRTPN*MPLC20FL | | | N | | 2 | |
| TRTPN*MPLC20FL | | | Y | | 2 | |

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL

BREXPIPRAZOLE

MMRM Output for Test on Treatment by (Intent to Treat Sample)

STAT-3.4.1

(Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY MPLC20FL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | 20%<br>Responder<br>Population<br>Flag in | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*MPLC20FL | | | N | | 3 | 1 |
| TRTPN*MPLC20FL | | | Y | | 3 | -1 |
| TRTPN*MPLC20FL | | | N | | 900 | -1 |
| TRTPN*MPLC20FL | | | Y | | 900 | 1 |
| AVISIT*TRTPN*MPLC20F | | | N | 3 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 3 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | N | 3 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 3 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | N | 3 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 3 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | N | 3 | 900 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 3 | 900 | |
| AVISIT*TRTPN*MPLC20F | | | N | 6 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 6 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | N | 6 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 6 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | N | 6 | 3 | |

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL

BREXPIPRAZOLE

STAT-3.4.1

MMRM Output for Test on Treatment by (Intent to Treat Sample)

(Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY MPLC20FL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Placebo<br>20%<br>Responder<br>Population<br>Flag in | | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*MPLC20F | | | Y | 6 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | N | 6 | 900 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 6 | 900 | |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 3 | 1 |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 3 | -1 |
| AVISIT*TRTPN*MPLC20F | | | N | 10 | 900 | -1 |
| AVISIT*TRTPN*MPLC20F | | | Y | 10 | 900 | 1 |
| AVISIT*TRTPN*MPLC20F | | | N | 12 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 12 | 1 | |
| AVISIT*TRTPN*MPLC20F | | | N | 12 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 12 | 2 | |
| AVISIT*TRTPN*MPLC20F | | | N | 12 | 3 | |
| AVISIT*TRTPN*MPLC20F | | | Y | 12 | 3 | |

FILE: stat2d1.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.1 FINAL



| BREXPIPRAZOLE PROTOCOL 331-201-00061 | _ | | | | | | | | 40 | OF 42 | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | MMRM Output | for Test on | Treatment by | 20 P | -3.4.1<br>ercent Impro<br>Treat Sample | | ubgroup Int | eraction | | | |
| | | | | Parameter | Code=CAPSTOT | | | | | | |
| The Mixed Procedure | | | | | | | | | | | |
| | | | | Esti | mates | | | | | | |
| I | Label | | | | Estimate | Standa<br>Err | | t Value | Pr > t | | |
| Ι | Dummy Y vs. Dum | my Z BY MPLC | 20FL AT Phase | В | 10.3139 | 4.09 | 37 238 | 2.52 | 0.0124 | | |
| | | | | Least Squ | ares Means | | | | | | |
| | Placebo | | | | | | | | | | |
| | 20%<br>Responder | Analysis | Planned | | | | | | | | |
| Effect | Population<br>Flag in | Visit<br>(N) | Treatment (N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISIT*TRTPN*MPLC20F | N | 3 | 1 | -6.5615 | 1.4085 | 284 | -4.66 | <.0001 | 0.05 | -9.3339 | -3.7891 |
| AVISIT*TRTPN*MPLC20F | Y | 3 | 1 | -6.0037 | 1.9400 | 282 | -3.09 | 0.0022 | 0.05 | -9.8224 | -2.1849 |
| AVISIT*TRTPN*MPLC20F | N | 3 | 2 | -3.4458 | 1.5811 | 288 | -2.18 | 0.0301 | 0.05 | -6.5578 | -0.3337 |
| AVISIT*TRTPN*MPLC20F | Y | 3 | 2 | -6.0500 | 1.9577 | 277 | -3.09 | 0.0022 | 0.05 | -9.9037 | -2.1962 |
| AVISIT*TRTPN*MPLC20F | N | 3 | 3 | -5.1128 | 1.4555 | 283 | -3.51 | 0.0005 | 0.05 | -7.9778 | -2.2479 |
| AVISIT*TRTPN*MPLC20F | Y | 3 | 3 | -7.8652 | 1.9022 | 277 | -4.13 | <.0001 | 0.05 | -11.6099 | -4.1205 |
| AVISIT*TRTPN*MPLC20F | N | 3 | 900 | -5.7150 | 1.4184 | 282 | -4.03 | <.0001 | 0.05 | -8.5071 | -2.9229 |
| AVISIT*TRTPN*MPLC20F | Y | 3 | 900 | -6.9412 | 1.8409 | 280 | -3.77 | 0.0002 | 0.05 | -10.5650 | -3.3173 |
| AVISIT*TRTPN*MPLC20F | N | 6 | 1 | -13.5581 | 1.7282 | 276 | -7.85 | <.0001 | 0.05 | -16.9601 | -10.1561 |

BREXPIPRAZOLE 41 OF 42 PROTOCOL 331-201-00061

STAT-3.4.1

MMRM Output for Test on Treatment by (Intent to Treat Sample)

.....

The Mixed Procedure

Least Squares Means

| | Placebo<br>20% | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Responder<br>Population | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
| Effect | Flag in | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISIT*TRTPN*MPLC20F | Y | 6 | 1 | -10.7737 | 2.3847 | 269 | -4.52 | <.0001 | 0.05 | -15.4687 | -6.0787 |
| AVISIT*TRTPN*MPLC20F | N | 6 | 2 | -9.0933 | 1.8693 | 279 | -4.86 | <.0001 | 0.05 | -12.7731 | -5.4136 |
| AVISIT*TRTPN*MPLC20F | Y | 6 | 2 | -5.5330 | 2.4967 | 285 | -2.22 | 0.0275 | 0.05 | -10.4474 | -0.6187 |
| AVISIT*TRTPN*MPLC20F | N | 6 | 3 | -7.8726 | 1.7683 | 288 | -4.45 | <.0001 | 0.05 | -11.3532 | -4.3921 |
| AVISIT*TRTPN*MPLC20F | Y | 6 | 3 | -13.2503 | 2.4170 | 270 | -5.48 | <.0001 | 0.05 | -18.0088 | -8.4919 |
| AVISIT*TRTPN*MPLC20F | N | 6 | 900 | -9.9567 | 1.6917 | 276 | -5.89 | <.0001 | 0.05 | -13.2870 | -6.6264 |
| AVISIT*TRTPN*MPLC20F | Y | 6 | 900 | -6.5873 | 2.2559 | 262 | -2.92 | 0.0038 | 0.05 | -11.0294 | -2.1452 |
| AVISIT*TRTPN*MPLC20F | N | 10 | 1 | -17.0866 | 1.8532 | 243 | -9.22 | <.0001 | 0.05 | -20.7369 | -13.4363 |
| AVISIT*TRTPN*MPLC20F | Y | 10 | 1 | -15.0059 | 2.6076 | 250 | -5.75 | <.0001 | 0.05 | -20.1416 | -9.8701 |
| AVISIT*TRTPN*MPLC20F | N | 10 | 2 | -12.3417 | 2.0363 | 261 | -6.06 | <.0001 | 0.05 | -16.3514 | -8.3320 |
| AVISIT*TRTPN*MPLC20F | Y | 10 | 2 | -11.7644 | 2.7677 | 268 | -4.25 | <.0001 | 0.05 | -17.2137 | -6.3152 |
| AVISIT*TRTPN*MPLC20F | N | 10 | 3 | -9.3241 | 1.8849 | 254 | -4.95 | <.0001 | 0.05 | -13.0362 | -5.6120 |
| AVISIT*TRTPN*MPLC20F | Y | 10 | 3 | -15.3750 | 2.6230 | 243 | -5.86 | <.0001 | 0.05 | -20.5417 | -10.2083 |
| AVISIT*TRTPN*MPLC20F | N | 10 | 900 | -11.8453 | 1.8076 | 253 | -6.55 | <.0001 | 0.05 | -15.4052 | -8.2855 |
| AVISIT*TRTPN*MPLC20F | Y | 10 | 900 | -7.5823 | 2.4699 | 240 | -3.07 | 0.0024 | 0.05 | -12.4477 | -2.7169 |
| AVISIT*TRTPN*MPLC20F | N | 12 | 1 | -17.2653 | 2.0451 | 247 | -8.44 | <.0001 | 0.05 | -21.2934 | -13.2371 |
| AVISIT*TRTPN*MPLC20F | Y | 12 | 1 | -17.2662 | 2.9034 | 259 | -5.95 | <.0001 | 0.05 | -22.9835 | -11.5490 |

| BREXPIPRAZOLE<br>PROTOCOL 331-201-00061 | | for Test on | Treatment by | 20 Pe | -3.4.1<br>ercent Improv<br>Freat Sample | | Subgroup Int | eraction | 42 | OF 42 | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | The Mixed | Procedure | | | | | | |
| | | | | Least Squa | ares Means | | | | | | |
| Effect | Placebo<br>20%<br>Responder<br>Population<br>Flag in | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISIT*TRTPN*MPLC20F | N<br>Y<br>N<br>Y<br>N | 12<br>12<br>12<br>12<br>12<br>12 | 2<br>2<br>3<br>3<br>900<br>900 | -13.4015<br>-9.9391<br>-13.5215<br>-17.6365<br>-12.6255<br>-9.6046 | 2.2279 3.0657 2.0656 2.8456 1.9587 2.8125 | 260<br>267<br>257<br>237<br>248<br>259 | -6.02<br>-3.24<br>-6.55<br>-6.20<br>-6.45<br>-3.41 | <.0001<br>0.0013<br><.0001<br><.0001<br><.0001<br>0.0007 | 0.05<br>0.05<br>0.05<br>0.05<br>0.05<br>0.05 | -17.7885<br>-15.9753<br>-17.5892<br>-23.2424<br>-16.4833<br>-15.1428 | -9.0146<br>-3.9030<br>-9.4537<br>-12.0305<br>-8.7677<br>-4.0664 |

BREXPIPRAZOLE 1 OF 42 PROTOCOL 331-201-00061 STAT-3.4.2 25 Percent Improvement Subgroup Interaction MMRM Output for Test on Treatment by (Intent to Treat Sample) The Mixed Procedure Model Information Data Set
Dependent Variable
Covariance Structure WORK.INDATA CHG Unstructured SUBJID Estimation Method REML Residual Variance Method None Fixed Effects SE Method Kenward-Roger Degrees of Freedom Method Kenward-Roger Class Level Information Class Levels Values AVISITN 4 3 6 10 12 TRTPN 4 POOLCNTR 10 COMBFL 2 NY

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL










BREXPIPRAZOLE 7 OF 42 PROTOCOL 331-201-00061 STAT-3.4.2 MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample) The Mixed Procedure Iteration History Iteration Evaluations -2 Res Log Like Criterion 0 1 7331.93442443 2 6868.02890783 0.00045719 1 6866.73189863 0.00001605 3 1 6866.68977151 0.00000002 1 6866.68970952 0.00000000 Convergence criteria met. Covariance Parameter Estimates Cov Parm Subject Estimate SUBJID 78.4737 UN(1,1) UN(2,1) SUBJID 51.8355 UN(2,2) SUBJID 111.08 UN(3,1) SUBJID 43.4739 UN(3,2) SUBJID 87.8417 UN(3,3) SUBJID 123.42 UN(4,1) SUBJID 48.3413

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

BREXPIPRAZOLE 8 OF 42 PROTOCOL 331-201-00061 STAT-3.4.2 25 Percent Improvement Subgroup Interaction MMRM Output for Test on Treatment by (Intent to Treat Sample) The Mixed Procedure Covariance Parameter Estimates Cov Parm Subject Estimate 88.5051 UN(4,2) SUBJID UN(4,3) SUBJID UN(4,4) SUBJID SUBJID 104.04 146.60 Fit Statistics -2 Res Log Likelihood 6866.7 AIC (Smaller is Better) 6886.7 AICC (Smaller is Better) 6886.9 BIC (Smaller is Better) 6923.7 Null Model Likelihood Ratio Test Chi-Square Pr > ChiSq

465.24

<.0001

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

BREXPIPRAZOLE

STAT-3.4.2

MMRM Output for Test on Treatment by (Intent to Treat Sample)

(Intent to Treat Sample)

The Mixed Procedure

Type 3 Tests of Fixed Effects

| Effect. | Num<br>DF | Den<br>DF | F Value | Pr > F |
|----------------------|-----------|-----------|---------|--------|
| FILECC | DE | DF | r value | F1 / F |
| POOLCNTR | 9 | 277 | 1.61 | 0.1112 |
| COMBFL | 1 | 278 | 3.20 | 0.0746 |
| AVISITN | 3 | 226 | 1.00 | 0.3942 |
| TRTPN | 3 | 266 | 3.14 | 0.0257 |
| AVISITN*TRTPN | 9 | 360 | 1.88 | 0.0541 |
| MPLC25FL | 1 | 272 | 0.54 | 0.4642 |
| AVISITN*MPLC25FL | 3 | 236 | 0.37 | 0.7716 |
| TRTPN*MPLC25FL | 3 | 267 | 2.63 | 0.0509 |
| AVISIT*TRTPN*MPLC25F | 9 | 360 | 0.93 | 0.4994 |
| BASE*AVISITN | 4 | 238 | 5.76 | 0.0002 |

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL



BREXPIPRAZOLE 11 OF 42 PROTOCOL 331-201-00061 STAT-3.4.2 MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy W vs. Dummy Z BY MPLC25FL AT Phase B Placebo Center Combat 25% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) (N) Row1 TRTPN 2 TRTPN TRTPN 900 TRTPN 3 AVISITN\*TRTPN 1 AVISITN\*TRTPN 2 AVISITN\*TRTPN AVISITN\*TRTPN 900 6 AVISITN\*TRTPN 1 6 AVISITN\*TRTPN 2 6 AVISITN\*TRTPN 6 900 AVISITN\*TRTPN AVISITN\*TRTPN 10 1 AVISITN\*TRTPN 10 2 AVISITN\*TRTPN 10 AVISITN\*TRTPN 10 900 AVISITN\*TRTPN 12

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

BREXPIPRAZOLE 12 OF 42 PROTOCOL 331-201-00061 STAT-3.4.2 MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy W vs. Dummy Z BY MPLC25FL AT Phase B Placebo Center Combat 25% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 12 2 AVISITN\*TRTPN 12 AVISITN\*TRTPN 900 AVISITN\*TRTPN 12 MPLC25FL N MPLC25FL Y AVISITN\*MPLC25FL N 3 AVISITN\*MPLC25FL AVISITN\*MPLC25FL N AVISITN\*MPLC25FL Y 6 AVISITN\*MPLC25FL N 10 Y 10 AVISITN\*MPLC25FL AVISITN\*MPLC25FL 12 N AVISITN\*MPLC25FL Y 12 TRTPN\*MPLC25FL N TRTPN\*MPLC25FL Y TRTPN\*MPLC25FL N

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

TRTPN\*MPLC25FL

BREXPIPRAZOLE 13 OF 42

STAT-3.4.2

MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY MPLC25FL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Placebo<br>25%<br>Responder<br>Population<br>Flag in | | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*MPLC25FL | | | N | | 3 | |
| TRTPN*MPLC25FL | | | Y | | 3 | |
| TRTPN*MPLC25FL | | | N | | 900 | -1 |
| TRTPN*MPLC25FL | | | Y | | 900 | 1 |
| AVISIT*TRTPN*MPLC25F | | | N | 3 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 3 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | N | 3 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 3 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | N | 3 | 3 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 3 | 3 | |
| AVISIT*TRTPN*MPLC25F | | | N | 3 | 900 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 3 | 900 | |
| AVISIT*TRTPN*MPLC25F | | | N | 6 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 6 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | N | 6 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 6 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | N | 6 | 3 | |

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

BREXPIPRAZOLE
\_\_\_\_STAT-3.4.2

MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY MPLC25FL AT Phase B

| ( | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | 25%<br>Responder<br>Population<br>Flag in | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*MPLC25F | | | Y | 6 | 3 | |
| AVISIT*TRTPN*MPLC25F | | | N | 6 | 900 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 6 | 900 | |
| AVISIT*TRTPN*MPLC25F | | | N | 10 | 1 | 1 |
| AVISIT*TRTPN*MPLC25F | | | Y | 10 | 1 | -1 |
| AVISIT*TRTPN*MPLC25F | | | N | 10 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 10 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | N | 10 | 3 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 10 | 3 | |
| AVISIT*TRTPN*MPLC25F | | | N | 10 | 900 | -1 |
| AVISIT*TRTPN*MPLC25F | | | Y | 10 | 900 | 1 |
| AVISIT*TRTPN*MPLC25F | | | N | 12 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 12 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | N | 12 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 12 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | N | 12 | 3 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 12 | 3 | |

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

BREXPIPRAZOLE 15 OF 42 PROTOCOL 331-201-00061 STAT-3.4.2 MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy W vs. Dummy Z BY MPLC25FL AT Phase B Placebo Center Combat 25% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) (N) Row1 900 12 AVISIT\*TRTPN\*MPLC25F Y 12 900 AVISIT\*TRTPN\*MPLC25F 3 BASE\*AVISITN 6 BASE\*AVISITN 10 BASE\*AVISITN BASE\*AVISITN 12

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL



BREXPIPRAZOLE 17 OF 42 PROTOCOL 331-201-00061 STAT-3.4.2 MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT --------The Mixed Procedure Coefficients for Dummy W vs. Dummy Y BY MPLC25FL AT Phase B Placebo Center Combat 25% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 TRTPN 2 TRTPN TRTPN 900 TRTPN 3 AVISITN\*TRTPN 1 AVISITN\*TRTPN 2 AVISITN\*TRTPN AVISITN\*TRTPN 900 6 AVISITN\*TRTPN 6 AVISITN\*TRTPN 2 6 AVISITN\*TRTPN 6 900 AVISITN\*TRTPN AVISITN\*TRTPN 10 1 AVISITN\*TRTPN 10 2 AVISITN\*TRTPN 10 AVISITN\*TRTPN 10 900 AVISITN\*TRTPN 12

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

BREXPIPRAZOLE 18 OF 42 PROTOCOL 331-201-00061 STAT-3.4.2 MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy W vs. Dummy Y BY MPLC25FL AT Phase B Placebo Center Combat 25% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 12 2 AVISITN\*TRTPN 12 AVISITN\*TRTPN 900 AVISITN\*TRTPN 12 MPLC25FL N MPLC25FL Y AVISITN\*MPLC25FL N 3 AVISITN\*MPLC25FL AVISITN\*MPLC25FL N AVISITN\*MPLC25FL Y 6 AVISITN\*MPLC25FL N 10 Y 10 AVISITN\*MPLC25FL AVISITN\*MPLC25FL 12 N Y AVISITN\*MPLC25FL 12 TRTPN\*MPLC25FL N TRTPN\*MPLC25FL Y TRTPN\*MPLC25FL N

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

TRTPN\*MPLC25FL

BREXPIPRAZOLE 19 OF 42 PROTOCOL 331-201-00061 STAT-3.4.2 MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ----- Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy W vs. Dummy Y BY MPLC25FL AT Phase B Placebo Center Combat 25% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 TRTPN\*MPLC25FL N -1 Υ TRTPN\*MPLC25FL 1 TRTPN\*MPLC25FL N 900 Y 900 TRTPN\*MPLC25FL 3 AVISIT\*TRTPN\*MPLC25F N 1 AVISIT\*TRTPN\*MPLC25F Y 1 AVISIT\*TRTPN\*MPLC25F AVISIT\*TRTPN\*MPLC25F Y AVISIT\*TRTPN\*MPLC25F N 3 Y AVISIT\*TRTPN\*MPLC25F 3 AVISIT\*TRTPN\*MPLC25F N 900

Y

N

Y

N

Y

3

6

6

6

6

900

1

1

2

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

AVISIT\*TRTPN\*MPLC25F

AVISIT\*TRTPN\*MPLC25F

AVISIT\*TRTPN\*MPLC25F

AVISIT\*TRTPN\*MPLC25F

AVISIT\*TRTPN\*MPLC25F

AVISIT\*TRTPN\*MPLC25F

BREXPIPRAZOLE
\_\_\_\_STAT-3.4.2

MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Placebo

Coefficients for Dummy W vs. Dummy Y BY MPLC25FL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | 25%<br>Responder<br>Population<br>Flag in | | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*MPLC25F | | | Y | 6 | 3 | |
| AVISIT*TRTPN*MPLC25F | | | N | 6 | 900 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 6 | 900 | |
| AVISIT*TRTPN*MPLC25F | | | N | 10 | 1 | 1 |
| AVISIT*TRTPN*MPLC25F | | | Y | 10 | 1 | -1 |
| AVISIT*TRTPN*MPLC25F | | | N | 10 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 10 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | N | 10 | 3 | -1 |
| AVISIT*TRTPN*MPLC25F | | | Y | 10 | 3 | 1 |
| AVISIT*TRTPN*MPLC25F | | | N | 10 | 900 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 10 | 900 | |
| AVISIT*TRTPN*MPLC25F | | | N | 12 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 12 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | N | 12 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 12 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | N | 12 | 3 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 12 | 3 | |

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

BREXPIPRAZOLE 21 OF 42 PROTOCOL 331-201-00061 STAT-3.4.2 MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy W vs. Dummy Y BY MPLC25FL AT Phase B Placebo Center Combat 25% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) (N) Row1 900 12 AVISIT\*TRTPN\*MPLC25F Y 12 900 AVISIT\*TRTPN\*MPLC25F 3 BASE\*AVISITN 6 BASE\*AVISITN 10 BASE\*AVISITN BASE\*AVISITN 12

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL



BREXPIPRAZOLE 23 OF 42 PROTOCOL 331-201-00061 STAT-3.4.2 MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy W vs. Dummy X BY MPLC25FL AT Phase B Placebo Center Combat 25% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 TRTPN 2 TRTPN TRTPN 3 900 TRTPN 3 AVISITN\*TRTPN 1 AVISITN\*TRTPN 2 AVISITN\*TRTPN AVISITN\*TRTPN 900 6 AVISITN\*TRTPN 1 6 AVISITN\*TRTPN 2 6 AVISITN\*TRTPN 6 900 AVISITN\*TRTPN AVISITN\*TRTPN 10 1 AVISITN\*TRTPN 10 2 AVISITN\*TRTPN 10 AVISITN\*TRTPN 10 900 AVISITN\*TRTPN 12

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

-1

-1

BREXPIPRAZOLE 24 OF 42 PROTOCOL 331-201-00061 STAT-3.4.2 MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy W vs. Dummy X BY MPLC25FL AT Phase B Placebo Center Combat 25% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 12 2 AVISITN\*TRTPN 12 AVISITN\*TRTPN 900 AVISITN\*TRTPN 12 MPLC25FL N MPLC25FL Y AVISITN\*MPLC25FL N 3 AVISITN\*MPLC25FL AVISITN\*MPLC25FL N AVISITN\*MPLC25FL Y 6 AVISITN\*MPLC25FL N 10 Y 10 AVISITN\*MPLC25FL AVISITN\*MPLC25FL 12 N AVISITN\*MPLC25FL Y 12 TRTPN\*MPLC25FL N

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

TRTPN\*MPLC25FL

TRTPN\*MPLC25FL

TRTPN\*MPLC25FL

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.

Y

N

BREXPIPRAZOLE

STAT-3.4.2

MMRM Output for Test on Treatment by (Intent to Treat Sample)

STAT-3.4.2

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY MPLC25FL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Placebo<br>25%<br>Responder<br>Population<br>Flag in | | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*MPLC25FL | | | N | | 3 | |
| TRTPN*MPLC25FL | | | Y | | 2 | |
| TRTPN*MPLC25FL | | | N | | 900 | |
| | | | N<br>Y | | | |
| TRTPN*MPLC25FL | | | = | 2 | 900 | |
| AVISIT*TRTPN*MPLC25F | | | N | 3 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 3 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | N | 3 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 3 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | N | 3 | 3 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 3 | 3 | |
| AVISIT*TRTPN*MPLC25F | | | N | 3 | 900 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 3 | 900 | |
| AVISIT*TRTPN*MPLC25F | | | N | 6 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 6 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | N | 6 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 6 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | N | 6 | 3 | |

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL


MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY MPLC25FL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Placebo<br>25%<br>Responder<br>Population<br>Flag in | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*M | PLC25F | | Y | 6 | 3 | |
| AVISIT*TRTPN*M | PLC25F | | N | 6 | 900 | |
| AVISIT*TRTPN*M | PLC25F | | Y | 6 | 900 | |
| AVISIT*TRTPN*M | PLC25F | | N | 10 | 1 | 1 |
| AVISIT*TRTPN*M | PLC25F | | Y | 10 | 1 | -1 |
| AVISIT*TRTPN*M | PLC25F | | N | 10 | 2 | -1 |
| AVISIT*TRTPN*M | PLC25F | | Y | 10 | 2 | 1 |
| AVISIT*TRTPN*M | PLC25F | | N | 10 | 3 | |
| AVISIT*TRTPN*M | PLC25F | | Y | 10 | 3 | |
| AVISIT*TRTPN*M | PLC25F | | N | 10 | 900 | |
| AVISIT*TRTPN*M | PLC25F | | Y | 10 | 900 | |
| AVISIT*TRTPN*M | PLC25F | | N | 12 | 1 | |
| AVISIT*TRTPN*M | PLC25F | | Y | 12 | 1 | |
| AVISIT*TRTPN*M | PLC25F | | N | 12 | 2 | |
| AVISIT*TRTPN*M | PLC25F | | Y | 12 | 2 | |
| AVISIT*TRTPN*M | PLC25F | | N | 12 | 3 | |
| AVISIT*TRTPN*M | PLC25F | | Y | 12 | 3 | |

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

BREXPIPRAZOLE 27 OF 42 PROTOCOL 331-201-00061 STAT-3.4.2 MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy W vs. Dummy X BY MPLC25FL AT Phase B Placebo Center Combat 25% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) (N) Row1 900 12 AVISIT\*TRTPN\*MPLC25F Y 12 900 AVISIT\*TRTPN\*MPLC25F BASE\*AVISITN 3 6 BASE\*AVISITN 10 BASE\*AVISITN BASE\*AVISITN 12

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL



BREXPIPRAZOLE 29 OF 42 PROTOCOL 331-201-00061 STAT-3.4.2 MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy X vs. Dummy Z BY MPLC25FL AT Phase B Placebo Center Combat 25% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 TRTPN 2 TRTPN TRTPN 900 TRTPN 3 AVISITN\*TRTPN 1 AVISITN\*TRTPN 2 AVISITN\*TRTPN AVISITN\*TRTPN 900 6 AVISITN\*TRTPN 6 AVISITN\*TRTPN 2 6 AVISITN\*TRTPN 6 900 AVISITN\*TRTPN AVISITN\*TRTPN 10 1 AVISITN\*TRTPN 10 2 AVISITN\*TRTPN 10 AVISITN\*TRTPN 10 900 AVISITN\*TRTPN 12

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

BREXPIPRAZOLE 30 OF 42 PROTOCOL 331-201-00061 STAT-3.4.2 MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT ------------The Mixed Procedure Coefficients for Dummy X vs. Dummy Z BY MPLC25FL AT Phase B Placebo Center Combat 25% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 12 2 AVISITN\*TRTPN 12 AVISITN\*TRTPN 900 AVISITN\*TRTPN 12 MPLC25FL N MPLC25FL Y AVISITN\*MPLC25FL N 3 AVISITN\*MPLC25FL AVISITN\*MPLC25FL N AVISITN\*MPLC25FL Y 6 AVISITN\*MPLC25FL N 10 Y 10 AVISITN\*MPLC25FL AVISITN\*MPLC25FL 12 N AVISITN\*MPLC25FL Y 12 TRTPN\*MPLC25FL N TRTPN\*MPLC25FL Y

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

TRTPN\*MPLC25FL

TRTPN\*MPLC25FL

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.

N

BREXPIPRAZOLE

MMRM Output for Test on Treatment by STAT-3.4.2
25 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

Parameter Code=CAPSTOT -----The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY MPLC25FL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Placebo<br>25%<br>Responder<br>Population<br>Flag in | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*MPLC25FL | | | N | | 3 | |
| TRTPN*MPLC25FL | | | Y | | 3 | |
| TRTPN*MPLC25FL | | | N | | 900 | -1 |
| TRTPN*MPLC25FL | | | Y | | 900 | 1 |
| AVISIT*TRTPN*MPLC25F | | | N | 3 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 3 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | N | 3 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 3 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | N | 3 | 3 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 3 | 3 | |
| AVISIT*TRTPN*MPLC25F | | | N | 3 | 900 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 3 | 900 | |
| AVISIT*TRTPN*MPLC25F | | | N | 6 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 6 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | N | 6 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 6 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | N | 6 | 3 | |

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

BREXPIPRAZOLE 32 OF 42 PROTOCOL 331-201-00061

MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY MPLC25FL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Placebo<br>25%<br>Responder<br>Population<br>Flag in | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*MPLC25F | | | Y | 6 | 3 | |
| AVISIT*TRTPN*MPLC25F | | | N | 6 | 900 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 6 | 900 | |
| AVISIT*TRTPN*MPLC25F | | | N | 10 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 10 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | N | 10 | 2 | 1 |
| AVISIT*TRTPN*MPLC25F | | | Y | 10 | 2 | -1 |
| AVISIT*TRTPN*MPLC25F | | | N | 10 | 3 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 10 | 3 | |
| AVISIT*TRTPN*MPLC25F | | | N | 10 | 900 | -1 |
| AVISIT*TRTPN*MPLC25F | | | Y | 10 | 900 | 1 |
| AVISIT*TRTPN*MPLC25F | | | N | 12 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 12 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | N | 12 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 12 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | N | 12 | 3 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 12 | 3 | |

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

BREXPIPRAZOLE 33 OF 42 PROTOCOL 331-201-00061 STAT-3.4.2 MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy X vs. Dummy Z BY MPLC25FL AT Phase B Placebo Center Combat 25% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) (N) Row1 900 12 AVISIT\*TRTPN\*MPLC25F Y 12 900 AVISIT\*TRTPN\*MPLC25F 3 BASE\*AVISITN 6 BASE\*AVISITN 10 BASE\*AVISITN BASE\*AVISITN 12

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL



BREXPIPRAZOLE 35 OF 42 PROTOCOL 331-201-00061 STAT-3.4.2 MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy Y vs. Dummy Z BY MPLC25FL AT Phase B Placebo Center Combat 25% (Pooled Related Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 TRTPN 2 TRTPN TRTPN 900 TRTPN 3 AVISITN\*TRTPN 1 AVISITN\*TRTPN 2 AVISITN\*TRTPN AVISITN\*TRTPN 900 6 AVISITN\*TRTPN 6 AVISITN\*TRTPN 2 6 AVISITN\*TRTPN 6 900 AVISITN\*TRTPN AVISITN\*TRTPN 10 1 AVISITN\*TRTPN 10 2 AVISITN\*TRTPN 10 AVISITN\*TRTPN 10 900 AVISITN\*TRTPN 12

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

| Coefficients | for | Dummy | Υ | vs. | Dummy | Z | BY | MPLC25FL | AΤ | Phase | В |
|---|---|---|---|---|---|---|---|---|---|---|---|

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Placebo<br>25%<br>Responder<br>Population<br>Flag in | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRIPN | | | | 12 | 3 | |
| AVISIIN"IRIPN<br>AVISITN*TRTPN | | | | 12 | 900 | |
| MPLC25FL | | | N | 12 | 900 | |
| MPLC25FL | | | Y<br>Y | | | |
| AVISITN*MPLC25FL | | | N | 3 | | |
| AVISITN*MPLC25FL | | | Y<br>Y | 3 | | |
| AVISITN*MPLC25FL | | | N | 6 | | |
| AVISITN MPLC25FL<br>AVISITN MPLC25FL | | | N<br>Y | 6 | | |
| | | | = | - | | |
| AVISITN*MPLC25FL | | | N | 10 | | |
| AVISITN*MPLC25FL | | | Y | 10 | | |
| AVISITN*MPLC25FL | | | N | 12 | | |
| AVISITN*MPLC25FL | | | Y | 12 | | |
| TRTPN*MPLC25FL | | | N | | 1 | |
| TRTPN*MPLC25FL | | | Y | | 1 | |
| TRTPN*MPLC25FL | | | N | | 2 | |
| TRTPN*MPLC25FL | | | Y | | 2 | |

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

BREXPIPRAZOLE 37 OF 42 PROTOCOL 331-201-00061 STAT-3.4.2 MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy Y vs. Dummy Z BY MPLC25FL AT Phase B Placebo Center Combat 25% Related (Pooled Responder Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag in (N) Row1 TRTPN\*MPLC25FL N Υ -1 TRTPN\*MPLC25FL -1 TRTPN\*MPLC25FL N 900 Y 900 1 TRTPN\*MPLC25FL 3 AVISIT\*TRTPN\*MPLC25F N 1 AVISIT\*TRTPN\*MPLC25F Y 1 AVISIT\*TRTPN\*MPLC25F AVISIT\*TRTPN\*MPLC25F Y N 3 3 AVISIT\*TRTPN\*MPLC25F Y AVISIT\*TRTPN\*MPLC25F 3

N

Y

N

Y

N

Y

900

900

1

1

2

3

6

6

6

6

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

AVISIT\*TRTPN\*MPLC25F

AVISIT\*TRTPN\*MPLC25F

AVISIT\*TRTPN\*MPLC25F

AVISIT\*TRTPN\*MPLC25F

AVISIT\*TRTPN\*MPLC25F

AVISIT\*TRTPN\*MPLC25F

AVISIT\*TRTPN\*MPLC25F

BREXPIPRAZOLE 38 OF 42 PROTOCOL 331-201-00061

MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Placebo

Coefficients for Dummy Y vs. Dummy Z BY MPLC25FL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | 25%<br>Responder<br>Population<br>Flag in | Visit | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*MPLC25F | | | Y | 6 | 3 | |
| AVISIT*TRTPN*MPLC25F | | | N | 6 | 900 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 6 | 900 | |
| AVISIT*TRTPN*MPLC25F | | | N | 10 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 10 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | N | 10 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 10 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | N | 10 | 3 | 1 |
| AVISIT*TRTPN*MPLC25F | | | Y | 10 | 3 | -1 |
| AVISIT*TRTPN*MPLC25F | | | N | 10 | 900 | -1 |
| AVISIT*TRTPN*MPLC25F | | | Y | 10 | 900 | 1 |
| AVISIT*TRTPN*MPLC25F | | | N | 12 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 12 | 1 | |
| AVISIT*TRTPN*MPLC25F | | | N | 12 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 12 | 2 | |
| AVISIT*TRTPN*MPLC25F | | | N | 12 | 3 | |
| AVISIT*TRTPN*MPLC25F | | | Y | 12 | 3 | |

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL



|---|---|---|---|---|---|---|---|---|---|---|---|
| FRO10001 331-201-00001 | | for Test on | Treatment by | 25 P | -3.4.2<br>ercent Impro<br>Treat Sample | | ubgroup Int | eraction | | | |
| | | | | Parameter ( | Code=CAPSTOT | | | | | | |
| | | | | The Mixed | Procedure | | | | | | |
| | | | | Esti | mates | | | | | | |
| I | Label | | | | Estimate | Standa:<br>Err | | t Value | Pr > t | | |
| I | Dummy Y vs. Dum | my Z BY MPLC | 25FL AT Phase | В | 10.7966 | 4.18 | 52 236 | 2.58 | 0.0105 | | |
| | | | | Least Squ | ares Means | | | | | | |
| | Placebo<br>25%<br>Responder | Analysis | Planned | | | | | | | | |
| Effect | Population<br>Flag in | Visit<br>(N) | Treatment (N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISIT*TRTPN*MPLC25F | N<br>Y<br>N<br>Y<br>N<br>Y | 3<br>3<br>3<br>3<br>3<br>3<br>3 | 1<br>1<br>2<br>2<br>3<br>3<br>900<br>900 | -7.2255<br>-4.4651<br>-4.6549<br>-4.0945<br>-5.6543<br>-7.3251<br>-6.8317<br>-4.7339 | 1.3324<br>2.1735<br>1.5127<br>2.1624<br>1.4457<br>1.9363<br>1.3494<br>2.0506 | 283<br>281<br>287<br>277<br>283<br>275<br>282<br>280 | -5.42<br>-2.05<br>-3.08<br>-1.89<br>-3.91<br>-3.78<br>-5.06<br>-2.31 | <.0001<br>0.0409<br>0.0023<br>0.0593<br>0.0001<br>0.0002<br><.0001 | 0.05<br>0.05<br>0.05<br>0.05<br>0.05<br>0.05<br>0.05 | -9.8481 -8.7434 -7.6324 -8.3514 -8.4999 -11.1369 -9.4879 -8.7705 | -4.6029<br>-0.1868<br>-1.6775<br>0.1623<br>-2.8088<br>-3.5133<br>-4.1755<br>-0.6974 |
| AVISIT*TRTPN*MPLC25F<br>AVISIT*TRTPN*MPLC25F | Y<br>N | 6 | 1 | -4.7339<br>-13.8787 | 1.6391 | 280 | -2.31<br>-8.47 | <.0001 | 0.05 | -8.7705<br>-17.1056 | -10.6518 |

MMRM Output for Test on Treatment by 25 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

------

The Mixed Procedure

Least Squares Means

| | Placebo<br>25% | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Responder<br>Population | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
| Effect | Flag in | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISIT*TRTPN*MPLC25F | Y | 6 | 1 | -9.5963 | 2.6507 | 263 | -3.62 | 0.0004 | 0.05 | -14.8156 | -4.3770 |
| AVISIT*TRTPN*MPLC25F | N | 6 | 2 | -9.5472 | 1.7916 | 280 | -5.33 | <.0001 | 0.05 | -13.0740 | -6.0205 |
| AVISIT*TRTPN*MPLC25F | Y | 6 | 2 | -4.1451 | 2.7626 | 282 | -1.50 | 0.1346 | 0.05 | -9.5831 | 1.2928 |
| AVISIT*TRTPN*MPLC25F | N | 6 | 3 | -8.2811 | 1.7534 | 285 | -4.72 | <.0001 | 0.05 | -11.7324 | -4.8298 |
| AVISIT*TRTPN*MPLC25F | Y | 6 | 3 | -12.9846 | 2.4771 | 266 | -5.24 | <.0001 | 0.05 | -17.8618 | -8.1074 |
| AVISIT*TRTPN*MPLC25F | N | 6 | 900 | -10.0084 | 1.6245 | 276 | -6.16 | <.0001 | 0.05 | -13.2064 | -6.8103 |
| AVISIT*TRTPN*MPLC25F | Y | 6 | 900 | -6.1814 | 2.4363 | 250 | -2.54 | 0.0118 | 0.05 | -10.9797 | -1.3831 |
| AVISIT*TRTPN*MPLC25F | N | 10 | 1 | -16.9313 | 1.7597 | 241 | -9.62 | <.0001 | 0.05 | -20.3976 | -13.4651 |
| AVISIT*TRTPN*MPLC25F | Y | 10 | 1 | -15.2122 | 2.9293 | 250 | -5.19 | <.0001 | 0.05 | -20.9814 | -9.4431 |
| AVISIT*TRTPN*MPLC25F | N | 10 | 2 | -13.2205 | 1.9706 | 269 | -6.71 | <.0001 | 0.05 | -17.1004 | -9.3407 |
| AVISIT*TRTPN*MPLC25F | Y | 10 | 2 | -9.7336 | 3.0571 | 262 | -3.18 | 0.0016 | 0.05 | -15.7532 | -3.7140 |
| AVISIT*TRTPN*MPLC25F | N | 10 | 3 | -9.2971 | 1.8724 | 253 | -4.97 | <.0001 | 0.05 | -12.9846 | -5.6097 |
| AVISIT*TRTPN*MPLC25F | Y | 10 | 3 | -15.9835 | 2.7007 | 241 | -5.92 | <.0001 | 0.05 | -21.3036 | -10.6633 |
| AVISIT*TRTPN*MPLC25F | N | 10 | 900 | -11.6997 | 1.7509 | 256 | -6.68 | <.0001 | 0.05 | -15.1477 | -8.2516 |
| AVISIT*TRTPN*MPLC25F | Y | 10 | 900 | -7.5894 | 2.6480 | 233 | -2.87 | 0.0045 | 0.05 | -12.8065 | -2.3724 |
| AVISIT*TRTPN*MPLC25F | N | 12 | 1 | -17.5147 | 1.9377 | 248 | -9.04 | <.0001 | 0.05 | -21.3313 | -13.6982 |
| AVISIT*TRTPN*MPLC25F | Y | 12 | 1 | -16.8118 | 3.2050 | 252 | -5.25 | <.0001 | 0.05 | -23.1239 | -10.4998 |

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

AVISIT\*TRTPN\*MPLC25F Y

| BREXPIPRAZOLE | | | | | | | | | 42 | OF 42 | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | | | | STAT- | -3.4.2 | | | | | | |
| | MMRM Output | for Test on | Treatment by | | ercent Impro | | ubgroup Int | eraction | | | |
| | | | | (Intent to ' | Treat Sample | ) | | | | | |
| | | | | - Parameter ( | Code=CAPSTOT | | | | | | |
| Parameter Code=CAPSTOT | | | | | | | | | | | |
| | The Mixed Procedure | | | | | | | | | | |
| | | | | Least Squa | ares Means | | | | | | |
| | Placebo | | | | | | | | | | |
| | 25% | | | | | | | | | | |
| | Responder | Analysis | Planned | | | | | | | | |
| | Population | Visit | Treatment | | Standard | | | | | _ | |
| Effect | Flag in | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISIT*TRTPN*MPLC25F | N | 12 | 2 | -14.0994 | 2.1461 | 268 | -6.57 | <.0001 | 0.05 | -18.3247 | -9.8741 |
| AVISIT*TRTPN*MPLC25F | Y | 12 | 2 | -7.8705 | 3.3613 | 261 | -2.34 | 0.0200 | 0.05 | -14.4891 | -1.2519 |
| AVISIT*TRTPN*MPLC25F | N | 12 | 3 | -13.5835 | 2.0386 | 256 | -6.66 | <.0001 | 0.05 | -17.5981 | -9.5690 |
| AVISIT*TRTPN*MPLC25F | Y | 12 | 3 | -17.9995 | 2.9117 | 235 | -6.18 | <.0001 | 0.05 | -23.7359 | -12.2631 |
| AVISIT*TRTPN*MPLC25F | N | 12 | 900 | -12.8520 | 1.8880 | 252 | -6.81 | <.0001 | 0.05 | -16.5704 | -9.1336 |

-8.8701

3.0061 254

-2.95

0.0035 0.05 -14.7901

-2.9501

FILE: stat2d2.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.2 FINAL

12

BREXPIPRAZOLE 1 OF 39 PROTOCOL 331-201-00061 MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction (Intent to Treat Sample) The Mixed Procedure Model Information Data Set
Dependent Variable
Covariance Structure WORK.INDATA CHG Unstructured SUBJID Estimation Method REML Residual Variance Method Fixed Effects SE Method Kenward-Roger Degrees of Freedom Method Kenward-Roger Class Level Information Class Levels Values AVISITN 4 3 6 10 12 1 2 3 900 TRTPN 4 POOLCNTR 10 COMBFL 2 NY

FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL



FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL





FILE: stat2d3.1is, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL



FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL





FILE: stat2d3.1is, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL



FILE: stat2d3.1is, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL

BREXPIPRAZOLE 7 OF 39 PROTOCOL 331-201-00061 STAT-3.4.3 MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction (Intent to Treat Sample) The Mixed Procedure Iteration History Iteration Evaluations -2 Res Log Like Criterion 7337.68028425 0 1 2 6868.62941909 0.00042848 1 6867.41753019 0.00001401 6867.38081232 3 1 0.00000002 6867.38076515 1 0.00000000 Convergence criteria met. Covariance Parameter Estimates Cov Parm Subject Estimate SUBJID 77.6215 UN(1,1) UN(2,1) SUBJID 51.7432 UN(2,2) SUBJID 112.81 UN(3,1) SUBJID 42.7606 UN(3,2) SUBJID 88.8408 UN(3,3) SUBJID 124.03 UN (4,1) SUBJID 47.7890

FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL

BREXPIPRAZOLE 8 OF 39 PROTOCOL 331-201-00061 STAT-3.4.3 MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction (Intent to Treat Sample) The Mixed Procedure Covariance Parameter Estimates Cov Parm Subject Estimate 89.4074 UN(4,2) SUBJID UN(4,3) SUBJID UN(4,4) SUBJID SUBJID 104.80 147.63 Fit Statistics -2 Res Log Likelihood 6867.4 AIC (Smaller is Better) 6887.4 AICC (Smaller is Better) 6887.6 BIC (Smaller is Better) 6924.4 Null Model Likelihood Ratio Test Chi-Square Pr > ChiSq

470.30

<.0001

FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL

BREXPIPRAZOLE

STAT-3.4.3

MMRM Output for Test on Treatment by (Intent to Treat Sample)

Parameter Code=CAPSTOT

Parameter Code=CAPSTOT

The Mixed Procedure

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|----------------------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| POOLCNTR | 9 | 278 | 1.71 | 0.0869 |
| COMBFL | 1 | 279 | 3.56 | 0.0601 |
| AVISITN | 3 | 227 | 0.97 | 0.4081 |
| TRTPN | 3 | 272 | 3.79 | 0.0109 |
| AVISITN*TRTPN | 9 | 360 | 1.60 | 0.1130 |
| MITTFL | 1 | 273 | 0.00 | 0.9968 |
| AVISITN*MITTFL | 3 | 237 | 0.18 | 0.9112 |
| TRTPN*MITTFL | 3 | 273 | 2.41 | 0.0674 |
| AVISITN*TRTPN*MITTFL | 9 | 360 | 0.34 | 0.9629 |
| BASE*AVISITN | 4 | 240 | 6.54 | <.0001 |

FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL



FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL

BREXPIPRAZOLE 11 OF 39 PROTOCOL 331-201-00061 STAT-3.4.3 MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy W vs. Dummy Z BY MITTFL AT Phase B Modified Center Combat (Pooled Related Planned ITT Analysis Population Population Visit Center) Treatment Effect for ITT Flag Flag (N) (N) Row1 TRTPN 2 TRTPN 900 TRTPN 3 AVISITN\*TRTPN 1 AVISITN\*TRTPN 3 2 AVISITN\*TRTPN 3 3 AVISITN\*TRTPN 3 900 AVISITN\*TRTPN AVISITN\*TRTPN 6 AVISITN\*TRTPN AVISITN\*TRTPN 6 900 10 AVISITN\*TRTPN 1 10 AVISITN\*TRTPN 2 AVISITN\*TRTPN 10 3 AVISITN\*TRTPN 10 900 AVISITN\*TRTPN 12 1

FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL

AVISITN\*TRTPN

AVISITN\*TRTPN

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.

12

12

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY MITTFL AT Phase B

| (Pooled Related ITT Analysis Planned Center) Population Population Visit Treatment Effect for ITT Flag Flag (N) (N) | Row1 |
|---|---|
| | Row1 |
| Effort for TEM Flor Flor (N) (N) | Row1 |
| Effect for its flag flag (N) (N) | |
| AVISITN*TRTPN 12 900 | |
| MITTFL | |
| MITTFL | |
| AVISITN*MITTFL N 3 | |
| AVISITN*MITTFL Y 3 | |
| AVISITN*MITTFL N 6 | |
| AVISITN*MITTFL Y 6 | |
| AVISITN*MITTFL N 10 | |
| AVISITN*MITTFL Y 10 | |
| AVISITN*MITTFL N 12 | |
| AVISITN*MITTFL Y 12 | |
| TRTPN*MITTFL N 1 | 1 |
| TRTPN*MITTFL Y 1 | -1 |
| TRTPN*MITTFL N 2 | |
| TRTPN*MITTFL Y 2 | |
| TRTPN*MITTFL N 3 | |
| TRTPN*MITTFL Y 3 | |
| TRTPN*MITTFL N 900 | -1 |

FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL

BREXPIPRAZOLE 13 OF 39
\_\_\_\_\_STAT-3.4.3

MMRM Output for Test on Treatment by (Intent to Treat Sample) (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY MITTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Modified<br>ITT<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*MITTFL | | | Y | | 900 | 1 |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 1 | |
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 1 | |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 2 | |
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 2 | |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 3 | |
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 3 | |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 900 | |
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 900 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 1 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 1 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 2 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 2 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 3 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 3 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 900 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 900 | |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 1 | 1 |

FILE: stat2d3.1is, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL


MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY MITTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Modified<br>ITT<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 1 | -1 |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 2 | |
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 2 | |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 3 | |
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 3 | |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 900 | -1 |
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 900 | 1 |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 1 | |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 1 | |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 2 | |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 2 | |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 3 | |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 3 | |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 900 | |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |

FILE: stat2d3.1is, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL



FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL



FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL

BREXPIPRAZOLE 17 OF 39 PROTOCOL 331-201-00061 STAT-3.4.3 MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy W vs. Dummy Y BY MITTFL AT Phase B Modified Center Combat (Pooled Related Planned ITT Analysis Center) Population Population Visit Treatment Effect for ITT Flag Flag (N) (N) Row1 AVISITN\*TRTPN 6 2 AVISITN\*TRTPN 6 6 900 AVISITN\*TRTPN AVISITN\*TRTPN 10 1 10 AVISITN\*TRTPN 2 AVISITN\*TRTPN 10 AVISITN\*TRTPN 10 900 AVISITN\*TRTPN 12 AVISITN\*TRTPN 12 12 AVISITN\*TRTPN 12 AVISITN\*TRTPN 900 MITTFL N

Y

N

Y

N

Y

3

3

6

6

10

FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL

MITTFL

AVISITN\*MITTFL

AVISITN\*MITTFL

AVISITN\*MITTFL

AVISITN\*MITTFL

AVISITN\*MITTFL


MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

\_\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY MITTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Modified<br>ITT<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*MITTFL | | | Y | 10 | | |
| AVISITN*MITTFL | | | N | 12 | | |
| AVISITN*MITTFL | | | Y | 12 | | |
| TRTPN*MITTFL | | | N | | 1 | 1 |
| TRTPN*MITTFL | | | Y | | 1 | -1 |
| TRTPN*MITTFL | | | N | | 2 | |
| TRTPN*MITTFL | | | Y | | 2 | |
| TRTPN*MITTFL | | | N | | 3 | -1 |
| TRTPN*MITTFL | | | Y | | 3 | 1 |
| TRTPN*MITTFL | | | N | | 900 | |
| TRTPN*MITTFL | | | Y | | 900 | |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 1 | |
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 1 | |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 2 | |
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 2 | |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 3 | |
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 3 | |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 900 | |

FILE: stat2d3.1is, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL

BREXPIPRAZOLE 19 OF 39

MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY MITTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Modified<br>ITT<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 900 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 1 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 1 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 2 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 2 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 3 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 3 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 900 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 900 | |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 1 | 1 |
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 1 | -1 |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 2 | |
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 2 | |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 3 | -1 |
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 3 | 1 |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 900 | |
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 900 | |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 1 | |

FILE: stat2d3.1is, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL


STAT-3.4.3

MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY MITTFL AT Phase B

| | Center | Combat | Modified | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | ITT | Analysis | Planned | |
| | Center) | Population | Population | Visit | Treatment | |
| Effect | for ITT | Flag | Flag | (N) | (N) | Row1 |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 1 | |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 2 | |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 2 | |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 3 | |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 3 | |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 900 | |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |
| BASE*AVISITN | | | | 12 | | |

FILE: stat2d3.1is, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL



FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL

BREXPIPRAZOLE 22 OF 39 PROTOCOL 331-201-00061 STAT-3.4.3 MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy W vs. Dummy X BY MITTFL AT Phase B Modified Center Combat (Pooled Related Planned ITT Analysis Population Population Visit Center) Treatment Effect for ITT Flag Flag (N) (N) Row1 TRTPN 2 TRTPN 900 TRTPN 3 AVISITN\*TRTPN 1 3 AVISITN\*TRTPN 2 AVISITN\*TRTPN 3 3 AVISITN\*TRTPN 3 900 AVISITN\*TRTPN AVISITN\*TRTPN 6 AVISITN\*TRTPN AVISITN\*TRTPN 6 900 10 AVISITN\*TRTPN 1

10

10

10

12

12

12

2

3

1

900

FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL

AVISITN\*TRTPN

AVISITN\*TRTPN

AVISITN\*TRTPN

AVISITN\*TRTPN

AVISITN\*TRTPN

AVISITN\*TRTPN

BREXPIPRAZOLE 23 OF 39 PROTOCOL 331-201-00061 STAT-3.4.3 MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy W vs. Dummy X BY MITTFL AT Phase B Center Combat Modified (Pooled Related Planned ITT Analysis Center) Population Population Visit Treatment Effect for ITT Flag Flag (N) (N) Row1 AVISITN\*TRTPN 12 900 MITTFL N Υ MITTFL 3 AVISITN\*MITTFL N AVISITN\*MITTFL Y 3 AVISITN\*MITTFL N 6 AVISITN\*MITTFL Y AVISITN\*MITTFL 10 Y AVISITN\*MITTFL 10 N 12 AVISITN\*MITTFL Y 12 AVISITN\*MITTFL TRTPN\*MITTFL N 1 Y -1 TRTPN\*MITTFL 1 TRTPN\*MITTFL N -1 Y TRTPN\*MITTFL TRTPN\*MITTFL N

FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL

TRTPN\*MITTFL

TRTPN\*MITTFL

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.

Y

900

BREXPIPRAZOLE 24 OF 39
\_\_\_\_\_STAT-3.4.3

MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY MITTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Modified<br>ITT<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*MITTFL | | | Y | | 900 | |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 1 | |
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 1 | |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 2 | |
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 2 | |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 3 | |
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 3 | |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 900 | |
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 900 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 1 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 1 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 2 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 2 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 3 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 3 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 900 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 900 | |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 1 | 1 |

FILE: stat2d3.1is, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL


MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY MITTFL AT Phase B

| | Center | Combat | Modified | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | ITT | Analysis | Planned | |
| | Center) | Population | Population | Visit | Treatment | |
| Effect | for ITT | Flag | Flag | (N) | (N) | Row1 |
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 1 | -1 |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 2 | -1 |
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 2 | 1 |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 3 | |
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 3 | |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 900 | |
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 900 | |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 1 | |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 1 | |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 2 | |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 2 | |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 3 | |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 3 | |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 900 | |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |

FILE: stat2d3.1is, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL



FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL



FILE: stat2d3.1is, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL

BREXPIPRAZOLE 28 OF 39 PROTOCOL 331-201-00061 STAT-3.4.3 MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy X vs. Dummy Z BY MITTFL AT Phase B Modified Center Combat (Pooled Related Planned ITT Analysis Center) Population Population Visit Treatment Effect for ITT Flag Flag (N) (N) Row1 AVISITN\*TRTPN 6 2 AVISITN\*TRTPN 6 6 900 AVISITN\*TRTPN AVISITN\*TRTPN 10 10 AVISITN\*TRTPN 2 AVISITN\*TRTPN 10 AVISITN\*TRTPN 10 900 AVISITN\*TRTPN 12 AVISITN\*TRTPN 12 12 AVISITN\*TRTPN 12 AVISITN\*TRTPN 900 MITTFL N Y MITTFL 3 AVISITN\*MITTFL N

FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL

AVISITN\*MITTFL

AVISITN\*MITTFL

AVISITN\*MITTFL

AVISITN\*MITTFL

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.

Y

N

Y

3

6

6

10

BREXPIPRAZOLE
STAT-3.4.3
MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction

(Intent to Treat Sample)

## The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY MITTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Modified<br>ITT<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*MITTFL | | | Y | 10 | | |
| AVISITN*MITTFL | | | N | 12 | | |
| AVISITN*MITTFL | | | Y | 12 | | |
| TRTPN*MITTFL | | | N | | 1 | |
| TRTPN*MITTFL | | | Y | | 1 | |
| TRTPN*MITTFL | | | N | | 2 | 1 |
| TRTPN*MITTFL | | | Y | | 2 | -1 |
| TRTPN*MITTFL | | | N | | 3 | |
| TRTPN*MITTFL | | | Y | | 3 | |
| TRTPN*MITTFL | | | N | | 900 | -1 |
| TRTPN*MITTFL | | | Y | | 900 | 1 |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 1 | |
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 1 | |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 2 | |
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 2 | |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 3 | |
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 3 | |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 900 | |

FILE: stat2d3.1is, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL


MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY MITTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Modified<br>ITT<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 900 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 1 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 1 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 2 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 2 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 3 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 3 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 900 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 900 | |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 1 | |
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 1 | |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 2 | 1 |
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 2 | -1 |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 3 | |
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 3 | |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 900 | -1 |
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 900 | 1 |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 1 | |

FILE: stat2d3.1is, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL

BREXPIPRAZOLE 31 OF 39
\_\_\_\_\_STAT-3.4.3

MMRM Output for Test on Treatment by (Intent to Treat Sample) (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY MITTFL AT Phase B

| | Center<br>(Pooled | Combat<br>Related | Modified<br>ITT | Analysis | Planned | |
|---|---|---|---|---|---|---|
| | Center) | Population | Population | Visit | Treatment | |
| Effect | for ITT | Flag | Flag | (N) | (N) | Row1 |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 1 | |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 2 | |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 2 | |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 3 | |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 3 | |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 900 | |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |
| BASE*AVISITN | | | | 12 | | |

FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL



FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL

BREXPIPRAZOLE 33 OF 39 PROTOCOL 331-201-00061 STAT-3.4.3 MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy Y vs. Dummy Z BY MITTFL AT Phase B Modified Center Combat (Pooled Related Planned ITT Analysis Population Population Visit Center) Treatment Effect for ITT Flag Flag (N) (N) Row1 TRTPN TRTPN 900 TRTPN 3 AVISITN\*TRTPN 1 3 AVISITN\*TRTPN 2 AVISITN\*TRTPN 3 3 AVISITN\*TRTPN 3 900 AVISITN\*TRTPN AVISITN\*TRTPN 6 AVISITN\*TRTPN AVISITN\*TRTPN 6 900 10 AVISITN\*TRTPN 1 10 AVISITN\*TRTPN 2 AVISITN\*TRTPN 10 3 AVISITN\*TRTPN 10 900 AVISITN\*TRTPN 12 1 AVISITN\*TRTPN 12

FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL

AVISITN\*TRTPN

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.

12

BREXPIPRAZOLE

STAT-3.4.3

MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

## Coefficients for Dummy Y vs. Dummy Z BY MITTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 12 | 900 | |
| MITTFL | | | N | | | |
| MITTFL | | | Y | | | |
| AVISITN*MITTFL | | | N | 3 | | |
| AVISITN*MITTFL | | | Y | 3 | | |
| AVISITN*MITTFL | | | N | 6 | | |
| AVISITN*MITTFL | | | Y | 6 | | |
| AVISITN*MITTFL | | | N | 10 | | |
| AVISITN*MITTFL | | | Y | 10 | | |
| AVISITN*MITTFL | | | N | 12 | | |
| AVISITN*MITTFL | | | Y | 12 | | |
| TRTPN*MITTFL | | | N | | 1 | |
| TRTPN*MITTFL | | | Y | | 1 | |
| TRTPN*MITTFL | | | N | | 2 | |
| TRTPN*MITTFL | | | Y | | 2 | |
| TRTPN*MITTFL | | | N | | 3 | 1 |
| TRTPN*MITTFL | | | Y | | 3 | -1 |
| TRTPN*MITTFL | | | N | | 900 | -1 |

FILE: stat2d3.1is, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL
BREXPIPRAZOLE

STAT-3.4.3

MMRM Output for Test on Treatment by (Intent to Treat Sample)

(Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY MITTFL AT Phase B

| | Center | Combat | Modified | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | ITT | Analysis | Planned | |
| | Center) | Population | Population | Visit | Treatment | |
| Effect | for ITT | Flag | Flag | (N) | (N) | Row1 |
| TRTPN*MITTFL | | | Y | | 900 | 1 |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 1 | |
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 1 | |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 2 | |
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 2 | |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 3 | |
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 3 | |
| AVISITN*TRTPN*MITTFL | | | N | 3 | 900 | |
| AVISITN*TRTPN*MITTFL | | | Y | 3 | 900 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 1 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 1 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 2 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 2 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 3 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 3 | |
| AVISITN*TRTPN*MITTFL | | | N | 6 | 900 | |
| AVISITN*TRTPN*MITTFL | | | Y | 6 | 900 | |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 1 | |

FILE: stat2d3.1is, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL


MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY MITTFL AT Phase B

| | Center | Combat | Modified | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | ITT | Analysis | Planned | |
| | Center) | Population | Population | Visit | Treatment | |
| Effect | for ITT | Flag | Flag | (N) | (N) | Row1 |
| 3111 G T WILL WO W D W L W T W W W T | | | ., | 1.0 | 1 | |
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 1 | |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 2 | |
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 2 | |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 3 | 1 |
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 3 | -1 |
| AVISITN*TRTPN*MITTFL | | | N | 10 | 900 | -1 |
| AVISITN*TRTPN*MITTFL | | | Y | 10 | 900 | 1 |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 1 | |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 1 | |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 2 | |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 2 | |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 3 | |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 3 | |
| AVISITN*TRTPN*MITTFL | | | N | 12 | 900 | |
| AVISITN*TRTPN*MITTFL | | | Y | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |

FILE: stat2d3.1is, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL



FILE: stat2d3.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.4.3 FINAL


MMRM Output for Test on Treatment by 30 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Least Squares Means

| | Modified | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | ITT | Analysis | Planned | | | | | | | | |
| | Population | Visit | Treatment | | Standard | | | | | | |
| Effect | Flag | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN*MITTFL | N | 3 | 1 | -6.3081 | 2.3377 | 281 | -2.70 | 0.0074 | 0.05 | -10.9098 | -1.7063 |
| AVISITN*TRTPN*MITTFL | Y | 3 | 1 | -6.4610 | 1.2810 | 283 | -5.04 | <.0001 | 0.05 | -8.9824 | -3.9395 |
| AVISITN*TRTPN*MITTFL | N | 3 | 2 | -4.6231 | 2.3455 | 277 | -1.97 | 0.0497 | 0.05 | -9.2405 | -0.00574 |
| AVISITN*TRTPN*MITTFL | Y | 3 | 2 | -4.5219 | 1.4479 | 286 | -3.12 | 0.0020 | 0.05 | -7.3718 | -1.6720 |
| AVISITN*TRTPN*MITTFL | N | 3 | 3 | -10.4830 | 2.4267 | 274 | -4.32 | <.0001 | 0.05 | -15.2604 | -5.7056 |
| AVISITN*TRTPN*MITTFL | Y | 3 | 3 | -4.9620 | 1.2964 | 282 | -3.83 | 0.0002 | 0.05 | -7.5137 | -2.4102 |
| AVISITN*TRTPN*MITTFL | N | 3 | 900 | -4.5495 | 2.3128 | 275 | -1.97 | 0.0502 | 0.05 | -9.1026 | 0.003519 |
| AVISITN*TRTPN*MITTFL | Y | 3 | 900 | -6.7297 | 1.2793 | 283 | -5.26 | <.0001 | 0.05 | -9.2479 | -4.2115 |
| AVISITN*TRTPN*MITTFL | N | 6 | 1 | -12.9429 | 2.9131 | 266 | -4.44 | <.0001 | 0.05 | -18.6785 | -7.2073 |
| AVISITN*TRTPN*MITTFL | Y | 6 | 1 | -12.5088 | 1.5915 | 272 | -7.86 | <.0001 | 0.05 | -15.6421 | -9.3755 |
| AVISITN*TRTPN*MITTFL | N | 6 | 2 | -5.4177 | 3.0993 | 287 | -1.75 | 0.0815 | 0.05 | -11.5180 | 0.6826 |
| AVISITN*TRTPN*MITTFL | Y | 6 | 2 | -8.8230 | 1.7357 | 278 | -5.08 | <.0001 | 0.05 | -12.2398 | -5.4062 |
| AVISITN*TRTPN*MITTFL | N | 6 | 3 | -14.1987 | 3.2353 | 270 | -4.39 | <.0001 | 0.05 | -20.5682 | -7.8291 |
| AVISITN*TRTPN*MITTFL | Y | 6 | 3 | -8.5272 | 1.5912 | 281 | -5.36 | <.0001 | 0.05 | -11.6595 | -5.3950 |
| AVISITN*TRTPN*MITTFL | N | 6 | 900 | -6.7102 | 2.8408 | 253 | -2.36 | 0.0189 | 0.05 | -12.3048 | -1.1156 |
| AVISITN*TRTPN*MITTFL | Y | 6 | 900 | -9.5101 | 1.5471 | 272 | -6.15 | <.0001 | 0.05 | -12.5559 | -6.4643 |
| AVISITN*TRTPN*MITTFL | N | 10 | 1 | -16.6564 | 3.2365 | 255 | -5.15 | <.0001 | 0.05 | -23.0301 | -10.2828 |
| AVISITN*TRTPN*MITTFL | Y | 10 | 1 | -16.3297 | 1.6978 | 242 | -9.62 | <.0001 | 0.05 | -19.6740 | -12.9854 |


STAT-3.4.3

MMRM Output for Test on Treatment by \_\_\_\_\_\_30 Percent Improvement Subgroup Interaction (Intent to Treat Sample)

------

The Mixed Procedure

Least Squares Means

| | Modified | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | ITT | Analysis | Planned | | | | | | | | |
| | Population | Visit | Treatment | | Standard | | | | | | |
| Effect | Flag | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN*MITTFL | N | 10 | 2 | -10.5106 | 3.3829 | 262 | -3.11 | 0.0021 | 0.05 | -17.1718 | -3.8494 |
| AVISITN*TRTPN*MITTFL | Y | 10 | 2 | -12.7414 | 1.9093 | 271 | -6.67 | <.0001 | 0.05 | -16.5004 | -8.9825 |
| AVISITN*TRTPN*MITTFL | N | 10 | 3 | -17.1670 | 3.5139 | 239 | -4.89 | <.0001 | 0.05 | -24.0891 | -10.2448 |
| AVISITN*TRTPN*MITTFL | Y | 10 | 3 | -9.9125 | 1.6933 | 253 | -5.85 | <.0001 | 0.05 | -13.2473 | -6.5776 |
| AVISITN*TRTPN*MITTFL | N | 10 | 900 | -6.9406 | 3.1049 | 240 | -2.24 | 0.0263 | 0.05 | -13.0569 | -0.8243 |
| AVISITN*TRTPN*MITTFL | Y | 10 | 900 | -11.5135 | 1.6552 | 252 | -6.96 | <.0001 | 0.05 | -14.7732 | -8.2538 |
| AVISITN*TRTPN*MITTFL | N | 12 | 1 | -17.3439 | 3.5556 | 257 | -4.88 | <.0001 | 0.05 | -24.3457 | -10.3420 |
| AVISITN*TRTPN*MITTFL | Y | 12 | 1 | -17.2586 | 1.8696 | 249 | -9.23 | <.0001 | 0.05 | -20.9409 | -13.5763 |
| AVISITN*TRTPN*MITTFL | N | 12 | 2 | -8.7967 | 3.7268 | 263 | -2.36 | 0.0190 | 0.05 | -16.1349 | -1.4585 |
| AVISITN*TRTPN*MITTFL | Y | 12 | 2 | -13.3994 | 2.0839 | 270 | -6.43 | <.0001 | 0.05 | -17.5022 | -9.2967 |
| AVISITN*TRTPN*MITTFL | N | 12 | 3 | -18.9200 | 3.8443 | 242 | -4.92 | <.0001 | 0.05 | -26.4925 | -11.3474 |
| AVISITN*TRTPN*MITTFL | Y | 12 | 3 | -13.9110 | 1.8371 | 253 | -7.57 | <.0001 | 0.05 | -17.5290 | -10.2931 |
| AVISITN*TRTPN*MITTFL | N | 12 | 900 | -8.3293 | 3.4638 | 252 | -2.40 | 0.0169 | 0.05 | -15.1509 | -1.5077 |
| AVISITN*TRTPN*MITTFL | Y | 12 | 900 | -12.6593 | 1.8062 | 253 | -7.01 | <.0001 | 0.05 | -16.2163 | -9.1022 |

BREXPIPRAZOLE 1 OF 37 PROTOCOL 331-201-00061

------

The Mixed Procedure

Model Information

Data Set WORK.INDATA
Dependent Variable CHG
Covariance Structure Unstructured
Subject Effect SUBJID
Estimation Method REML
Residual Variance Method None

Fixed Effects SE Method Kenward-Roger Degrees of Freedom Method Kenward-Roger

Class Level Information

| Class | Levels | Values |
|------------------|--------|------------------------|
| AVISITN<br>TRTPN | 4<br>4 | 3 6 10 12<br>1 2 3 900 |
| POOLCNTR | 10 | |
| COMBFL | 2 | N Y |

FILE: stat2e.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.5 FINAL

BREXPIPRAZOLE
STAT-3.5

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

------

The Mixed Procedure



FILE: stat2e.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.5 FINAL

BREXPIPRAZOLE

STAT-3.5

MMRM Output for Test on Treatment by Type of Trauma Interaction
(Intent to Treat Sample)

The Mixed Procedure



FILE: stat2e.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.5 FINAL

BREXPIPRAZOLE 5 OF 37 PROTOCOL 331-201-00061

MMRM Output for Test on Treatment by Type of Trauma Interaction
(Intent to Treat Sample)

The Mixed Procedure



FILE: stat2e.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.5 FINAL

BREXPIPRAZOLE 6 OF 37 PROTOCOL 331-201-00061 MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample) The Mixed Procedure COMBFL 2 NY Dimensions Covariance Parameters 10 Columns in X 89 Columns in Z 0 299 Subjects Max Obs per Subject Number of Observations 996 Number of Observations Read 996 Number of Observations Used Number of Observations Not Used

FILE: stat2e.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.5 FINAL

BREXPIPRAZOLE 7 OF 37 PROTOCOL 331-201-00061

STAT-3.5

MMRM Output for Test on Treatment by Type of Trauma Interaction

(Intent to Treat Sample)

.....

The Mixed Procedure

Iteration History

| Criterion | -2 Res Log Like | Evaluations | Iteration |
|------------|-----------------|-------------|-----------|
| | 7329.71676721 | 1 | 0 |
| 0.00163324 | 6852.58631754 | 2 | 1 |
| 0.00016830 | 6847.71408270 | 1 | 2 |
| 0.00000244 | 6847.25354259 | 1 | 3 |
| 0.0000000 | 6847.24725471 | 1 | 4 |

Convergence criteria met.

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | 78.2606 |
| UN(2,1) | SUBJID | 52.8071 |
| UN(2,2) | SUBJID | 113.16 |
| UN(3,1) | SUBJID | 43.3385 |
| UN(3,2) | SUBJID | 90.7080 |
| UN(3,3) | SUBJID | 121.79 |
| UN(4,1) | SUBJID | 47.2805 |

FILE: stat2e.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.5 FINAL

BREXPIPRAZOLE 8 OF 37 PROTOCOL 331-201-00061

STAT-3.5

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN (4,2) | SUBJID | 89.4682 |
| UN (4,3) | SUBJID | 103.52 |
| UN (4,4) | SUBJID | 145.27 |

Fit Statistics

| -2 Res Log Likelihood | 6847.2 |
|--------------------------|--------|
| AIC (Smaller is Better) | 6867.2 |
| AICC (Smaller is Better) | 6867.5 |
| BIC (Smaller is Better) | 6904.3 |

Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSc |
|----|------------|------------|
| 9 | 482.47 | <.0001 |

BREXPIPRAZOLE 9 OF 37 PROTOCOL 331-201-00061 STAT-3.5 MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample) The Mixed Procedure Type 3 Tests of Fixed Effects Num Den Effect DF DF F Value Pr > F POOLCNTR 9 1.71 0.0866 COMBFL 1 283 1.93 0.1661 AVISITN 3 230 0.94 0.4225 3 276 TRTPN 2.45 0.0636 AVISITN\*TRTPN 9 367 1.84 0.0596 AVISITN\*COMBFL 3 243 2.95 0.0336 TRTPN\*COMBFL 3 277 1.00 0.3943 AVISITN\*TRTPN\*COMBFL 9 367 1.97 0.0421 BASE\*AVISITN 4 240 15.22 <.0001 Coefficients for Dummy W vs. Dummy Z BY COMBFL AT Phase B Center Combat (Pooled Related Analysis Planned Center) Population Visit Treatment

for ITT

FILE: stat2e.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.5 FINAL

Effect

Intercept POOLCNTR

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.

Flag (N)

(N)

Row1



FILE: stat2e.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.5 FINAL

BREXPIPRAZOLE 11 OF 37 PROTOCOL 331-201-00061

STAT-3.5

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY COMBFL AT Phase B

Center Combat

| | (Pooled<br>Center) | Related<br>Population | | Treatment | _ 1 |
|---|---|---|---|---|---|
| Effect | for ITT | Flag | (N) | (N) | Row1 |
| TRTPN | | | | 900 | |
| AVISITN*TRTPN | | | 3 | 1 | |
| AVISITN*TRTPN | | | 3 | 2 | |
| AVISITN*TRTPN | | | 3 | 3 | |
| AVISITN*TRTPN | | | 3 | 900 | |
| AVISITN*TRTPN | | | 6 | 1 | |
| AVISITN*TRTPN | | | 6 | 2 | |
| AVISITN*TRTPN | | | 6 | 3 | |
| AVISITN*TRTPN | | | 6 | 900 | |
| AVISITN*TRTPN | | | 10 | 1 | |
| AVISITN*TRTPN | | | 10 | 2 | |
| | | | | 3 | |
| AVISITN*TRTPN | | | 10 | - | |
| AVISITN*TRTPN | | | 10 | 900 | |
| AVISITN*TRTPN | | | 12 | 1 | |
| AVISITN*TRTPN | | | 12 | 2 | |
| AVISITN*TRTPN | | | 12 | 3 | |
| AVISITN*TRTPN | | | 12 | 900 | |
| AVISITN*COMBFL | | N | 3 | | |

FILE: stat2e.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.5 FINAL

BREXPIPRAZOLE 12 OF 37 PROTOCOL 331-201-00061

STAT-3

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY COMBFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|
| AVISITN*COMBFL | | Y | 3 | | |
| AVISITN*COMBFL | | N | 6 | | |
| AVISITN*COMBFL | | Y | 6 | | |
| AVISITN*COMBFL | | N | 10 | | |
| AVISITN*COMBFL | | Y | 10 | | |
| AVISITN*COMBFL | | N | 12 | | |
| AVISITN*COMBFL | | Y | 12 | | |
| TRTPN*COMBFL | | N | | 1 | 1 |
| TRTPN*COMBFL | | Y | | 1 | -1 |
| TRTPN*COMBFL | | N | | 2 | |
| TRTPN*COMBFL | | Y | | 2 | |
| TRTPN*COMBFL | | N | | 3 | |
| TRTPN*COMBFL | | Y | | 3 | |
| TRTPN*COMBFL | | N | | 900 | -1 |
| TRTPN*COMBFL | | Y | | 900 | 1 |
| AVISITN*TRTPN*COMBFL | | N | 3 | 1 | |
| AVISITN*TRTPN*COMBFL | | Y | 3 | 1 | |
| AVISITN*TRTPN*COMBFL | | N | 3 | 2 | |

BREXPIPRAZOLE 13 OF 37 PROTOCOL 331-201-00061

STAT-3.

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY COMBFL AT Phase B

| | Center | Combat | | | |
|---|---|---|---|---|---|
| | (Pooled | Related | Analysis | Planned | |
| | Center) | Population | Visit | Treatment | |
| Effect | for ITT | Flag | (N) | (N) | Row1 |
| ALLE CEMPLE MEDITE COMPLET | | ., | 2 | 2 | |
| AVISITN*TRTPN*COMBFL | | Y | 3 | 2 | |
| AVISITN*TRTPN*COMBFL | | N | 3 | 3 | |
| AVISITN*TRTPN*COMBFL | | Y | 3 | 3 | |
| AVISITN*TRTPN*COMBFL | | N | 3 | 900 | |
| AVISITN*TRTPN*COMBFL | | Y | 3 | 900 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 1 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 1 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 2 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 2 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 3 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 3 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 900 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 900 | |
| AVISITN*TRTPN*COMBFL | | N | 10 | 1 | 1 |
| AVISITN*TRTPN*COMBFL | | Y | 10 | 1 | -1 |
| AVISITN*TRTPN*COMBFL | | N | 10 | 2 | |
| AVISITN*TRTPN*COMBFL | | Y | 10 | 2 | |
| AVISITN*TRTPN*COMBFL | | N | 10 | 3 | |

FILE: stat2e.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.5 FINAL

BREXPIPRAZOLE 14 OF 37 PROTOCOL 331-201-00061

STAT-3.

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY COMBFL AT Phase B

| | Center | Combat | | | |
|---|---|---|---|---|---|
| | (Pooled | Related | Analysis | Planned | |
| | Center) | Population | Visit | Treatment | |
| Effect | for ITT | Flag | (N) | (N) | Row1 |
| | | = | | | |
| AVISITN*TRTPN*COMBFL | | N | 10 | 900 | -1 |
| AVISITN*TRTPN*COMBFL | | Y | 10 | 900 | 1 |
| AVISITN*TRTPN*COMBFL | | N | 12 | 1 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 1 | |
| AVISITN*TRTPN*COMBFL | | N | 12 | 2 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 2 | |
| AVISITN*TRTPN*COMBFL | | N | 12 | 3 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 3 | |
| AVISITN*TRTPN*COMBFL | | N | 12 | 900 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 900 | |
| BASE*AVISITN | | | 3 | | |
| BASE*AVISITN | | | 6 | | |
| BASE*AVISITN | | | 10 | | |
| BASE*AVISITN | | | 12 | | |
| | AVISITN*TRTPN*COMBFL BASE*AVISITN BASE*AVISITN BASE*AVISITN BASE*AVISITN | Effect (Pooled Center) Effect for ITT AVISITN*TRTPN*COMBFL BASE*AVISITN BASE*AVISITN BASE*AVISITN BASE*AVISITN | (Pooled Related Center) Population for ITT Flag AVISITN*TRTPN*COMBFL Y AVISITN*TRTPN*COMBFL N AVISITN*TRTPN*COMBFL Y AVISITN*TRTPN*COMBFL N AVISITN*TRTPN*COMBFL N AVISITN*TRTPN*COMBFL Y AVISITN*TRTPN*COMBFL N AVISITN*TRTPN*COMBFL N AVISITN*TRTPN*COMBFL N AVISITN*TRTPN*COMBFL Y AVISITN*TRTPN*COMBFL N AVISITN*TRTPN*COMBFL N AVISITN*TRTPN*COMBFL N AVISITN*TRTPN*COMBFL Y BASE*AVISITN BASE*AVISITN BASE*AVISITN BASE*AVISITN | Pooled Center | Planned Center |



FILE: stat2e.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.5 FINAL

BREXPIPRAZOLE 16 OF 37 PROTOCOL 331-201-00061

STAT-3.5

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY COMBFL AT Phase B

| | Center | Combat | | | |
|---------------|---------|------------|----------|-----------|------|
| | (Pooled | Related | Analysis | Planned | |
| | Center) | Population | Visit | Treatment | |
| Effect | for ITT | Flag | (N) | (N) | Row1 |
| TRTPN | | | | 2 | |
| TRTPN | | | | 3 | |
| TRTPN | | | | 900 | |
| AVISITN*TRTPN | | | 3 | 1 | |
| AVISITN*TRTPN | | | 3 | 2 | |
| AVISITN*TRTPN | | | 3 | 3 | |
| AVISITN*TRTPN | | | 3 | 900 | |
| AVISITN*TRTPN | | | 6 | 1 | |
| AVISITN*TRTPN | | | 6 | 2 | |
| AVISITN*TRTPN | | | 6 | 3 | |
| AVISITN*TRTPN | | | 6 | 900 | |
| AVISITN*TRTPN | | | 10 | 1 | |
| AVISITN*TRTPN | | | 10 | 2 | |
| AVISITN*TRTPN | | | 10 | 3 | |
| AVISITN*TRTPN | | | 10 | 900 | |
| AVISITN*TRTPN | | | 12 | 1 | |
| AVISITN*TRTPN | | | 12 | 2 | |
| AVISITN*TRTPN | | | 12 | 3 | |

FILE: stat2e.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.5 FINAL

BREXPIPRAZOLE 17 OF 37 PROTOCOL 331-201-00061

STAT-3.

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

.\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY COMBFL AT Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|
| AVISITN*TRTPN | | | 12 | 900 | |
| AVISITN*COMBFL | | N | 3 | | |
| AVISITN*COMBFL | | Y | 3 | | |
| AVISITN*COMBFL | | N | 6 | | |
| AVISITN*COMBFL | | Y | 6 | | |
| AVISITN*COMBFL | | N | 10 | | |
| AVISITN*COMBFL | | Y | 10 | | |
| AVISITN*COMBFL | | N | 12 | | |
| AVISITN*COMBFL | | Y | 12 | | |
| TRTPN*COMBFL | | N | | 1 | 1 |
| TRTPN*COMBFL | | Y | | 1 | -1 |
| TRTPN*COMBFL | | N | | 2 | |
| TRTPN*COMBFL | | Y | | 2 | |
| TRTPN*COMBFL | | N | | 3 | -1 |
| TRTPN*COMBFL | | Y | | 3 | 1 |
| TRTPN*COMBFL | | N | | 900 | |
| TRTPN*COMBFL | | Y | | 900 | |
| AVISITN*TRTPN*COMBFL | | N | 3 | 1 | |

BREXPIPRAZOLE 18 OF 37 PROTOCOL 331-201-00061

STAT-3.

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY COMBFL AT Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|
| AVISITN*TRTPN*COMBFL | | Υ | 3 | 1 | |
| AVISITN*TRTPN*COMBFL | | N | 2 | 2 | |
| | | | 3 | = | |
| AVISITN*TRTPN*COMBFL | | Y | 3 | 2 | |
| AVISITN*TRTPN*COMBFL | | N | 3 | 3 | |
| AVISITN*TRTPN*COMBFL | | Y | 3 | 3 | |
| AVISITN*TRTPN*COMBFL | | N | 3 | 900 | |
| AVISITN*TRTPN*COMBFL | | Y | 3 | 900 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 1 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 1 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 2 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 2 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 3 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 3 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 900 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 900 | |
| AVISITN*TRTPN*COMBFL | | N | 10 | 1 | 1 |
| AVISITN*TRTPN*COMBFL | | Y | 10 | 1 | -1 |
| AVISITN*TRTPN*COMBFL | | N | 10 | 2 | |

BREXPIPRAZOLE 19 OF 37 PROTOCOL 331-201-00061

STAT-3.5

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY COMBFL AT Phase B

| | Center | Combat | | | |
|----------------------|---------|------------|----------|-----------|------|
| | (Pooled | Related | Analysis | Planned | |
| | Center) | Population | Visit | Treatment | |
| Effect | for ITT | Flag | (N) | (N) | Row1 |
| AVISITN*TRTPN*COMBFL | | Y | 10 | 2 | |
| AVISITN*TRTPN*COMBFL | | N | 10 | 3 | -1 |
| AVISITN*TRTPN*COMBFL | | Y | 10 | 3 | 1 |
| AVISITN*TRTPN*COMBFL | | N | 10 | 900 | |
| AVISITN*TRTPN*COMBFL | | Y | 10 | 900 | |
| AVISITN*TRTPN*COMBFL | | N | 12 | 1 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 1 | |
| AVISITN*TRTPN*COMBFL | | N | 12 | 2 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 2 | |
| AVISITN*TRTPN*COMBFL | | N | 12 | 3 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 3 | |
| AVISITN*TRTPN*COMBFL | | N | 12 | 900 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 900 | |
| BASE*AVISITN | | | 3 | | |
| BASE*AVISITN | | | 6 | | |
| BASE*AVISITN | | | 10 | | |
| BASE*AVISITN | | | 12 | | |



FILE: stat2e.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.5 FINAL

BREXPIPRAZOLE 21 OF 37 PROTOCOL 331-201-00061

STAT-3.

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY COMBFL AT Phase B

| | Center | Combat | | | |
|---------------|---------|------------|----------|-----------|------|
| | (Pooled | Related | Analysis | Planned | |
| | Center) | Population | Visit | Treatment | |
| Effect | for ITT | Flag | (N) | (N) | Row1 |
| TRTPN | | | | 2 | |
| | | | | 3 | |
| TRTPN | | | | | |
| TRTPN | | | | 900 | |
| AVISITN*TRTPN | | | 3 | 1 | |
| AVISITN*TRTPN | | | 3 | 2 | |
| AVISITN*TRTPN | | | 3 | 3 | |
| AVISITN*TRTPN | | | 3 | 900 | |
| AVISITN*TRTPN | | | 6 | 1 | |
| AVISITN*TRTPN | | | 6 | 2 | |
| AVISITN*TRTPN | | | 6 | 3 | |
| AVISITN*TRTPN | | | 6 | 900 | |
| AVISITN*TRTPN | | | 10 | 1 | |
| AVISITN*TRTPN | | | 10 | 2 | |
| AVISITN*TRTPN | | | 10 | 3 | |
| AVISITN*TRTPN | | | 10 | 900 | |
| AVISITN*TRTPN | | | 12 | 1 | |
| AVISITN*TRTPN | | | 12 | 2 | |
| AVISITN*TRTPN | | | 12 | 3 | |

BREXPIPRAZOLE 22 OF 37 PROTOCOL 331-201-00061

STAT-3.

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY COMBFL AT Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|
| AVISITN*TRTPN | | | 12 | 900 | |
| AVISITN*COMBFL | | N | 3 | | |
| AVISITN*COMBFL | | Y | 3 | | |
| AVISITN*COMBFL | | N | 6 | | |
| AVISITN*COMBFL | | Y | 6 | | |
| AVISITN*COMBFL | | N | 10 | | |
| AVISITN*COMBFL | | Y | 10 | | |
| AVISITN*COMBFL | | N | 12 | | |
| AVISITN*COMBFL | | Y | 12 | | |
| TRTPN*COMBFL | | N | | 1 | 1 |
| TRTPN*COMBFL | | Y | | 1 | -1 |
| TRTPN*COMBFL | | N | | 2 | -1 |
| TRTPN*COMBFL | | Y | | 2 | 1 |
| TRTPN*COMBFL | | N | | 3 | |
| TRTPN*COMBFL | | Y | | 3 | |
| TRTPN*COMBFL | | N | | 900 | |
| TRTPN*COMBFL | | Y | | 900 | |
| AVISITN*TRTPN*COMBFL | | N | 3 | 1 | |

BREXPIPRAZOLE 23 OF 37 PROTOCOL 331-201-00061

STAT-3

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY COMBFL AT Phase B

| Effect | (Pooled<br>Center)<br>for ITT | | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|
| 222000 | 101 111 | 1 109 | (21) | (21) | 110111 |
| AVISITN*TRTPN*COMBFL | | Y | 3 | 1 | |
| AVISITN*TRTPN*COMBFL | | N | 3 | 2 | |
| AVISITN*TRTPN*COMBFL | | Y | 3 | 2 | |
| AVISITN*TRTPN*COMBFL | | N | 3 | 3 | |
| AVISITN*TRTPN*COMBFL | | Y | 3 | 3 | |
| AVISITN*TRTPN*COMBFL | | N | 3 | 900 | |
| AVISITN*TRTPN*COMBFL | | Y | 3 | 900 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 1 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 1 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 2 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 2 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 3 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 3 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 900 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 900 | |
| AVISITN*TRTPN*COMBFL | | N | 10 | 1 | 1 |
| AVISITN*TRTPN*COMBFL | | Y | 10 | 1 | -1 |
| AVISITN*TRTPN*COMBFL | | N | 10 | 2 | -1 |

BREXPIPRAZOLE 24 OF 37 PROTOCOL 331-201-00061

STAT-3.5

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

-----

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY COMBFL AT Phase B

| | Center<br>(Pooled | Combat<br>Related | Analysis | | |
|---|---|---|---|---|---|
| | Center) | Population | Visit | Treatment | |
| Effect | for ITT | Flag | (N) | (N) | Row1 |
| | | | 1.0 | ^ | |
| AVISITN*TRTPN*COMBFL | | Y | 10 | 2 | 1 |
| AVISITN*TRTPN*COMBFL | | N | 10 | 3 | |
| AVISITN*TRTPN*COMBFL | | Y | 10 | 3 | |
| AVISITN*TRTPN*COMBFL | | N | 10 | 900 | |
| AVISITN*TRTPN*COMBFL | | Y | 10 | 900 | |
| AVISITN*TRTPN*COMBFL | | N | 12 | 1 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 1 | |
| AVISITN*TRTPN*COMBFL | | N | 12 | 2 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 2 | |
| AVISITN*TRTPN*COMBFL | | N | 12 | 3 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 3 | |
| AVISITN*TRTPN*COMBFL | | N | 12 | 900 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 900 | |
| BASE*AVISITN | | | 3 | | |
| BASE*AVISITN | | | 6 | | |
| BASE*AVISITN | | | 10 | | |
| BASE*AVISITN | | | 12 | | |



FILE: stat2e.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.5 FINAL

BREXPIPRAZOLE 26 OF 37 PROTOCOL 331-201-00061

STAT-3.5

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY COMBFL AT Phase B

| | Center | Combat | | | |
|---------------|---------|------------|----------|-----------|------|
| | (Pooled | Related | Analysis | Planned | |
| | Center) | Population | Visit | Treatment | |
| Effect | for ITT | Flag | (N) | (N) | Row1 |
| TRTPN | | | | 2 | |
| TRTPN | | | | 3 | |
| TRTPN | | | | 900 | |
| AVISITN*TRTPN | | | 3 | 1 | |
| AVISITN*TRTPN | | | 3 | 2 | |
| AVISITN*TRTPN | | | 3 | 3 | |
| AVISITN*TRTPN | | | 3 | 900 | |
| AVISITN*TRTPN | | | 6 | 1 | |
| AVISITN*TRTPN | | | 6 | 2 | |
| AVISITN*TRTPN | | | 6 | 3 | |
| AVISITN*TRTPN | | | 6 | 900 | |
| AVISITN*TRTPN | | | 10 | 1 | |
| AVISITN*TRTPN | | | 10 | 2 | |
| AVISITN*TRTPN | | | 10 | 3 | |
| AVISITN*TRTPN | | | 10 | 900 | |
| AVISITN*TRTPN | | | 12 | 1 | |
| AVISITN*TRTPN | | | 12 | 2 | |
| AVISITN*TRTPN | | | 12 | 3 | |

BREXPIPRAZOLE 27 OF 37 PROTOCOL 331-201-00061

STAT-3.

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY COMBFL AT Phase B

| | Center | Combat | | | |
|----------------------|---------|------------|----------|-----------|------|
| | (Pooled | Related | Analysis | Planned | |
| | Center) | Population | Visit | Treatment | |
| Effect | for ITT | Flag | (N) | (N) | Row1 |
| AVISITN*TRTPN | | | 12 | 900 | |
| AVISITN*COMBFL | | N | 3 | | |
| AVISITN*COMBFL | | Y | 3 | | |
| AVISITN*COMBFL | | N | 6 | | |
| AVISITN*COMBFL | | Y | 6 | | |
| AVISITN*COMBFL | | N | 10 | | |
| AVISITN*COMBFL | | Y | 10 | | |
| AVISITN*COMBFL | | N | 12 | | |
| AVISITN*COMBFL | | Y | 12 | | |
| TRTPN*COMBFL | | N | | 1 | |
| TRTPN*COMBFL | | Y | | 1 | |
| TRTPN*COMBFL | | N | | 2 | 1 |
| TRTPN*COMBFL | | Y | | 2 | -1 |
| TRTPN*COMBFL | | N | | 3 | |
| TRTPN*COMBFL | | Y | | 3 | |
| TRTPN*COMBFL | | N | | 900 | -1 |
| TRTPN*COMBFL | | Y | | 900 | 1 |
| AVISITN*TRTPN*COMBFL | | N | 3 | 1 | |

BREXPIPRAZOLE 28 OF 37 PROTOCOL 331-201-00061

STAT-3.5

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY COMBFL AT Phase B

| Effect | , | Related<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|
| AVISITN*TRTPN*COMBFL | | Υ | 3 | 1 | |
| AVISITN*TRTPN*COMBFL | | N | 3 | 2 | |
| AVISITN*TRTPN*COMBFL | | Y | 3 | 2 | |
| AVISITN*TRTPN*COMBFL | | N | 3 | 3 | |
| AVISITN*TRTPN*COMBFL | | Y | 3 | 3 | |
| AVISITN*TRTPN*COMBFL | | N | 3 | 900 | |
| AVISITN*TRTPN*COMBFL | | Y | 3 | 900 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 1 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 1 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 2 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 2 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 3 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 3 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 900 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 900 | |
| AVISITN*TRTPN*COMBFL | | N | 10 | 1 | |
| AVISITN*TRTPN*COMBFL | | Y | 10 | 1 | |
| AVISITN*TRTPN*COMBFL | | N | 10 | 2 | 1 |

BREXPIPRAZOLE 29 OF 37 PROTOCOL 331-201-00061

STAT-3.5

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY COMBFL AT Phase B

| | Center | enter Combat | | | |
|----------------------|---------|--------------|----------|-----------|------|
| | (Pooled | Related | Analysis | Planned | |
| | Center) | Population | Visit | Treatment | |
| Effect | for ITT | Flag | (N) | (N) | Row1 |
| AVISITN*TRTPN*COMBFL | | Y | 10 | 2 | -1 |
| AVISITN*TRTPN*COMBFL | | N | 10 | 3 | |
| AVISITN*TRTPN*COMBFL | | Y | 10 | 3 | |
| AVISITN*TRTPN*COMBFL | | N | 10 | 900 | -1 |
| AVISITN*TRTPN*COMBFL | | Y | 10 | 900 | 1 |
| AVISITN*TRTPN*COMBFL | | N | 12 | 1 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 1 | |
| AVISITN*TRTPN*COMBFL | | N | 12 | 2 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 2 | |
| AVISITN*TRTPN*COMBFL | | N | 12 | 3 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 3 | |
| AVISITN*TRTPN*COMBFL | | N | 12 | 900 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 900 | |
| BASE*AVISITN | | | 3 | | |
| BASE*AVISITN | | | 6 | | |
| BASE*AVISITN | | | 10 | | |
| BASE*AVISITN | | | 12 | | |



FILE: stat2e.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.5 FINAL

BREXPIPRAZOLE 31 OF 37 PROTOCOL 331-201-00061

STAT-3.5

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

-----

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY COMBFL AT Phase B

| Center | Combat | | | |
|---|---|---|---|---|
| (Pooled | Related | Analysis | Planned | |
| Center) | Population | Visit | Treatment | |
| for ITT | Flag | (N) | (N) | Row1 |
| | | | 2 | |
| | | | 3 | |
| | | | 900 | |
| | | 3 | 1 | |
| | | 3 | 2 | |
| | | 3 | 3 | |
| | | 3 | 900 | |
| | | 6 | 1 | |
| | | 6 | 2 | |
| | | 6 | 3 | |
| | | 6 | 900 | |
| | | 10 | 1 | |
| | | 10 | 2 | |
| | | 10 | 3 | |
| | | 10 | 900 | |
| | | 12 | 1 | |
| | | 12 | 2 | |
| | | 12 | 3 | |
| | Center) | (Pooled Related<br>Center) Population | (Pooled Related Analysis Center) Population Visit for ITT Flag (N) 3 3 3 3 6 6 6 6 10 10 10 10 10 10 12 12 | (Pooled Center) Related Population Flag Analysis Visit Treatment (N) Treatment (N) for ITT Flag (N) (N) |
BREXPIPRAZOLE 32 OF 37 PROTOCOL 331-201-00061

STAT-3.5

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY COMBFL AT Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|
| AVISITN*TRTPN | | | 12 | 900 | |
| AVISITN*COMBFL | | N | 3 | | |
| AVISITN*COMBFL | | Y | 3 | | |
| AVISITN*COMBFL | | N | 6 | | |
| AVISITN*COMBFL | | Y | 6 | | |
| AVISITN*COMBFL | | N | 10 | | |
| AVISITN*COMBFL | | Y | 10 | | |
| AVISITN*COMBFL | | N | 12 | | |
| AVISITN*COMBFL | | Y | 12 | | |
| TRTPN*COMBFL | | N | | 1 | |
| TRTPN*COMBFL | | Y | | 1 | |
| TRTPN*COMBFL | | N | | 2 | |
| TRTPN*COMBFL | | Y | | 2 | |
| TRTPN*COMBFL | | N | | 3 | 1 |
| TRTPN*COMBFL | | Y | | 3 | -1 |
| TRTPN*COMBFL | | N | | 900 | -1 |
| TRTPN*COMBFL | | Y | | 900 | 1 |
| AVISITN*TRTPN*COMBFL | | N | 3 | 1 | |

BREXPIPRAZOLE 33 OF 37 PROTOCOL 331-201-00061

STAT-3.5

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY COMBFL AT Phase B

| | Center | Combat | | | |
|---|---|---|---|---|---|
| | (Pooled | Related | Analysis | Planned | |
| | Center) | Population | Visit | Treatment | |
| Effect | for ITT | Flag | (N) | (N) | Row1 |
| | | = | - | 1 | |
| AVISITN*TRTPN*COMBFL | | N | 3 | 2 | |
| AVISITN*TRTPN*COMBFL | | Y | 3 | 2 | |
| AVISITN*TRTPN*COMBFL | | N | 3 | 3 | |
| AVISITN*TRTPN*COMBFL | | Y | 3 | 3 | |
| AVISITN*TRTPN*COMBFL | | N | 3 | 900 | |
| AVISITN*TRTPN*COMBFL | | Y | 3 | 900 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 1 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 1 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 2 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 2 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 3 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 3 | |
| AVISITN*TRTPN*COMBFL | | N | 6 | 900 | |
| AVISITN*TRTPN*COMBFL | | Y | 6 | 900 | |
| AVISITN*TRTPN*COMBFL | | N | 10 | 1 | |
| AVISITN*TRTPN*COMBFL | | Y | 10 | 1 | |
| AVISITN*TRTPN*COMBFL | | N | 10 | 2 | |
| | AVISITN*TRTPN*COMBFL | CPOOLED CENTER) Effect AVISITN*TRTPN*COMBFL | (Pooled Related Center) Population Effect (Pooled Related Center) Population for ITT Flag AVISITN*TRTPN*COMBFL Y AVISITN*TRTPN*COMBFL N AVISITN*TRTPN*COMBFL N AVISITN*TRTPN*COMBFL N AVISITN*TRTPN*COMBFL Y AVISITN*TRTPN*COMBFL N AVISITN*TRTPN*COMBFL N AVISITN*TRTPN*COMBFL Y AVISITN*TRTPN*COMBFL N AVISITN*TRTPN*COMBFL N AVISITN*TRTPN*COMBFL Y AVISITN*TRTPN*COMBFL N | Pooled Related Analysis | Planned Center |

BREXPIPRAZOLE 34 OF 37 PROTOCOL 331-201-00061

STAT-3.

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

\_\_\_\_\_

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY COMBFL AT Phase B

| | Center | Combat | | | |
|----------------------|---------|------------|----------|-----------|------|
| | (Pooled | Related | Analysis | Planned | |
| | Center) | Population | Visit | Treatment | |
| Effect | for ITT | Flag | (N) | (N) | Row1 |
| AVISITN*TRTPN*COMBFL | | Y | 10 | 2 | |
| AVISITN*TRTPN*COMBFL | | N | 10 | 3 | 1 |
| AVISITN*TRTPN*COMBFL | | Y | 10 | 3 | -1 |
| AVISITN*TRTPN*COMBFL | | N | 10 | 900 | -1 |
| AVISITN*TRTPN*COMBFL | | Y | 10 | 900 | 1 |
| AVISITN*TRTPN*COMBFL | | N | 12 | 1 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 1 | |
| AVISITN*TRTPN*COMBFL | | N | 12 | 2 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 2 | |
| AVISITN*TRTPN*COMBFL | | N | 12 | 3 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 3 | |
| AVISITN*TRTPN*COMBFL | | N | 12 | 900 | |
| AVISITN*TRTPN*COMBFL | | Y | 12 | 900 | |
| BASE*AVISITN | | | 3 | | |
| BASE*AVISITN | | | 6 | | |
| BASE*AVISITN | | | 10 | | |
| BASE*AVISITN | | | 12 | | |

BREXPIPRAZOLE 35 OF 37 PROTOCOL 331-201-00061

STAT-3.5

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

The Mixed Procedure

Estimates

| | | Standard | | | |
|---|---|---|---|---|---|
| Label | Estimate | Error | DF | t Value | Pr > t |
| Dummy W vs. Dummy Z BY COMBFL AT Phase B | -1.2786 | 4.4667 | 234 | -0.29 | 0.7749 |
| Dummy W vs. Dummy Y BY COMBFL AT Phase B | -9.1358 | 4.7247 | 239 | -1.93 | 0.0543 |
| Dummy W vs. Dummy X BY COMBFL AT Phase B | -4.6175 | 5.7957 | 277 | -0.80 | 0.4263 |
| Dummy X vs. Dummy Z BY COMBFL AT Phase B | 3.3389 | 5.7779 | 276 | 0.58 | 0.5638 |
| Dummy Y vs. Dummy Z BY COMBFL AT Phase B | 7.8572 | 4.6952 | 237 | 1.67 | 0.0956 |

Least Squares Means

| Effect | Combat<br>Related<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN*COMBFL | N | 3 | 1 | -5.4540 | 1.1912 | 281 | -4.58 | <.0001 | 0.05 | -7.7987 | -3.1092 |
| AVISITN*TRTPN*COMBFL | Y | 3 | 1 | -6.8538 | 2.1684 | 285 | -3.16 | 0.0017 | 0.05 | -11.1219 | -2.5856 |
| AVISITN*TRTPN*COMBFL | N | 3 | 2 | -2.9761 | 1.2129 | 282 | -2.45 | 0.0147 | 0.05 | -5.3635 | -0.5886 |
| AVISITN*TRTPN*COMBFL | Y | 3 | 2 | -7.6297 | 2.6776 | 274 | -2.85 | 0.0047 | 0.05 | -12.9010 | -2.3585 |
| AVISITN*TRTPN*COMBFL | N | 3 | 3 | -4.2773 | 1.1856 | 280 | -3.61 | 0.0004 | 0.05 | -6.6112 | -1.9434 |
| AVISITN*TRTPN*COMBFL | Y | 3 | 3 | -10.1529 | 2.2995 | 275 | -4.42 | <.0001 | 0.05 | -14.6799 | -5.6260 |

BREXPIPRAZOLE 36 OF 37 PROTOCOL 331-201-00061

STAT-3.5

MMRM Output for Test on Treatment by Type of Trauma Interaction (Intent to Treat Sample)

| Effect | Combat<br>Related<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN*COMBFL | N | 3 | 900 | -5.1726 | 1.1632 | 278 | -4.45 | <.0001 | 0.05 | -7.4624 | -2.8828 |
| AVISITN*TRTPN*COMBFL | Y | 3 | 900 | -6.7476 | 2.1589 | 275 | -3.13 | 0.0020 | 0.05 | -10.9976 | -2.4975 |
| AVISITN*TRTPN*COMBFL | N | 6 | 1 | -10.4557 | 1.4952 | 269 | -6.99 | <.0001 | 0.05 | -13.3995 | -7.5119 |
| AVISITN*TRTPN*COMBFL | Y | 6 | 1 | -16.6958 | 2.6125 | 258 | -6.39 | <.0001 | 0.05 | -21.8402 | -11.5513 |
| AVISITN*TRTPN*COMBFL | N | 6 | 2 | -6.5897 | 1.4640 | 261 | -4.50 | <.0001 | 0.05 | -9.4724 | -3.7071 |
| AVISITN*TRTPN*COMBFL | Y | 6 | 2 | -9.8529 | 3.9562 | 295 | -2.49 | 0.0133 | 0.05 | -17.6388 | -2.0669 |
| AVISITN*TRTPN*COMBFL | N | 6 | 3 | -8.2770 | 1.4793 | 269 | -5.60 | <.0001 | 0.05 | -11.1895 | -5.3645 |
| AVISITN*TRTPN*COMBFL | Y | 6 | 3 | -11.3745 | 2.9953 | 277 | -3.80 | 0.0002 | 0.05 | -17.2709 | -5.4781 |
| AVISITN*TRTPN*COMBFL | N | 6 | 900 | -8.3156 | 1.4333 | 260 | -5.80 | <.0001 | 0.05 | -11.1380 | -5.4932 |
| AVISITN*TRTPN*COMBFL | Y | 6 | 900 | -7.8831 | 2.6189 | 250 | -3.01 | 0.0029 | 0.05 | -13.0410 | -2.7251 |
| AVISITN*TRTPN*COMBFL | N | 10 | 1 | -16.9149 | 1.5914 | 246 | -10.63 | <.0001 | 0.05 | -20.0495 | -13.7803 |
| AVISITN*TRTPN*COMBFL | Y | 10 | 1 | -12.5091 | 2.7575 | 234 | -4.54 | <.0001 | 0.05 | -17.9419 | -7.0763 |
| AVISITN*TRTPN*COMBFL | N | 10 | 2 | -11.0599 | 1.5761 | 250 | -7.02 | <.0001 | 0.05 | -14.1640 | -7.9559 |
| AVISITN*TRTPN*COMBFL | Y | 10 | 2 | -11.2716 | 4.5968 | 298 | -2.45 | 0.0148 | 0.05 | -20.3178 | -2.2254 |
| AVISITN*TRTPN*COMBFL | N | 10 | 3 | -9.6659 | 1.5697 | 245 | -6.16 | <.0001 | 0.05 | -12.7578 | -6.5740 |
| AVISITN*TRTPN*COMBFL | Y | 10 | 3 | -14.3958 | 3.1301 | 242 | -4.60 | <.0001 | 0.05 | -20.5615 | -8.2301 |
| AVISITN*TRTPN*COMBFL | N | 10 | 900 | -10.5054 | 1.5308 | 244 | -6.86 | <.0001 | 0.05 | -13.5206 | -7.4902 |
| AVISITN*TRTPN*COMBFL | Y | 10 | 900 | -7.3782 | 2.7598 | 230 | -2.67 | 0.0080 | 0.05 | -12.8159 | -1.9405 |

BREXPIPRAZOLE 37 OF 37 PROTOCOL 331-201-00061

STAT-3.5

MMRM Output for Test on Treatment by Type of Trauma Interaction

(Intent to Treat Sample)

The Mixed Procedure

Least Squares Means

| | Combat | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Related | Analysis | Planned | | | | | | | | |
| | Population | Visit | Treatment | | Standard | | | | | | |
| Effect | Flag | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN*COMBFL | N | 12 | 1 | -16.3362 | 1.7475 | 243 | -9.35 | <.0001 | 0.05 | -19.7785 | -12.8939 |
| AVISITN*TRTPN*COMBFL | Y | 12 | 1 | -17.6543 | 3.1212 | 245 | -5.66 | <.0001 | 0.05 | -23.8021 | -11.5066 |
| AVISITN*TRTPN*COMBFL | N | 12 | 2 | -11.0683 | 1.7448 | 249 | -6.34 | <.0001 | 0.05 | -14.5047 | -7.6319 |
| AVISITN*TRTPN*COMBFL | Y | 12 | 2 | -11.9169 | 4.8874 | 264 | -2.44 | 0.0154 | 0.05 | -21.5400 | -2.2938 |
| AVISITN*TRTPN*COMBFL | N | 12 | 3 | -12.5249 | 1.7188 | 242 | -7.29 | <.0001 | 0.05 | -15.9106 | -9.1392 |
| AVISITN*TRTPN*COMBFL | Y | 12 | 3 | -20.8155 | 3.4460 | 240 | -6.04 | <.0001 | 0.05 | -27.6037 | -14.0273 |
| AVISITN*TRTPN*COMBFL | N | 12 | 900 | -11.3141 | 1.6739 | 239 | -6.76 | <.0001 | 0.05 | -14.6115 | -8.0167 |
| AVISITN*TRTPN*COMBFL | Y | 12 | 900 | -9.7796 | 3.1245 | 243 | -3.13 | 0.0020 | 0.05 | -15.9342 | -3.6250 |

BREXPIPRAZOLE 1 OF 39

STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction

(Intent to Treat Sample)

The Mixed Procedure

Model Information

Data Set WORK.INDATA
Dependent Variable CHG
Covariance Structure Unstructured
Subject Effect SUBJID
Estimation Method REML

Residual Variance Method None Fixed Effects SE Method Kenward-Roger

Fixed Effects SE Method Kenward-Roger Degrees of Freedom Method Kenward-Roger

Class Level Information


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Class Level Information

Class Levels Values

SUBJID 299



FILE: stat2f.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.6 FINAL

BREXPIPRAZOLE 3 OF 39

 $$\tt STAT-3.6$$  MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction

(Intent to Treat Sample)

.....

The Mixed Procedure



FILE: stat2f.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.6 FINAL

BREXPIPRAZOLE 4 OF 39

STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

-----

The Mixed Procedure



FILE: stat2f.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.6 FINAL

BREXPIPRAZOLE 5 OF 39

STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure



FILE: stat2f.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.6 FINAL

BREXPIPRAZOLE 6 OF 39 PROTOCOL 331-201-00061 STAT-3.6 MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample) The Mixed Procedure NY PSYCHFL 2 Dimensions Covariance Parameters 10 Columns in X 91 Columns in Z 0 299 Subjects Max Obs per Subject Number of Observations 996 Number of Observations Read 996 Number of Observations Used Number of Observations Not Used

FILE: stat2f.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.6 FINAL

BREXPIPRAZOLE 7 OF 39

STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 7347.29266401 | |
| 1 | 2 | 6871.95746428 | 0.00046015 |
| 2 | 1 | 6870.65074164 | 0.00001625 |
| 3 | 1 | 6870.60806155 | 0.00000002 |
| 4 | 1 | 6870.60799804 | 0.00000000 |

Convergence criteria met.

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | 78.0946 |
| UN(2,1) | SUBJID | 51.6582 |
| UN(2,2) | SUBJID | 112.64 |
| UN(3,1) | SUBJID | 43.7333 |
| UN(3,2) | SUBJID | 89.6240 |
| UN(3,3) | SUBJID | 125.14 |
| UN(4,1) | SUBJID | 48.6156 |

BREXPIPRAZOLE 8 OF 39 PROTOCOL 331-201-00061

STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction

(Intent to Treat Sample)

The Mixed Procedure

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(4,2) | SUBJID | 90.8869 |
| UN(4,3) | SUBJID | 107.04 |
| UN (4,4) | SUBJID | 149.19 |

Fit Statistics

| -2 Res Log Likelihood | 6870.6 |
|--------------------------|--------|
| AIC (Smaller is Better) | 6890.6 |
| AICC (Smaller is Better) | 6890.8 |
| BIC (Smaller is Better) | 6927.6 |

Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|----|------------|------------|
| 9 | 476.68 | <.0001 |

FILE: stat2f.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC STAT/stat2.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.6 FINAL

BREXPIPRAZOLE 9 OF 39

STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|----------------------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| POOLCNTR | 9 | 277 | 1.65 | 0.1002 |
| COMBFL | 1 | 278 | 4.02 | 0.0460 |
| AVISITN | 3 | 228 | 1.04 | 0.3774 |
| TRTPN | 3 | 262 | 3.34 | 0.0199 |
| AVISITN*TRTPN | 9 | 358 | 1.91 | 0.0491 |
| PSYCHFL | 1 | 280 | 0.62 | 0.4325 |
| AVISITN*PSYCHFL | 3 | 235 | 0.96 | 0.4119 |
| TRTPN*PSYCHFL | 3 | 264 | 0.85 | 0.4671 |
| AVISIT*TRTPN*PSYCHFL | 9 | 358 | 0.87 | 0.5500 |
| BASE*AVISITN | 4 | 241 | 15.47 | <.0001 |



FILE: stat2f.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.6 FINAL


## STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)



\_\_\_\_\_\_

## The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY PSYCHFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Psychotherapy<br>received<br>Population | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY PSYCHFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Psychotherapy<br>received<br>Population | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 12 | 900 | |
| PSYCHFL | | | N | | | |
| PSYCHFL | | | Y | | | |
| AVISITN*PSYCHFL | | | N | 3 | | |
| AVISITN*PSYCHFL | | | Y | 3 | | |
| AVISITN*PSYCHFL | | | N | 6 | | |
| AVISITN*PSYCHFL | | | Y | 6 | | |
| AVISITN*PSYCHFL | | | N | 10 | | |
| AVISITN*PSYCHFL | | | Y | 10 | | |
| AVISITN*PSYCHFL | | | N | 12 | | |
| AVISITN*PSYCHFL | | | Y | 12 | | |
| TRTPN*PSYCHFL | | | N | | 1 | 1 |
| TRTPN*PSYCHFL | | | Y | | 1 | -1 |
| TRTPN*PSYCHFL | | | N | | 2 | |
| TRTPN*PSYCHFL | | | Y | | 2 | |
| TRTPN*PSYCHFL | | | N | | 3 | |
| TRTPN*PSYCHFL | | | Y | | 3 | |
| TRTPN*PSYCHFL | | | N | | 900 | -1 |


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY PSYCHFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Psychotherapy<br>received<br>Population | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*PSYCHFL | | | Y | | 900 | 1 |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 1 | 1 |


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

.\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY PSYCHFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Psychotherapy<br>received<br>Population | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 1 | -1 |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 900 | -1 |
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 900 | 1 |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |



BREXPIPRAZOLE 16 OF 39 PROTOCOL 331-201-00061 STAT-3.6 MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy W vs. Dummy Y BY PSYCHFL AT Phase B Center Combat E-TRIP (Pooled Related Psychotherapy Analysis Planned Visit Center) Population received Treatment Effect for ITT Flag Population (N) Row1 POOLCNTR POOLCNTR POOLCNTR COMBFL Ν Υ COMBFL 3 AVISITN AVISITN 6 AVISITN 10 AVISITN 12 1 TRTPN TRTPN 2 3 TRTPN TRTPN 900 AVISITN\*TRTPN 3 1 3 2 AVISITN\*TRTPN AVISITN\*TRTPN 3 3 AVISITN\*TRTPN 3 900 AVISITN\*TRTPN

FILE: stat2f.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.6 FINAL


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY PSYCHFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Psychotherapy<br>received<br>Population | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |
| AVISITN*TRTPN | | | | 12 | 900 | |
| PSYCHFL | | | N | | | |
| PSYCHFL | | | Y | | | |
| AVISITN*PSYCHFL | | | N | 3 | | |
| AVISITN*PSYCHFL | | | Y | 3 | | |
| AVISITN*PSYCHFL | | | N | 6 | | |
| AVISITN*PSYCHFL | | | Y | 6 | | |
| AVISITN*PSYCHFL | | | N | 10 | | |


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY PSYCHFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Psychotherapy<br>received<br>Population | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*PSYCHFL | | | Y | 10 | | |
| AVISITN*PSYCHFL | | | N | 12 | | |
| AVISITN*PSYCHFL | | | Y | 12 | | |
| TRTPN*PSYCHFL | | | N | | 1 | 1 |
| TRTPN*PSYCHFL | | | Y | | 1 | -1 |
| TRTPN*PSYCHFL | | | N | | 2 | |
| TRTPN*PSYCHFL | | | Y | | 2 | |
| TRTPN*PSYCHFL | | | N | | 3 | -1 |
| TRTPN*PSYCHFL | | | Y | | 3 | 1 |
| TRTPN*PSYCHFL | | | N | | 900 | |
| TRTPN*PSYCHFL | | | Y | | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 900 | |


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

to freat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY PSYCHFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Psychotherapy<br>received<br>Population | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 1 | 1 |
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 1 | -1 |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 3 | -1 |
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 3 | 1 |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 1 | |


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY PSYCHFL AT Phase B

| | Center<br>(Pooled | Combat<br>Related | E-TRIP<br>Psychotherapy | Analysis | Planned | |
|---|---|---|---|---|---|---|
| | Center) | Population | received | Visit | Treatment | |
| Effect | for ITT | Flag | Population | (N) | (N) | Row1 |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |
| BASE*AVISITN | | | | 12 | | |



FILE: stat2f.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.6 FINAL


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

-----

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY PSYCHFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Psychotherapy<br>received<br>Population | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

.\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY PSYCHFL AT Phase B

| | Center | Combat | E-TRIP | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | Psychotherapy | Analysis | Planned | |
| | Center) | Population | received | Visit | Treatment | |
| Effect | for ITT | Flag | Population | (N) | (N) | Row1 |
| AVISITN*TRTPN | | | | 12 | 900 | |
| PSYCHFL | | | N | | | |
| PSYCHFL | | | Y | | | |
| AVISITN*PSYCHFL | | | N | 3 | | |
| AVISITN*PSYCHFL | | | Y | 3 | | |
| AVISITN*PSYCHFL | | | N | 6 | | |
| AVISITN*PSYCHFL | | | Y | 6 | | |
| AVISITN*PSYCHFL | | | N | 10 | | |
| AVISITN*PSYCHFL | | | Y | 10 | | |
| AVISITN*PSYCHFL | | | N | 12 | | |
| AVISITN*PSYCHFL | | | Y | 12 | | |
| TRTPN*PSYCHFL | | | N | | 1 | 1 |
| TRTPN*PSYCHFL | | | Y | | 1 | -1 |
| TRTPN*PSYCHFL | | | N | | 2 | -1 |
| TRTPN*PSYCHFL | | | Y | | 2 | 1 |
| TRTPN*PSYCHFL | | | N | | 3 | |
| TRTPN*PSYCHFL | | | Y | | 3 | |
| TRTPN*PSYCHFL | | | N | | 900 | |


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)



The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY PSYCHFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Psychotherapy<br>received<br>Population | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*PSYCHFL | | | Y | | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 1 | 1 |


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY PSYCHFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Psychotherapy<br>received<br>Population | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 1 | -1 |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 2 | -1 |
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 2 | 1 |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |



FILE: stat2f.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.6 FINAL

BREXPIPRAZOLE 27 OF 39 PROTOCOL 331-201-00061 STAT-3.6 MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy X vs. Dummy Z BY PSYCHFL AT Phase B Center Combat E-TRIP (Pooled Related Psychotherapy Analysis Planned Visit Center) Population received Treatment Effect for ITT Flag Population (N) Row1 POOLCNTR POOLCNTR POOLCNTR COMBFL Ν Υ COMBFL 3 AVISITN AVISITN 6 AVISITN 10 AVISITN 12 1 TRTPN TRTPN 2 3 TRTPN TRTPN 900 AVISITN\*TRTPN 3 1 3 2 AVISITN\*TRTPN AVISITN\*TRTPN 3 3 AVISITN\*TRTPN 3 900 AVISITN\*TRTPN

FILE: stat2f.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.6 FINAL


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY PSYCHFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Psychotherapy<br>received<br>Population | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |
| AVISITN*TRTPN | | | | 12 | 900 | |
| PSYCHFL | | | N | | | |
| PSYCHFL | | | Y | | | |
| AVISITN*PSYCHFL | | | N | 3 | | |
| AVISITN*PSYCHFL | | | Y | 3 | | |
| AVISITN*PSYCHFL | | | N | 6 | | |
| AVISITN*PSYCHFL | | | Y | 6 | | |
| AVISITN*PSYCHFL | | | N | 10 | | |


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY PSYCHFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Psychotherapy<br>received<br>Population | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*PSYCHFL | | | Y | 10 | | |
| AVISITN*PSYCHFL | | | N | 12 | | |
| AVISITN*PSYCHFL | | | Y | 12 | | |
| TRTPN*PSYCHFL | | | N | | 1 | |
| TRTPN*PSYCHFL | | | Y | | 1 | |
| TRTPN*PSYCHFL | | | N | | 2 | 1 |
| TRTPN*PSYCHFL | | | Y | | 2 | -1 |
| TRTPN*PSYCHFL | | | N | | 3 | |
| TRTPN*PSYCHFL | | | Y | | 3 | |
| TRTPN*PSYCHFL | | | N | | 900 | -1 |
| TRTPN*PSYCHFL | | | Y | | 900 | 1 |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 900 | |


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY PSYCHFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Psychotherapy<br>received<br>Population | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 2 | 1 |
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 2 | -1 |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 900 | -1 |
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 900 | 1 |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 1 | |

STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY PSYCHFL AT Phase B

| | Center<br>(Pooled | Combat<br>Related | E-TRIP | Analusis | Planned | |
|---|---|---|---|---|---|---|
| | (POOLEG<br>Center) | Population | Psychotherapy<br>received | Analysis<br>Visit | Treatment | |
| Effect | for ITT | Flag | Population | (N) | (N) | Row1 |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |
| BASE*AVISITN | | | | 12 | | |



FILE: stat2f.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.6 FINAL


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY PSYCHFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Psychotherapy<br>received<br>Population | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |

FILE: stat2f.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.6 FINAL


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)



The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY PSYCHFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Psychotherapy<br>received<br>Population | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 12 | 900 | |
| PSYCHFL | | | N | | | |
| PSYCHFL | | | Y | | | |
| AVISITN*PSYCHFL | | | N | 3 | | |
| AVISITN*PSYCHFL | | | Y | 3 | | |
| AVISITN*PSYCHFL | | | N | 6 | | |
| AVISITN*PSYCHFL | | | Y | 6 | | |
| AVISITN*PSYCHFL | | | N | 10 | | |
| AVISITN*PSYCHFL | | | Y | 10 | | |
| AVISITN*PSYCHFL | | | N | 12 | | |
| AVISITN*PSYCHFL | | | Y | 12 | | |
| TRTPN*PSYCHFL | | | N | | 1 | |
| TRTPN*PSYCHFL | | | Y | | 1 | |
| TRTPN*PSYCHFL | | | N | | 2 | |
| TRTPN*PSYCHFL | | | Y | | 2 | |
| TRTPN*PSYCHFL | | | N | | 3 | 1 |
| TRTPN*PSYCHFL | | | Y | | 3 | -1 |
| TRTPN*PSYCHFL | | | N | | 900 | -1 |


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY PSYCHFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Psychotherapy<br>received<br>Population | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*PSYCHFL | | | Y | | 900 | 1 |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 3 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 3 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 6 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 6 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 1 | |


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY PSYCHFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Psychotherapy<br>received<br>Population | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 3 | 1 |
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 3 | -1 |
| AVISIT*TRTPN*PSYCHFL | | | N | 10 | 900 | -1 |
| AVISIT*TRTPN*PSYCHFL | | | Y | 10 | 900 | 1 |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 1 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 2 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 3 | |
| AVISIT*TRTPN*PSYCHFL | | | N | 12 | 900 | |
| AVISIT*TRTPN*PSYCHFL | | | Y | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |

BREXPIPRAZOLE 37 OF 39 PROTOCOL 331-201-00061 STAT-3.6 MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample) ------ Parameter Code=CAPSTOT -------The Mixed Procedure Coefficients for Dummy Y vs. Dummy Z BY PSYCHFL AT Phase B Center Combat E-TRIP (Pooled Related Psychotherapy Analysis Planned Center) Population received Visit Treatment Effect for ITT Flag Population (N) (N) Row1 BASE\*AVISITN 12 Estimates Standard Label Estimate Error DF t Value Pr > |t| 4.0198 235 0.35 0.7267 Dummy W vs. Dummy Z BY PSYCHFL AT Phase B 1.4065 Dummy W vs. Dummy Y BY PSYCHFL AT Phase B 2.4487 4.0839 238 0.60 0.5493 4.2667 239 1.37 5.8348 Dummy W vs. Dummy X BY PSYCHFL AT Phase B 0.1728 -4.4283 4.2406 243 -1.04 0.2974 Dummy X vs. Dummy Z BY PSYCHFL AT Phase B Dummy Y vs. Dummy Z BY PSYCHFL AT Phase B -1.0422 4.0383 239 -0.26 0.7966


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Least Squares Means

| Effect | E-TRIP<br>Psychotherapy<br>received<br>Population | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|---|
| AVISIT*TRTPN*PSYCHFL | N | 3 | 1 | -6.1372 | 1.3503 | 284 | -4.55 | <.0001 | 0.05 | -8.7950 | -3.4795 |
| AVISIT*TRTPN*PSYCHFL | Y | 3 | 1 | -6.9434 | 1.8105 | 286 | -3.83 | 0.0002 | 0.05 | -10.5071 | -3.3797 |
| AVISIT*TRTPN*PSYCHFL | N | 3 | 2 | -6.1027 | 1.4475 | 287 | -4.22 | <.0001 | 0.05 | -8.9518 | -3.2536 |
| AVISIT*TRTPN*PSYCHFL | Y | 3 | 2 | -1.8493 | 1.8811 | 278 | -0.98 | 0.3264 | 0.05 | -5.5522 | 1.8536 |
| AVISIT*TRTPN*PSYCHFL | N | 3 | 3 | -5.6929 | 1.4210 | 283 | -4.01 | <.0001 | 0.05 | -8.4900 | -2.8958 |
| AVISIT*TRTPN*PSYCHFL | Y | 3 | 3 | -6.9042 | 1.6863 | 278 | -4.09 | <.0001 | 0.05 | -10.2237 | -3.5847 |
| AVISIT*TRTPN*PSYCHFL | N | 3 | 900 | -6.4863 | 1.3364 | 282 | -4.85 | <.0001 | 0.05 | -9.1169 | -3.8557 |
| AVISIT*TRTPN*PSYCHFL | Y | 3 | 900 | -5.6811 | 1.7378 | 278 | -3.27 | 0.0012 | 0.05 | -9.1020 | -2.2602 |
| AVISIT*TRTPN*PSYCHFL | N | 6 | 1 | -11.9025 | 1.6729 | 280 | -7.11 | <.0001 | 0.05 | -15.1957 | -8.6094 |
| AVISIT*TRTPN*PSYCHFL | Y | 6 | 1 | -13.8684 | 2.1890 | 273 | -6.34 | <.0001 | 0.05 | -18.1779 | -9.5589 |
| AVISIT*TRTPN*PSYCHFL | N | 6 | 2 | -9.8421 | 1.7652 | 289 | -5.58 | <.0001 | 0.05 | -13.3164 | -6.3678 |
| AVISIT*TRTPN*PSYCHFL | Y | 6 | 2 | -4.5722 | 2.3491 | 272 | -1.95 | 0.0526 | 0.05 | -9.1969 | 0.05248 |
| AVISIT*TRTPN*PSYCHFL | N | 6 | 3 | -9.3668 | 1.7605 | 285 | -5.32 | <.0001 | 0.05 | -12.8321 | -5.9015 |
| AVISIT*TRTPN*PSYCHFL | Y | 6 | 3 | -10.0468 | 2.1052 | 271 | -4.77 | <.0001 | 0.05 | -14.1914 | -5.9022 |
| AVISIT*TRTPN*PSYCHFL | N | 6 | 900 | -9.9468 | 1.6157 | 268 | -6.16 | <.0001 | 0.05 | -13.1278 | -6.7658 |
| AVISIT*TRTPN*PSYCHFL | Y | 6 | 900 | -6.9034 | 2.1181 | 263 | -3.26 | 0.0013 | 0.05 | -11.0739 | -2.7328 |
| AVISIT*TRTPN*PSYCHFL | N | 10 | 1 | -16.1671 | 1.8153 | 252 | -8.91 | <.0001 | 0.05 | -19.7421 | -12.5920 |
| AVISIT*TRTPN*PSYCHFL | Y | 10 | 1 | -16.8136 | 2.3126 | 239 | -7.27 | <.0001 | 0.05 | -21.3694 | -12.2578 |

E MDID


STAT-3.6

MMRM Output for Test on Treatment by Psychosocial Support at Baseline Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Least Squares Means

| | E-TRIP<br>Psychotherapy | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | received | Visit | Treatment | | Standard | | | | | | |
| Effect | Population | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISIT*TRTPN*PSYCHFL | N | 10 | 2 | -14.0019 | 1.9371 | 276 | -7.23 | <.0001 | 0.05 | -17.8151 | -10.1886 |
| AVISIT*TRTPN*PSYCHFL | Y | 10 | 2 | -8.8136 | 2.6020 | 259 | -3.39 | 0.0008 | 0.05 | -13.9374 | -3.6898 |
| AVISIT*TRTPN*PSYCHFL | N | 10 | 3 | -12.0719 | 1.8954 | 257 | -6.37 | <.0001 | 0.05 | -15.8045 | -8.3394 |
| AVISIT*TRTPN*PSYCHFL | Y | 10 | 3 | -10.2698 | 2.2463 | 240 | -4.57 | <.0001 | 0.05 | -14.6946 | -5.8449 |
| AVISIT*TRTPN*PSYCHFL | N | 10 | 900 | -10.7352 | 1.7357 | 243 | -6.18 | <.0001 | 0.05 | -14.1542 | -7.3162 |
| AVISIT*TRTPN*PSYCHFL | Y | 10 | 900 | -9.9752 | 2.3036 | 249 | -4.33 | <.0001 | 0.05 | -14.5122 | -5.4383 |
| AVISIT*TRTPN*PSYCHFL | N | 12 | 1 | -17.2254 | 1.9928 | 258 | -8.64 | <.0001 | 0.05 | -21.1495 | -13.3013 |
| AVISIT*TRTPN*PSYCHFL | Y | 12 | 1 | -17.3662 | 2.5482 | 244 | -6.81 | <.0001 | 0.05 | -22.3855 | -12.3468 |
| AVISIT*TRTPN*PSYCHFL | N | 12 | 2 | -12.3917 | 2.1219 | 274 | -5.84 | <.0001 | 0.05 | -16.5690 | -8.2145 |
| AVISIT*TRTPN*PSYCHFL | Y | 12 | 2 | -11.7277 | 2.8526 | 261 | -4.11 | <.0001 | 0.05 | -17.3448 | -6.1106 |
| AVISIT*TRTPN*PSYCHFL | N | 12 | 3 | -13.9717 | 2.0651 | 258 | -6.77 | <.0001 | 0.05 | -18.0384 | -9.9051 |
| AVISIT*TRTPN*PSYCHFL | Y | 12 | 3 | -16.2002 | 2.4506 | 243 | -6.61 | <.0001 | 0.05 | -21.0274 | -11.3730 |
| AVISIT*TRTPN*PSYCHFL | N | 12 | 900 | -12.1535 | 1.9208 | 252 | -6.33 | <.0001 | 0.05 | -15.9363 | -8.3708 |
| AVISIT*TRTPN*PSYCHFL | Y | 12 | 900 | -10.7332 | 2.4790 | 244 | -4.33 | <.0001 | 0.05 | -15.6162 | -5.8502 |

BREXPIPRAZOLE 1 OF 39

STAT-3.7

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Model Information

Data Set WORK.INDATA
Dependent Variable CHG
Covariance Structure Unstructured
Subject Effect SUBJID
Estimation Method REML

Estimation Method REML
Residual Variance Method None
Fixed Effects SE Method Kenward

Fixed Effects SE Method Kenward-Roger Degrees of Freedom Method Kenward-Roger

Class Level Information



FILE: stat2g.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.7 FINAL

BREXPIPRAZOLE

3 OF 39

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

------

The Mixed Procedure



BREXPIPRAZOLE

STAT-3.7

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

The Mixed Procedure



FILE: stat2g.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.7 FINAL

BREXPIPRAZOLE 5 OF 39

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

------

The Mixed Procedure



FILE: stat2g.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.7 FINAL

BREXPIPRAZOLE 6 OF 39 PROTOCOL 331-201-00061 STAT-3.7 MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample) The Mixed Procedure ΝΥ PREMEDFL 2 Dimensions Covariance Parameters 10 Columns in X 91 Columns in Z 0 299 Subjects Max Obs per Subject Number of Observations 996 Number of Observations Read Number of Observations Used 996 Number of Observations Not Used

FILE: stat2g.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.7 FINAL

BREXPIPRAZOLE 7 OF 39

STAT-3.7

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)



The Mixed Procedure

Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 7350.10732814 | |
| 1 | 2 | 6874.16683915 | 0.00059842 |
| 2 | 1 | 6872.44878479 | 0.00002676 |
| 3 | 1 | 6872.37799072 | 0.0000007 |
| 4 | 1 | 6872.37782002 | 0.00000000 |

Convergence criteria met.

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | 78.4556 |
| UN(2,1) | SUBJID | 53.7623 |
| UN(2,2) | SUBJID | 114.95 |
| UN(3,1) | SUBJID | 45.2487 |
| UN(3,2) | SUBJID | 91.1453 |
| UN(3,3) | SUBJID | 125.08 |
| UN(4,1) | SUBJID | 49.9731 |

BREXPIPRAZOLE 8 OF 39

STAT-3.7

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN (4,2) | SUBJID | 91.1421 |
| UN (4,3) | SUBJID | 105.71 |
| UN (4,4) | SUBJID | 148.31 |

Fit Statistics

| -2 Res Log Likelihood | 6872.4 |
|--------------------------|--------|
| AIC (Smaller is Better) | 6892.4 |
| AICC (Smaller is Better) | 6892.6 |
| BIC (Smaller is Better) | 6929.4 |

Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|----|------------|------------|
| 9 | 477.73 | <.0001 |

FILE: stat2g.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.7 FINAL

BREXPIPRAZOLE 9 OF 39

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction

(Intent to Treat Sample)

The Mixed Procedure

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|----------------------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| POOLCNTR | 9 | 277 | 1.60 | 0.1137 |
| COMBFL | 1 | 278 | 4.09 | 0.0441 |
| AVISITN | 3 | 228 | 0.70 | 0.5533 |
| TRTPN | 3 | 263 | 2.90 | 0.0355 |
| AVISITN*TRTPN | 9 | 357 | 1.74 | 0.0795 |
| PREMEDFL | 1 | 270 | 1.92 | 0.1672 |
| AVISITN*PREMEDFL | 3 | 234 | 2.49 | 0.0609 |
| TRTPN*PREMEDFL | 3 | 265 | 0.15 | 0.9284 |
| AVISIT*TRTPN*PREMEDF | 9 | 357 | 0.57 | 0.8251 |
| BASE*AVISITN | 4 | 240 | 14.94 | <.0001 |



FILE: stat2g.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.7 FINAL


STAT-3.7

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

------

The Mixed Procedure

------ Parameter Code=CAPSTOT ------

Coefficients for Dummy W vs. Dummy Z BY PREMEDFL AT Phase B

| | Center | Combat | E-TRIP | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | Prescription | Analysis | Planned | |
| | Center) | Population | Medication | Visit | Treatment | |
| Effect | for ITT | Flag | Usage Pop | (N) | (N) | Row1 |
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |


MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY PREMEDFL AT Phase B

| Effect | Center) | | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|
| AVISITN*TRTPN PREMEDFL PREMEDFL AVISITN*PREMEDFL | | N Y | 3<br>3<br>6<br>6<br>10<br>10<br>12<br>12 | 900 | 1 |
| TRTPN*PREMEDFL | | N | | 1 | 1 |
| TRTPN*PREMEDFL TRTPN*PREMEDFL | | Y<br>N | | 1 2 | -1 |
| TRTPN*PREMEDEL | | Y | | 2 | |
| TRTPN*PREMEDFL | | N | | 3 | |
| TRTPN*PREMEDFL | | Y | | 3 | |
| TRTPN*PREMEDFL | | N | | 900 | -1 |

BREXPIPRAZOLE 13 OF 39


MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY PREMEDFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Prescription<br>Medication<br>Usage Pop | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*PREMEDFL | | | Y | | 900 | 1 |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 1 | 1 |


STAT-3.7

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY PREMEDFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Prescription<br>Medication<br>Usage Pop | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 1 | -1 |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 900 | -1 |
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 900 | 1 |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |



FILE: stat2g.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.7 FINAL

| BREXPIPRAZOLE<br>PROTOCOL 331-20 | 1 00061 | | | | | | 16 OF 39 |
|---|---|---|---|---|---|---|---|
| | MMRM Output for Test on Treatr | ment by Previc | us Pharmacolog | AT-3.7<br>yical Treatment I<br>Treat Sample) | ntervention | for PTSD Inter | raction |
| | | | The Mixed | l Procedure | | | |
| | Coeff | icients for Du | mmy W vs. Dumn | ny Y BY PREMEDFL | AT Phase B | | |
| | Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Prescription<br>Medication<br>Usage Pop | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
| | POOLCNTR POOLCNTR POOLCNTR COMBFL COMBFL AVISITN AVISITN AVISITN TRTPN TRTPN TRTPN TRTPN TRTPN AVISITN*TRTPN | | N<br>Y | | 3<br>6<br>10<br>12<br>3<br>3<br>3<br>3<br>3<br>6 | 1<br>2<br>3<br>900<br>1<br>2<br>3<br>900<br>1 | |

FILE: stat2g.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.7 FINAL


STAT-3.7

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

------

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY PREMEDFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Prescription<br>Medication<br>Usage Pop | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |
| AVISITN*TRTPN | | | | 12 | 900 | |
| PREMEDFL | | | N | | | |
| PREMEDFL | | | Y | | | |
| AVISITN*PREMEDFL | | | N | 3 | | |
| AVISITN*PREMEDFL | | | Y | 3 | | |
| AVISITN*PREMEDFL | | | N | 6 | | |
| AVISITN*PREMEDFL | | | Y | 6 | | |
| AVISITN*PREMEDFL | | | N | 10 | | |


STAT-3.7

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY PREMEDFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Prescription<br>Medication<br>Usage Pop | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*PREMEDFL | | | Y | 10 | | |
| AVISITN*PREMEDFL | | | N | 12 | | |
| AVISITN*PREMEDFL | | | Y | 12 | | |
| TRTPN*PREMEDFL | | | N | | 1 | 1 |
| TRTPN*PREMEDFL | | | Y | | 1 | -1 |
| TRTPN*PREMEDFL | | | N | | 2 | |
| TRTPN*PREMEDFL | | | Y | | 2 | |
| TRTPN*PREMEDFL | | | N | | 3 | -1 |
| TRTPN*PREMEDFL | | | Y | | 3 | 1 |
| TRTPN*PREMEDFL | | | N | | 900 | |
| TRTPN*PREMEDFL | | | Y | | 900 | |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 900 | |

BREXPIPRAZOLE 19 OF 39


MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY PREMEDFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Prescription<br>Medication<br>Usage Pop | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 1 | 1 |
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 1 | -1 |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 3 | -1 |
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 3 | 1 |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 1 | |

BREXPIPRAZOLE 20 OF 39


MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

-----

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY PREMEDFL AT Phase B

| | Center | Combat | E-TRIP | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | Prescription | Analysis | Planned | |
| | Center) | Population | Medication | Visit | Treatment | |
| Effect | for ITT | Flag | Usage Pop | (N) | (N) | Row1 |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 2 | |
| | | | | | 2 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |
| BASE*AVISITN | | | | 12 | | |



FILE: stat2g.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.7 FINAL

BREXPIPRAZOLE 22 OF 39


MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY PREMEDFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | E-TRIP<br>Prescription<br>Medication<br>Usage Pop | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|
| TRTPN | | | | 2 | |
| TRTPN | | | | 3 | |
| TRTPN | | | | 900 | |
| AVISITN*TRTPN | | | 3 | 1 | |
| AVISITN*TRTPN | | | 3 | 2 | |
| AVISITN*TRTPN | | | 3 | 3 | |
| AVISITN*TRTPN | | | 3 | 900 | |
| AVISITN*TRTPN | | | 6 | 1 | |
| AVISITN*TRTPN | | | 6 | 2 | |
| AVISITN*TRTPN | | | 6 | 3 | |
| AVISITN*TRTPN | | | 6 | 900 | |
| AVISITN*TRTPN | | | 10 | 1 | |
| AVISITN*TRTPN | | | 10 | 2 | |
| AVISITN*TRTPN | | | 10 | 3 | |
| AVISITN*TRTPN | | | 10 | 900 | |
| AVISITN*TRTPN | | | 12 | 1 | |
| AVISITN*TRTPN | | | 12 | 2 | |
| AVISITN*TRTPN | | | 12 | 3 | |

BREXPIPRAZOLE 23 OF 39

STAT-3.7

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY PREMEDFL AT Phase B

| Effect | • | Combat<br>Related<br>Population<br>Flag | * | | | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN PREMEDFL PREMEDFL AVISITN*PREMEDFL | | | N<br>Y<br>N<br>Y<br>N<br>Y | 12<br>3<br>3<br>6<br>6<br>10 | 900 | |
| AVISITN*PREMEDFL | | | N | 12 | | |
| AVISITN*PREMEDFL | | | Y | 12 | | |
| TRTPN*PREMEDFL | | | N | | 1 | 1 |
| TRTPN*PREMEDFL | | | Y | | 1 | -1 |
| TRTPN*PREMEDFL TRTPN*PREMEDFL | | | N<br>Y | | 2 2 | -1 |
| TRTPN*PREMEDEL | | | N | | 3 | 1 |
| TRTPN*PREMEDFL | | | Y | | 3 | |
| TRTPN*PREMEDFL | | | N | | 900 | |


STAT-3.7

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY PREMEDFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Prescription<br>Medication<br>Usage Pop | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*PREMEDFL | | | Y | | 900 | |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 1 | 1 |


STAT-3.7

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY PREMEDFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Prescription<br>Medication<br>Usage Pop | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 1 | -1 |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 2 | -1 |
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 2 | 1 |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |



FILE: stat2g.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.7 FINAL



FILE: stat2g.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.7 FINAL
BREXPIPRAZOLE 28 OF 39


MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY PREMEDFL AT Phase B

| Effect | E-TRIP<br>Prescription<br>Medication<br>Usage Pop | | | Row1 |
|---|---|---|---|---|
| AVISITN*TRTPN | | 6 | 2 | |
| AVISITN*TRTPN | | 6 | 3 | |
| AVISITN*TRTPN | | 6 | 900 | |
| AVISITN*TRTPN | | 10 | 1 | |
| AVISITN*TRTPN | | 10 | 2 | |
| AVISITN*TRTPN | | 10 | 3 | |
| AVISITN*TRTPN | | 10 | 900 | |
| AVISITN*TRTPN | | 12 | 1 | |
| AVISITN*TRTPN | | 12 | 2 | |
| AVISITN*TRTPN | | 12 | 3 | |
| AVISITN*TRTPN | | 12 | 900 | |
| PREMEDFL | N | | | |
| PREMEDFL | Y | | | |
| AVISITN*PREMEDFL | N | 3 | | |
| AVISITN*PREMEDFL | Y | 3 | | |
| AVISITN*PREMEDFL | N | 6 | | |
| AVISITN*PREMEDFL | Y | 6 | | |
| AVISITN*PREMEDFL | N | 10 | | |


STAT-3.7

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

-----

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY PREMEDFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*PREMEDFL | | | Y | 10 | | |
| AVISITN*PREMEDFL | | | N | 12 | | |
| AVISITN*PREMEDFL | | | Y | 12 | | |
| TRTPN*PREMEDFL | | | N | | 1 | |
| TRTPN*PREMEDFL | | | Y | | 1 | |
| TRTPN*PREMEDFL | | | N | | 2 | 1 |
| TRTPN*PREMEDFL | | | Y | | 2 | -1 |
| TRTPN*PREMEDFL | | | N | | 3 | |
| TRTPN*PREMEDFL | | | Y | | 3 | |
| TRTPN*PREMEDFL | | | N | | 900 | -1 |
| TRTPN*PREMEDFL | | | Y | | 900 | 1 |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 900 | |


STAT-3.7

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

-----

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY PREMEDFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Prescription<br>Medication<br>Usage Pop | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 2 | 1 |
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 2 | -1 |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 900 | -1 |
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 900 | 1 |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 1 | |

BREXPIPRAZOLE 31 OF 39


MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

.\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY PREMEDFL AT Phase B

| | Center | Combat | E-TRIP | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | Prescription | Analysis | Planned | |
| | Center) | Population | Medication | Visit | Treatment | |
| Effect | for ITT | Flag | Usage Pop | (N) | (N) | Row1 |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |
| BASE*AVISITN | | | | 12 | | |



FILE: stat2g.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.7 FINAL

BREXPIPRAZOLE 33 OF 39


MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

.\_\_\_\_\_

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY PREMEDFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Prescription<br>Medication<br>Usage Pop | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |


STAT-3.7

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

-----

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY PREMEDFL AT Phase B

| Effect | Center) | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Prescription<br>Medication<br>Usage Pop | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 12 | 900 | |
| PREMEDFL | | | N | | | |
| PREMEDFL | | | Y | | | |
| AVISITN*PREMEDFL | | | N | 3 | | |
| AVISITN*PREMEDFL | | | Y | 3 | | |
| AVISITN*PREMEDFL | | | N | 6 | | |
| AVISITN*PREMEDFL | | | Y | 6 | | |
| AVISITN*PREMEDFL | | | N | 10 | | |
| AVISITN*PREMEDFL | | | Y | 10 | | |
| AVISITN*PREMEDFL | | | N | 12 | | |
| AVISITN*PREMEDFL | | | Y | 12 | | |
| TRTPN*PREMEDFL | | | N | | 1 | |
| TRTPN*PREMEDFL | | | Y | | 1 | |
| TRTPN*PREMEDFL | | | N | | 2 | |
| TRTPN*PREMEDFL | | | Y | | 2 | |
| TRTPN*PREMEDFL | | | N | | 3 | 1 |
| TRTPN*PREMEDFL | | | Y | | 3 | -1 |
| TRTPN*PREMEDFL | | | N | | 900 | -1 |


STAT-3.7

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)



The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY PREMEDFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | E-TRIP<br>Prescription<br>Medication<br>Usage Pop | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*PREMEDFL | | | Y | | 900 | 1 |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | N | 3 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 3 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | N | 6 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 6 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 1 | |


STAT-3.7

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY PREMEDFL AT Phase B

| | Center | Combat | E-TRIP | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | Prescription | Analysis | Planned | |
| | Center) | Population | Medication | Visit | Treatment | |
| Effect | for ITT | Flag | Usage Pop | (N) | (N) | Row1 |
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 1 | |
| | | | | | 1 | |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 3 | 1 |
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 3 | -1 |
| AVISIT*TRTPN*PREMEDF | | | N | 10 | 900 | -1 |
| AVISIT*TRTPN*PREMEDF | | | Y | 10 | 900 | 1 |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 1 | |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 2 | |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 3 | |
| AVISIT*TRTPN*PREMEDF | | | N | 12 | 900 | |
| AVISIT*TRTPN*PREMEDF | | | Y | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | 37 OF 39 |
|---|---|---|---|---|---|---|
| MMRM Output for Test on Treatmen | t by Previous | STAT<br>Pharmacologi<br>(Intent to T | cal Treatment I | ntervention | for PTSD Intera | ction |
| | | - Parameter C | ode=CAPSTOT | | | |
| | | The Mixed | Procedure | | | |
| Coeffici | ents for Dumm | y Y vs. Dummy | Z BY PREMEDFL | AT Phase B | | |
| | | Combat | E-TRIP | | | |
| | • | Related<br>Population | Prescription<br>Medication | Analysis<br>Visit | Planned<br>Treatment | |
| Effect | | Flag | Usage Pop | (N) | (N) | Row1 |
| BASE*AVISITN | | | | 12 | | |
| | | Estin | ates | | | |
| | | | St | andard | | |
| Label | | | Estimate | Error | DF t Value | Pr > t |
| Dummy W vs. Dummy Z BY PREM<br>Dummy W vs. Dummy Y BY PREM | | | | | 41 -0.65<br>39 -1.19 | 0.5185<br>0.2358 |
| Dummy W vs. Dummy X BY PREM | | | | | 49 -0.41 | 0.6804 |
| Dummy X vs. Dummy Z BY PREM | | | | | 41 -0.19 | 0.8494 |
| Dummy Y vs. Dummy Z BY PREM | EDFL AT Phase | В | 2.2118 | 3.8943 2 | 36 0.57 | 0.5706 |


STAT-3.

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

.\_\_\_\_\_

The Mixed Procedure

Least Squares Means

| Effect | E-TRIP<br>Prescription<br>Medication<br>Usage Pop | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|---|
| AVISIT*TRTPN*PREMEDF | N | 3 | 1 | -5.9586 | 1.4528 | 284 | -4.10 | <.0001 | 0.05 | -8.8183 | -3.0989 |
| AVISIT*TRTPN*PREMEDF | Y | 3 | 1 | -7.1843 | 1.5970 | 284 | -4.50 | <.0001 | 0.05 | -10.3277 | -4.0409 |
| AVISIT*TRTPN*PREMEDF | N | 3 | 2 | -5.3257 | 1.4509 | 286 | -3.67 | 0.0003 | 0.05 | -8.1813 | -2.4700 |
| AVISIT*TRTPN*PREMEDF | Y | 3 | 2 | -3.2959 | 1.8974 | 283 | -1.74 | 0.0835 | 0.05 | -7.0308 | 0.4390 |
| AVISIT*TRTPN*PREMEDF | N | 3 | 3 | -6.0331 | 1.5188 | 280 | -3.97 | <.0001 | 0.05 | -9.0227 | -3.0434 |
| AVISIT*TRTPN*PREMEDF | Y | 3 | 3 | -6.4722 | 1.5379 | 280 | -4.21 | <.0001 | 0.05 | -9.4996 | -3.4448 |
| AVISIT*TRTPN*PREMEDF | N | 3 | 900 | -5.2659 | 1.4825 | 280 | -3.55 | 0.0004 | 0.05 | -8.1842 | -2.3476 |
| AVISIT*TRTPN*PREMEDF | Y | 3 | 900 | -7.3272 | 1.5014 | 280 | -4.88 | <.0001 | 0.05 | -10.2826 | -4.3718 |
| AVISIT*TRTPN*PREMEDF | N | 6 | 1 | -13.5175 | 1.8602 | 291 | -7.27 | <.0001 | 0.05 | -17.1786 | -9.8564 |
| AVISIT*TRTPN*PREMEDF | Y | 6 | 1 | -11.8145 | 1.9044 | 255 | -6.20 | <.0001 | 0.05 | -15.5649 | -8.0641 |
| AVISIT*TRTPN*PREMEDF | N | 6 | 2 | -8.2573 | 1.7743 | 290 | -4.65 | <.0001 | 0.05 | -11.7494 | -4.7652 |
| AVISIT*TRTPN*PREMEDF | Y | 6 | 2 | -7.6094 | 2.3669 | 273 | -3.21 | 0.0015 | 0.05 | -12.2690 | -2.9498 |
| AVISIT*TRTPN*PREMEDF | N | 6 | 3 | -10.1851 | 1.9237 | 278 | -5.29 | <.0001 | 0.05 | -13.9719 | -6.3982 |
| AVISIT*TRTPN*PREMEDF | Y | 6 | 3 | -9.2714 | 1.9102 | 274 | -4.85 | <.0001 | 0.05 | -13.0318 | -5.5109 |
| AVISIT*TRTPN*PREMEDF | N | 6 | 900 | -9.2920 | 1.8273 | 271 | -5.09 | <.0001 | 0.05 | -12.8895 | -5.6945 |
| AVISIT*TRTPN*PREMEDF | Y | 6 | 900 | -8.5329 | 1.8245 | 258 | -4.68 | <.0001 | 0.05 | -12.1258 | -4.9401 |
| AVISIT*TRTPN*PREMEDF | N | 10 | 1 | -19.0715 | 1.9707 | 256 | -9.68 | <.0001 | 0.05 | -22.9524 | -15.1906 |
| AVISIT*TRTPN*PREMEDF | Y | 10 | 1 | -13.6610 | 2.0425 | 237 | -6.69 | <.0001 | 0.05 | -17.6847 | -9.6373 |


STAT-3.

MMRM Output for Test on Treatment by Previous Pharmacological Treatment Intervention for PTSD Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Least Squares Means

| | E-TRIP | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| <b>-</b> | Prescription<br>Medication | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
| Effect | Usage Pop | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISIT*TRTPN*PREMEDF | N | 10 | 2 | -13.5968 | 1.9479 | 284 | -6.98 | <.0001 | 0.05 | -17.4309 | -9.7628 |
| AVISIT*TRTPN*PREMEDF | Y | 10 | 2 | -9.9327 | 2.5490 | 250 | -3.90 | 0.0001 | 0.05 | -14.9529 | -4.9125 |
| AVISIT*TRTPN*PREMEDF | N | 10 | 3 | -11.7285 | 2.0469 | 249 | -5.73 | <.0001 | 0.05 | -15.7598 | -7.6971 |
| AVISIT*TRTPN*PREMEDF | Y | 10 | 3 | -11.0617 | 2.0291 | 245 | -5.45 | <.0001 | 0.05 | -15.0583 | -7.0650 |
| AVISIT*TRTPN*PREMEDF | N | 10 | 900 | -11.9431 | 1.9566 | 251 | -6.10 | <.0001 | 0.05 | -15.7965 | -8.0897 |
| AVISIT*TRTPN*PREMEDF | Y | 10 | 900 | -9.0645 | 1.9476 | 239 | -4.65 | <.0001 | 0.05 | -12.9011 | -5.2278 |
| AVISIT*TRTPN*PREMEDF | N | 12 | 1 | -19.5557 | 2.1581 | 261 | -9.06 | <.0001 | 0.05 | -23.8051 | -15.3062 |
| AVISIT*TRTPN*PREMEDF | Y | 12 | 1 | -14.9362 | 2.2502 | 242 | -6.64 | <.0001 | 0.05 | -19.3687 | -10.5036 |
| AVISIT*TRTPN*PREMEDF | N | 12 | 2 | -12.8805 | 2.1286 | 280 | -6.05 | <.0001 | 0.05 | -17.0706 | -8.6903 |
| AVISIT*TRTPN*PREMEDF | Y | 12 | 2 | -11.1719 | 2.7840 | 249 | -4.01 | <.0001 | 0.05 | -16.6550 | -5.6887 |
| AVISIT*TRTPN*PREMEDF | N | 12 | 3 | -15.7175 | 2.2111 | 244 | -7.11 | <.0001 | 0.05 | -20.0728 | -11.3622 |
| AVISIT*TRTPN*PREMEDF | Y | 12 | 3 | -14.1342 | 2.2280 | 250 | -6.34 | <.0001 | 0.05 | -18.5223 | -9.7462 |
| AVISIT*TRTPN*PREMEDF | N | 12 | 900 | -13.1450 | 2.1214 | 247 | -6.20 | <.0001 | 0.05 | -17.3234 | -8.9666 |
| AVISIT*TRTPN*PREMEDF | Y | 12 | 900 | -10.2577 | 2.1553 | 249 | -4.76 | <.0001 | 0.05 | -14.5028 | -6.0127 |

BREXPIPRAZOLE 1 OF 39

 $$\tt STAT-3.8$$  MMRM Output for Test on Treatment by Use of Wearable Device Interaction

(Intent to Treat Sample)

The Mixed Procedure

Model Information

Data Set WORK.INDATA
Dependent Variable CHG
Covariance Structure Unstructured
Subject Effect SUBJID
Estimation Method REML
Residual Variance Method None

Fixed Effects SE Method Kenward-Roger Degrees of Freedom Method Kenward-Roger

Class Level Information

BREXPIPRAZOLE

STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

The Mixed Procedure
Class Level Information

Class Levels Values

SUBJID 299

FILE: stat2h.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.8 FINAL

BREXPIPRAZOLE 3 OF 39

 $$\tt STAT-3.8$$  MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure



FILE: stat2h.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.8 FINAL

BREXPIPRAZOLE

STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction
(Intent to Treat Sample)

The Mixed Procedure



FILE: stat2h.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.8 FINAL

BREXPIPRAZOLE

STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction
(Intent to Treat Sample)

The Mixed Procedure



FILE: stat2h.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.8 FINAL

BREXPIPRAZOLE 6 OF 39 PROTOCOL 331-201-00061 STAT-3.8 MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample) The Mixed Procedure ACTFL 2 NY Dimensions Covariance Parameters 10 Columns in X 91 Columns in Z 0 299 Subjects Max Obs per Subject Number of Observations 996 Number of Observations Read 996 Number of Observations Used Number of Observations Not Used

FILE: stat2h.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.8 FINAL

BREXPIPRAZOLE 7 OF 39

STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

The Mixed Procedure

Iteration History

| Criterion | -2 Res Log Like | Evaluations | Iteration |
|------------|-----------------|-------------|-----------|
| | 7339.70119712 | 1 | 0 |
| 0.00097377 | 6874.98262651 | 2 | 1 |
| 0.00006613 | 6872.12913247 | 1 | 2 |
| 0.00000039 | 6871.95142830 | 1 | 3 |
| 0.00000000 | 6871.95041291 | 1 | 4 |

Convergence criteria met.

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | 78.9311 |
| UN(2,1) | SUBJID | 53.3500 |
| UN(2,2) | SUBJID | 114.65 |
| UN(3,1) | SUBJID | 44.7163 |
| UN(3,2) | SUBJID | 90.3579 |
| UN(3,3) | SUBJID | 125.18 |
| UN(4,1) | SUBJID | 48.5868 |

BREXPIPRAZOLE 8 OF 39

STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Covariance Parameter Estimates

| Cov Parm Subject | Estimate |
|------------------|----------|
| UN(4,2) SUBJID | 89.8766 |
| UN(4,3) SUBJID | 104.28 |
| UN(4,4) SUBJID | 144.74 |

Fit Statistics

| -2 Res Log Likelihood | 6872.0 |
|--------------------------|--------|
| AIC (Smaller is Better) | 6892.0 |
| AICC (Smaller is Better) | 6892.2 |
| BIC (Smaller is Better) | 6929.0 |

Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|----|------------|------------|
| 9 | 467.75 | <.0001 |

BREXPIPRAZOLE 9 OF 39

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

-----

The Mixed Procedure

Type 3 Tests of Fixed Effects

| Num | Den | | |
|---|---|---|---|
| DF | DF | F Value | Pr > F |
| ^ | 0.7.7 | 1 60 | 0 0016 |
| 9 | 2// | 1.68 | 0.0946 |
| 1 | 278 | 3.85 | 0.0508 |
| 3 | 226 | 0.76 | 0.5187 |
| 3 | 270 | 2.10 | 0.1003 |
| 9 | 361 | 1.02 | 0.4226 |
| 1 | 298 | 2.40 | 0.1224 |
| 3 | 235 | 2.48 | 0.0619 |
| 3 | 271 | 0.04 | 0.9904 |
| 9 | 361 | 0.32 | 0.9679 |
| 4 | 240 | 13.44 | <.0001 |
| | DF 9 1 3 3 9 1 3 3 9 9 | DF DF 9 277 1 278 3 226 3 270 9 361 1 298 3 271 9 361 | DF DF F Value 9 277 1.68 1 278 3.85 3 226 0.76 3 270 2.10 9 361 1.02 1 298 2.40 3 235 2.48 3 271 0.04 9 361 0.32 |



FILE: stat2h.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.8 FINAL


STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

\_\_\_\_\_

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY ACTFL AT Phase B

| | | Center | Combat | Actiwatch | | | |
|---|---|---|---|---|---|---|---|
| | | (Pooled | Related | Usage | Analysis | Planned | |
| | | Center) | Population | Population | Visit | Treatment | |
| Effect | | for ITT | Flag | Flag | (N) | (N) | Row1 |
| TRTPN | | | | | | 2 | |
| TRTPN | | | | | | 3 | |
| TRTPN | | | | | | 900 | |
| AVISITN*TRTE | N | | | | 3 | 1 | |
| AVISITN*TRTE | N | | | | 3 | 2 | |
| AVISITN*TRTE | N | | | | 3 | 3 | |
| AVISITN*TRTE | N | | | | 3 | 900 | |
| AVISITN*TRTE | N | | | | 6 | 1 | |
| AVISITN*TRTE | N | | | | 6 | 2 | |
| AVISITN*TRTE | N | | | | 6 | 3 | |
| AVISITN*TRTE | N | | | | 6 | 900 | |
| AVISITN*TRTE | N | | | | 10 | 1 | |
| AVISITN*TRTE | N | | | | 10 | 2 | |
| AVISITN*TRTE | N | | | | 10 | 3 | |
| AVISITN*TRTE | N | | | | 10 | 900 | |
| AVISITN*TRTE | N | | | | 12 | 1 | |
| AVISITN*TRTE | | | | | 12 | 2 | |
| AVISITN*TRTE | | | | | 12 | 3 | |
| 11 1 1 1 1 1 1 1 1 1 1 1 1 | 7.4 | | | | 14 | 9 | |


STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

.\_\_\_\_\_

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY ACTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Actiwatch<br>Usage<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 12 | 900 | |
| ACTFL | | | N | | | |
| ACTFL | | | Y | | | |
| AVISITN*ACTFL | | | N | 3 | | |
| AVISITN*ACTFL | | | Y | 3 | | |
| AVISITN*ACTFL | | | N | 6 | | |
| AVISITN*ACTFL | | | Y | 6 | | |
| AVISITN*ACTFL | | | N | 10 | | |
| AVISITN*ACTFL | | | Y | 10 | | |
| AVISITN*ACTFL | | | N | 12 | | |
| AVISITN*ACTFL | | | Y | 12 | | |
| TRTPN*ACTFL | | | N | | 1 | 1 |
| TRTPN*ACTFL | | | Y | | 1 | -1 |
| TRTPN*ACTFL | | | N | | 2 | |
| TRTPN*ACTFL | | | Y | | 2 | |
| TRTPN*ACTFL | | | N | | 3 | |
| TRTPN*ACTFL | | | Y | | 3 | |
| TRTPN*ACTFL | | | N | | 900 | -1 |


STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY ACTFL AT Phase B

| | Center | Combat | Actiwatch | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | Usage | Analysis | Planned | |
| | Center) | Population | Population | Visit | Treatment | |
| Effect | for ITT | Flag | Flag | (N) | (N) | Row1 |
| TRTPN*ACTFL | | | Y | | 900 | 1 |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 1 | |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 1 | |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 2 | |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 2 | |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 3 | |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 3 | |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 900 | |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 900 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 1 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 1 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 2 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 2 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 3 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 3 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 900 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 900 | |
| AVISITN*TRTPN*ACTFL | | | N | 10 | 1 | 1 |


STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

\_\_\_\_\_

------Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Z BY ACTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Actiwatch<br>Usage<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN*ACTFL | | | Y | 10 | 1 | -1 |
| AVISITN*TRTPN*ACTFL | | | N | 10 | 2 | |
| AVISITN*TRTPN*ACTFL | | | Y | 10 | 2 | |
| AVISITN*TRTPN*ACTFL | | | N | 10 | 3 | |
| AVISITN*TRTPN*ACTFL | | | Y | 10 | 3 | |
| AVISITN*TRTPN*ACTFL | | | N | 10 | 900 | -1 |
| AVISITN*TRTPN*ACTFL | | | Y | 10 | 900 | 1 |
| AVISITN*TRTPN*ACTFL | | | N | 12 | 1 | |
| AVISITN*TRTPN*ACTFL | | | Y | 12 | 1 | |
| AVISITN*TRTPN*ACTFL | | | N | 12 | 2 | |
| AVISITN*TRTPN*ACTFL | | | Y | 12 | 2 | |
| AVISITN*TRTPN*ACTFL | | | N | 12 | 3 | |
| AVISITN*TRTPN*ACTFL | | | Y | 12 | 3 | |
| AVISITN*TRTPN*ACTFL | | | N | 12 | 900 | |
| AVISITN*TRTPN*ACTFL | | | Y | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |



FILE: stat2h.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.8 FINAL

BREXPIPRAZOLE 16 OF 39 PROTOCOL 331-201-00061 STAT-3.8 MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy W vs. Dummy Y BY ACTFL AT Phase B Center Combat Actiwatch (Pooled Related Usage Analysis Planned Population Population Visit Center) Treatment Effect for ITT Flag Flag (N) (N) Row1 POOLCNTR POOLCNTR POOLCNTR COMBFL N COMBFL 3 AVISITN AVISITN AVISITN 10 AVISITN 12 1 TRTPN TRTPN 2 TRTPN 900 TRTPN AVISITN\*TRTPN 3 1 AVISITN\*TRTPN 3 2 AVISITN\*TRTPN 3 AVISITN\*TRTPN 3 900 AVISITN\*TRTPN 1

FILE: stat2h.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.8 FINAL


MMRM Output for Test on Treatment by Use of Wearable Device Interaction

(Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY ACTFL AT Phase B

| | Center | Combat | Actiwatch | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | Usage | Analysis | Planned | |
| | Center) | Population | Population | Visit | Treatment | |
| Effect | for ITT | Flag | Flag | (N) | (N) | Row1 |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |
| AVISITN*TRTPN | | | | 12 | 900 | |
| ACTFL | | | N | | | |
| ACTFL | | | Y | | | |
| AVISITN*ACTFL | | | N | 3 | | |
| AVISITN*ACTFL | | | Y | 3 | | |
| AVISITN*ACTFL | | | N | 6 | | |
| AVISITN*ACTFL | | | Y | 6 | | |
| AVISITN*ACTFL | | | N | 10 | | |


STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY ACTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Actiwatch<br>Usage<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*ACTFL | | | Y | 10 | | |
| AVISITN*ACTFL | | | N | 12 | | |
| AVISITN*ACTFL | | | Y | 12 | | |
| TRTPN*ACTFL | | | N | | 1 | 1 |
| TRTPN*ACTFL | | | Y | | 1 | -1 |
| TRTPN*ACTFL | | | N | | 2 | |
| TRTPN*ACTFL | | | Y | | 2 | |
| TRTPN*ACTFL | | | N | | 3 | -1 |
| TRTPN*ACTFL | | | Y | | 3 | 1 |
| TRTPN*ACTFL | | | N | | 900 | |
| TRTPN*ACTFL | | | Y | | 900 | |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 1 | |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 1 | |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 2 | |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 2 | |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 3 | |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 3 | |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 900 | |


STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

-----

The Mixed Procedure

------ Parameter Code=CAPSTOT ------

Coefficients for Dummy W vs. Dummy Y BY ACTFL AT Phase B

| | Center | Combat | Actiwatch | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | Usage | Analysis | Planned | |
| | Center) | Population | Population | Visit | Treatment | |
| Effect | for ITT | Flag | Flag | (N) | (N) | Row1 |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 900 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 1 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 1 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 2 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 2 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 3 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 3 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 900 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 900 | |
| AVISITN*TRTPN*ACTFL | | | N | 10 | 1 | 1 |
| AVISITN*TRTPN*ACTFL | | | Y | 10 | 1 | -1 |
| AVISITN*TRTPN*ACTFL | | | N | 10 | 2 | |
| AVISITN*TRTPN*ACTFL | | | Y | 10 | 2 | |
| AVISITN*TRTPN*ACTFL | | | N | 10 | 3 | -1 |
| AVISITN*TRTPN*ACTFL | | | Y | 10 | 3 | 1 |
| AVISITN*TRTPN*ACTFL | | | N | 10 | 900 | |
| AVISITN*TRTPN*ACTFL | | | Y | 10 | 900 | |
| AVISITN*TRTPN*ACTFL | | | N | 12 | 1 | |


STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy Y BY ACTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Actiwatch<br>Usage<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| Filect | 101 111 | riag | riag | (IV) | (11) | ROWI |
| AVISITN*TRTPN*ACTFL | | | Y | 12 | 1 | |
| AVISITN*TRTPN*ACTFL | | | N | 12 | 2 | |
| AVISITN*TRTPN*ACTFL | | | Y | 12 | 2 | |
| AVISITN*TRTPN*ACTFL | | | N | 12 | 3 | |
| AVISITN*TRTPN*ACTFL | | | Y | 12 | 3 | |
| AVISITN*TRTPN*ACTFL | | | N | 12 | 900 | |
| AVISITN*TRTPN*ACTFL | | | Y | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |
| BASE*AVISITN | | | | 12 | | |



FILE: stat2h.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.8 FINAL


STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY ACTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Actiwatch<br>Usage<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |

FILE: stat2h.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.8 FINAL


 $$\operatorname{\mathtt{STAT-3.8}}$$  MMRM Output for Test on Treatment by Use of Wearable Device Interaction

(Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY ACTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Actiwatch<br>Usage<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 12 | 900 | |
| ACTFL | | | N | | | |
| ACTFL | | | Y | | | |
| AVISITN*ACTFL | | | N | 3 | | |
| AVISITN*ACTFL | | | Y | 3 | | |
| AVISITN*ACTFL | | | N | 6 | | |
| AVISITN*ACTFL | | | Y | 6 | | |
| AVISITN*ACTFL | | | N | 10 | | |
| AVISITN*ACTFL | | | Y | 10 | | |
| AVISITN*ACTFL | | | N | 12 | | |
| AVISITN*ACTFL | | | Y | 12 | | |
| TRTPN*ACTFL | | | N | | 1 | 1 |
| TRTPN*ACTFL | | | Y | | 1 | -1 |
| TRTPN*ACTFL | | | N | | 2 | -1 |
| TRTPN*ACTFL | | | Y | | 2 | 1 |
| TRTPN*ACTFL | | | N | | 3 | |
| TRTPN*ACTFL | | | Y | | 3 | |
| TRTPN*ACTFL | | | N | | 900 | |


STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

\_\_\_\_\_

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY ACTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Actiwatch<br>Usage<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*ACTFL | | | Y | | 900 | |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 1 | |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 1 | |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 2 | |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 2 | |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 3 | |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 3 | |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 900 | |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 900 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 1 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 1 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 2 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 2 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 3 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 3 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 900 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 900 | |
| AVISITN*TRTPN*ACTFL | | | N | 10 | 1 | 1 |

STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

.\_\_\_\_\_

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy W vs. Dummy X BY ACTFL AT Phase B

| (Pooled Related Usage Analysis Planned | |
|-----------------------------------------------|------|
| Center) Population Population Visit Treatment | |
| Effect for ITT Flag Flag (N) (N) | Row1 |
| AVISITN*TRTPN*ACTFL Y 10 1 | -1 |
| AVISITN TRIFIN ACTEL N 10 2 | -1 |
| | _ |
| AVISITN*TRTPN*ACTFL Y 10 2 | 1 |
| AVISITN*TRTPN*ACTFL N 10 3 | |
| AVISITN*TRTPN*ACTFL Y 10 3 | |
| AVISITN*TRTPN*ACTFL N 10 900 | |
| AVISITN*TRTPN*ACTFL Y 10 900 | |
| AVISITN*TRTPN*ACTFL N 12 1 | |
| AVISITN*TRTPN*ACTFL Y 12 1 | |
| AVISITN*TRTPN*ACTFL N 12 2 | |
| AVISITN*TRTPN*ACTFL Y 12 2 | |
| AVISITN*TRTPN*ACTFL N 12 3 | |
| AVISITN*TRTPN*ACTFL Y 12 3 | |
| AVISITN*TRTPN*ACTFL N 12 900 | |
| AVISITN*TRTPN*ACTFL Y 12 900 | |
| BASE*AVISITN 3 | |
| BASE*AVISITN 6 | |
| BASE*AVISITN 10 | |



FILE: stat2h.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.8 FINAL

BREXPIPRAZOLE 27 OF 39 PROTOCOL 331-201-00061 STAT-3.8 MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy X vs. Dummy Z BY ACTFL AT Phase B Center Combat Actiwatch (Pooled Related Usage Analysis Planned Population Population Visit Center) Treatment Effect for ITT Flag Flag (N) (N) Row1 POOLCNTR POOLCNTR POOLCNTR COMBFL N COMBFL 3 AVISITN AVISITN AVISITN 10 AVISITN 12 1 TRTPN TRTPN 2 TRTPN 900 TRTPN AVISITN\*TRTPN 3 1 AVISITN\*TRTPN 3 2

FILE: stat2h.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.8 FINAL

AVISITN\*TRTPN

AVISITN\*TRTPN

AVISITN\*TRTPN

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.

3

1

900

3


STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction

(Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY ACTFL AT Phase B

| | Center | Combat | Actiwatch | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | Usage | Analysis | Planned | |
| | Center) | Population | Population | Visit | Treatment | |
| Effect | for ITT | Flag | Flag | (N) | (N) | Row1 |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |
| AVISITN*TRTPN | | | | 12 | 900 | |
| ACTFL | | | N | | | |
| ACTFL | | | Y | | | |
| AVISITN*ACTFL | | | N | 3 | | |
| AVISITN*ACTFL | | | Y | 3 | | |
| AVISITN*ACTFL | | | N | 6 | | |
| AVISITN*ACTFL | | | Y | 6 | | |
| AVISITN*ACTFL | | | N | 10 | | |
| AVISITN*TRTPN AVISITN*TRTPN ACTFL ACTFL AVISITN*ACTFL AVISITN*ACTFL AVISITN*ACTFL AVISITN*ACTFL AVISITN*ACTFL | | | Y<br>N<br>Y<br>N<br>Y | 12<br>12<br>3<br>3<br>6<br>6 | 3 | |


STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

-----

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY ACTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Actiwatch<br>Usage<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*ACTFL | | | Y | 10 | | |
| AVISITN*ACTFL | | | N | 12 | | |
| AVISITN*ACTFL | | | Y | 12 | | |
| TRTPN*ACTFL | | | N | | 1 | |
| TRTPN*ACTFL | | | Y | | 1 | |
| TRTPN*ACTFL | | | N | | 2 | 1 |
| TRTPN*ACTFL | | | Y | | 2 | -1 |
| TRTPN*ACTFL | | | N | | 3 | |
| TRTPN*ACTFL | | | Y | | 3 | |
| TRTPN*ACTFL | | | N | | 900 | -1 |
| TRTPN*ACTFL | | | Y | | 900 | 1 |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 1 | |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 1 | |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 2 | |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 2 | |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 3 | |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 3 | |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 900 | |


STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

-----

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY ACTFL AT Phase B

| | Center | Combat | Actiwatch | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | Usage | Analysis | Planned | |
| | Center) | Population | Population | Visit | Treatment | |
| Effect | for ITT | Flag | Flag | (N) | (N) | Row1 |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 900 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 1 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 1 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 2 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 2 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 3 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 3 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 900 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 900 | |
| AVISITN*TRTPN*ACTFL | | | N | 10 | 1 | |
| AVISITN*TRTPN*ACTFL | | | Y | 10 | 1 | |
| AVISITN*TRTPN*ACTFL | | | N | 10 | 2 | 1 |
| AVISITN*TRTPN*ACTFL | | | Y | 10 | 2 | -1 |
| AVISITN*TRTPN*ACTFL | | | N | 10 | 3 | |
| AVISITN*TRTPN*ACTFL | | | Y | 10 | 3 | |
| AVISITN*TRTPN*ACTFL | | | N | 10 | 900 | -1 |
| AVISITN*TRTPN*ACTFL | | | Y | 10 | 900 | 1 |
| AVISITN*TRTPN*ACTFL | | | N | 12 | 1 | |


STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

.\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs. Dummy Z BY ACTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Actiwatch<br>Usage<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN*ACTFL | | | Υ | 12 | 1 | |
| AVISITN*TRTPN*ACTFL | | | N | 12 | 2 | |
| AVISITN*TRTPN*ACTFL | | | Y | 12 | 2 | |
| AVISITN*TRTPN*ACTFL | | | N | 12 | 3 | |
| AVISITN*TRTPN*ACTFL | | | Y | 12 | 3 | |
| AVISITN*TRTPN*ACTFL | | | N | 12 | 900 | |
| AVISITN*TRTPN*ACTFL | | | Y | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |
| BASE*AVISITN | | | | 12 | | |



FILE: stat2h.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.8 FINAL


STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

.\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY ACTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Actiwatch<br>Usage<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |


STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY ACTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Actiwatch<br>Usage<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 12 | 900 | |
| ACTFL | | | N | | | |
| ACTFL | | | Y | | | |
| AVISITN*ACTFL | | | N | 3 | | |
| AVISITN*ACTFL | | | Y | 3 | | |
| AVISITN*ACTFL | | | N | 6 | | |
| AVISITN*ACTFL | | | Y | 6 | | |
| AVISITN*ACTFL | | | N | 10 | | |
| AVISITN*ACTFL | | | Y | 10 | | |
| AVISITN*ACTFL | | | N | 12 | | |
| AVISITN*ACTFL | | | Υ | 12 | | |
| TRTPN*ACTFL | | | N | | 1 | |
| TRTPN*ACTFL | | | Y | | 1 | |
| TRTPN*ACTFL | | | N | | 2 | |
| TRTPN*ACTFL | | | Y | | 2 | |
| TRTPN*ACTFL | | | N | | 3 | 1 |
| TRTPN*ACTFL | | | Y | | 3 | -1 |
| TRTPN*ACTFL | | | N | | 900 | -1 |


STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY ACTFL AT Phase B

| | Center | Combat | Actiwatch | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | Usage | Analysis | Planned | |
| | Center) | Population | Population | Visit | Treatment | |
| Effect | for ITT | Flag | Flag | (N) | (N) | Row1 |
| | | | | | 222 | |
| TRTPN*ACTFL | | | Y | _ | 900 | 1 |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 1 | |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 1 | |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 2 | |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 2 | |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 3 | |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 3 | |
| AVISITN*TRTPN*ACTFL | | | N | 3 | 900 | |
| AVISITN*TRTPN*ACTFL | | | Y | 3 | 900 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 1 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 1 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 2 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 2 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 3 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 3 | |
| AVISITN*TRTPN*ACTFL | | | N | 6 | 900 | |
| AVISITN*TRTPN*ACTFL | | | Y | 6 | 900 | |
| AVISITN*TRTPN*ACTFL | | | N | 10 | 1 | |


 $$\tt STAT-3.8$$  MMRM Output for Test on Treatment by Use of Wearable Device Interaction

(Intent to Treat Sample)

.\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy Y vs. Dummy Z BY ACTFL AT Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Actiwatch<br>Usage<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN*ACTFL | | | Y | 10 | 1 | |
| AVISITN*TRTPN*ACTFL | | | N | 10 | 2 | |
| AVISITN*TRTPN*ACTFL | | | Y | 10 | 2 | |
| AVISITN*TRTPN*ACTFL | | | N | 10 | 3 | 1 |
| AVISITN*TRTPN*ACTFL | | | Y | 10 | 3 | -1 |
| AVISITN*TRTPN*ACTFL | | | N | 10 | 900 | -1 |
| AVISITN*TRTPN*ACTFL | | | Y | 10 | 900 | 1 |
| AVISITN*TRTPN*ACTFL | | | N | 12 | 1 | |
| AVISITN*TRTPN*ACTFL | | | Y | 12 | 1 | |
| AVISITN*TRTPN*ACTFL | | | N | 12 | 2 | |
| AVISITN*TRTPN*ACTFL | | | Y | 12 | 2 | |
| AVISITN*TRTPN*ACTFL | | | N | 12 | 3 | |
| AVISITN*TRTPN*ACTFL | | | Y | 12 | 3 | |
| AVISITN*TRTPN*ACTFL | | | N | 12 | 900 | |
| AVISITN*TRTPN*ACTFL | | | Y | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |




STAT-3.8

MMRM Output for Test on Treatment by Use of Wearable Device Interaction (Intent to Treat Sample)

-----

The Mixed Procedure

Least Squares Means

| Effect | Actiwatch<br>Usage<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN*ACTFL | N | 3 | 1 | -7.9435 | 2.1206 | 284 | -3.75 | 0.0002 | 0.05 | -12.1176 | -3.7693 |
| AVISITN*TRTPN*ACTFL | Y | 3 | 1 | -5.9863 | 1.2849 | 286 | -4.66 | <.0001 | 0.05 | -8.5154 | -3.4573 |
| AVISITN*TRTPN*ACTFL | N | 3 | 2 | -3.5042 | 2.0389 | 284 | -1.72 | 0.0868 | 0.05 | -7.5174 | 0.5090 |
| AVISITN*TRTPN*ACTFL | Y | 3 | 2 | -5.1180 | 1.4112 | 286 | -3.63 | 0.0003 | 0.05 | -7.8956 | -2.3404 |
| AVISITN*TRTPN*ACTFL | N | 3 | 3 | -5.6913 | 1.9165 | 277 | -2.97 | 0.0032 | 0.05 | -9.4641 | -1.9186 |
| AVISITN*TRTPN*ACTFL | Y | 3 | 3 | -6.4961 | 1.3592 | 284 | -4.78 | <.0001 | 0.05 | -9.1715 | -3.8208 |
| AVISITN*TRTPN*ACTFL | N | 3 | 900 | -5.4811 | 1.9443 | 279 | -2.82 | 0.0052 | 0.05 | -9.3084 | -1.6537 |
| AVISITN*TRTPN*ACTFL | Y | 3 | 900 | -6.5675 | 1.2908 | 282 | -5.09 | <.0001 | 0.05 | -9.1084 | -4.0266 |
| AVISITN*TRTPN*ACTFL | N | 6 | 1 | -11.9700 | 2.7777 | 291 | -4.31 | <.0001 | 0.05 | -17.4369 | -6.5032 |
| AVISITN*TRTPN*ACTFL | Y | 6 | 1 | -12.8305 | 1.5449 | 272 | -8.30 | <.0001 | 0.05 | -15.8720 | -9.7890 |
| AVISITN*TRTPN*ACTFL | N | 6 | 2 | -7.4242 | 2.4665 | 274 | -3.01 | 0.0029 | 0.05 | -12.2798 | -2.5685 |
| AVISITN*TRTPN*ACTFL | Y | 6 | 2 | -8.2664 | 1.7407 | 287 | -4.75 | <.0001 | 0.05 | -11.6924 | -4.8404 |
| AVISITN*TRTPN*ACTFL | N | 6 | 3 | -9.0108 | 2.4003 | 265 | -3.75 | 0.0002 | 0.05 | -13.7369 | -4.2847 |
| AVISITN*TRTPN*ACTFL | Y | 6 | 3 | -10.0441 | 1.6821 | 292 | -5.97 | <.0001 | 0.05 | -13.3547 | -6.7336 |
| AVISITN*TRTPN*ACTFL | N | 6 | 900 | -7.2664 | 2.3780 | 263 | -3.06 | 0.0025 | 0.05 | -11.9489 | -2.5840 |
| AVISITN*TRTPN*ACTFL | Y | 6 | 900 | -9.5807 | 1.5605 | 272 | -6.14 | <.0001 | 0.05 | -12.6530 | -6.5085 |
| AVISITN*TRTPN*ACTFL | N | 10 | 1 | -13.4038 | 3.0528 | 264 | -4.39 | <.0001 | 0.05 | -19.4147 | -7.3929 |
| AVISITN*TRTPN*ACTFL | Y | 10 | 1 | -17.2135 | 1.6338 | 245 | -10.54 | <.0001 | 0.05 | -20.4316 | -13.9953 |


 $$\tt STAT-3.8$$  MMRM Output for Test on Treatment by Use of Wearable Device Interaction

(Intent to Treat Sample)

The Mixed Procedure

Least Squares Means

| Effect | Actiwatch<br>Usage<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN*ACTFL | N | 10 | 2 | -10.2150 | 2.6569 | 254 | -3.84 | 0.0002 | 0.05 | -15.4473 | -4.9826 |
| AVISITN*TRTPN*ACTFL | Y | 10 | 2 | -13.1389 | 1.9171 | 279 | -6.85 | <.0001 | 0.05 | -16.9128 | -9.3650 |
| AVISITN*TRTPN*ACTFL | N | 10 | 3 | -10.7035 | 2.6193 | 247 | -4.09 | <.0001 | 0.05 | -15.8625 | -5.5445 |
| AVISITN*TRTPN*ACTFL | Y | 10 | 3 | -11.7100 | 1.7693 | 256 | -6.62 | <.0001 | 0.05 | -15.1942 | -8.2258 |
| AVISITN*TRTPN*ACTFL | N | 10 | 900 | -9.0686 | 2.6623 | 264 | -3.41 | 0.0008 | 0.05 | -14.3107 | -3.8266 |
| AVISITN*TRTPN*ACTFL | Y | 10 | 900 | -11.0841 | 1.6435 | 245 | -6.74 | <.0001 | 0.05 | -14.3214 | -7.8469 |
| AVISITN*TRTPN*ACTFL | N | 12 | 1 | -13.8921 | 3.2980 | 265 | -4.21 | <.0001 | 0.05 | -20.3857 | -7.3986 |
| AVISITN*TRTPN*ACTFL | Y | 12 | 1 | -18.1845 | 1.7699 | 254 | -10.27 | <.0001 | 0.05 | -21.6699 | -14.6990 |
| AVISITN*TRTPN*ACTFL | N | 12 | 2 | -8.4998 | 2.9027 | 263 | -2.93 | 0.0037 | 0.05 | -14.2153 | -2.7843 |
| AVISITN*TRTPN*ACTFL | Y | 12 | 2 | -14.0508 | 2.0523 | 275 | -6.85 | <.0001 | 0.05 | -18.0910 | -10.0107 |
| AVISITN*TRTPN*ACTFL | N | 12 | 3 | -11.9079 | 2.8635 | 255 | -4.16 | <.0001 | 0.05 | -17.5471 | -6.2687 |
| AVISITN*TRTPN*ACTFL | Y | 12 | 3 | -16.1860 | 1.8861 | 256 | -8.58 | <.0001 | 0.05 | -19.9002 | -12.4718 |
| AVISITN*TRTPN*ACTFL | N | 12 | 900 | -8.6752 | 2.8453 | 262 | -3.05 | 0.0025 | 0.05 | -14.2778 | -3.0727 |
| AVISITN*TRTPN*ACTFL | Y | 12 | 900 | -12.8390 | 1.7772 | 252 | -7.22 | <.0001 | 0.05 | -16.3390 | -9.3390 |

BREXPIPRAZOLE 1 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

The Mixed Procedure

Model Information

Data Set WORK.INDATA
Dependent Variable CHG
Covariance Structure Unstructured
Subject Effect SUBJID
Estimation Method REML
Residual Variance Method None

Fixed Effects SE Method Kenward-Roger Degrees of Freedom Method Kenward-Roger

Class Level Information

FILE: stat2i.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.9 FINAL

BREXPIPRAZOLE


STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure



FILE: stat2i.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.9 FINAL

BREXPIPRAZOLE 4 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

------

The Mixed Procedure



FILE: stat2i.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.9 FINAL

BREXPIPRAZOLE 5 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

-----

The Mixed Procedure



FILE: stat2i.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.9 FINAL

BREXPIPRAZOLE


STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

The Mixed Procedure

IEDURGRP 3 IEDURGRP1: <5 IEDURGRP2: >=5 -

<10 IEDURGRP3: >=10

Dimensions

Covariance Parameters 10
Columns in X 116
Columns in Z 0
Subjects 297
Max Obs per Subject 4

Number of Observations

Number of Observations Read 996
Number of Observations Used 988
Number of Observations Not Used 8

FILE: stat2i.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.9 FINAL

BREXPIPRAZOLE 7 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Iteration History

| Criterion | -2 Res Log Like | Evaluations | Iteration |
|------------|-----------------|-------------|-----------|
| | 7181.92830375 | 1 | 0 |
| 0.00081044 | 6732.11084333 | 2 | 1 |
| 0.00004736 | 6729.79975003 | 1 | 2 |
| 0.00000021 | 6729.67570335 | 1 | 3 |
| 0.00000000 | 6729.67518003 | 1 | 4 |

Convergence criteria met.

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | 77.3339 |
| UN(2,1) | SUBJID | 53.4661 |
| UN(2,2) | SUBJID | 115.65 |
| UN(3,1) | SUBJID | 42.3834 |
| UN(3,2) | SUBJID | 89.8338 |
| UN(3,3) | SUBJID | 121.60 |
| UN(4,1) | SUBJID | 46.9018 |

BREXPIPRAZOLE


STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Covariance Parameter Estimates

| Cov Parm Subj | |
|-------------------------------------------------|-----------|
| UN (4,2) SUBJ<br>UN (4,3) SUBJ<br>UN (4,4) SUBJ | ID 101.45 |

Fit Statistics

| -2 Res Log Likelihood | 6729.7 |
|--------------------------|--------|
| AIC (Smaller is Better) | 6749.7 |
| AICC (Smaller is Better) | 6749.9 |
| BIC (Smaller is Better) | 6786.6 |

Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|----|------------|------------|
| 9 | 452.25 | <.0001 |

BREXPIPRAZOLE 9 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

.....

------Parameter Code=CAPSTOT ------

The Mixed Procedure

Type 3 Tests of Fixed Effects

| Num | Den | | |
|---|---|---|---|
| DF | DF | F Value | Pr > F |
| 9 | 270 | 2.05 | 0.0345 |
| 1 | 273 | 4.81 | 0.0291 |
| 3 | 222 | 0.64 | 0.5878 |
| 3 | 258 | 2.96 | 0.0327 |
| 9 | 351 | 1.90 | 0.0511 |
| 2 | 267 | 1.39 | 0.2521 |
| 6 | 301 | 2.13 | 0.0500 |
| 6 | 260 | 1.21 | 0.2989 |
| 18 | 437 | 1.04 | 0.4164 |
| 4 | 235 | 13.86 | <.0001 |
| | DF<br>9<br>1<br>3<br>3<br>9<br>2<br>6<br>6<br>6 | DF DF 9 270 1 273 3 222 3 258 9 351 2 267 6 301 6 260 18 437 | DF DF F Value 9 270 2.05 1 273 4.81 3 222 0.64 3 258 2.96 9 351 1.90 2 267 1.39 6 301 2.13 6 260 1.21 18 437 1.04 |



FILE: stat2i.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.9 FINAL

BREXPIPRAZOLE 11 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs Dummy Z by GRP1 vs GRP2 at Phase B

| | (Pooled | Related | | Analysis | Planned | |
|---|---|---|---|---|---|---|
| | Center) | Population | | Visit | Treatment | |
| Effect | for ITT | Flag | IEDURGRP | (N) | (N) | Row1 |
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |

BREXPIPRAZOLE 12 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

-----

The Mixed Procedure

Coefficients for Dummy W vs Dummy Z by GRP1 vs GRP2 at Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | IEDURGRP | | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | | 12 | 900 | |
| IEDURGRP | | | IEDURGRP1: | <5 | | | |
| IEDURGRP | | | IEDURGRP2: | >=5 - <10 | | | |
| IEDURGRP | | | IEDURGRP3: | >=10 | | | |
| AVISITN*IEDURGRP | | | <pre>IEDURGRP1:</pre> | <5 | 3 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | 3 | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: | >=10 | 3 | | |
| AVISITN*IEDURGRP | | | IEDURGRP1: | <5 | 6 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: | | 6 | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: | >=10 | 6 | | |
| AVISITN*IEDURGRP | | | IEDURGRP1: | <5 | 10 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | 10 | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: | >=10 | 10 | | |
| AVISITN*IEDURGRP | | | IEDURGRP1: | <5 | 12 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | 12 | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: | >=10 | 12 | | |
| TRTPN*IEDURGRP | | | <pre>IEDURGRP1:</pre> | <5 | | 1 | 1 |
| TRTPN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | | 1 | -1 |

BREXPIPRAZOLE 13 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

------

The Mixed Procedure

Coefficients for Dummy W vs Dummy Z by GRP1 vs GRP2 at Phase B

| | Center | Combat | | | | | |
|---|---|---|---|---|---|---|---|
| | (Pooled | Related | | | Analysis | Planned | |
| | Center) | Population | | | Visit | Treatment | |
| Effect | for ITT | Flag | IEDURGRP | | (N) | (N) | Row1 |
| TRTPN*IEDURGRP | | | IEDURGRP3: | >=10 | | 1 | |
| TRTPN*IEDURGRP | | | <pre>IEDURGRP1:</pre> | <5 | | 2 | |
| TRTPN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | | 2 | |
| TRTPN*IEDURGRP | | | IEDURGRP3: | >=10 | | 2 | |
| TRTPN*IEDURGRP | | | IEDURGRP1: | <5 | | 3 | |
| TRTPN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | | 3 | |
| TRTPN*IEDURGRP | | | IEDURGRP3: | >=10 | | 3 | |
| TRTPN*IEDURGRP | | | IEDURGRP1: | <5 | | 900 | -1 |
| TRTPN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | | 900 | 1 |
| TRTPN*IEDURGRP | | | IEDURGRP3: | >=10 | | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 3 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 3 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 3 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 3 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 3 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 3 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 3 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 3 | 3 | |

BREXPIPRAZOLE 14 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs Dummy Z by GRP1 vs GRP2 at Phase B

| | Center<br>(Pooled | Combat<br>Related | | | Analysis | Planned | |
|---|---|---|---|---|---|---|---|
| | Center) | Population | | | Visit | Treatment | |
| Effect | for ITT | Flag | IEDURGRP | | (N) | (N) | Row1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 3 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | | 3 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | | 3 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | | 3 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | | 6 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | TEDURGRP2: | | 6 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 6 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | | 6 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | | 6 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 6 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 6 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 6 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 6 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | | 6 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 6 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 6 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 10 | 1 | 1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | | 10 | 1 | -1 |

BREXPIPRAZOLE 15 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

•

The Mixed Procedure

Coefficients for Dummy W vs Dummy Z by GRP1 vs GRP2 at Phase B

| | Center | Combat | | | | | |
|---|---|---|---|---|---|---|---|
| | (Pooled | Related | | | Analysis | Planned | |
| | Center) | Population | | | Visit | Treatment | |
| Effect | for ITT | Flag | IEDURGRP | | (N) | (N) | Row1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 10 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | <pre>IEDURGRP1:</pre> | <5 | 10 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 10 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 10 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 10 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 10 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 10 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 10 | 900 | -1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 10 | 900 | 1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 10 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 12 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 12 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 12 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 12 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 12 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 12 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 12 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 12 | 3 | |

BREXPIPRAZOLE 16 OF 48


STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction

(Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs Dummy Z by GRP1 vs GRP2 at Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | IEDURGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*TEDURGR | | | TEDURGRP3: >=10 | 12 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 12 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 - <10 | 12 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |
| BASE*AVISITN | | | | 12 | | |



FILE: stat2i.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.9 FINAL

BREXPIPRAZOLE 18 OF 48


 $$\tt STAT-3.9$$  MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Coefficients for Dummy W vs Dummy Y by GRP1 vs GRP2 at Phase B

| | (Pooled | Related | | Analysis | Planned | |
|---|---|---|---|---|---|---|
| | Center) | Population | | Visit | Treatment | |
| T C C | • | | TERMOOR | | | D . 1 |
| Effect | for ITT | Flag | IEDURGRP | (N) | (N) | Row1 |
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |

BREXPIPRAZOLE 19 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

-----

The Mixed Procedure

Coefficients for Dummy W vs Dummy Y by GRP1 vs GRP2 at Phase B

| | (Pooled | Related | | Analysis | Planned | |
|---|---|---|---|---|---|---|
| | | Population | | Visit | | |
| Effect | for ITT | Flag | IEDURGRP | (N) | (N) | Row1 |
| AVISITN*TRTPN | | | | 12 | 900 | |
| IEDURGRP | | | IEDURGRP1: <5 | | | |
| IEDURGRP | | | IEDURGRP2: >=5 - <10 | | | |
| IEDURGRP | | | IEDURGRP3: >=10 | | | |
| AVISITN*IEDURGRP | | | IEDURGRP1: <5 | 3 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: >=5 - <10 | | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: >=10 | 3 | | |
| AVISITN*IEDURGRP | | | IEDURGRP1: <5 | 6 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: >=5 - <10 | | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: >=10 | 6 | | |
| AVISITN*IEDURGRP | | | IEDURGRP1: <5 | 10 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: >=5 - <10 | 10 | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: >=10 | 10 | | |
| AVISITN*IEDURGRP | | | IEDURGRP1: <5 | 12 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: >=5 - <10 | 12 | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: >=10 | 12 | | |
| TRTPN*IEDURGRP | | | IEDURGRP1: <5 | | 1 | 1 |
| TRTPN*IEDURGRP | | | IEDURGRP2: >=5 - <10 | | 1 | -1 |

BREXPIPRAZOLE 20 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

Interaction

------

The Mixed Procedure

Coefficients for Dummy W vs Dummy Y by GRP1 vs GRP2 at Phase B

| | | Combat<br>Related<br>Population | | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | IEDURGRP | | (N) | (N) | Row1 |
| TRTPN*IEDURGRP | | | IEDURGRP3: | >=10 | | 1 | |
| TRTPN*IEDURGRP | | | IEDURGRP1: | <5 | | 2 | |
| TRTPN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | | 2 | |
| TRTPN*IEDURGRP | | | IEDURGRP3: | >=10 | | 2 | |
| TRTPN*IEDURGRP | | | IEDURGRP1: | <5 | | 3 | -1 |
| TRTPN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | | 3 | 1 |
| TRTPN*IEDURGRP | | | IEDURGRP3: | >=10 | | 3 | |
| TRTPN*IEDURGRP | | | <pre>IEDURGRP1:</pre> | <5 | | 900 | |
| TRTPN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | | 900 | |
| TRTPN*IEDURGRP | | | IEDURGRP3: | >=10 | | 900 | |
| AVISIT*TRTPN*IEDURGR | | | <pre>IEDURGRP1:</pre> | <5 | 3 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 3 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 3 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | <pre>IEDURGRP1:</pre> | <5 | 3 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 3 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 3 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | <pre>IEDURGRP1:</pre> | <5 | 3 | 3 | |

IEDURGRP2: >=5 - <10 3

FILE: stat2i.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.9 FINAL

AVISIT\*TRTPN\*IEDURGR

BREXPIPRAZOLE 21 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

\_\_\_\_\_

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Coefficients for Dummy W vs Dummy Y by GRP1 vs GRP2 at Phase B

| Effect. | | Related<br>Population<br>Flag | IEDURGRP | | Analysis<br>Visit<br>(N) | | Row1 |
|---|---|---|---|---|---|---|---|
| FILECT | 101 111 | riag | IEDURGRE | | (11) | (IV) | KOWI |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 3 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 3 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 3 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 3 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 6 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 6 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 6 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 6 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 6 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 6 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 6 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 6 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 6 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 6 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 6 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 6 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | <pre>IEDURGRP1:</pre> | <5 | 10 | 1 | 1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 10 | 1 | -1 |
BREXPIPRAZOLE 22 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs Dummy Y by GRP1 vs GRP2 at Phase B

| Effect | (Pooled | Related | IEDURGRP | | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|---|
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 10 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 10 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 10 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 10 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 10 | 3 | -1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 10 | 3 | 1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 10 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 10 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 10 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 10 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 12 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 12 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 12 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 12 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 12 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 12 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 12 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 12 | 3 | |
| | AVISIT*TRTPN*IEDURGR | Effect Center) AVISIT*TRTPN*IEDURGR | (Pooled Related Center) Population for ITT Flag AVISIT*TRTPN*IEDURGR | (Pooled Related Center) Population for ITT Flag IEDURGRP AVISIT*TRTPN*IEDURGR IEDURGRP1: AVISIT*TRTPN*IEDURGR IEDURGRP2: AVISIT*TRTPN*IEDURGR IEDURGRP3: AVISIT*TRTPN*IEDURGR IEDURGRP3: AVISIT*TRTPN*IEDURGR IEDURGRP3: AVISIT*TRTPN*IEDURGR IEDURGRP1: AVIS | (Pooled Center) Population Effect Flag IEDURGRP AVISIT*TRTPN*IEDURGR IEDURGRP1: <5 AVISIT*TRTPN*IEDURGR IEDURGRP2: >=5 - <10 AVISIT*TRTPN*IEDURGR IEDURGRP3: >=10 AVISIT*TRTPN*IEDURGR IEDURGRP3: >=10 AVISIT*TRTPN*IEDURGR IEDURGRP1: <5 AVISIT*TRTPN*IEDURGR IEDURGRP1: <5 AVISIT*TRTPN*IEDURGR IEDURGRP1: <5 AVISIT*TRTPN*IEDURGR IEDURGRP3: >=10 AVISIT*TRTPN*IEDURGR IEDURGRP1: <5 IEDURGRP1: <5 IEDURGRP1: <5 IEDURGRP1: <5 IEDURGRP3: >=10 AVISIT*TRTPN*IEDURGR IEDURGRP1: <5 IEDURGRP1: <5 | Related Center) Population Flag IEDURGRP Visit Effect Flag IEDURGRP (N) AVISIT*TRTPN*IEDURGR IEDURGRP1: <5 10 AVISIT*TRTPN*IEDURGR IEDURGRP2: >=5 - <10 10 AVISIT*TRTPN*IEDURGR IEDURGRP1: <5 12 AVISIT*TRTPN*IEDURGR IEDURGRP1: <5 12 | Related Related Center Population Flag IEDURGRP IEDURGRP Visit Treatment Visit Visit Treatment Visit Visit |

BREXPIPRAZOLE 23 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs Dummy Y by GRP1 vs GRP2 at Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | IEDURGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 12 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 12 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 - <10 | 12 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |
| BASE*AVISITN | | | | 12 | | |



FILE: stat2i.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.9 FINAL

TRTPN
TRTPN
TRTPN
AVISITN\*TRTPN

AVISITN\*TRTPN

AVISITN\*TRTPN AVISITN\*TRTPN

AVISITN\*TRTPN

AVISITN\*TRTPN

AVISITN\*TRTPN

BREXPIPRAZOLE 25 OF 48


STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)



2

3

1

900

10

10

10

12

12 12

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs Dummy X by GRP1 vs GRP2 at Phase B

| Center | Combat | | | | |
|---------|------------|----------|----------|-----------|------|
| (Pooled | Related | | Analysis | Planned | |
| Center) | Population | | Visit | Treatment | |
| for ITT | Flag | IEDURGRP | (N) | (N) | Row1 |
| | | | | 2 | |
| | | | | 3 | |
| | | | | 900 | |
| | | | 3 | 1 | |
| | | | 3 | 2 | |
| | | | 3 | 3 | |
| | | | 3 | 900 | |
| | | | 6 | 1 | |
| | | | 6 | 2 | |
| | | | 6 | 3 | |
| | | | 6 | 900 | |
| | | | 10 | 1 | |

BREXPIPRAZOLE 26 OF 48

PROTOCOL 331-201-00061 STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs Dummy X by GRP1 vs GRP2 at Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | IEDURGRP | | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | | 12 | 900 | |
| IEDURGRP | | | IEDURGRP1: | <5 | | | |
| IEDURGRP | | | IEDURGRP2: | >=5 - <10 | | | |
| IEDURGRP | | | IEDURGRP3: | >=10 | | | |
| AVISITN*IEDURGRP | | | IEDURGRP1: | <5 | 3 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | 3 | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: | >=10 | 3 | | |
| AVISITN*IEDURGRP | | | <pre>IEDURGRP1:</pre> | <5 | 6 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: | | 6 | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: | >=10 | 6 | | |
| AVISITN*IEDURGRP | | | <pre>IEDURGRP1:</pre> | <5 | 10 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | 10 | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: | >=10 | 10 | | |
| AVISITN*IEDURGRP | | | <pre>IEDURGRP1:</pre> | <5 | 12 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | 12 | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: | >=10 | 12 | | |
| TRTPN*IEDURGRP | | | <pre>IEDURGRP1:</pre> | <5 | | 1 | 1 |
| TRTPN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | | 1 | -1 |

BREXPIPRAZOLE 27 OF 48 PROTOCOL 331-201-00061

STAT-3.9

Center

Combat

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs Dummy X by GRP1 vs GRP2 at Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | IEDURGRP | | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|---|
| TRTPN*IEDURGRP | | | IEDURGRP3: | >=10 | | 1 | |
| TRTPN*IEDURGRP | | | IEDURGRP1: | <5 | | 2 | -1 |
| TRTPN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | | 2 | 1 |
| TRTPN*IEDURGRP | | | IEDURGRP3: | >=10 | | 2 | |
| TRTPN*IEDURGRP | | | IEDURGRP1: | <5 | | 3 | |
| TRTPN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | | 3 | |
| TRTPN*IEDURGRP | | | IEDURGRP3: | >=10 | | 3 | |
| TRTPN*IEDURGRP | | | IEDURGRP1: | <5 | | 900 | |
| TRTPN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | | 900 | |
| TRTPN*IEDURGRP | | | IEDURGRP3: | >=10 | | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 3 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 3 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 3 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 3 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 3 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 3 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 3 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 3 | 3 | |

BREXPIPRAZOLE 28 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

-----

The Mixed Procedure

Coefficients for Dummy W vs Dummy X by GRP1 vs GRP2 at Phase B

| | Center<br>(Pooled<br>Center) | Combat<br>Related<br>Population | | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | IEDURGRP | | (N) | (N) | Row1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 3 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 3 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 3 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 3 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 6 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 6 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 6 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | <pre>IEDURGRP1:</pre> | <5 | 6 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 6 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 6 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | <pre>IEDURGRP1:</pre> | <5 | 6 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 6 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 6 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | <pre>IEDURGRP1:</pre> | <5 | 6 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 6 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 6 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | <pre>IEDURGRP1:</pre> | <5 | 10 | 1 | 1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 10 | 1 | -1 |

BREXPIPRAZOLE 29 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs Dummy X by GRP1 vs GRP2 at Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | IEDURGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 10 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 10 | 2 | -1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 - <10 | 10 | 2 | 1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 10 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 10 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 - <10 | 10 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 10 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 10 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 - <10 | 10 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 10 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 12 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 - <10 | 12 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 12 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 12 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 - <10 | 12 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 12 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 12 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 - <10 | 12 | 3 | |

BREXPIPRAZOLE 30 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

-----

The Mixed Procedure

Coefficients for Dummy W vs Dummy X by GRP1 vs GRP2 at Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | IEDURGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 12 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 12 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 - <10 | 12 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |
| BASE*AVISITN | | | | 12 | | |



FILE: stat2i.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.9 FINAL

BREXPIPRAZOLE 32 OF 48


STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)



Planned

------

The Mixed Procedure

Coefficients for Dummy X vs Dummy Z by GRP1 vs GRP2 at Phase B

| CICHED I | LOI | Danany | 21 00 | Daning | 2 2 | 01(11 | ٧.5 | OIGL | u c | Inabe | ב | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Center | | Comba | at | | | | | | | | | |
| (Pooled | ŀ | Rela | ted | | | | | | | Anal | ysi | s |
| Center) | | Popu. | latio | n | | | | | | Visi | t | |
| C T T | - | T 2 | | т. | DDIID | TD D | | | | (37) | | |

| | Center) | Population | | Visit | Treatment | |
|---------------|---------|------------|----------|-------|-----------|------|
| Effect | for ITT | Flag | IEDURGRP | (N) | (N) | Row1 |
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |

BREXPIPRAZOLE 33 OF 48 PROTOCOL 331-201-00061

STAT-3.9

(Intent to Treat Sample)

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction

The Mixed Procedure

Coefficients for Dummy X vs Dummy Z by GRP1 vs GRP2 at Phase B

| | Center | Combat | | | | | |
|---|---|---|---|---|---|---|---|
| | (Pooled | Related | | | Analysis | Planned | |
| | Center) | Population | | | Visit | Treatment | |
| Effect | for ITT | Flag | IEDURGRP | | (N) | (N) | Row1 |
| AVISITN*TRTPN | | | | | 12 | 900 | |
| IEDURGRP | | | IEDURGRP1: | | | | |
| IEDURGRP | | | IEDURGRP2: | >=5 - <10 | | | |
| IEDURGRP | | | IEDURGRP3: | >=10 | | | |
| AVISITN*IEDURGRP | | | IEDURGRP1: | <5 | 3 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | 3 | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: | >=10 | 3 | | |
| AVISITN*IEDURGRP | | | IEDURGRP1: | <5 | 6 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | 6 | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: | >=10 | 6 | | |
| AVISITN*IEDURGRP | | | IEDURGRP1: | <5 | 10 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | 10 | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: | >=10 | 10 | | |
| AVISITN*IEDURGRP | | | IEDURGRP1: | <5 | 12 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | 12 | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: | >=10 | 12 | | |
| TRTPN*IEDURGRP | | | IEDURGRP1: | <5 | | 1 | |
| TRTPN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | | 1 | |

FILE: stat2i.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC STAT/stat2.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.9 FINAL

BREXPIPRAZOLE


STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Coefficients for Dummy X vs Dummy Z by GRP1 vs GRP2 at Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | IEDURGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*IEDURGRP | | | IEDURGRP3: >=10 | | 1 | |
| TRTPN*IEDURGRP | | | IEDURGRP1: <5 | | 2 | 1 |
| TRTPN*IEDURGRP | | | IEDURGRP2: >=5 - <10 | | 2 | -1 |
| TRTPN*IEDURGRP | | | IEDURGRP3: >=10 | | 2 | |
| TRTPN*IEDURGRP | | | IEDURGRP1: <5 | | 3 | |
| TRTPN*IEDURGRP | | | IEDURGRP2: >=5 - <10 | | 3 | |
| TRTPN*IEDURGRP | | | IEDURGRP3: >=10 | | 3 | |
| TRTPN*IEDURGRP | | | IEDURGRP1: <5 | | 900 | -1 |
| TRTPN*IEDURGRP | | | IEDURGRP2: >=5 - <10 | | 900 | 1 |
| TRTPN*IEDURGRP | | | IEDURGRP3: >=10 | | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 3 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 - <10 | 3 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 3 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 3 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 - <10 | 3 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 3 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 3 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 - <10 | 3 | 3 | |

FILE: stat2i.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.9 FINAL

BREXPIPRAZOLE 35 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

\_\_\_

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs Dummy Z by GRP1 vs GRP2 at Phase B

| 0101100 101 | Daning II vo Da | 2 2 2 01.22 | 01.12 40 | 111400 5 | |
|-------------|-----------------|-------------|----------|----------|----------|
| Center | Combat | | | | |
| (Pooled | Related | | | Analysis | Planned |
| Center) | Population | | | Visit | Treatmen |
| for ITT | Flag | IEDURGRP | | (N) | (N) |

| | Center) | Population | | | Visit | Treatment | |
|---|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | IEDURGRP | | (N) | (N) | Row1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | ) | 3 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | | 3 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 | - <10 | 3 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | ) | 3 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | | 6 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 | - <10 | 6 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | ) | 6 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | | 6 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 | - <10 | 6 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | ) | 6 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | | 6 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | <pre>IEDURGRP2: &gt;=5</pre> | - <10 | 6 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | ) | 6 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | | 6 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 | - <10 | 6 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | ) | 6 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | | 10 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 | - <10 | 10 | 1 | |

BREXPIPRAZOLE 36 OF 48

PROTOCOL 331-201-00061 STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs Dummy Z by GRP1 vs GRP2 at Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | IEDURGRP | Analysis<br>Visit<br>(N) | | Row1 |
|---|---|---|---|---|---|---|
| BIICCC | 101 111 | 1149 | IBBORORE | (14) | (11) | 110W1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 10 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 10 | 2 | 1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 - <10 | 10 | 2 | -1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 10 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 10 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 - <10 | 10 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 10 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 10 | 900 | -1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 - <10 | 10 | 900 | 1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 10 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 12 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: $>=5$ - $<10$ | 12 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 12 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 12 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: $>=5$ - $<10$ | 12 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 12 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 12 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 - <10 | 12 | 3 | |

Effect

BASE\*AVISITN BASE\*AVISITN

BASE\*AVISITN

AVISIT\*TRTPN\*IEDURGR AVISIT\*TRTPN\*IEDURGR AVISIT\*TRTPN\*IEDURGR AVISIT\*TRTPN\*IEDURGR BASE\*AVISITN

BREXPIPRAZOLE 37 OF 48


STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction

(Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy X vs Dummy Z by GRP1 vs GRP2 at Phase B

| Center<br>(Pooled<br>Center) | Combat<br>Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|
| for ITT | Flag | IEDURGRP | (N) | (N) | Row1 |
| | | IEDURGRP3: >=10 | 12 | 3 | |
| | | IEDURGRP1: <5 | 12 | 900 | |
| | | IEDURGRP2: >=5 - <1 | .0 12 | 900 | |
| | | IEDURGRP3: >=10 | 12 | 900 | |
| | | | 3 | | |

6

10

12



FILE: stat2i.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.9 FINAL

BREXPIPRAZOLE 39 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Coefficients for Dummy Y vs Dummy Z by GRP1 vs GRP2 at Phase B

| | Center | Combat | | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | | Analysis | Planned | |
| | Center) | Population | | Visit | Treatment | |
| Effect | for ITT | Flag | IEDURGRP | (N) | (N) | Row1 |
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |

FILE: stat2i.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.9 FINAL

BREXPIPRAZOLE 40 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

.\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy Y vs Dummy Z by GRP1 vs GRP2 at Phase B  $\,$ 

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | IEDURGRP | | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | .5 | 12 | 900 | |
| IEDURGRP | | | IEDURGRP1: | | | | |
| IEDURGRP | | | IEDURGRP2: | | | | |
| IEDURGRP | | | IEDURGRP3: | | | | |
| AVISITN*IEDURGRP | | | IEDURGRP1: | | 3 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: | | 3 | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: | | 3 | | |
| AVISITN*IEDURGRP | | | IEDURGRP1: | | 6 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: | | 6 | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: | >=10 | 6 | | |
| AVISITN*IEDURGRP | | | IEDURGRP1: | <5 | 10 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | 10 | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: | >=10 | 10 | | |
| AVISITN*IEDURGRP | | | IEDURGRP1: | <5 | 12 | | |
| AVISITN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | 12 | | |
| AVISITN*IEDURGRP | | | IEDURGRP3: | >=10 | 12 | | |
| TRTPN*IEDURGRP | | | IEDURGRP1: | <5 | | 1 | |
| TRTPN*IEDURGRP | | | IEDURGRP2: | >=5 - <10 | | 1 | |

BREXPIPRAZOLE 41 OF 48 PROTOCOL 331-201-00061

STAT-3.9

Center Combat

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

.\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy Y vs Dummy Z by GRP1 vs GRP2 at Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | IEDURGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| Ellect | TOT ITT | riag | IEDURGRP | (N) | (N) | ROWI |
| TRTPN*IEDURGRP | | | IEDURGRP3: >=10 | | 1 | |
| TRTPN*IEDURGRP | | | IEDURGRP1: <5 | | 2 | |
| TRTPN*IEDURGRP | | | IEDURGRP2: >=5 - <10 | | 2 | |
| TRTPN*IEDURGRP | | | IEDURGRP3: >=10 | | 2 | |
| TRTPN*IEDURGRP | | | IEDURGRP1: <5 | | 3 | 1 |
| TRTPN*IEDURGRP | | | IEDURGRP2: >=5 - <10 | | 3 | -1 |
| TRTPN*IEDURGRP | | | IEDURGRP3: >=10 | | 3 | |
| TRTPN*IEDURGRP | | | IEDURGRP1: <5 | | 900 | -1 |
| TRTPN*IEDURGRP | | | IEDURGRP2: >=5 - <10 | | 900 | 1 |
| TRTPN*IEDURGRP | | | IEDURGRP3: >=10 | | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 3 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 - <10 | 3 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 3 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 3 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 - <10 | 3 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: >=10 | 3 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: <5 | 3 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: >=5 - <10 | 3 | 3 | |

BREXPIPRAZOLE 42 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Coefficients for Dummy Y vs Dummy Z by GRP1 vs GRP2 at Phase B

| | Center | Combat | | | | | |
|---|---|---|---|---|---|---|---|
| | (Pooled | Related | | | Analysis | Planned | |
| | Center) | Population | | | Visit | Treatment | |
| Effect | for ITT | Flag | IEDURGRP | | (N) | (N) | Row1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: > | | 3 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: < | <5 | 3 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | <pre>IEDURGRP2: &gt;</pre> | >=5 - <10 | 3 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: > | >=10 | 3 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: < | <5 | 6 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: > | >=5 - <10 | 6 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: > | >=10 | 6 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: < | <5 | 6 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: > | >=5 - <10 | 6 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: > | >=10 | 6 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: < | <5 | 6 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: > | >=5 - <10 | 6 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: > | >=10 | 6 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | <pre>IEDURGRP1: &lt;</pre> | <5 | 6 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | <pre>IEDURGRP2: &gt;</pre> | >=5 - <10 | 6 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: > | >=10 | 6 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: < | <5 | 10 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: > | >=5 - <10 | 10 | 1 | |

BREXPIPRAZOLE 43 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy Y vs Dummy Z by GRP1 vs GRP2 at Phase B

| | Center<br>(Pooled<br>Center) | Combat<br>Related<br>Population | | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | IEDURGRP | | (N) | (N) | Row1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 10 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 10 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 10 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 10 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 10 | 3 | 1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 10 | 3 | -1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 10 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | <pre>IEDURGRP1:</pre> | <5 | 10 | 900 | -1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 10 | 900 | 1 |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 10 | 900 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 12 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 12 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 12 | 1 | |
| AVISIT*TRTPN*IEDURGR | | | <pre>IEDURGRP1:</pre> | <5 | 12 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 12 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP3: | >=10 | 12 | 2 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP1: | <5 | 12 | 3 | |
| AVISIT*TRTPN*IEDURGR | | | IEDURGRP2: | >=5 - <10 | 12 | 3 | |

FILE: stat2i.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.9 FINAL

BREXPIPRAZOLE 44 OF 48 PROTOCOL 331-201-00061 STAT-3.9 MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy Y vs Dummy Z by GRP1 vs GRP2 at Phase B Center Combat (Pooled Related Analysis Planned Center) Population Visit Treatment Effect for ITT Flag IEDURGRP (N) (N) Row1 AVISIT\*TRTPN\*IEDURGR IEDURGRP3: >=10 12 3 900 AVISIT\*TRTPN\*IEDURGR IEDURGRP1: <5 12 IEDURGRP2: >=5 - <10 12 900 AVISIT\*TRTPN\*IEDURGR AVISIT\*TRTPN\*IEDURGR IEDURGRP3: >=10 12 900 3 BASE\*AVISITN BASE\*AVISITN 6 BASE\*AVISITN 10 BASE\*AVISITN 12 Estimates Standard Label DF t Value Pr > |t| Estimate Error Dummy W vs Dummy Z by GRP1 vs GRP2 at Phase B 4.0987 4.8391 229 0.85 0.3979 234 Dummy W vs Dummy Y by GRP1 vs GRP2 at Phase B -4.3930 4.8986 -0.90 0.3708 Dummy W vs Dummy X by GRP1 vs GRP2 at Phase B -5.6979 4.9432 238 -1.15 0.2502

FILE: stat2i.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.9 FINAL

BREXPIPRAZOLE 45 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

## The Mixed Procedure

## Estimates

| | | Standard | | | |
|---|---|---|---|---|---|
| Label | Estimate | Error | DF | t Value | Pr > t |
| | 0 7065 | 4 6700 | 000 | 0.10 | 0 0071 |
| Dummy X vs Dummy Z by GRP1 vs GRP2 at Phase B | 9.7965 | 4.6722 | 230 | 2.10 | 0.0371 |
| Dummy Y vs Dummy Z by GRP1 vs GRP2 at Phase B | 8.4917 | 4.6296 | 227 | 1.83 | 0.0679 |
| Dummy W vs Dummy Z by GRP1 vs GRP3 at Phase B | -6.3581 | 4.5607 | 228 | -1.39 | 0.1646 |
| Dummy W vs Dummy Y by GRP1 vs GRP3 at Phase B | -7.6990 | 4.8791 | 232 | -1.58 | 0.1159 |
| Dummy W vs Dummy X by GRP1 vs GRP3 at Phase B | -5.6627 | 5.1608 | 237 | -1.10 | 0.2736 |
| Dummy X vs Dummy Z by GRP1 vs GRP3 at Phase B | -0.6954 | 5.2318 | 246 | -0.13 | 0.8944 |
| Dummy Y vs Dummy Z by GRP1 vs GRP3 at Phase B | 1.3409 | 4.9193 | 237 | 0.27 | 0.7854 |
| Dummy W vs Dummy Z by GRP2 vs GRP3 at Phase B | -10.4568 | 5.0012 | 225 | -2.09 | 0.0377 |
| Dummy W vs Dummy Y by GRP2 vs GRP3 at Phase B | -3.3060 | 5.5472 | 232 | -0.60 | 0.5518 |
| Dummy W vs Dummy X by GRP2 vs GRP3 at Phase B | 0.03516 | 5.5043 | 234 | 0.01 | 0.9949 |
| Dummy X vs Dummy Z by GRP2 vs GRP3 at Phase B | -10.4919 | 5.3725 | 238 | -1.95 | 0.0520 |
| Dummy Y vs Dummy Z by GRP2 vs GRP3 at Phase B | -7.1508 | 5.3525 | 230 | -1.34 | 0.1829 |

BREXPIPRAZOLE 46 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

\_\_\_\_\_

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Contrasts

| Num | Den | | DF | F Value | Pr > F | TRT BY IEDURGRP AT Phase B | 6 | 233 | 1.66 | 0.1326

Least Squares Means

| | | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | IEDURGRP | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISIT*TRTPN*IEDURGR | IEDURGRP1: <5 | 3 | 1 | -9.9445 | 1.7514 | 283 | -5.68 | <.0001 | 0.05 | -13.3918 | -6.4971 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP2: >=5 - <10 | 3 | 1 | -5.4672 | 2.0143 | 275 | -2.71 | 0.0071 | 0.05 | -9.4326 | -1.5018 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP3: >=10 | 3 | 1 | -3.9250 | 1.8188 | 267 | -2.16 | 0.0318 | 0.05 | -7.5060 | -0.3440 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP1: <5 | 3 | 2 | -5.7579 | 1.7681 | 280 | -3.26 | 0.0013 | 0.05 | -9.2383 | -2.2774 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP2: >=5 - <10 | 3 | 2 | -5.1226 | 1.9348 | 272 | -2.65 | 0.0086 | 0.05 | -8.9318 | -1.3134 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP3: >=10 | 3 | 2 | -1.9152 | 2.3174 | 276 | -0.83 | 0.4093 | 0.05 | -6.4771 | 2.6468 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP1: <5 | 3 | 3 | -5.3893 | 1.5461 | 276 | -3.49 | 0.0006 | 0.05 | -8.4329 | -2.3456 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP2: >=5 - <10 | 3 | 3 | -8.5774 | 1.9793 | 269 | -4.33 | <.0001 | 0.05 | -12.4743 | -4.6805 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP3: >=10 | 3 | 3 | -6.2676 | 2.3712 | 275 | -2.64 | 0.0087 | 0.05 | -10.9357 | -1.5995 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP1: <5 | 3 | 900 | -7.3896 | 1.6878 | 275 | -4.38 | <.0001 | 0.05 | -10.7123 | -4.0669 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP2: >=5 - <10 | 3 | 900 | -5.3994 | 1.9831 | 276 | -2.72 | 0.0069 | 0.05 | -9.3033 | -1.4955 |

FILE: stat2i.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.9 FINAL

BREXPIPRAZOLE 47 OF 48 PROTOCOL 331-201-00061

STAT-3.9

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Least Squares Means

| | | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | IEDURGRP | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISIT*TRTPN*IEDURGR | IEDURGRP3: >=10 | 3 | 900 | -6.1366 | 1.8423 | 269 | -3.33 | 0.0010 | 0.05 | -9.7638 | -2.5094 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP1: <5 | 6 | 1 | -13.8396 | 2.1289 | 275 | -6.50 | <.0001 | 0.05 | -18.0307 | -9.6486 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP2: >=5 - <10 | 6 | 1 | -12.7875 | 2.7147 | 286 | -4.71 | <.0001 | 0.05 | -18.1307 | -7.4442 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP3: >=10 | 6 | 1 | -12.2938 | 2.2637 | 248 | -5.43 | <.0001 | 0.05 | -16.7523 | -7.8352 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP1: <5 | 6 | 2 | -7.1646 | 2.1749 | 274 | -3.29 | 0.0011 | 0.05 | -11.4462 | -2.8830 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP2: >=5 - <10 | 6 | 2 | -8.3548 | 2.3873 | 267 | -3.50 | 0.0005 | 0.05 | -13.0552 | -3.6543 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP3: >=10 | 6 | 2 | -10.0506 | 3.0427 | 274 | -3.30 | 0.0011 | 0.05 | -16.0406 | -4.0605 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP1: <5 | 6 | 3 | -9.6547 | 1.9523 | 293 | -4.95 | <.0001 | 0.05 | -13.4970 | -5.8123 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP2: >=5 - <10 | 6 | 3 | -9.5093 | 2.5318 | 259 | -3.76 | 0.0002 | 0.05 | -14.4948 | -4.5237 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP3: >=10 | 6 | 3 | -11.3311 | 2.9232 | 256 | -3.88 | 0.0001 | 0.05 | -17.0876 | -5.5745 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP1: <5 | 6 | 900 | -9.8040 | 2.1099 | 275 | -4.65 | <.0001 | 0.05 | -13.9576 | -5.6503 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP2: >=5 - <10 | 6 | 900 | -7.0710 | 2.3580 | 248 | -3.00 | 0.0030 | 0.05 | -11.7153 | -2.4266 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP3: >=10 | 6 | 900 | -10.0749 | 2.3071 | 258 | -4.37 | <.0001 | 0.05 | -14.6181 | -5.5318 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP1: <5 | 10 | 1 | -20.3259 | 2.2844 | 257 | -8.90 | <.0001 | 0.05 | -24.8244 | -15.8274 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP2: >=5 - <10 | 10 | 1 | -15.6312 | 2.8358 | 238 | -5.51 | <.0001 | 0.05 | -21.2176 | -10.0447 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP3: >=10 | 10 | 1 | -13.7442 | 2.3302 | 212 | -5.90 | <.0001 | 0.05 | -18.3375 | -9.1509 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP1: <5 | 10 | 2 | -12.2574 | 2.3812 | 269 | -5.15 | <.0001 | 0.05 | -16.9455 | -7.5692 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP2: >=5 - <10 | 10 | 2 | -13.2605 | 2.5071 | 243 | -5.29 | <.0001 | 0.05 | -18.1989 | -8.3220 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP3: >=10 | 10 | 2 | -11.3384 | 3.3073 | 248 | -3.43 | 0.0007 | 0.05 | -17.8525 | -4.8243 |

BREXPIPRAZOLE 48 OF 48 PROTOCOL 331-201-00061

STAT-3.

MMRM Output for Test on Treatment by Years Since Index Traumatic Event Interaction (Intent to Treat Sample)

(-110010 00 12000 0000,

The Mixed Procedure

Least Squares Means

| | | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | IEDURGRP | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| HITECC | IEDONGNI | (14) | (14) | E3CIMACE | BITOI | DI | c varue | 11 > 0 | Aipiid | HOWEL | opper |
| AVISIT*TRTPN*IEDURGR | IEDURGRP1: <5 | 10 | 3 | -11.4784 | 2.0289 | 252 | -5.66 | <.0001 | 0.05 | -15.4741 | -7.4827 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP2: >=5 - <10 | 10 | 3 | -11.1766 | 2.6541 | 227 | -4.21 | <.0001 | 0.05 | -16.4065 | -5.9467 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP3: >=10 | 10 | 3 | -12.5957 | 3.1208 | 237 | -4.04 | <.0001 | 0.05 | -18.7437 | -6.4476 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP1: <5 | 10 | 900 | -13.4531 | 2.2224 | 247 | -6.05 | <.0001 | 0.05 | -17.8303 | -9.0759 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP2: >=5 - <10 | 10 | 900 | -4.6596 | 2.4634 | 224 | -1.89 | 0.0598 | 0.05 | -9.5140 | 0.1947 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP3: >=10 | 10 | 900 | -13.2295 | 2.4429 | 236 | -5.42 | <.0001 | 0.05 | -18.0421 | -8.4169 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP1: <5 | 12 | 1 | -20.0500 | 2.4640 | 257 | -8.14 | <.0001 | 0.05 | -24.9022 | -15.1978 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP2: >=5 - <10 | 12 | 1 | -18.5732 | 3.1983 | 255 | -5.81 | <.0001 | 0.05 | -24.8717 | -12.2747 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP3: >=10 | 12 | 1 | -14.4185 | 2.5562 | 220 | -5.64 | <.0001 | 0.05 | -19.4563 | -9.3806 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP1: <5 | 12 | 2 | -13.0938 | 2.5687 | 262 | -5.10 | <.0001 | 0.05 | -18.1518 | -8.0359 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP2: >=5 - <10 | 12 | 2 | -12.0585 | 2.7662 | 249 | -4.36 | <.0001 | 0.05 | -17.5067 | -6.6104 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP3: >=10 | 12 | 2 | -12.0022 | 3.6062 | 249 | -3.33 | 0.0010 | 0.05 | -19.1047 | -4.8996 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP1: <5 | 12 | 3 | -15.4052 | 2.1930 | 256 | -7.02 | <.0001 | 0.05 | -19.7238 | -11.0865 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP2: >=5 - <10 | 12 | 3 | -12.2437 | 2.9138 | 235 | -4.20 | <.0001 | 0.05 | -17.9842 | -6.5031 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP3: >=10 | 12 | 3 | -18.5335 | 3.3496 | 230 | -5.53 | <.0001 | 0.05 | -25.1334 | -11.9335 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP1: <5 | 12 | 900 | -15.7377 | 2.4310 | 254 | -6.47 | <.0001 | 0.05 | -20.5252 | -10.9502 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP2: >=5 - <10 | 12 | 900 | -5.1931 | 2.7322 | 238 | -1.90 | 0.0586 | 0.05 | -10.5755 | 0.1893 |
| AVISIT*TRTPN*IEDURGR | IEDURGRP3: >=10 | 12 | 900 | -13.6051 | 2.6073 | 230 | -5.22 | <.0001 | 0.05 | -18.7425 | -8.4677 |


STAT-3.10

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction

(Intent to Treat Sample)

The Mixed Procedure

Model Information

Data Set WORK.INDATA
Dependent Variable CHG
Covariance Structure Unstructured
Subject Effect SUBJID
Estimation Method REML

Estimation Method REML
Residual Variance Method None

Fixed Effects SE Method Kenward-Roger Degrees of Freedom Method Kenward-Roger

Class Level Information

FILE: stat2j.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.10 FINAL

FILE: stat2j.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.10 FINAL

BREXPIPRAZOLE


MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure



FILE: stat2j.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.10 FINAL


MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure



FILE: stat2j.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.10 FINAL


MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

.....

The Mixed Procedure



FILE: stat2j.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.10 FINAL

BREXPIPRAZOLE 6 OF 48 PROTOCOL 331-201-00061

 $$\tt STAT-3.10$  MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction

(Intent to Treat Sample)

The Mixed Procedure

AGEGRP2 3 AGEGRP 1: <30 AGEGRP 2: >=30 -

<40 AGEGRP 3: >=40

Dimensions

Covariance Parameters 10
Columns in X 116
Columns in Z 0
Subjects 299
Max Obs per Subject 4

Number of Observations

Number of Observations Read 996
Number of Observations Used 996
Number of Observations Not Used 0

FILE: stat2j.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.10 FINAL


STAT-3.10

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 7253.29512935 | |
| U | 1 | | |
| 1 | 2 | 6792.07841993 | 0.00034866 |
| 2 | 1 | 6791.10843333 | 0.00000952 |
| 3 | 1 | 6791.08379983 | 0.0000001 |

Convergence criteria met.

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|---|---|---|
| UN (1,1)<br>UN (2,1)<br>UN (2,2)<br>UN (3,1)<br>UN (3,2)<br>UN (3,3)<br>UN (4,1) | SUBJID<br>SUBJID<br>SUBJID<br>SUBJID<br>SUBJID<br>SUBJID | 78.6821<br>53.1196<br>111.64<br>43.6449<br>89.4337<br>125.38<br>48.5602 |
| UN(4,2) | SUBJID | 88.0055 |

BREXPIPRAZOLE


STAT-3.10

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction

(Intent to Treat Sample)

The Mixed Procedure

Covariance Parameter Estimates

Cov Parm Subject Estimate

UN(4,3) SUBJID 104.89

UN(4,4) SUBJID 146.59

Fit Statistics

-2 Res Log Likelihood 6791.1
AIC (Smaller is Better) 6811.1
AICC (Smaller is Better) 6811.3
BIC (Smaller is Better) 6848.1

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 9 462.21 <.0001


MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|----------------------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| POOLCNTR | 9 | 274 | 1.77 | 0.0748 |
| COMBFL | 1 | 274 | 4.09 | 0.0442 |
| AVISITN | 3 | 222 | 0.74 | 0.5315 |
| TRTPN | 3 | 261 | 3.57 | 0.0147 |
| AVISITN*TRTPN | 9 | 355 | 1.97 | 0.0417 |
| AGEGRP2 | 2 | 267 | 0.21 | 0.8077 |
| AVISITN*AGEGRP2 | 6 | 304 | 1.59 | 0.1492 |
| TRTPN*AGEGRP2 | 6 | 264 | 1.28 | 0.2674 |
| AVISIT*TRTPN*AGEGRP2 | 18 | 441 | 0.86 | 0.6339 |
| BASE*AVISITN | 4 | 234 | 15.42 | <.0001 |


FILE: stat2j.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.10 FINAL

BREXPIPRAZOLE 11 OF 48


MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs Dummy Z by GRP1 vs GRP2 at Phase B

| | (Pooled | Related | | Analysis<br>Visit | Planned | |
|---|---|---|---|---|---|---|
| | | Population | _ | | Treatment | |
| Effect | for ITT | Flag | AGEGRP2 | (N) | (N) | Row1 |
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |

FILE: stat2j.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.10 FINAL


STAT-3.10

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

------

The Mixed Procedure

Coefficients for Dummy W vs Dummy Z by GRP1 vs GRP2 at Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | AGEGRP2 | | sit | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 12 | | 900 | |
| AGEGRP2 | | | AGEGRP 1: <30 | | | | |
| AGEGRP2 | | | AGEGRP 2: >=30 - <4 | 40 | | | |
| AGEGRP2 | | | AGEGRP 3: >=40 | | | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 1 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <4 | 40 3 | 1 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | i | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <4 | 40 6 | i | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | i | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <4 | 40 10 | ı | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <4 | 40 12 | | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | | | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | | 1 | 1 |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <4 | 40 | | 1 | -1 |


STAT-3.10

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

------

The Mixed Procedure

Coefficients for Dummy W vs Dummy Z by GRP1 vs GRP2 at Phase B

| | Center<br>(Pooled<br>Center) | Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | AGEGRP2 | (N) | (N) | Row1 |
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 1 | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | 2 | |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | 2 | |
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 2 | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | 3 | |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | 3 | |
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 3 | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | 900 | -1 |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | 900 | 1 |
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | 3 | |


STAT-3.1

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

------

The Mixed Procedure

Coefficients for Dummy W vs Dummy Z by GRP1 vs GRP2 at Phase B

| | Center | Combat | | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | | Analysis | Planned | |
| | Center) | Population | | Visit | Treatment | |
| Effect | for ITT | Flag | AGEGRP2 | (N) | (N) | Row1 |
| | | | | 2 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | 1 | 1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | 1 | -1 |


STAT-3.1

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs Dummy Z by GRP1 vs GRP2 at Phase B

| | Center<br>(Pooled<br>Center) | Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | AGEGRP2 | (N) | (N) | Row1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | 900 | -1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | 900 | 1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | 3 | |

BREXPIPRAZOLE 16 OF 48


MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs Dummy Z by GRP1 vs GRP2 at Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | AGEGRP2 | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | 3 | |
| AVISIT^TRTPN^AGEGRPZ | | | AGEGRP 3: >=40 | | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |
| BASE*AVISITN | | | | 12 | | |



FILE: stat2j.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.10 FINAL

BREXPIPRAZOLE 18 OF 48 PROTOCOL 331-201-00061

STAT-3.1

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs Dummy Y by GRP1 vs GRP2 at Phase B

| (Pooled | Polated | | Analucic | Plannod | |
|---|---|---|---|---|---|
| | | | 4 | | |
| | | ACECDD2 | | | Row1 |
| 101 111 | riag | AGEGNE 2 | (14) | (14) | KOWI |
| | | | | 2 | |
| | | | | 3 | |
| | | | | 900 | |
| | | | 3 | 1 | |
| | | | 3 | 2 | |
| | | | 3 | 3 | |
| | | | 3 | 900 | |
| | | | 6 | 1 | |
| | | | 6 | 2 | |
| | | | 6 | 3 | |
| | | | 6 | 900 | |
| | | | 10 | 1 | |
| | | | 10 | 2 | |
| | | | 10 | 3 | |
| | | | 10 | 900 | |
| | | | 12 | 1 | |
| | | | 12 | 2 | |
| | | | 12 | 3 | |
| | Center<br>(Pooled<br>Center)<br>for ITT | (Pooled Related Center) Population | (Pooled Related<br>Center) Population | (Pooled Related Analysis Center) Population Visit for ITT Flag AGEGRP2 (N) | (Pooled Center) Related Population for ITT Analysis Treatment (N) for ITT Flag AGEGRP2 (N) (N) 2 3 900 3 1 3 2 3 3 2 3 3 3 900 6 1 6 2 6 3 6 900 10 1 10 2 10 3 10 900 12 1 12 1 12 2 1 12 2 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |

FILE: stat2j.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.10 FINAL


STAT-3.10

Combat

Center

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

------

The Mixed Procedure

Coefficients for Dummy W vs Dummy Y by GRP1 vs GRP2 at Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | AGEGRP2 | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 12 | 900 | |
| AGEGRP2 | | | AGEGRP 1: <30 | | | |
| AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | | |
| AGEGRP2 | | | AGEGRP 3: >=40 | | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | 1 | 1 |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | 1 | -1 |


MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs Dummy Y by GRP1 vs GRP2 at Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | AGEGRP2 | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 1 | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | 2 | |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | 2 | |
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 2 | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | 3 | -1 |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | 3 | 1 |
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 3 | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | 900 | |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | 900 | |
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | 3 | |


STAT-3.10

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction

(Intent to Treat Sample)

------

The Mixed Procedure

Coefficients for Dummy W vs Dummy Y by GRP1 vs GRP2 at Phase B

| | Center | Combat | | | D1 1 | |
|---|---|---|---|---|---|---|
| | (Pooled<br>Center) | Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | |
| TIGG: | , | * | 3.000000 | | | n. 1 |
| Effect | for ITT | Flag | AGEGRP2 | (N) | (N) | Row1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | 1 | 1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | 1 | -1 |


STAT-3.1

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs Dummy Y by GRP1 vs GRP2 at Phase B

| | Center<br>(Pooled | Combat<br>Related | | Analysis | Planned | |
|---|---|---|---|---|---|---|
| | Center) | Population | 0 | Visit | Treatment | |
| Effect | for ITT | Flag | AGEGRP2 | (N) | (N) | Row1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | 3 | -1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | 3 | 1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | 3 | |

BREXPIPRAZOLE 23 OF 48


STAT-3.10

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction

(Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs Dummy Y by GRP1 vs GRP2 at Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | AGEGRP2 | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |
| BASE*AVISITN | | | | 12 | | |



FILE: stat2j.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.10 FINAL

BREXPIPRAZOLE 25 OF 48 PROTOCOL 331-201-00061

STAT-3.1

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs Dummy X by GRP1 vs GRP2 at Phase B

| (Pooled | Polated | | Analysis | Plannod | |
|---|---|---|---|---|---|
| • | | | 4 | | |
| | | ACECPD2 | | | Row1 |
| 101 111 | riag | AGEGILI Z | (14) | (14) | NOWI |
| | | | | 2 | |
| | | | | 3 | |
| | | | | 900 | |
| | | | 3 | 1 | |
| | | | 3 | 2 | |
| | | | 3 | 3 | |
| | | | 3 | 900 | |
| | | | 6 | 1 | |
| | | | 6 | 2 | |
| | | | 6 | 3 | |
| | | | 6 | 900 | |
| | | | 10 | 1 | |
| | | | 10 | 2 | |
| | | | 10 | 3 | |
| | | | 10 | 900 | |
| | | | 12 | 1 | |
| | | | 12 | 2 | |
| | | | 12 | 3 | |
| | (Pooled<br>Center)<br>for ITT | (Pooled Related Center) Population | (Pooled Related<br>Center) Population | (Pooled Related Analysis Center) Population Visit for ITT Flag AGEGRP2 (N) | (Pooled Center) Related Population for ITT Analysis Treatment (N) for ITT Flag AGEGRP2 (N) (N) 2 3 900 3 1 3 2 3 3 3 2 3 3 3 3 900 6 1 6 2 6 3 6 900 10 1 10 2 10 3 10 900 10 1 10 900 10 1 10 900 12 1 12 1 12 2 1 12 2 1 12 2 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 2 1 1 |

BREXPIPRAZOLE 26 OF 48 PROTOCOL 331-201-00061

STAT-3.10

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

------

The Mixed Procedure

Coefficients for Dummy W vs Dummy X by GRP1 vs GRP2 at Phase B

Center Combat

| | Center) | Related<br>Population<br>Flag | AGEGRP2 | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | | 12 | 900 | |
| AGEGRP2 | | | AGEGRP 1: <30 | | | |
| AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | | |
| AGEGRP2 | | | AGEGRP 3: >=40 | | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | 1 | 1 |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | 1 | -1 |


STAT-3.1

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

.....

The Mixed Procedure

Coefficients for Dummy W vs Dummy X by GRP1 vs GRP2 at Phase B

| | Center | COMDAC | | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | | Analysis | Planned | |
| | Center) | Population | | Visit | Treatment | |
| Effect | for ITT | Flag | AGEGRP2 | (N) | (N) | Row1 |
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 1 | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | 2 | -1 |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | 2 | 1 |
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 2 | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | 3 | |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | 3 | |
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 3 | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | 900 | |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | 900 | |
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | 3 | |


STAT-3.1

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs Dummy X by GRP1 vs GRP2 at Phase B

| Effect | (Pooled<br>(Center)<br>for ITT | Related<br>Population<br>Flag | AGEGRP2 | Analysis<br>Visit<br>(N) | | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 2 | 3 | |
| | | | | 3 | | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | 1 | 1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | 1 | -1 |


STAT-3.10

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy W vs Dummy X by GRP1 vs GRP2 at Phase B

| | • | Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | AGEGRP2 | (N) | (N) | Row1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | 2 | -1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | 2 | 1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | 3 | |

BREXPIPRAZOLE 30 OF 48


MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy W vs Dummy X by GRP1 vs GRP2 at Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | AGEGRP2 | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| | | | | , , | , , | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |
| BASE*AVISITN | | | | 12 | | |



FILE: stat2j.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.10 FINAL

BREXPIPRAZOLE 32 OF 48


MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs Dummy Z by GRP1 vs GRP2 at Phase B

| | (Pooled<br>Center) | Related<br>Population | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | AGEGRP2 | (N) | (N) | Row1 |
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |


STAT-3.1

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy X vs Dummy Z by GRP1 vs GRP2 at Phase B

| | Center<br>(Pooled | Combat<br>Related | | Analysis | Planned | |
|---|---|---|---|---|---|---|
| | Center) | Population | | Visit | Treatment | |
| Effect | for ITT | Flag | AGEGRP2 | (N) | (N) | Row1 |
| AVISITN*TRTPN | | | | 12 | 900 | |
| AGEGRP2 | | | AGEGRP 1: <30 | 12 | 900 | |
| AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | | |
| AGEGRP2 | | | AGEGRP 3: >=40 | | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | 1 | |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | 1 | |

BREXPIPRAZOLE


STAT-3.1

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

------

The Mixed Procedure

Coefficients for Dummy X vs Dummy Z by GRP1 vs GRP2 at Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | AGEGRP2 | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 1 | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | 2 | 1 |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | 2 | -1 |
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 2 | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | 3 | |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | 3 | |
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 3 | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | 900 | -1 |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | 900 | 1 |
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | 3 | |


STAT-3.1

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

-----

The Mixed Procedure

Coefficients for Dummy X vs Dummy Z by GRP1 vs GRP2 at Phase B

| Effect. | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | AGEGRP2 | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| ETTECL | TOT ITT | riay | AGEGREZ | (1/1) | (IN) | KOMI |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | 1 | |

BREXPIPRAZOLE


STAT-3.10

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy X vs Dummy Z by GRP1 vs GRP2 at Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | AGEGRP2 | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | 2 | 1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | 2 | -1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | 900 | -1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | 900 | 1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | 3 | |

BREXPIPRAZOLE 37 OF 48


MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy X vs Dummy Z by GRP1 vs GRP2 at Phase B

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | AGEGRP2 | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | 900 | |
| BASE*AVISITN | | | | 3 | | |
| BASE*AVISITN | | | | 6 | | |
| BASE*AVISITN | | | | 10 | | |
| BASE*AVISITN | | | | 12 | | |



FILE: stat2j.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.10 FINAL

BREXPIPRAZOLE 39 OF 48


MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy Y vs Dummy Z by GRP1 vs GRP2 at Phase B

| | (Pooled | Related | | Analysis | Planned | |
|---|---|---|---|---|---|---|
| | Center) | Population | | Visit | Treatment | |
| T.C.C. | , | | 3.000000 | | | D . 1 |
| Effect | for ITT | Flag | AGEGRP2 | (N) | (N) | Row1 |
| TRTPN | | | | | 2 | |
| TRTPN | | | | | 3 | |
| TRTPN | | | | | 900 | |
| AVISITN*TRTPN | | | | 3 | 1 | |
| AVISITN*TRTPN | | | | 3 | 2 | |
| AVISITN*TRTPN | | | | 3 | 3 | |
| AVISITN*TRTPN | | | | 3 | 900 | |
| AVISITN*TRTPN | | | | 6 | 1 | |
| AVISITN*TRTPN | | | | 6 | 2 | |
| AVISITN*TRTPN | | | | 6 | 3 | |
| AVISITN*TRTPN | | | | 6 | 900 | |
| AVISITN*TRTPN | | | | 10 | 1 | |
| AVISITN*TRTPN | | | | 10 | 2 | |
| AVISITN*TRTPN | | | | 10 | 3 | |
| AVISITN*TRTPN | | | | 10 | 900 | |
| AVISITN*TRTPN | | | | 12 | 1 | |
| AVISITN*TRTPN | | | | 12 | 2 | |
| AVISITN*TRTPN | | | | 12 | 3 | |


STAT-3.10

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

------

The Mixed Procedure

Coefficients for Dummy Y vs Dummy Z by GRP1 vs GRP2 at Phase B

| | Center | Combat | | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | | Analysis | Planned | |
| | Center) | Population | | Visit | Treatment | |
| Effect | for ITT | Flag | AGEGRP2 | (N) | (N) | Row1 |
| AVISITN*TRTPN | | | | 12 | 900 | |
| AGEGRP2 | | | AGEGRP 1: <30 | | | |
| AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | | |
| AGEGRP2 | | | AGEGRP 3: >=40 | | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 6 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 6 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 6 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | | |
| AVISITN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | 1 | |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | 1 | |


STAT-3.1

Center Combat

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy Y vs Dummy Z by GRP1 vs GRP2 at Phase B

| Effect | (Pooled<br>Center)<br>for ITT | Related<br>Population<br>Flag | AGEGRP2 | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|---|
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 1 | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | 2 | |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | 2 | |
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 2 | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | 3 | 1 |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | 3 | -1 |
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 3 | |
| TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | | 900 | -1 |
| TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | | 900 | 1 |
| TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 3 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 3 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 3 | 3 | |


MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

The Mixed Procedure

Coefficients for Dummy Y vs Dummy Z by GRP1 vs GRP2 at Phase B

| Effect | <br>Combat<br>Related<br>Population<br>Flag | AGEGRP2 | Analysis<br>Visit<br>(N) | | Row1 |
|---|---|---|---|---|---|
| AVISIT*TRTPN*AGEGRP2 | | AGEGRP 3: >=40 | 3 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | AGEGRP 1: <30 | 3 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | AGEGRP 2: >=30 - <40 | - | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | AGEGRP 3: >=40 | 3 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | AGEGRP 1: <30 | 6 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | AGEGRP 2: >=30 - <40 | 6 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | AGEGRP 3: >=40 | 6 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | AGEGRP 1: <30 | 6 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | AGEGRP 2: >=30 - <40 | 6 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | AGEGRP 3: >=40 | 6 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | AGEGRP 1: <30 | 6 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | AGEGRP 2: >=30 - <40 | 6 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | AGEGRP 3: >=40 | 6 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | AGEGRP 1: <30 | 6 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | AGEGRP 2: >=30 - <40 | 6 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | AGEGRP 3: >=40 | 6 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | AGEGRP 1: <30 | 10 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | AGEGRP 2: >=30 - <40 | 10 | 1 | |


STAT-3.1

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for Dummy Y vs Dummy Z by GRP1 vs GRP2 at Phase B

| | Center | Combat | | | | |
|---|---|---|---|---|---|---|
| | (Pooled | Related | | Analysis | Planned | |
| | Center) | Population | | Visit | Treatment | |
| Effect | for ITT | Flag | AGEGRP2 | (N) | (N) | Row1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | 3 | 1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | 3 | -1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 10 | 900 | -1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 10 | 900 | 1 |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 10 | 900 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | 1 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 3: >=40 | 12 | 2 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 1: <30 | 12 | 3 | |
| AVISIT*TRTPN*AGEGRP2 | | | AGEGRP 2: >=30 - <40 | 12 | 3 | |

BREXPIPRAZOLE 44 OF 48 PROTOCOL 331-201-00061 STAT-3.10 MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample) The Mixed Procedure Coefficients for Dummy Y vs Dummy Z by GRP1 vs GRP2 at Phase B Center Combat (Pooled Related Analysis Planned Center) Population Visit Treatment Effect for ITT Flag AGEGRP2 (N) (N) Row1 AVISIT\*TRTPN\*AGEGRP2 AGEGRP 3: >=40 12 3 900 AVISIT\*TRTPN\*AGEGRP2 AGEGRP 1: <30 12 AGEGRP 2: >=30 - <40 12 900 AVISIT\*TRTPN\*AGEGRP2 AGEGRP 3: >=40 AVISIT\*TRTPN\*AGEGRP2 12 900 3 BASE\*AVISITN BASE\*AVISITN 6 BASE\*AVISITN 10 BASE\*AVISITN 12 Estimates Standard Label DF t Value Pr > |t| Estimate Error Dummy W vs Dummy Z by GRP1 vs GRP2 at Phase B -8.0993 5.5169 233 -1.47 0.1434 Dummy W vs Dummy Y by GRP1 vs GRP2 at Phase B -7.5352 5.6239 238 248 -1.34 0.1816 Dummy W vs Dummy X by GRP1 vs GRP2 at Phase B -6.7764 5.7919 -1.17 0.2431

FILE: stat2j.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.10 FINAL


STAT-3.10

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

The Mixed Procedure

## Estimates

| | | Standard | | | |
|---|---|---|---|---|---|
| Label | Estimate | Error | DF | t Value | Pr > t |
| Dummy X vs Dummy Z by GRP1 vs GRP2 at Phase B | -1.3229 | 5.9550 | 242 | -0.22 | 0.8244 |
| Dummy Y vs Dummy Z by GRP1 vs GRP2 at Phase B | -0.5641 | 5.8225 | 236 | -0.10 | 0.9229 |
| Dummy W vs Dummy Z by GRP1 vs GRP3 at Phase B | -9.7301 | 5.3417 | 228 | -1.82 | 0.0698 |
| Dummy W vs Dummy Y by GRP1 vs GRP3 at Phase B | -9.9839 | 5.2575 | 234 | -1.90 | 0.0588 |
| Dummy W vs Dummy X by GRP1 vs GRP3 at Phase B | -3.3795 | 5.5924 | 245 | -0.60 | 0.5462 |
| Dummy X vs Dummy Z by GRP1 vs GRP3 at Phase B | -6.3506 | 5.5451 | 240 | -1.15 | 0.2532 |
| Dummy Y vs Dummy Z by GRP1 vs GRP3 at Phase B | 0.2538 | 5.2474 | 235 | 0.05 | 0.9615 |
| Dummy W vs Dummy Z by GRP2 vs GRP3 at Phase B | -1.6308 | 4.4276 | 234 | -0.37 | 0.7130 |
| Dummy W vs Dummy Y by GRP2 vs GRP3 at Phase B | -2.4487 | 4.6629 | 230 | -0.53 | 0.6000 |
| Dummy W vs Dummy X by GRP2 vs GRP3 at Phase B | 3.3969 | 4.6771 | 237 | 0.73 | 0.4684 |
| Dummy X vs Dummy Z by GRP2 vs GRP3 at Phase B | -5.0277 | 4.6396 | 240 | -1.08 | 0.2796 |
| Dummy Y vs Dummy Z by GRP2 vs GRP3 at Phase B | 0.8179 | 4.6172 | 232 | 0.18 | 0.8595 |

STAT-3.10

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

.\_\_\_\_\_

The Mixed Procedure

Contrasts

Least Squares Means

| | | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | AGEGRP2 | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 1: <30 | 3 | 1 | -9.6327 | 2.2552 | 274 | -4.27 | <.0001 | 0.05 | -14.0725 | -5.1929 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 2: >=30 - <40 | 3 | 1 | -4.8803 | 1.6447 | 276 | -2.97 | 0.0033 | 0.05 | -8.1180 | -1.6427 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 3: >=40 | 3 | 1 | -6.3674 | 1.7746 | 282 | -3.59 | 0.0004 | 0.05 | -9.8606 | -2.8742 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 1: <30 | 3 | 2 | -4.0192 | 2.4594 | 273 | -1.63 | 0.1034 | 0.05 | -8.8610 | 0.8226 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 2: >=30 - <40 | 3 | 2 | -4.8855 | 1.9219 | 273 | -2.54 | 0.0116 | 0.05 | -8.6692 | -1.1019 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 3: >=40 | 3 | 2 | -4.6841 | 1.7029 | 285 | -2.75 | 0.0063 | 0.05 | -8.0360 | -1.3323 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 1: <30 | 3 | 3 | -5.9120 | 2.1981 | 281 | -2.69 | 0.0076 | 0.05 | -10.2388 | -1.5852 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 2: >=30 - <40 | 3 | 3 | -4.0711 | 2.1422 | 271 | -1.90 | 0.0584 | 0.05 | -8.2885 | 0.1463 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 3: >=40 | 3 | 3 | -7.4602 | 1.5101 | 274 | -4.94 | <.0001 | 0.05 | -10.4330 | -4.4874 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 1: <30 | 3 | 900 | -4.6844 | 2.5915 | 280 | -1.81 | 0.0717 | 0.05 | -9.7856 | 0.4169 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 2: >=30 - <40 | 3 | 900 | -5.6220 | 1.7513 | 272 | -3.21 | 0.0015 | 0.05 | -9.0699 | -2.1741 |

FILE: stat2j.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.10 FINAL


STAT-3.1

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Least Squares Means

| Effect | AGEGRP2 | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|---|
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 3: >=40 | 3 | 900 | -7.2208 | 1.5521 | 277 | -4.65 | <.0001 | 0.05 | -10.2763 | -4.1654 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 1: <30 | 6 | 1 | -16.3627 | 2.9100 | 281 | -5.62 | <.0001 | 0.05 | -22.0909 | -10.6345 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 2: >=30 - <40 | 6 | 1 | -12.8370 | 1.9778 | 251 | -6.49 | <.0001 | 0.05 | -16.7323 | -8.9418 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 3: >=40 | 6 | 1 | -10.2105 | 2.1547 | 271 | -4.74 | <.0001 | 0.05 | -14.4526 | -5.9684 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 1: <30 | 6 | 2 | -2.9996 | 3.0323 | 268 | -0.99 | 0.3234 | 0.05 | -8.9696 | 2.9705 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 2: >=30 - <40 | 6 | 2 | -10.8046 | 2.4704 | 282 | -4.37 | <.0001 | 0.05 | -15.6673 | -5.9419 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 3: >=40 | 6 | 2 | -8.3290 | 1.9954 | 265 | -4.17 | <.0001 | 0.05 | -12.2579 | -4.4001 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 1: <30 | 6 | 3 | -6.4684 | 2.8121 | 284 | -2.30 | 0.0222 | 0.05 | -12.0035 | -0.9332 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 2: >=30 - <40 | 6 | 3 | -8.7999 | 2.5819 | 248 | -3.41 | 0.0008 | 0.05 | -13.8851 | -3.7147 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 3: >=40 | 6 | 3 | -11.5405 | 1.8683 | 279 | -6.18 | <.0001 | 0.05 | -15.2182 | -7.8628 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 1: <30 | 6 | 900 | -7.3593 | 2.9847 | 244 | -2.47 | 0.0144 | 0.05 | -13.2383 | -1.4802 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 2: >=30 - <40 | 6 | 900 | -10.8294 | 2.1850 | 258 | -4.96 | <.0001 | 0.05 | -15.1320 | -6.5268 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 3: >=40 | 6 | 900 | -8.2133 | 1.8542 | 272 | -4.43 | <.0001 | 0.05 | -11.8636 | -4.5630 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 1: <30 | 10 | 1 | -20.9788 | 3.0702 | 233 | -6.83 | <.0001 | 0.05 | -27.0278 | -14.9299 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 2: >=30 - <40 | 10 | 1 | -15.8923 | 2.1973 | 236 | -7.23 | <.0001 | 0.05 | -20.2210 | -11.5635 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 3: >=40 | 10 | 1 | -14.3246 | 2.3143 | 236 | -6.19 | <.0001 | 0.05 | -18.8839 | -9.7654 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 1: <30 | 10 | 2 | -13.5275 | 3.5320 | 276 | -3.83 | 0.0002 | 0.05 | -20.4805 | -6.5745 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 2: >=30 - <40 | 10 | 2 | -15.2174 | 2.7361 | 255 | -5.56 | <.0001 | 0.05 | -20.6056 | -9.8291 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 3: >=40 | 10 | 2 | -10.2528 | 2.1766 | 245 | -4.71 | <.0001 | 0.05 | -14.5400 | -5.9656 |

FILE: stat2j.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.10 FINAL


STAT-3.1

MMRM Output for Test on Treatment by Age (<30 vs 30-40 vs >=40) Interaction (Intent to Treat Sample)

\_\_\_\_\_

The Mixed Procedure

Least Squares Means

| Effect | AGEGRP2 | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|---|
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 1: <30 | 10 | 3 | -9.0130 | 3.1252 | 255 | -2.88 | 0.0043 | 0.05 | -15.1675 | -2.8584 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 2: >=30 - <40 | 10 | 3 | -11.4616 | 2.8529 | 235 | -4.02 | <.0001 | 0.05 | -17.0822 | -5.8410 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 3: >=40 | 10 | 3 | -12.3427 | 1.9725 | 235 | -6.26 | <.0001 | 0.05 | -16.2289 | -8.4565 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 1: <30 | 10 | 900 | -7.9754 | 3.2587 | 229 | -2.45 | 0.0151 | 0.05 | -14.3963 | -1.5545 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 2: >=30 - <40 | 10 | 900 | -10.9881 | 2.4402 | 241 | -4.50 | <.0001 | 0.05 | -15.7949 | -6.1813 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 3: >=40 | 10 | 900 | -11.0513 | 1.9753 | 244 | -5.59 | <.0001 | 0.05 | -14.9421 | -7.1604 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 1: <30 | 12 | 1 | -20.7564 | 3.3785 | 245 | -6.14 | <.0001 | 0.05 | -27.4109 | -14.1018 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 2: >=30 - <40 | 12 | 1 | -18.2342 | 2.3978 | 238 | -7.60 | <.0001 | 0.05 | -22.9579 | -13.5105 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 3: >=40 | 12 | 1 | -14.2673 | 2.5224 | 246 | -5.66 | <.0001 | 0.05 | -19.2355 | -9.2991 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 1: <30 | 12 | 2 | -13.7542 | 3.8897 | 274 | -3.54 | 0.0005 | 0.05 | -21.4116 | -6.0968 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 2: >=30 - <40 | 12 | 2 | -14.2271 | 2.9780 | 255 | -4.78 | <.0001 | 0.05 | -20.0917 | -8.3626 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 3: >=40 | 12 | 2 | -10.9756 | 2.3568 | 245 | -4.66 | <.0001 | 0.05 | -15.6178 | -6.3333 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 1: <30 | 12 | 3 | -10.8895 | 3.4445 | 266 | -3.16 | 0.0018 | 0.05 | -17.6714 | -4.1076 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 2: >=30 - <40 | 12 | 3 | -14.3849 | 3.0599 | 229 | -4.70 | <.0001 | 0.05 | -20.4141 | -8.3558 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 3: >=40 | 12 | 3 | -16.7603 | 2.1294 | 239 | -7.87 | <.0001 | 0.05 | -20.9552 | -12.5654 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 1: <30 | 12 | 900 | -8.4619 | 3.6991 | 254 | -2.29 | 0.0230 | 0.05 | -15.7469 | -1.1770 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 2: >=30 - <40 | 12 | 900 | -14.0999 | 2.6556 | 243 | -5.31 | <.0001 | 0.05 | -19.3308 | -8.8690 |
| AVISIT*TRTPN*AGEGRP2 | AGEGRP 3: >=40 | 12 | 900 | -11.2824 | 2.1187 | 245 | -5.33 | <.0001 | 0.05 | -15.4556 | -7.1093 |

FILE: stat2j.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-3.10 FINAL

BREXPIPRAZOLE 1 OF 14 PROTOCOL 331-201-00061 Proc Mixed Output for Change in CAPS-5 Total Score, MMRM (UN), DDFM=KENWARDROGER (Intent to Treat Sample) The Mixed Procedure Model Information Data Set
Dependent Variable
Covariance Structure WORK.INDATA CHG Unstructured SUBJID Estimation Method REML Residual Variance Method None Fixed Effects SE Method Kenward-Roger Degrees of Freedom Method Kenward-Roger Class Level Information Class Levels Values 4 AVISITN 3 6 10 12 1 2 3 900 TRTPN 4 POOLCNTR 10 COMBFL 2 NY

SOURCE: MMRMOUT; TABLE: statlaa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.1 FINAL



SOURCE: MMRMOUT; TABLE: statlaa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.1 FINAL





SOURCE: MMRMOUT; TABLE: statlaa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.1 FINAL





SOURCE: MMRMOUT; TABLE: statlaa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.1 FINAL





SOURCE: MMRMOUT; TABLE: statlaa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.1 FINAL

BREXPIPRAZOLE 6 OF 14 PROTOCOL 331-201-00061 Proc Mixed Output for Change in CAPS-5 Total Score, MMRM (UN), DDFM=KENWARDROGER (Intent to Treat Sample) The Mixed Procedure Dimensions 10 Covariance Parameters Columns in X 41 Columns in Z Ω 299 Subjects Max Obs per Subject Number of Observations Number of Observations Read 996 Number of Observations Used 996 Number of Observations Not Used

SOURCE: MMRMOUT; TABLE: statlaa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.1 FINAL

BREXPIPRAZOLE 7 OF 14 PROTOCOL 331-201-00061 Proc Mixed Output for Change in CAPS-5 Total Score, MMRM (UN), DDFM=KENWARDROGER (Intent to Treat Sample) The Mixed Procedure Iteration History Iteration Evaluations -2 Res Log Like Criterion 0 1 7419.63261777 2 6942.08156810 0.00073594 1 6939.93600307 0.00003899 6939.83150668 3 1 0.00000014 1 6939.83114836 0.00000000 Convergence criteria met. Covariance Parameter Estimates Cov Parm Subject Estimate SUBJID 78.1269 UN(1,1) UN(2,1) SUBJID 52.5499 UN(2,2) SUBJID 113.08 UN(3,1) SUBJID 43.8955 UN(3,2) SUBJID 89.6163 UN(3,3) SUBJID 124.63 UN(4,1) SUBJID 48.3003

SOURCE: MMRMOUT; TABLE: statlaa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.1 FINAL

BREXPIPRAZOLE 8 OF 14 PROTOCOL 331-201-00061 Proc Mixed Output for Change in CAPS-5 Total Score, MMRM (UN), DDFM=KENWARDROGER (Intent to Treat Sample) The Mixed Procedure Covariance Parameter Estimates Cov Parm Subject Estimate UN(4,2) SUBJID 89.7025 UN(4,3) UN(4,4) SUBJID 105.06 SUBJID 146.78 Fit Statistics -2 Res Log Likelihood 6939.8 AIC (Smaller is Better) 6959.8 AICC (Smaller is Better) 6960.1 BIC (Smaller is Better) 6996.8 Null Model Likelihood Ratio Test Pr > ChiSq Chi-Square 479.80 <.0001

SOURCE: MMRMOUT; TABLE: statlaa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.1 FINAL

BREXPIPRAZOLE 9 OF 14 PROTOCOL 331-201-00061

> Proc Mixed Output for Change in CAPS-5 Total Score, MMRM (UN), DDFM=KENWARDROGER (Intent to Treat Sample)

## The Mixed Procedure

## Solution for Fixed Effects

| | Center<br>(Pooled<br>Center) | Combat<br>Related<br>Population | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | (N) | (N) | Estimate | Error | DF | t Value | Pr > t |
| Intercept | | | | | 3.8537 | 3.4109 | 345 | 1.13 | 0.2593 |
| AVISITN | | | 3 | | 0.6901 | 2.5973 | 250 | 0.27 | 0.7907 |
| AVISITN | | | 6 | | -0.2730 | 2.1267 | 217 | -0.13 | 0.8980 |
| AVISITN | | | 10 | | 1.0916 | 1.8901 | 214 | 0.58 | 0.5642 |
| AVISITN | | | 12 | | 0 | | | | |
| TRTPN | | | | 1 | -5.6267 | 2.1147 | 241 | -2.66 | 0.0083 |
| TRTPN | | | | 2 | -0.5710 | 2.1994 | 247 | -0.26 | 0.7954 |
| TRTPN | | | | 3 | -3.2353 | 2.1222 | 240 | -1.52 | 0.1287 |
| TRTPN | | | | 900 | 0 | | | | |
| AVISITN*TRTPN | | | 3 | 1 | 5.3923 | 2.0073 | 252 | 2.69 | 0.0077 |
| AVISITN*TRTPN | | | 3 | 2 | 2.2048 | 2.0904 | 259 | 1.05 | 0.2925 |
| AVISITN*TRTPN | | | 3 | 3 | 3.2522 | 2.0062 | 247 | 1.62 | 0.1063 |
| AVISITN*TRTPN | | | 3 | 900 | 0 | | | | |
| AVISITN*TRTPN | | | 6 | 1 | 1.8609 | 1.6533 | 223 | 1.13 | 0.2616 |
| AVISITN*TRTPN | | | 6 | 2 | 1.4711 | 1.7360 | 225 | 0.85 | 0.3977 |
| AVISITN*TRTPN | | | 6 | 3 | 2.4279 | 1.6511 | 219 | 1.47 | 0.1429 |
| AVISITN*TRTPN | | | 6 | 900 | 0 | | | | |
| AVISITN*TRTPN | | | 10 | 1 | -0.3608 | 1.4658 | 216 | -0.25 | 0.8058 |

SOURCE: MMRMOUT; TABLE: statlaa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.1 FINAL

BREXPIPRAZOLE

STAT-4.1.1
Proc Mixed Output for Change
(Intent to Treat Sample)

Parameter Code=CAPSTOT

The Mixed Procedure

# Solution for Fixed Effects

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | 10 | 2 | -1.1719 | 1.5456 | 217 | -0.76 | 0.4491 |
| AVISITN*TRTPN | | | 10 | 3 | 2.3246 | 1.4625 | 214 | 1.59 | 0.1134 |
| AVISITN*TRTPN | | | 10 | 900 | 0 | | | | |
| AVISITN*TRTPN | | | 12 | 1 | 0 | | | | |
| AVISITN*TRTPN | | | 12 | 2 | 0 | | | | |
| AVISITN*TRTPN | | | 12 | 3 | 0 | | | | |
| AVISITN*TRTPN | | | 12 | 900 | 0 | | | | |
| POOLCNTR | | | | | 0.9907 | 3.0086 | 279 | 0.33 | 0.7422 |
| POOLCNTR | | | | | -0.7991 | 2.9472 | 281 | -0.27 | 0.7865 |
| POOLCNTR | | | | | 0.1817 | 2.4770 | 281 | 0.07 | 0.9416 |
| POOLCNTR | | | | | 0.3656 | 2.2129 | 285 | 0.17 | 0.8689 |
| POOLCNTR | | | | | -1.7756 | 2.3317 | 282 | -0.76 | 0.4470 |
| POOLCNTR | | | | | -3.9197 | 2.3813 | 285 | -1.65 | 0.1009 |
| POOLCNTR | | | | | -2.3470 | 2.3914 | 285 | -0.98 | 0.3272 |
| POOLCNTR | | | | | -4.6066 | 2.4078 | 280 | -1.91 | 0.0567 |
| POOLCNTR | | | | | -3.8650 | 2.4765 | 284 | -1.56 | 0.1197 |
| POOLCNTR | | | | | 0 | | | | |
| COMBFL | | N | | | 2.4761 | 1.2332 | 282 | 2.01 | 0.0456 |

SOURCE: MMRMOUT; TABLE: statlaa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.1 FINAL

BREXPIPRAZOLE 11 OF 14 PROTOCOL 331-201-00061

STAT-4.1.1 Proc Mixed Output for Change in

in CAPS-5 Total Score, MMRM (UN), DDFM=KENWARDROGER

(Intent to Treat Sample)

------

The Mixed Procedure

Solution for Fixed Effects

| | Center<br>(Pooled<br>Center) | Combat<br>Related<br>Population | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | for ITT | Flag | (N) | (N) | Estimate | Error | DF | t Value | Pr > t |
| COMBFL | | Y | | | 0 | | | | |
| BASE*AVISITN | | | 3 | | -0.2945 | 0.04717 | 285 | -6.24 | <.0001 |
| BASE*AVISITN | | | 6 | | -0.3423 | 0.05752 | 269 | -5.95 | <.0001 |
| BASE*AVISITN | | | 10 | | -0.4252 | 0.06194 | 247 | -6.86 | <.0001 |
| BASE*AVISITN | | | 12 | | -0.4287 | 0.06757 | 250 | -6.34 | < .0001 |

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|---------------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| AVISITN | 3 | 230 | 0.80 | 0.4940 |
| TRTPN | 3 | 268 | 2.87 | 0.0370 |
| AVISITN*TRTPN | 9 | 365 | 1.91 | 0.0487 |
| POOLCNTR | 9 | 281 | 1.68 | 0.0934 |
| COMBFL | 1 | 282 | 4.03 | 0.0456 |
| BASE*AVISITN | 4 | 243 | 15.03 | <.0001 |

SOURCE: MMRMOUT; TABLE: statlaa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.1 FINAL

BREXPIPRAZOLE 12 OF 14

STAT-4.1.1

Ctandard

Proc Mixed Output for Change in CAPS-5 Total Score, MMRM (UN), DDFM=KENWARDROGER (Intent to Treat Sample)

\_\_\_\_\_

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Estimates

| | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| WEEK3 1 vs 900 | -0.2343 | 1.4361 | 280 | -0.16 | 0.8705 | 0.05 | -3.0612 | 2.5925 |
| WEEK6 1 vs 900 | -3.7658 | 1.7875 | 262 | -2.11 | 0.0361 | 0.05 | -7.2855 | -0.2460 |
| WEEK10 1 vs 900 | -5.9875 | 1.9283 | 237 | -3.10 | 0.0021 | 0.05 | -9.7864 | -2.1885 |
| WEEK12 1 vs 900 | -5.6267 | 2.1147 | 241 | -2.66 | 0.0083 | 0.05 | -9.7922 | -1.4611 |
| WEEK3 1 vs 2 | -1.8682 | 1.4949 | 282 | -1.25 | 0.2125 | 0.05 | -4.8107 | 1.0744 |
| WEEK6 1 vs 2 | -4.6659 | 1.8691 | 267 | -2.50 | 0.0131 | 0.05 | -8.3458 | -0.9859 |
| WEEK10 1 vs 2 | -4.2446 | 2.0394 | 247 | -2.08 | 0.0384 | 0.05 | -8.2614 | -0.2277 |
| WEEK12 1 vs 2 | -5.0557 | 2.2352 | 249 | -2.26 | 0.0246 | 0.05 | -9.4580 | -0.6534 |
| WEEK3 1 vs 3 | -0.2512 | 1.4560 | 281 | -0.17 | 0.8631 | 0.05 | -3.1172 | 2.6148 |
| WEEK6 1 vs 3 | -2.9583 | 1.8330 | 266 | -1.61 | 0.1077 | 0.05 | -6.5672 | 0.6507 |
| WEEK10 1 vs 3 | -5.0767 | 1.9703 | 237 | -2.58 | 0.0106 | 0.05 | -8.9582 | -1.1952 |
| WEEK12 1 vs 3 | -2.3913 | 2.1550 | 241 | -1.11 | 0.2682 | 0.05 | -6.6364 | 1.8537 |
| WEEK3 2 vs 900 | 1.6338 | 1.4809 | 280 | 1.10 | 0.2709 | 0.05 | -1.2814 | 4.5490 |
| WEEK6 2 vs 900 | 0.9001 | 1.8390 | 263 | 0.49 | 0.6249 | 0.05 | -2.7208 | 4.5211 |
| WEEK10 2 vs 900 | -1.7429 | 2.0102 | 246 | -0.87 | 0.3868 | 0.05 | -5.7022 | 2.2164 |
| WEEK12 2 vs 900 | -0.5710 | 2.1994 | 247 | -0.26 | 0.7954 | 0.05 | -4.9030 | 3.7611 |
| WEEK3 3 vs 900 | 0.01689 | 1.4412 | 279 | 0.01 | 0.9907 | 0.05 | -2.8202 | 2.8540 |
| WEEK6 3 vs 900 | -0.8075 | 1.8057 | 262 | -0.45 | 0.6551 | 0.05 | -4.3630 | 2.7481 |
| WEEK10 3 vs 900 | -0.9108 | 1.9445 | 237 | -0.47 | 0.6399 | 0.05 | -4.7416 | 2.9200 |
| WEEK12 3 vs 900 | -3.2353 | 2.1222 | 240 | -1.52 | 0.1287 | 0.05 | -7.4158 | 0.9451 |

SOURCE: MMRMOUT; TABLE: statlaa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.1 FINAL

BREXPIPRAZOLE 13 OF 14 PROTOCOL 331-201-00061

Proc Mixed Output for Change in CAPS-5 Total Score, MMRM (UN), DDFM=KENWARDROGER (Intent to Treat Sample)

The Mixed Procedure

Least Squares Means

| | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 3 | 1 | -6.4581 | 1.0908 | 290 | -5.92 | <.0001 | 0.05 | -8.6049 | -4.3112 |
| AVISITN*TRTPN | 3 | 2 | -4.5899 | 1.1749 | 291 | -3.91 | 0.0001 | 0.05 | -6.9023 | -2.2775 |
| AVISITN*TRTPN | 3 | 3 | -6.2068 | 1.1067 | 286 | -5.61 | <.0001 | 0.05 | -8.3850 | -4.0286 |
| AVISITN*TRTPN | 3 | 900 | -6.2237 | 1.0787 | 286 | -5.77 | <.0001 | 0.05 | -8.3469 | -4.1006 |
| AVISITN*TRTPN | 6 | 1 | -12.6460 | 1.3343 | 281 | -9.48 | <.0001 | 0.05 | -15.2725 | -10.0195 |
| AVISITN*TRTPN | 6 | 2 | -7.9801 | 1.4338 | 300 | -5.57 | <.0001 | 0.05 | -10.8018 | -5.1585 |
| AVISITN*TRTPN | 6 | 3 | -9.6877 | 1.3688 | 291 | -7.08 | <.0001 | 0.05 | -12.3817 | -6.9938 |
| AVISITN*TRTPN | 6 | 900 | -8.8803 | 1.3025 | 276 | -6.82 | <.0001 | 0.05 | -11.4444 | -6.3161 |
| AVISITN*TRTPN | 10 | 1 | -16.4384 | 1.4287 | 251 | -11.51 | <.0001 | 0.05 | -19.2522 | -13.6247 |
| AVISITN*TRTPN | 10 | 2 | -12.1939 | 1.5685 | 285 | -7.77 | <.0001 | 0.05 | -15.2812 | -9.1065 |
| AVISITN*TRTPN | 10 | 3 | -11.3617 | 1.4604 | 258 | -7.78 | <.0001 | 0.05 | -14.2374 | -8.4860 |
| AVISITN*TRTPN | 10 | 900 | -10.4510 | 1.3976 | 254 | -7.48 | <.0001 | 0.05 | -13.2033 | -7.6986 |
| AVISITN*TRTPN | 12 | 1 | -17.2944 | 1.5619 | 259 | -11.07 | <.0001 | 0.05 | -20.3700 | -14.2188 |
| AVISITN*TRTPN | 12 | 2 | -12.2387 | 1.7024 | 283 | -7.19 | <.0001 | 0.05 | -15.5897 | -8.8878 |
| AVISITN*TRTPN | 12 | 3 | -14.9031 | 1.5808 | 260 | -9.43 | <.0001 | 0.05 | -18.0160 | -11.7902 |
| AVISITN*TRTPN | 12 | 900 | -11.6677 | 1.5210 | 260 | -7.67 | <.0001 | 0.05 | -14.6627 | -8.6728 |

SOURCE: MMRMOUT; TABLE: statlaa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.1 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201 | -00061 | | | | | | 14 OF 14 |
|---|---|---|---|---|---|---|---|
| | Proc Mixed Output for Change | | ST<br>(Intent t | | CAPS-5 | Total Scor | e, MMRM (UN), DDFM=KENWARDROGER |
| | | | Paramete | | | | |
| | | | The Mix | ked Proce | edure | | |
| | | | Tests of | f Effect | Slices | | |
| | | | Analysis<br>Visit | Num | Den | | |
| | Effec | ct | (N) | DF | DF | F Value | Pr > F |
| | | ITN*TRTPN<br>ITN*TRTPN | 3 | 3<br>3 | 280<br>264 | 0.65<br>2.42 | 0.5864<br>0.0667 |
| | | ITN*TRTPN<br>ITN*TRTPN | 10<br>12 | 3 | 241<br>244 | 3.70<br>2.90 | 0.0123<br>0.0356 |

SOURCE: MMRMOUT; TABLE: statlaa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.1 FINAL

BREXPIPRAZOLE 1 OF 12 PROTOCOL 331-201-00061 Proc Mixed Output for Change in CAPS-5 Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Intent to Treat Sample) The Mixed Procedure Model Information Data Set
Dependent Variable
Covariance Structure WORK.INDATA CHG Unstructured SUBJID Estimation Method REML Residual Variance Method None Model-Based Fixed Effects SE Method Degrees of Freedom Method Satterthwaite Class Level Information Class Levels Values AVISITN 4 3 6 10 12 1 2 3 900 TRTPN 4 POOLCNTR 10 COMBFL 2 NY

SOURCE: MMRMOUT; TABLE: statlab.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.2 FINAL



SOURCE: MMRMOUT; TABLE: statlab.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.2 FINAL





SOURCE: MMRMOUT; TABLE: statlab.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.2 FINAL





SOURCE: MMRMOUT; TABLE: statlab.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.2 FINAL





SOURCE: MMRMOUT; TABLE: statlab.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.2 FINAL

BREXPIPRAZOLE 6 OF 12 PROTOCOL 331-201-00061 in CAPS-5 Total Score, MMRM (UN), DDFM=SATTERTHWAITE Proc Mixed Output for Change (Intent to Treat Sample) The Mixed Procedure Dimensions 10 Covariance Parameters Columns in X 41 Columns in Z Ω 299 Subjects Max Obs per Subject Number of Observations Number of Observations Read 996 Number of Observations Used 996 Number of Observations Not Used

SOURCE: MMRMOUT; TABLE: statlab.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.2 FINAL

BREXPIPRAZOLE 7 OF 12 PROTOCOL 331-201-00061 Proc Mixed Output for Change in CAPS-5 Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Intent to Treat Sample) The Mixed Procedure Iteration History Iteration Evaluations -2 Res Log Like Criterion 0 1 7419.63261777 2 6942.08156810 0.00073594 1 6939.93600307 0.00003899 6939.83150668 3 1 0.00000014 1 6939.83114836 0.00000000 Convergence criteria met. Covariance Parameter Estimates Cov Parm Subject Estimate SUBJID 78.1269 UN(1,1) UN(2,1) SUBJID 52.5499 UN(2,2) SUBJID 113.08 UN(3,1) SUBJID 43.8955 UN(3,2) SUBJID 89.6163 UN(3,3) SUBJID 124.63 UN(4,1) SUBJID 48.3003

SOURCE: MMRMOUT; TABLE: statlab.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.2 FINAL

BREXPIPRAZOLE 8 OF 12 PROTOCOL 331-201-00061 STAT-4.1.2 Proc Mixed Output for Change in CAPS-5 Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Intent to Treat Sample) The Mixed Procedure Covariance Parameter Estimates Cov Parm Subject Estimate UN(4,2) SUBJID 89.7025 UN (4,3) UN (4,4) SUBJID 105.06 SUBJID 146.78 Fit Statistics -2 Res Log Likelihood 6939.8 AIC (Smaller is Better) 6959.8 AICC (Smaller is Better) 6960.1 BIC (Smaller is Better) 6996.8 Null Model Likelihood Ratio Test Chi-Square Pr > ChiSq

479.80

<.0001

SOURCE: MMRMOUT; TABLE: statlab.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.2 FINAL

BREXPIPRAZOLE 9 OF 12 PROTOCOL 331-201-00061 in CAPS-5 Total Score, MMRM (UN), DDFM=SATTERTHWAITE Proc Mixed Output for Change (Intent to Treat Sample) The Mixed Procedure Type 3 Tests of Fixed Effects Num Den Effect DF DF F Value Pr > F AVISITN 234 0.81 0.4893 TRTPN 3 268 2.87 0.0369 AVISITN\*TRTPN 9 240 1.94 0.0469 9 POOLCNTR 281 1.72 0.0840 282 0.0433 COMBFL 1 4.12 BASE\*AVISITN 4 250 15.26 <.0001 Estimates Standard Label Estimate DF t Value Error Pr > |t| Alpha Lower Upper WEEK3 1 vs 900 -0.2343 1.4358 280 -0.16 0.8705 -3.0606 0.05 2.5919 WEEK6 1 vs 900 -3.7658 -2.11 0.0360 -7.2836 -0.2479 1.7865 262 0.05 WEEK10 1 vs 900 -5.9875 1.9265 237 -3.11 0.0021 0.05 -9.7827 -2.1922 -2.66 -1.25 -2.50 WEEK12 1 vs 900 -5.6267 2.1121 -9.7872 241 0.0082 0.05 -1.4661 282 267 WEEK3 1 vs 2 -1.8682 1.4943 0.2123 0.05 -4.8096 1.0733 WEEK6 1 vs 2 -4.6659 1.8678 0.0131 0.05 -8.3432 -0.9885 WEEK10 1 vs 2 -4.2446 2.0368 247 -2.08 0.0382 0.05 -8.2562 -0.2329

SOURCE: MMRMOUT; TABLE: statlab.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.2 FINAL

BREXPIPRAZOLE 10 OF 12 PROTOCOL 331-201-00061

Proc Mixed Output for Change in CAPS-5 Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Intent to Treat Sample)

------ Parameter Code=CAPSTOT ------

### The Mixed Procedure

#### Estimates

| | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| WEEK12 1 vs 2 | -5.0557 | 2.2318 | 249 | -2.27 | 0.0244 | 0.05 | -9.4513 | -0.6600 |
| WEEK3 1 vs 3 | -0.2512 | 1.4556 | 281 | -0.17 | 0.8631 | 0.05 | -3.1164 | 2.6140 |
| WEEK6 1 vs 3 | -2.9583 | 1.8317 | 266 | -1.62 | 0.1075 | 0.05 | -6.5647 | 0.6481 |
| WEEK10 1 vs 3 | -5.0767 | 1.9683 | 237 | -2.58 | 0.0105 | 0.05 | -8.9542 | -1.1991 |
| WEEK12 1 vs 3 | -2.3913 | 2.1524 | 241 | -1.11 | 0.2677 | 0.05 | -6.6314 | 1.8487 |
| WEEK3 2 vs 900 | 1.6338 | 1.4805 | 280 | 1.10 | 0.2707 | 0.05 | -1.2805 | 4.5481 |
| WEEK6 2 vs 900 | 0.9001 | 1.8379 | 263 | 0.49 | 0.6247 | 0.05 | -2.7188 | 4.5191 |
| WEEK10 2 vs 900 | -1.7429 | 2.0076 | 246 | -0.87 | 0.3862 | 0.05 | -5.6973 | 2.2114 |
| WEEK12 2 vs 900 | -0.5710 | 2.1963 | 247 | -0.26 | 0.7951 | 0.05 | -4.8968 | 3.7548 |
| WEEK3 3 vs 900 | 0.01689 | 1.4411 | 279 | 0.01 | 0.9907 | 0.05 | -2.8199 | 2.8536 |
| WEEK6 3 vs 900 | -0.8075 | 1.8048 | 262 | -0.45 | 0.6549 | 0.05 | -4.3611 | 2.7462 |
| WEEK10 3 vs 900 | -0.9108 | 1.9427 | 237 | -0.47 | 0.6396 | 0.05 | -4.7378 | 2.9163 |
| WEEK12 3 vs 900 | -3.2353 | 2.1199 | 240 | -1.53 | 0.1283 | 0.05 | -7.4112 | 0.9406 |

SOURCE: MMRMOUT; TABLE: statlab.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.2 FINAL

BREXPIPRAZOLE 11 OF 12 PROTOCOL 331-201-00061

Proc Mixed Output for Change in CAPS-5 Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Intent to Treat Sample)

The Mixed Procedure

Least Squares Means

| | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 3 | 1 | -6.4581 | 1.0890 | 290 | -5.93 | <.0001 | 0.05 | -8.6014 | -4.3147 |
| AVISITN*TRTPN | 3 | 2 | -4.5899 | 1.1726 | 291 | -3.91 | 0.0001 | 0.05 | -6.8978 | -2.2821 |
| AVISITN*TRTPN | 3 | 3 | -6.2068 | 1.1049 | 286 | -5.62 | <.0001 | 0.05 | -8.3816 | -4.0321 |
| AVISITN*TRTPN | 3 | 900 | -6.2237 | 1.0770 | 286 | -5.78 | <.0001 | 0.05 | -8.3436 | -4.1038 |
| AVISITN*TRTPN | 6 | 1 | -12.6460 | 1.3324 | 281 | -9.49 | <.0001 | 0.05 | -15.2687 | -10.0233 |
| AVISITN*TRTPN | 6 | 2 | -7.9801 | 1.4312 | 300 | -5.58 | <.0001 | 0.05 | -10.7966 | -5.1637 |
| AVISITN*TRTPN | 6 | 3 | -9.6877 | 1.3666 | 291 | -7.09 | <.0001 | 0.05 | -12.3774 | -6.9981 |
| AVISITN*TRTPN | 6 | 900 | -8.8803 | 1.3008 | 276 | -6.83 | <.0001 | 0.05 | -11.4410 | -6.3195 |
| AVISITN*TRTPN | 10 | 1 | -16.4384 | 1.4264 | 251 | -11.52 | <.0001 | 0.05 | -19.2476 | -13.6293 |
| AVISITN*TRTPN | 10 | 2 | -12.1939 | 1.5647 | 285 | -7.79 | <.0001 | 0.05 | -15.2737 | -9.1140 |
| AVISITN*TRTPN | 10 | 3 | -11.3617 | 1.4578 | 258 | -7.79 | <.0001 | 0.05 | -14.2324 | -8.4910 |
| AVISITN*TRTPN | 10 | 900 | -10.4510 | 1.3952 | 254 | -7.49 | <.0001 | 0.05 | -13.1986 | -7.7033 |
| AVISITN*TRTPN | 12 | 1 | -17.2944 | 1.5590 | 259 | -11.09 | <.0001 | 0.05 | -20.3644 | -14.2244 |
| AVISITN*TRTPN | 12 | 2 | -12.2387 | 1.6982 | 283 | -7.21 | <.0001 | 0.05 | -15.5815 | -8.8959 |
| AVISITN*TRTPN | 12 | 3 | -14.9031 | 1.5781 | 260 | -9.44 | <.0001 | 0.05 | -18.0107 | -11.7955 |
| AVISITN*TRTPN | 12 | 900 | -11.6677 | 1.5183 | 260 | -7.68 | <.0001 | 0.05 | -14.6574 | -8.6781 |

SOURCE: MMRMOUT; TABLE: statlab.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.2 FINAL

BREXPIPRAZOLE

12 OF 12

PROTOCOL 331-201-00061 Proc Mixed Output for Change in CAPS-5 Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Intent to Treat Sample) The Mixed Procedure

Tests of Effect Slices

Analmaia

| | Allalysis | | | | |
|---------------|-----------|-----|-----|---------|--------|
| | Visit | Num | Den | | |
| Effect | (N) | DF | DF | F Value | Pr > F |
| AVISITN*TRTPN | 3 | 3 | 280 | 0.65 | 0.5861 |
| AVISITN*TRTPN | 6 | 3 | 264 | 2.42 | 0.0664 |
| AVISITN*TRTPN | 10 | 3 | 241 | 3.71 | 0.0122 |
| AVISITN*TRTPN | 12 | 3 | 244 | 2.91 | 0.0353 |

SOURCE: MMRMOUT; TABLE: statlab.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.1.2 FINAL

| BREXPIPRAZOLE<br>PROTOCOL 331-201-00061 | Proc GLM Output for Change | STAT-4.2 (Intent to Treat Sample) | 1 OF 6 in CAPS-5 Total Score, LOCF |
|---|---|---|---|
| | Parameter Co | ode=CAPSTOT Analysis Visit | (N) = 10 |
| | | The GLM Procedure | |
| | C. | lass Level Information | |
| | Class Levels | Values | |
| | TRTPN 4 | 1 2 3 900 | |
| | POOLCNTR 10 | | |
| | COMBFL 2 | N Y | |
| | | | 307<br>307 |

SOURCE: GLMOUT; TABLE: statlb.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.2 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | 2 OF 6 |
|---|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | Proc GLM Output for Change | | STAT-4.2 | in | n CAPS-5 Tot | al Score, LOCF | |
| | | | tent to Treat S | | | · | |
| | F | arameter Cod | e=CAPSTOT Analy | sis Visit (N)=10 | ) | | |
| | | | The GLM Procedu | re | | | |
| | De | pendent Vari | able: CHG Cha | nge from Baselin | ne | | |
| | | | Sum of | | | | |
| | Source | DF | Squares | Mean Square | F Value | Pr > F | |
| | Model | 14 | 9591.13489 | 685.08106 | 5.67 | <.0001 | |
| | Error | 292 | 35268.22668 | 120.78160 | | | |
| | Corrected Total | 306 | 44859.36156 | | | | |
| | R-Sc | uare Coe | ff Var Roo | t MSE CHG M | lean | | |
| | 0.21 | 3805 -10 | 0.3256 10. | 99007 -10.95 | 5440 | | |
| | Source | DF | Type III SS | Mean Square | F Value | Pr > F | |
| | TRTPN<br>POOLCNTR<br>COMBFL | 3<br>9<br>1 | 1146.283220<br>2023.768218<br>4.280406 | 382.094407<br>224.863135<br>4.280406 | 3.16<br>1.86<br>0.04 | 0.0249<br>0.0574<br>0.8508 | |
| | BASE | 1 | 5480.115400 | 5480.115400 | 45.37 | <.0001 | |

SOURCE: GLMOUT; TABLE: statlb.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.2 FINAL

BREXPIPRAZOLE

Proc GLM Output for Change in CAPS-5 Total Score, LOCF

\_\_\_\_\_

## The GLM Procedure

| Level of | | CHC | G | BASE | |
|----------|----|-------------|------------|------------|------------|
| TRTPN | N | Mean | Std Dev | Mean | Std Dev |
| 1 | 78 | -14.0641026 | 13.3039783 | 35.6410256 | 11.4551348 |
| 2 | 72 | -10.0416667 | 11.5300434 | 34.1805556 | 13.2157891 |
| 3 | 77 | -10.4285714 | 11.0005126 | 36.7662338 | 10.2017750 |
| 900 | 80 | -9.2500000 | 12.0793788 | 35.2625000 | 10.5826987 |

SOURCE: GLMOUT; TABLE: statlb.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.2 FINAL

| BREXPIPRAZOLE | | | | | | 4 OF 6 |
|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | | | STAT-4.2 | | | |
| | Proc GLM Output for Cha | | | | in CAPS-5 Total Score, | LOCF |
| | | (Inte | ent to Treat Sam | ple) | | |
| | | - Parameter Code= | -CAPSTOT Analysi | s Visit (N)= | 10 | |
| | | | - | | | |
| | | | ne GLM Procedure<br>Ast Squares Mear | | | |
| | | пес | isc squares mean | | | |
| | | | Standard | | LSMEAN | |
| | TRTPN | CHG LSMEAN | Error | Pr > t | Number | |
| | 1 | -14.2497820 | 1.3315680 | <.0001 | 1 | |
| | 2 | -10.7317336 | 1.4251581 | <.0001 | 2 | |
| | 3 | -9.8128458 | 1.3613721 | <.0001 | 3 | |
| | 900 | -9.3462805 | 1.3329065 | <.0001 | 4 | |
| | | T | | C | | |
| | | | res Means for ef<br>or HO: LSMean(i) | | | |
| | | Dener | ndent Variable: | CHC | | |
| | | Deper | ident variable. | CIIG | | |
| | i/j | 1 | 2 | 3 | 4 | |
| | 1 | | 0.0526 | 0.0131 | 0.0055 | |
| | 2 | 0.0526 | | 0.6138 | 0.4402 | |
| | 3 | 0.0131 | 0.6138 | | 0.7912 | |
| | 4 | 0.0055 | 0.4402 | 0.7912 | | |

SOURCE: GLMOUT; TABLE: statlb.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.2 FINAL

BREXPIPRAZOLE 5 OF 6 PROTOCOL 331-201-00061 in CAPS-5 Total Score, LOCF Proc GLM Output for Change (Intent to Treat Sample) ------ Parameter Code=CAPSTOT Analysis Visit (N)=10 ------The GLM Procedure Least Squares Means TRTPN CHG LSMEAN 95% Confidence Limits -14.249782 1 -16.870469 -11.629095 -13.536618 -7.926849 -12.492191 -7.133500 2 -10.731734 -9.812846 900 -9.346281 -11.969602 -6.722959 Least Squares Means for Effect TRTPN Difference Between 95% Confidence Limits for i j Means LSMean(i)-LSMean(j) 2 -3.518048 -7.076422 0.040325 -4.436936 -7.934242 -0.939630 -8.352735 -1.454268 1 4 -4.903501 2 3 -4.498991 2.661216 -0.918888 -1.385453 -4.912988 2.142082 2 4 3 -0.466565 -3.931224 2.998093

NOTE: To ensure overall protection level, only probabilities associated with pre-planned comparisons should be used.

SOURCE: GLMOUT; TABLE: statlb.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.2 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | Proc GLM Output for Change | STAT- | | in CAPS | -5 Total Score, | 6 OF 6 |
|---|---|---|---|---|---|---|
| | | The GLM Properties of the The GLM Properties of the The GLM Properties of the The T | ocedure | | | |
| | Parameter | Estimate | Standard<br>Error | t Value | Pr > t | |
| | 1 vs 900<br>1 vs 3<br>1 vs 2<br>2 vs 900<br>3 vs 900 | -4.90350146<br>-4.43693620<br>-3.51804843<br>-1.38545304<br>-0.46656526 | 1.75255116<br>1.77697680<br>1.80800508<br>1.79233627<br>1.76038849 | -2.80<br>-2.50<br>-1.95<br>-0.77<br>-0.27 | 0.0055<br>0.0131<br>0.0526<br>0.4402<br>0.7912 | |

SOURCE: GLMOUT; TABLE: statlb.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.2 FINAL

BREXPIPRAZOLE 1 OF 6 PROTOCOL 331-201-00061 STAT-4.3 Proc GLM Output for Change in CAPS-5 Total Score, OC (Intent to Treat Sample) The GLM Procedure Class Level Information Levels Values Class TRTPN 4 1 2 3 900 Number of Observations Read 307 Number of Observations Used 307

SOURCE: GLMOUT; TABLE: stat1c.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.3 FINAL
|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | tal Score, OC | | | | | |
| | Pa | rameter Cod | de=CAPSTOT Analys | sis Visit (N)=10 | | |
| | | | The GLM Procedu | re | | |
| | Dep | endent Vari | able: CHG Char | nge from Baselin | e | |
| | Source | DF | Sum of<br>Squares | Mean Square | F Value | Pr > F |
| | Model | 4 | 7566.86549 | 1891.71637 | 15.32 | <.0001 |
| | Error | 302 | 37292.49607 | 123.48509 | | |
| | Corrected Total | 306 | 44859.36156 | | | |
| | R-Squ | are Coe | eff Var Root | t MSE CHG M | lean | |
| | 0.168 | 680 -10 | )1.4422 11.3 | 11238 -10.95 | 440 | |
| | Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| | TRTPN<br>BASE | 3<br>1 | 1027.098016<br>6498.915555 | 342.366005<br>6498.915555 | 2.77<br>52.63 | 0.0417 |

BREXPIPRAZOLE 3 OF 6 PROTOCOL 331-201-00061 Proc GLM Output for Change in CAPS-5 Total Score, OC (Intent to Treat Sample) The GLM Procedure Level of -----CHG----------BASE-----Std Dev Mean Std Dev TRTPN N Mean -14.0641026 13.3039783 -10.0416667 11.5300434 -10.4285714 11.0005126 -9.2500000 12.0793788 35.6410256 11.4551348 78 1 34.1805556 36.7662338 13.2157891 2 72 77 10.2017750 900 80 35.2625000 10.5826987

SOURCE: GLMOUT; TABLE: stat1c.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.3 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | 4 OF 6 |
|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | | | STAT-4.3 | | | |
| | Proc GLM Output for Ch | | ent to Treat Sam | | in CAPS-5 Total Score, O | С |
| | | - Parameter Code= | -CAPSTOT Analysi | s Visit (N)=1 | .0 | |
| | | | ne GLM Procedure<br>ast Squares Mear | | | |
| | | | Standard | | LSMEAN | |
| | TRTPN | CHG LSMEAN | Error | Pr > t | Number | |
| | 1 | -13.9994374 | 1.2582613 | <.0001 | 1 | |
| | 2 | -10.5711945 | 1.3116396 | <.0001 | 2 | |
| | 3 | -9.9061147 | 1.2684199 | <.0001 | 3 | |
| | 900 | -9.3393381 | 1.2424634 | <.0001 | 4 | |
| | | | res Means for ef<br>or H0: LSMean(i) | | | |
| | | Depen | ndent Variable: | CHG | | |
| | i/j | 1 | 2 | 3 | 4 | |
| | 1<br>2 | 0.0603 | 0.0603 | 0.0226<br>0.7162 | 0.0088<br>0.4957 | |
| | 3 | 0.0226 | 0.7162 | 0.7102 | 0.7499 | |
| | 4 | 0.0088 | 0.4957 | 0.7499 | - · · · | |

BREXPIPRAZOLE 5 OF 6 PROTOCOL 331-201-00061 STAT-4.3 in CAPS-5 Total Score, OC Proc GLM Output for Change (Intent to Treat Sample) The GLM Procedure Least Squares Means TRTPN CHG LSMEAN 95% Confidence Limits 1 -13.999437 -16.475507 -11.523367 -7.990084 -7.410054 2 -10.571194 -13.152305 -9.906115 -12.402175 900 -9.339338 -11.784320 -6.894356 Least Squares Means for Effect TRTPN Difference Between 95% Confidence Limits for i j Means LSMean(i)-LSMean(j) 2 -3.428243 -7.005685 0.149199 -4.093323 -7.608471 -0.578174 -8.140000 -1.180199 1 4 -4.660099 2 3 -0.665080 -4.261350 2.931190 -1.231856 -4.786164 2.322452 2 4 3 4 -0.566777 -4.061790 2.928237

NOTE: To ensure overall protection level, only probabilities associated with pre-planned comparisons should be used.

SOURCE: GLMOUT; TABLE: stat1c.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.3 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | Proc GLM Output for Change | STAT- | | in CAF | S-5 Total Score, | 6 OF 6 |
|---|---|---|---|---|---|---|
| | Par | rameter Code=CAPSTOT in | - | (N)=10 | | |
| | Depe | endent Variable: CHG | Change from B | Baseline | | |
| | Parameter | Estimate | Standard<br>Error | t Value | Pr > t | |
| | 1 vs 900<br>1 vs 3<br>1 vs 2<br>2 vs 900<br>3 vs 900 | -4.66009920<br>-4.09332267<br>-3.42824286<br>-1.23185635<br>-0.56677654 | 1.76837676<br>1.78628851<br>1.81794426<br>1.80618824<br>1.77605684 | -2.64<br>-2.29<br>-1.89<br>-0.68<br>-0.32 | 0.0088<br>0.0226<br>0.0603<br>0.4957<br>0.7499 | |

BREXPIPRAZOLE 1 OF 2 PROTOCOL 331-201-00061 Proc GLM Output for Treatment by Center Interaction in CAPS-5 Total Score, LOCF (Intent to Treat Sa The GLM Procedure Class Level Information Class Levels Values TRTPN 4 1 2 3 900 POOLCNTR 10 2 COMBFL NY Number of Observations Read 307 Number of Observations Used

SOURCE: GLMCNTR; TABLE: stat1d.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.4 FINAL

BREXPIPRAZOLE 2 OF 2 PROTOCOL 331-201-00061

STAT-4.4

Proc GLM Output for Treatment by Center Interaction in CAPS-5 Total Score, LOCF (Intent to Treat Sa

The GLM Procedure

Dependent Variable: CHG Change from Baseline

Sum of

| Source | | DF | Squar | es Mear | Square | F Value | Pr > F |
|---|---|---|---|---|---|---|---|
| Model | | 41 | 11141.848 | 74 27 | 71.75241 | 2.14 | 0.0002 |
| Error | | 265 | 33717.512 | 82 12 | 27.23590 | | |
| Corrected Total | | 306 | 44859.361 | 56 | | | |
| | R-Square | Coei | f Var | Root MSE | CHG Me | ean | |
| | 0.248373 | -102 | .9713 | 11.27989 | -10.954 | 140 | |
| Source | | DF | Type III | SS Mear | n Square | F Value | Pr > F |
| TRTPN<br>POOLCNTR | | 3<br>9 | 972.1076<br>1863.9265 | | 1.035883 | 2.55<br>1.63 | 0.0564<br>0.1073 |
| TRTPN*POOLCNTR | | 27 | 1550.7138 | | 7.433847 | 0.45 | 0.9922 |
| COMBFL | | 1 | 13.7061 | 00 13 | 3.706100 | 0.11 | 0.7430 |

1 5385.659316 5385.659316 42.33 <.0001

SOURCE: GLMCNTR; TABLE: stat1d.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.4 FINAL

BASE

BREXPIPRAZOLE 1 OF 3

STAT-4.5.1

Summary of Mean Change in CAPS-5 Total Score
By Center - LOCF (Intent to Treat Sample)

CAPS-5 TOTAL SCORE BREX SERT TREATMENT N LS MEAN (SE) N LS MEAN (SE) N LS MEAN (SE) COMPARISON LS MEAN DIFFERENCE<sup>1</sup> CENTER N LS MEAN (SE) OVERALL 78 -14.2 (1.33) 72 -10.7 (1.43) 77 -9.81 (1.36) 80 -9.35 (1.33) BREX+SERT VS. BREX -3.52 (-7.08, 0.04) BREX+SERT VS. SERT -4.44 (-7.93, -0.94) BREX+SERT VS. PLACEBO -4.90 (-8.35, -1.45) BREX VS. PLACEBO -1.39 (-4.91, 2.14) SERT VS. PLACEBO -0.47 (-3.93, 3.00) 3 -10.8 (6.52) BREX+SERT VS. BREX 5.60 (-11.4, 22.60) BREX+SERT VS. SERT -4.37 (-21.3, 12.61) 4 -8.36 (5.65) 3 -14.0 (6.52) 3 -4.00 (6.52) BREX+SERT VS. PLACEBO 2.43 (-14.5, 19.40) BREX VS. PLACEBO -3.17 (-21.3, 14.98) SERT VS. PLACEBO 6.79 (-11.3, 24.93) 4 -15.0 (5.66) 4 -4.30 (5.66) 3 -9.06 (6.52) 4 -10.6 (5.66) BREX+SERT VS. BREX -10.7 (-26.4, 5.05) BREX+SERT VS. SERT -5.89 (-22.9, 11.07) BREX+SERT VS. PLACEBO -4.35 (-20.1, 11.35) BREX VS. PLACEBO 6.30 (-9.40, 22.01) SERT VS. PLACEBO 1.54 (-15.4, 18.51) 7 -12.1 (4.34) 8 -10.8 (4.04) 7 -15.9 (4.33) 7 -8.01 (4.30) BREX+SERT VS. BREX -1.28 (-12.8, 10.23) BREX+SERT VS. SERT 3.82 (-8.05, 15.69) BREX+SERT VS. PLACEBO -4.08 (-16.0, 7.84) BREX VS. PLACEBO -2.80 (-14.3, 8.70) -7.90 (-19.8, 4.01) SERT VS. PLACEBO 14 -12.3 (3.12) 13 -8.20 (3.22) 16 -6.02 (2.87) 15 -6.81 (2.98) BREX+SERT VS. BREX -4.14 (-12.7, 4.42) BREX+SERT VS. SERT -6.32 (-14.5, 1.83)

FILE: centera.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/center.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.5.1 FINAL

BREXPIPRAZOLE 2 OF 3

STAT-4 5 1

Summary of Mean Change in CAPS-5 Total Score

By Center - LOCF (Intent to Treat Sample)

CAPS-5 TOTAL SCORE BREX SERT PLACEBO TREATMENT CENTER N LS MEAN (SE) N LS MEAN (SE) N LS MEAN (SE) N LS MEAN (SE) COMPARISON LS MEAN DIFFERENCE<sup>1</sup> 14 -12.3 (3.12) 13 -8.20 (3.22) 16 -6.02 (2.87) 15 -6.81 (2.98) BREX+SERT VS. PLACEBO -5.53 (-13.8, 2.74) BREX VS. PLACEBO -1.39 (-9.81, 7.04) SERT VS. PLACEBO 0.80 (-7.21, 8.80) 13 -10.6 (3.14) 9 -10.8 (3.82) 7 -9.05 (4.31) 10 -8.06 (3.62) BREX+SERT VS. BREX 0.21 (-9.51, 9.93) BREX+SERT VS. SERT -1.58 (-12.0, 8.89) BREX+SERT VS. PLACEBO -2.56 (-11.9, 6.82) BREX VS. PLACEBO -2.77 (-13.0, 7.48) SERT VS. PLACEBO -0.99 (-11.9, 9.96) 7 -14.6 (4.32) 10 -15.8 (3.63) 9 -9.98 (3.82) 9 -11.4 (3.79) BREX+SERT VS. BREX 1.17 (-9.79, 12.14) BREX+SERT VS. SERT -4.63 (-15.8, 6.56) BREX+SERT VS. PLACEBO -3.22 (-14.4, 8.01) BREX VS. PLACEBO -4.39 (-14.6, 5.82) SERT VS. PLACEBO 1.42 (-9.08, 11.91) 9 -16.2 (3.77) 8 -7.83 (4.02) 8 -10.5 (4.05) 10 -7.91 (3.58) BREX+SERT VS. BREX -8.36 (-19.2, 2.47) BREX+SERT VS. SERT -5.73 (-16.6, 5.14) BREX+SERT VS. PLACEBO -8.28 (-18.5, 1.94) BREX VS. PLACEBO 0.08 (-10.5, 10.62) SERT VS. PLACEBO -2.55 (-13.1, 8.01)

FILE: centera.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/center.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.5.1 FINAL

BREXPIPRAZOLE 3 OF 3 PROTOCOL 331-201-00061

STAT-4.5.1

Summary of Mean Change in CAPS-5 Total Score
By Center - LOCF (Intent to Treat Sample)

------

| | | CAPS-5 TO | TAL SCORE | | | |
|---|---|---|---|---|---|---|
| CENTER | BREX+SERT N LS MEAN (SE) | BREX<br>N LS MEAN (SE) | SERT<br>N LS MEAN (SE) | PLACEBO SE) | TREATMENT<br>COMPARISON | LS MEAN DIFFERENCE <sup>1</sup> |
| | 8 -20.6 (4.01) | 6 -16.8 (4.64) | 11 -16.3 (3.44) | 10 -14.0 (3.64) | BREX+SERT VS. BREX | -3.81 (-15.8, 8.19) |
| | 7 -13.9 (4.30) | 7 -9.63 (4.37) | 7 -12.5 (4.27) | 7 -12.0 (4.32) | BREX+SERT VS. SERT<br>BREX+SERT VS. PLACEBO<br>BREX VS. PLACEBO<br>SERT VS. PLACEBO<br>BREX+SERT VS. BREX | -4.29 (-14.6, 6.04)<br>-6.60 (-17.2, 3.96)<br>-2.78 (-14.3, 8.69)<br>-2.31 (-12.1, 7.44)<br>-4.30 (-16.3, 7.68) |
| | | | | | BREX+SERT VS. SERT<br>BREX+SERT VS. PLACEBO<br>BREX VS. PLACEBO<br>SERT VS. PLACEBO | -1.42 (-13.3, 10.49)<br>-1.87 (-13.8, 10.08)<br>2.42 (-9.46, 14.31)<br>-0.45 (-12.4, 11.52) |
| | 5 -20.8 (5.07) | 4 -9.09 (5.66) | 6 -4.10 (4.61) | 5 -8.00 (5.09) | BREX+SERT VS. BREX<br>BREX+SERT VS. SERT<br>BREX+SERT VS. PLACEBO<br>BREX VS. PLACEBO<br>SERT VS. PLACEBO | -11.7 (-26.6, 3.22)<br>-16.7 (-30.1, -3.22)<br>-12.8 (-26.9, 1.33)<br>-1.09 (-16.0, 13.83)<br>3.89 (-9.61, 17.40) |

1

FILE: centera.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/center.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.5.1 FINA

BREXPIPRAZOLE 1 OF 1

STAT-4.5.2

Differences in Unadjusted Mean Changes of CAPS-5 Total Score

By Center - LOCF (Intent to Treat

Among Treatment Groups

| | | _BRE | X+SERT_ | | BREX | | SERT | PI | ACEBO | BREX+SERT<br>VS. PLACEB<br>O | BREX+SERT<br>VS. SERT | BREX+SERT<br>VS. BREX | BREX VS. P<br>LACEBO | SERT Vs. P |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CENTER | COUNTRY | N | MEAN1 | N | MEAN¹ | N | MEAN <sup>1</sup> | N | MEAN¹ | DIFF <sup>2</sup> | DIFF <sup>2</sup> | DIFF <sup>2</sup> | DIFF <sup>2</sup> | DIFF <sup>2</sup> |
| | USA<br>USA | 5<br>9 | -21.80<br>-15.00 | 4 8 | -8.25<br>-9.38 | 6 | -4.83<br>-13.00 | | -4.80<br>-8.70 | -17.00<br>-6.30 | -16.97<br>-2.00 | -13.55<br>-5.63 | -3.45<br>-0.68 | -0.03<br>-4.30 |
| | USA<br>USA<br>USA | 7<br>7<br>14 | -14.29<br>-16.71<br>-10.14 | | -4.71<br>-15.90<br>-6.31 | 7<br>9<br>16 | -13.43<br>-11.56<br>-5.63 | 9 | -8.14<br>-10.78<br>-4.53 | -6.14<br>-5.94<br>-5.61 | -0.86<br>-5.16<br>-4.52 | -9.57<br>-0.81<br>-3.84 | 3.43<br>-5.12<br>-1.77 | -5.29<br>-0.78<br>-1.09 |
| | USA<br>USA<br>USA | 8<br>4<br>13 | -21.13<br>-16.75<br>-12.00 | 6<br>4<br>9 | -18.50<br>-6.50<br>-10.11 | 11<br>3<br>7 | -15.45<br>-10.67<br>-10.57 | 4 | -16.10<br>-12.50<br>-10.30 | -5.02<br>-4.25<br>-1.70 | -5.67<br>-6.08<br>-1.43 | -2.63<br>-10.25<br>-1.89 | -2.40<br>6.00<br>0.19 | 0.65<br>1.83<br>-0.27 |
| | USA<br>USA | 7<br>4 | -8.57<br>-10.50 | 8 | -9.25<br>-13.00 | 7<br>3 | -12.86<br>-5.33 | 7<br>3 | -7.86<br>-12.67 | -0.71<br>2.17 | 4.29<br>-5.17 | 0.68<br>2.50 | -1.39<br>-0.33 | -5.00<br>7.33 |

--\_----

FILE: centerb.lis, RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/center.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.5.2 FINAL

| BREXPIPRAZOLE | | | | | | | | 1 OF 40 |
|---|---|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | Unadjusted Me | ean Change | (Int | STAT-4 | Phase B by | / Study Week | CAPS-5 Total Score | e, LOCF |
| | | | Analy | vsis Visit | (N)=3 | | | |
| | | | The T | TEST Proced | dure | | | |
| | | Vā | ariable: CHG | G (Change | from Baseline | e) | | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| | 1<br>900<br>Diff | | -5.6250 | | 1.2533<br>1.0792<br>1.6477 | -33.0000<br>-37.0000 | 36.0000<br>12.0000 | |
| | TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev | |
| | 1<br>900<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -5.9467<br>-5.6250<br>-0.3217 | | -3.4769<br>2.9334 | 10.8539<br>9.6527<br>10.2513 | 9.3520 12.9352<br>8.3539 11.4333<br>9.2200 11.5443 | |
| | | Method | Variance | es DI | f t Value | Pr > t | | |
| | | Pooled<br>Satterthwaite | Equal<br>Unequal | 153<br>148.13 | | | | |

BREXPIPRAZOLE

STAT-4.6
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 74 79 1.26 0.3055

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | | 3 OF 40 |
|---|---|---|---|---|---|---|---|---|
| | Unadjusted Mean | Change | (Inter | STAT-4.6<br>F<br>nt to Treat | | udy Week CAP: | G-5 Total | Score, LOCF |
| | | | Anai | lysis Visit | (N)=6 | | | |
| | | | The | TTEST Proce | dure | | | |
| | | | Variable: CF | HG (Change | from Baselin | e) | | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| | 1<br>900<br>Diff | 78<br>80<br>(1-2) | -10.5769<br>-8.0500<br>-2.5269 | 12.3357<br>11.1252<br>11.7383 | 1.3967<br>1.2438<br>1.8678 | -47.0000<br>-33.0000 | 23.0000<br>24.0000 | |
| | TRTPN | Method | Mean | 95% CI | Mean | Std Dev | 95% CL 3 | Std Dev |
| | 1<br>900<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -10.5769<br>-8.0500<br>-2.5269<br>-2.5269 | -13.3582<br>-10.5258<br>-6.2165<br>-6.2218 | -5.5742<br>1.1626 | 11.1252 | 10.6575<br>9.6283<br>10.5677 | 13.1775 |
| | | Method | Variand | ces D | F t Value | Pr > t | | |
| | | Pooled<br>Satterthwai | Equal<br>te Unequal | | | | | |

BREXPIPRAZOLE

STAT-4.6
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 77 79 1.23 0.3629

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | | 5 OF 40 |
|---|---|---|---|---|---|---|---|---|
| | Jnadjusted Mean ( | Change | | STAT-4.6 | hase B by St | udv Week CAP: | S-5 Total | Score, LOCE |
| | onaajassea nean ( | siidiige | (Inten | t to Treat | | aay woon one | 3 0 10001 | 20010, 2001 |
| | | | Analy | sis Visit ( | (N) =10 | | | |
| | | | The | TTEST Proce | edure | | | |
| | | V | Variable: CH | G (Change | from Baselin | e) | | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | 1 |
| | 1 | | | 13.3040 | 1.5064 | -47.0000 | 15.0000 | |
| | 900<br>Diff | 80<br>(1-2) | | 12.0794<br>12.6986 | 1.3505<br>2.0207 | -45.0000 | 13.0000 | |
| | TRTPN | Method | Mean | 95% CI | Mean | Std Dev | 95% CL | Std Dev |
| | 1<br>900 | | -14.0641<br>-9.2500 | | | | 11.4941 | |
| | 900<br>Diff (1-2) | Pooled | | -8.8055 | | | 10.4541 | |
| | Diff (1-2) | Satterthwaite | -4.8141 | | -0.8174 | | | |
| | | Method | Varianc | es I | F t Value | Pr > t | | |
| | | Pooled | Equal | 15 | | | | |
| | | Satterthwait | e Unequal | 153.7 | '3 -2.38 | 0.0186 | | |

BREXPIPRAZOLE

STAT-4.6
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 77 79 1.21 0.3949

SOURCE: TTESTLOCF; TABLE: stat1h.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | | 7 OF 40 |
|---|---|---|---|---|---|---|---|---|
| | Unadjusted Mean ( | Change | | | Phase B by St | udy Week CAP | S-5 Total | Score, LOCF |
| | | | (Inter | nt to Treat | Sample) | | | |
| | | | Analy | ysis Visit | (N)=12 | | | |
| | | | The | TTEST Proc | edure | | | |
| | | | Variable: CH | HG (Change | from Baselin | e) | | |
| | TRTP | ı N | Mean | Std Dev | Std Err | Minimum | Maximum | 1 |
| | 1<br>900 | 78<br>80<br>(1-2) | | 13.0908<br>13.3892<br>13.2427 | 1.4822<br>1.4970<br>2.1072 | -47.0000<br>-43.0000 | 18.0000<br>18.0000 | |
| | TRTPN | Method | Mean | | L Mean | Std Dev | 95% CL | Std Dev |
| | 1<br>900<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -14.7308<br>-10.0875<br>-4.6433<br>-4.6433 | -13.0671<br>-8.8057 | -7.1079 | 13.3892 | 11.3099<br>11.5877<br>11.9221 | 15.8591 |
| | | Method | Variano | | DF t Value | | | |
| | | Pooled<br>Satterthwai | Equal<br>te Unequal | 1 1 | 56 -2.20<br>56 -2.20 | | | |

BREXPIPRAZOLE

STAT-4.6
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 79 77 1.05 0.8435

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | 9 OF 40 |
|---|---|---|---|---|---|---|---|
| | Unadjusted Mean Cha | ange | (Intent | STAT-4.6 Pt to Treat | | udy Week CAPS | -5 Total Score, LOCF |
| | | | Analy | ysis Visit | (N)=3 | | |
| | | | The T | TEST Proce | dure | | |
| | | Va | riable: CHG | G (Change | from Baselin | e) | |
| | TRTPN | N | Mean | Std Dev | Std Err | Minimum | Maximum |
| | 1<br>3<br>Diff (1 | 76 | | 10.8539<br>8.6217<br>9.7941 | 1.2533<br>0.9890<br>1.5941 | -33.0000<br>-33.0000 | 36.0000<br>17.0000 |
| | TRTPN N | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| | , , | Pooled<br>Satterthwaite | -5.9467<br>-6.0132<br>0.0665<br>0.0665 | -8.4439<br>-7.9833<br>-3.0835<br>-3.0897 | -4.0430<br>3.2165 | 10.8539<br>8.6217<br>9.7941 | 9.3520 12.9352<br>7.4354 10.2618<br>8.7971 11.0480 |
| | | Method | Variance | es D | F t Value | Pr > t | |
| | | Pooled<br>Satterthwaite | Equal<br>Unequal | | | | |

BREXPIPRAZOLE

STAT-4.6
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 74 75 1.58 0.0484

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | | 11 OF 40 |
|---|---|---|---|---|---|---|---|---|
| | Unadjusted Mean ( | Change | (Inten | STAT-4.6 | | cudy Week CAP | S-5 Total S | core, LOCF |
| | | | Anal | ysis Visit | (N)=6 | | | |
| | | | The | TTEST Proce | dure | | | |
| | | V | ariable: CH | IG (Change | from Baselin | ne) | | |
| | TRTPI | N N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| | 1<br>3<br>Diff | | | 12.3357<br>10.1390<br>11.2980 | 1.3967<br>1.1554<br>1.8150 | -47.0000<br>-46.0000 | 23.0000<br>12.0000 | |
| | TRTPN | Method | Mean | 95% CI | Mean | Std Dev | 95% CL St | d Dev |
| | 1<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -10.5769<br>-8.8701<br>-1.7068<br>-1.7068 | -5.2925 | -6.5689 | 12.3357<br>10.1390<br>11.2980 | 10.6575 1<br>8.7519 1<br>10.1615 1 | 2.0526 |
| | | Method | Varianc | es D | F t Value | Pr > t | | |
| | | Pooled<br>Satterthwait | Equal<br>e Unequal | 15<br>. 148.1 | | | | |

BREXPIPRAZOLE

STAT-4.6
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 77 76 1.48 0.0886

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | | 13 OF 40 |
|---|---|---|---|---|---|---|---|---|
| | Unadjusted Mean | Change | (Inten | STAT-4.6<br>F<br>t to Treat | S-5 Total | Score, LOCF | | |
| | | | Analy | sis Visit | (N) =10 | | | |
| | | | The | TTEST Proce | edure | | | |
| | | V | ariable: CH | G (Change | from Baselir | ne) | | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | ı |
| | 1<br>3<br>Diff | | -10.4286 | 13.3040<br>11.0005<br>12.2142 | 1.5064<br>1.2536<br>1.9622 | -47.0000<br>-38.0000 | 15.0000<br>12.0000 | |
| | TRTPN | Method | Mean | 95% CI | Mean | Std Dev | 95% CL | Std Dev |
| | 1<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -14.0641<br>-10.4286<br>-3.6355<br>-3.6355 | -7.5120 | -7.9318<br>0.2409 | | 11.4941<br>9.4956<br>10.9855 | 13.0768 |
| | | Method | Varianc | es I | F t Value | Pr > t | | |
| | | Pooled<br>Satterthwait | Equal<br>e Unequal | 15<br>148.4 | | | | |

BREXPIPRAZOLE

STAT-4.6
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 77 76 1.46 0.0987

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | | 15 OF 40 |
|---|---|---|---|---|---|---|---|---|
| | Unadjusted Mean ( | Change | (Inter | STAT-4.6 | Phase B by St<br>Sample) | udy Week CAP | S-5 Total S | Score, LOCF |
| | | | Analy | sis Visit | (N) =12 | | | |
| The TTEST Procedure | | | | | | | | |
| | | | Variable: CH | IG (Change | from Baselin | ie) | | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| | 1<br>3<br>Diff | 77 | -13.1558 | 13.0908<br>12.3257<br>12.7165 | 1.4822<br>1.4046<br>2.0429 | | 18.0000<br>12.0000 | |
| | TRTPN | Method | Mean | 95% CI | L Mean | Std Dev | 95% CL St | ed Dev |
| | 1<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -1.5749 | -15.9534<br>-5.6108 | -10.3583 | 12.3257 | 11.3099 1<br>10.6395 1<br>11.4373 1 | 14.6521 |
| | | Method | Variano | es I | OF t Value | Pr > t | | |
| | | Pooled<br>Satterthwai | Equal<br>te Unequal | 152.6 | | 0.4419 | | |

BREXPIPRAZOLE

STAT-4.6
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 77 76 1.13 0.6001

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | 17 OF 40 |
|---|---|---|---|---|---|---|---|
| | Jnadjusted Mean C | hange | | STAT-4.6 | hase B hv Sti | udv Week CAPS | 3-5 Total Score, LOCF |
| | maajustea mean c | mange | (Intent | to Treat | | udy week CAID | of a focal score, hoci |
| | | | Analy | sis Visit | (N)=3 | | |
| | | | The I | TEST Proce | dure | | |
| | | Vā | ariable: CHG | G (Change | from Baseline | e) | |
| | TRTPN | N N | Mean | Std Dev | Std Err | Minimum | Maximum |
| | 1 | | | 10.8539 | 1.2533 | -33.0000 | 36.0000 |
| | 2<br>Diff | | | 8.7019<br>9.8979 | 1.0631<br>1.6639 | -24.0000 | 17.0000 |
| | TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| | 1 | | -5.9467 | -8.4439 | | 10.8539 | 9.3520 12.9352 |
| | 2 | | -3.3731 | | | | 7.4374 10.4883 |
| | Diff (1-2) | Pooled | -2.5735 | -5.8631 | | 9.8979 | 8.8618 11.2104 |
| | Diff (1-2) | Satterthwaite | -2.5735 | -5.8231 | 0.6760 | | |
| | | Method | Variance | es D | F t Value | Pr > t | |
| | | Pooled | Equal | 14 | 0 -1.55 | 0.1242 | |
| | | Satterthwaite | | | | | |

BREXPIPRAZOLE

STAT-4.6
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 74 66 1.56 0.0688

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | | 19 OF 40 |
|---|---|---|---|---|---|---|---|---|
| | Unadjusted Mean C | thange | (Inter | STAT-4.6 Int to Treat | | udy Week CAP | S-5 Total | l Score, LOCF |
| | | | Anal | ysis Visit | (N)=6 | | | |
| | | | The | TTEST Proce | edure | | | |
| | | V | ariable: CH | IG (Change | from Baselin | ie) | | |
| | TRTPN | I N | Mean | Std Dev | Std Err | Minimum | Maximum | n |
| | 1<br>2<br>Diff | 72 | | | 1.3967<br>1.3430<br>1.9439 | -47.0000<br>-29.0000 | 23.0000<br>29.0000 | |
| | TRTPN | Method | Mean | 95% CI | L Mean | Std Dev | 95% CL | Std Dev |
| | 1<br>2<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -10.5769<br>-6.0694<br>-4.5075<br>-4.5075 | -8.7474<br>-8.3488 | -3.3915 | 12.3357<br>11.3960<br>11.8942 | 9.7908 | 14.6460<br>13.6356<br>13.4227 |
| | | Method | Variano | ces I | OF t Value | Pr > t | | |
| | | Pooled<br>Satterthwait | Equal<br>e Unequal | 14 | | | | |

BREXPIPRAZOLE

STAT-4.6
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 77 71 1.17 0.5000

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | | 21 OF 40 |
|---|---|---|---|---|---|---|---|---|
| | Unadjusted Mean ( | Change | (Inten | STAT-4.6 | | udy Week CAP | S-5 Total | l Score, LOCF |
| | | | Analy | sis Visit ( | (N) =10 | | | |
| | | | The | TTEST Proce | edure | | | |
| | | 7 | /ariable: CH | IG (Change | from Baselin | ie) | | |
| | TRTPI | N N | Mean | Std Dev | Std Err | Minimum | Maximum | n |
| | 1<br>2<br>Diff | | | 13.3040<br>11.5300<br>12.4845 | 1.5064<br>1.3588<br>2.0403 | -47.0000<br>-37.0000 | 15.0000<br>29.0000 | |
| | TRTPN | Method | Mean | 95% CI | Mean | Std Dev | 95% CL | Std Dev |
| | 1<br>2<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -4.0224 | -17.0637<br>-12.7511<br>-8.0544<br>-8.0315 | -7.3322 | 13.3040<br>11.5300<br>12.4845 | 9.9060 | 15.7957<br>13.7960<br>14.0889 |
| | | Method | Variano | es I | F t Value | Pr > t | | |
| | | Pooled<br>Satterthwait | Equal<br>ce Unequal | 147.4 | | | | |

BREXPIPRAZOLE

STAT-4.6
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 77 71 1.33 0.2231

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE | | | | | | | | 23 OF 40 |
|---|---|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | Unadjusted Mean | Change | (Inten | STAT-4.6 | | B by Study Week CAPS-5 Total Score, LOCF<br>e) | | |
| | | | Analy | sis Visit ( | N)=12 | | | |
| | | | The | TTEST Proce | dure | | | |
| | | | Variable: CH | G (Change | from Baselin | e) | | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | ı |
| | 1<br>2<br>Diff | 78<br>72<br>(1-2) | -9.8611 | | 1.4822<br>1.5030<br>2.1132 | -47.0000<br>-40.0000 | 18.0000<br>29.0000 | |
| | TRTPN | Method | Mean | 95% CI | Mean | Std Dev | 95% CL | Std Dev |
| | 1<br>2<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | | -12.8581<br>-9.0456 | -6.8641<br>-0.6938 | 12.7537 | 11.3099<br>10.9573<br>11.6099 | 15.2601 |
| | | Method | Varianc | es D | F t Value | Pr > t | | |
| | | Pooled<br>Satterthwai | Equal<br>te Unequal | | | | | |

BREXPIPRAZOLE

STAT-4.6
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 77 71 1.05 0.8257

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE<br>PROTOCOL 331-201-00061 | | | | | | | 25 OF 40 |
|---|---|---|---|---|---|---|---|
| | Unadjusted Mean ( | Change | | STAT-4.6 | hase B by St | udy Week CAPS | S-5 Total Score, LOCF |
| | | | (Intent | to Treat | Sample) | | |
| | | | Analy | ysis Visit | (N)=3 | | |
| | | | The T | TTEST Proce | dure | | |
| Variable: CHG (Change from Baseline) | | | | | | | |
| | TRTPI | N N | Mean | Std Dev | Std Err | Minimum | Maximum |
| | 2<br>900 | 80 | | | 1.0631<br>1.0792 | -24.0000<br>-37.0000 | 17.0000<br>12.0000 |
| | Diff | (1-2)<br>Method | 2.2519<br>Mean | 9.2320<br>95% CL | 1.5289<br>Mean | Std Dev | 95% CL Std Dev |
| | 2 | | -3.3731 | -5.4957 | -1.2506 | 8.7019 | 7.4374 10.4883 |
| | 900<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -5.6250<br>2.2519<br>2.2519 | -7.7731<br>-0.7699<br>-0.7424 | 5.2736 | 9.6527<br>9.2320 | 8.3539 11.4333<br>8.2807 10.4322 |
| | | Method | Variance | es D | F t Value | Pr > t | |
| | | Pooled<br>Satterthwaite | Equal<br>Unequal | 14<br>144.1 | | | |
BREXPIPRAZOLE

STAT-4.6
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 79 66 1.23 0.3866

SOURCE: TTESTLOCF; TABLE: stat1h.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | | 27 OF 40 |
|---|---|---|---|---|---|---|---|---|
| | Jnadjusted Mean C | hange | | STAT-4.6 | STAT-4.6 Phase B by Study Week CAPS-5 Total Score, LOCF | | | |
| | | | (Inten | t to Treat | Sample) | | | |
| | | | Anal | ysis Visit | (N)=6 | | | |
| | | | The | -<br>TTEST Proce | dure | | | |
| | | Va | riable: CH | G (Change | from Baselin | e) | | |
| | TRTPN | N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| | 2<br>900<br>Diff | 80 | -8.0500 | 11.3960<br>11.1252<br>11.2542 | 1.3430<br>1.2438<br>1.8282 | -29.0000<br>-33.0000 | 29.0000<br>24.0000 | |
| | TRTPN | Method | Mean | 95% CL | | Std Dev | 95% CL | Std Dev |
| | 2<br>900<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -6.0694<br>-8.0500<br>1.9806<br>1.9806 | -10.5258<br>-1.6318 | -5.5742 | | 9.7908<br>9.6283<br>10.1120 | |
| | | Method | Varianc | es D | F t Value | Pr > t | | |
| | | Pooled<br>Satterthwaite | Equal<br>Unequal | 15<br>147. | | | | |

SOURCE: TTESTLOCF; TABLE: stat1h.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

BREXPIPRAZOLE

STAT-4.6
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 71 79 1.05 0.8325

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | | 29 OF 40 |
|---|---|---|---|---|---|---|---|---|
| | Unadjusted Mean | Change | (Inter | STAT-4.6 | | udy Week CAP | S-5 Total | l Score, LOCF |
| | | | Analy | sis Visit ( | (N) =10 | | | |
| | | | The | TTEST Proce | dure | | | |
| | | V | ariable: CH | IG (Change | from Baselir | ie) | | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | α |
| | 2<br>900<br>Diff | | | 11.5300<br>12.0794<br>11.8225 | 1.3588<br>1.3505<br>1.9205 | -37.0000<br>-45.0000 | 29.0000<br>13.0000 | |
| | TRTPN | Method | Mean | 95% CI | Mean | Std Dev | 95% CL | Std Dev |
| | 2<br>900<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -10.0417<br>-9.2500<br>-0.7917<br>-0.7917 | -4.5865 | -6.5619 | | 10.4541 | 13.7960<br>14.3077<br>13.3304 |
| | | Method | Variano | es I | F t Value | Pr > t | | |
| | | Pooled<br>Satterthwait | Equal<br>e Unequal | 15<br>. 149.4 | | | | |

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

BREXPIPRAZOLE

STAT-4 6
Unadjusted Mean Change

Unadjusted Mean Change

One of the to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 79 71 1.10 0.6916

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | | 31 OF 40 |
|---|---|---|---|---|---|---|---|---|
| | Unadjusted Mean ( | Change | (Inten | STAT-4.6 P | | udy Week CAP | S-5 Total | L Score, LOCF |
| | | | Analy | rsis Visit ( | N)=12 | | | |
| | | | The | TTEST Proce | dure | | | |
| | | 7 | Variable: CH | G (Change | from Baselin | e) | | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | n |
| | 2<br>900<br>Diff | 72<br>80<br>(1-2) | | 12.7537<br>13.3892<br>13.0922 | 1.5030<br>1.4970<br>2.1268 | -40.0000<br>-43.0000 | 29.0000<br>18.0000 | |
| | TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL | Std Dev |
| | 2<br>900<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -9.8611<br>-10.0875<br>0.2264<br>0.2264 | -12.8581<br>-13.0671<br>-3.9759<br>-3.9653 | -7.1079<br>4.4287 | | 11.5877 | 15.2601<br>15.8591<br>14.7621 |
| | | Method | Varianc | es D | F t Value | Pr > t | | |
| | | Pooled<br>Satterthwait | | 15<br>149.5 | | | | |

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

BREXPIPRAZOLE

STAT-4.6
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 79 71 1.10 0.6785

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE | | | | | | | | 33 OF 40 |
|---|---|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | Unadjusted Mean | Change | 3-5 Total Score, LOG | CF | | | | |
| | | | Analys | sis Visit | (N)=3 | | | |
| | | | The T | TEST Proced | dure | | | |
| | | V | ariable: CHG | (Change i | from Baseline | e) | | |
| | TRT | PN N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| | 3<br>900<br>Dif | | | | 0.9890<br>1.0792<br>1.4681 | | 17.0000<br>12.0000 | |
| | TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev | |
| | 3<br>900<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -6.0132<br>-5.6250<br>-0.3882<br>-0.3882 | | -3.4769<br>2.5120 | 8.6217<br>9.6527<br>9.1651 | 7.4354 10.2618<br>8.3539 11.4333<br>8.2458 10.3168 | |
| | | Method | Variance | s DI | f t Value | Pr > t | | |
| | | Pooled<br>Satterthwaite | Equal<br>e Unequal | 154<br>153.43 | | | | |

SOURCE: TTESTLOCF; TABLE: stat1h.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

BREXPIPRAZOLE

STAT-4.6
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 79 75 1.25 0.3253

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | | 35 OF 40 |
|---|---|---|---|---|---|---|---|---|
| | Unadjusted Mean ( | Change | | STAT-4.6 | hase R hv St | udv Week CAPS | :-5 Total | l Score IOCF |
| | onaujuseed neun ( | Sirange | (Inten | it to Treat | 4 | day week enre | , 3 10001 | i secie, Ecci |
| | | | Anal | ysis Visit | (N)=6 | | | |
| | | | The | TTEST Proce | dure | | | |
| | | V | ariable: CH | IG (Change | from Baselir | ne) | | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | n |
| | 3 | 77 | -8.8701 | 10.1390 | 1.1554 | -46.0000 | 12.0000 | |
| | 900<br>Diff | 80<br>(1-2) | -8.0500<br>-0.8201 | 11.1252<br>10.6530 | 1.2438<br>1.7007 | -33.0000 | 24.0000 | 0 |
| | TRTPN | Method | Mean | 95% CI | Mean | Std Dev | 95% CL | Std Dev |
| | 3<br>900 | | -8.8701<br>-8.0500 | -11.1714<br>-10.5258 | | 10.1390<br>11.1252 | | 12.0526<br>13.1775 |
| | Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -0.8201<br>-0.8201 | -4.1797<br>-4.1738 | 2.5394 | 10.6530 | | 11.9869 |
| | | Method | Variano | es D | F t Value | e Pr > t | | |
| | | Pooled<br>Satterthwait | Equal<br>e Unequal | 15<br>. 154.5 | | | | |

SOURCE: TTESTLOCF; TABLE: stat1h.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

BREXPIPRAZOLE

STAT-4.6
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 79 76 1.20 0.4169

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | | 37 OF 40 |
|---|---|---|---|---|---|---|---|---|
| | | | | STAT-4.6 | | | | |
| | Unadjusted Mean C | Change | (Inten | t to Treat | | udy Week CAP | S-5 Total | Score, LOCF |
| | | | Anals | raia Wisit ( | N) =10 | | | |
| | | | Analy | SIS AISIC ( | N)=10 | | | |
| | | | The | TTEST Proce | dure | | | |
| | | • | Variable: CH | G (Change | from Baselin | e) | | |
| | TRTPN | I N | Mean | Std Dev | Std Err | Minimum | Maximum | n |
| | 3 | 77 | -10.4286 | 11.0005 | 1.2536 | -38.0000 | 12.0000 | ) |
| | 900 | | | | 1.3505 | -45.0000 | 13.0000 | ) |
| | Diff | (1-2) | -1.1786 | 11.5630 | 1.8460 | | | |
| | TRTPN | Method | Mean | 95% CI | Mean | Std Dev | 95% CL | Std Dev |
| | 3 | | -10.4286 | -12.9254 | -7.9318 | 11.0005 | 9.4956 | 13.0768 |
| | 900 | | -9.2500 | -11.9381 | -6.5619 | 12.0794 | 10.4541 | 14.3077 |
| | Diff (1-2) | Pooled | -1.1786 | -4.8251 | 2.4680 | 11.5630 | 10.4066 | 13.0108 |
| | Diff (1-2) | Satterthwaite | -1.1786 | -4.8187 | 2.4615 | | | |
| | | Method | Varianc | es D | F t Value | Pr > t | | |
| | | Pooled | Equal | 15 | 5 -0.64 | 0.5241 | | |
| | | Satterthwai | te Unequal | 154.5 | -0.64 | 0.5234 | | |

SOURCE: TTESTLOCF; TABLE: stat1h.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

BREXPIPRAZOLE

STAT-4.6
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 79 76 1.21 0.4132

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | | 39 OF 40 |
|---|---|---|---|---|---|---|---|---|
| 11010001 331 201 00001 | Unadjusted Mean ( | Change | | STAT-4.6 | Phase B by St | udv Week CAP | S-5 Total | Score, LOCF |
| | onaujuseed nean v | Silarige | (Inter | nt to Treat | | day week en | 0 0 10001 | Beere, Eeer |
| | | | Analy | sis Visit | (N)=12 | | | |
| | | | The | TTEST Proce | edure | | | |
| | | | Variable: CF | IG (Change | from Baselin | ie) | | |
| | TRTPI | N N | Mean | Std Dev | Std Err | Minimum | Maximum | 1 |
| | 3<br>900<br>Diff | 77<br>80<br>(1-2) | | | 1.4046<br>1.4970<br>2.0560 | -50.0000<br>-43.0000 | 12.0000<br>18.0000 | |
| | TRTPN | Method | Mean | 95% CI | L Mean | Std Dev | 95% CL | Std Dev |
| | 3<br>900<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -13.1558<br>-10.0875<br>-3.0683<br>-3.0683 | -13.0671<br>-7.1298 | -7.1079 | 12.3257<br>13.3892<br>12.8787 | 10.6395<br>11.5877<br>11.5907 | 15.8591 |
| | | Method<br>Pooled<br>Satterthwai | Variand<br>Equal<br>te Unequal | 1 | | 0.1376 | | |

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

BREXPIPRAZOLE

STAT-4 6
Unadjusted Mean Change

Unadjusted Mean Change

One of the phase B by Study Week CAPS-5 Total Score, LOCF
(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 79 76 1.18 0.4692

SOURCE: TTESTLOCF; TABLE: statlh.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.6 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | | 1 OF 40 |
|---|---|---|---|---|---|---|---|---|
| | Unadjusted Mean Change Phase B by Study Week CAPS-5 Total Score, OC (Intent to Treat Sample) | | | | | | | |
| | | | Anal | ysis Visit | (N)=3 | | | |
| | | | The | TTEST Proce | dure | | | |
| | | V | ariable: CH | G (Change | from Baselin | ie) | | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| | 1<br>900<br>Diff | 74<br>77<br>(1-2) | -5.6623 | 10.9125<br>9.7732<br>10.3471 | 1.2685<br>1.1138<br>1.6844 | -33.0000<br>-37.0000 | 36.0000<br>12.0000 | |
| | TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev | |
| | 1<br>900<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -6.0135<br>-5.6623<br>-0.3512<br>-0.3512 | -8.5417<br>-7.8806<br>-3.6796<br>-3.6875 | -3.4441<br>2.9772 | 10.9125<br>9.7732<br>10.3471 | 9.3936 13.0219<br>8.4362 11.6179<br>9.2938 11.6717 | |
| | | Method | Varianc | es D | F t Value | Pr > t | | |
| | | Pooled<br>Satterthwait | Equal<br>e Unequal | 14<br>145.7 | | | | |

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

BREXPIPRAZOLE

STAT-4.7
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 73 76 1.25 0.3423

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

|---|---|---|---|---|---|---|---|
| Unadjusted Mean | al Score, OC | | | | | | |
| | | Anal | ysis Visit | (N)=6 | | | |
| | | The | TTEST Proce | edure | | | |
| | , | Variable: CH | IG (Change | from Baselin | ie) | | |
| TRTPN | N | Mean | Std Dev | Std Err | Minimum | Maximum | α |
| 1<br>900<br>Diff | | | 12.9123<br>11.1205<br>12.0091 | 1.6140<br>1.3292<br>2.0769 | -47.0000<br>-29.0000 | 23.0000<br>24.0000 | |
| TRTPN | Method | Mean | 95% CI | Mean | Std Dev | 95% CL | Std Dev |
| 1<br>900<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -11.5469<br>-7.7571<br>-3.7897<br>-3.7897 | -7.8981 | -5.1056 | | 9.5349 | 15.6384<br>13.3435<br>13.6555 |
| | Method<br>Pooled | Varianc<br>Equal | 13 | | 0.0703 | | |
| | Satterthwai | te Unequal | 124.9 | 95 -1.81 | 0.0723 | | |

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

BREXPIPRAZOLE

STAT-4.7
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 63 69 1.35 0.2255

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

|---|---|---|---|---|---|---|---|---|
| FR010C0L 331-201-00001 | Unadjusted Mea | - Channa | | STAT-4.7 | Dh D h 0 | +d W1- 03 | DC E M-+- | 1 0 00 |
| | unadjusted Mea | n Change | (Inten | t to Treat | | tudy Week CA | P5-5 TOLA | i score, oc |
| | | | Analy | sis Visit ( | N)=10 | | | |
| | | | The | TTEST Proce | dure | | | |
| | | V | ariable: CH | G (Change | from Baselin | e) | | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| | 1 | | | 14.2178 | 1.8510 | -47.0000 | 15.0000 | |
| | 900<br>Diff | 62 | | 12.3919<br>13.3132 | 1.5738<br>2.4213 | -45.0000 | 13.0000 | |
| | TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL | Std Dev |
| | 1 | | -15.4237 | -19.1289 | -11.7186 | 14.2178 | 12.0358 | 17.3735 |
| | 900 | | -9.6935 | -12.8405 | | | 10.5302 | |
| | Diff (1-2) | Pooled | -5.7302 | -10.5246 | -0.9357 | 13.3132 | 11.8153 | 15.2494 |
| | Diff (1-2) | Satterthwaite | -5.7302 | -10.5427 | -0.9176 | | | |
| | | Method | Varianc | es D | F t Value | Pr > t | | |
| | | Pooled | Equal | 11 | 9 -2.37 | 0.0196 | | |
| | | Satterthwait | | | 2 -2.36 | 0.0200 | | |

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

BREXPIPRAZOLE

STAT-4.7

Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 58 61 1.32 0.2904

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

|---|---|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | Unadjusted Mean | .1 Score, OC | | | | | | |
| | | | Analy | sis Visit ( | N)=12 | | | |
| | | | The | TTEST Proce | dure | | | |
| | | V | ariable: CH | G (Change | from Baselin | e) | | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | ı |
| | 1<br>900<br>Diff | | -11.1148 | 13.7643<br>13.6920<br>13.7269 | 1.8231<br>1.7531<br>2.5288 | -47.0000<br>-43.0000 | 18.0000<br>18.0000 | |
| | TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL | Std Dev |
| | 1<br>900<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -5.6045 | | -7.6081<br>-0.5960 | 13.6920 | 11.6206<br>11.6205<br>12.1650 | 16.6691 |
| | | Method | Varianc | es D | F t Value | Pr > t | | |
| | | Pooled<br>Satterthwait | * | 11<br>115.3 | | | | |

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

BREXPIPRAZOLE

Unadjusted Mean Change

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 56 60 1.01 0.9657

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

| BREXPIPRAZOLE | | | | | 9 OF 40 | | | |
|---|---|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | Unadjusted Mea | n Change | | | | tudy Week CAF | S-5 Total Score, OC | : |
| | | | (Intent | to Treat | Sample) | | | |
| | | | Analy | sis Visit | (N)=3 | | | |
| | | | The T | TEST Proce | dure | | | |
| | | Va | riable: CHG | (Change | from Baselin | e) | | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| | 1 | 74 | -6.0135 | 10.9125 | 1.2685 | -33.0000 | 36.0000 | |
| | 3 | | | | 1.0155 | -33.0000 | 17.0000 | |
| | Diff | (1-2) | 0.0270 | 9.8842 | 1.6250 | | | |
| | TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev | |
| | 1 | | -6.0135 | -8.5417 | -3.4853 | 10.9125 | 9.3936 13.0219 | |
| | 3 | | -6.0405 | | | | 7.5198 10.4244 | |
| | Diff (1-2) | Pooled | 0.0270 | -3.1844 | 3.2385 | 9.8842 | 8.8688 11.1642 | |
| | Diff (1-2) | Satterthwaite | 0.0270 | -3.1857 | 3.2398 | | | |
| | | Method | Variance | s D | F t Value | Pr > t | | |
| | | Pooled | Equal | 14 | 6 0.02 | 0.9868 | | |
| | | Satterthwaite | Unequal | 139.3 | 3 0.02 | 0.9868 | | |

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

BREXPIPRAZOLE

Unadjusted Mean Change

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 73 73 1.56 0.0592

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

|---|---|---|---|---|---|---|---|---|
| | Unadjusted Mea | n Change | (Inter | STAT-4.7 | | Study Week CA | PS-5 Tota | al Score, OC |
| | | | Anal | ysis Visit | (N)=6 | | | |
| | | | The | TTEST Proce | edure | | | |
| Variable: CHG (Change from Baseline) | | | | | | | | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | α |
| | 1<br>3<br>Diff | 64<br>62<br>(1-2) | -11.5469<br>-9.3387<br>-2.2082 | 12.9123<br>10.4394<br>11.7610 | 1.6140<br>1.3258<br>2.0958 | -47.0000<br>-46.0000 | 23.0000 | |
| | TRTPN | Method | Mean | 95% CI | Mean | Std Dev | 95% CL | Std Dev |
| | 1<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -11.5469<br>-9.3387<br>-2.2082<br>-2.2082 | -14.7723<br>-11.9898<br>-6.3563<br>-6.3437 | -6.6876<br>1.9399 | | | 15.6384<br>12.6867<br>13.4317 |
| | | Method | Variano | ces I | F t Value | Pr > t | | |
| | | Pooled<br>Satterthwai | Equal<br>te Unequal | | | | | |

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

BREXPIPRAZOLE

Unadjusted Mean Change

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 63 61 1.53 0.0974

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

|---|---|---|---|---|---|---|---|---|
| | Unadjusted Mea | n Change | (Inten | STAT-4.7 | Phase B by S<br>Sample) | tudy Week CA | ?S-5 Tota | l Score, OC |
| | | | Analy | sis Visit ( | N)=10 | | | |
| | | | The | TTEST Proce | dure | | | |
| Variable: CHG (Change from Baseline) | | | | | | | | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | 1 |
| | 1<br>3<br>Diff | | -11.3448 | 14.2178<br>9.9852<br>12.3032 | 1.8510<br>1.3111<br>2.2750 | -47.0000<br>-38.0000 | 15.0000<br>10.0000 | |
| | TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL | Std Dev |
| | 1<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -15.4237<br>-11.3448<br>-4.0789<br>-4.0789 | -19.1289<br>-13.9703<br>-8.5851<br>-8.5770 | -8.7194<br>0.4273 | | 12.0358<br>8.4415<br>10.8979 | 12.2250 |
| | | Method | Varianc | es D | F t Value | Pr > t | | |
| | | Pooled<br>Satterthwait | Equal<br>e Unequal | 11<br>104.1 | | | | |

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

BREXPIPRAZOLE

STAT-4.7
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 58 57 2.03 0.0083

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

|---|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | Unadjusted Mean Change | (Ir | STAT-4.7 | | cudy Week CAP | S-5 Total | Score, OC |
| | | Ar | nalysis Visit (N | i)=12 | | | |
| | | 7 | The TTEST Proced | lure | | | |
| | | Variable: | CHG (Change f | rom Baseline | <b>)</b> | | |
| | TRTPN | N Mean | Std Dev | Std Err | Minimum | Maximum | |
| | 1<br>3<br>Diff (1-2) | 57 -16.7193<br>58 -15.0517<br>-1.6676 | 11.7852 | | -47.0000<br>-50.0000 | 18.0000<br>12.0000 | |
| | TRTPN Method | Mea | an 95% CL | Mean | Std Dev | 95% CL S | td Dev |
| | 1<br>3<br>Diff (1-2) Pooled<br>Diff (1-2) Sattert | | -18.1505 -<br>76 -6.3988 | 11.9530<br>3.0637 | 11.7852 | 11.6206<br>9.9633<br>11.3304 | 14.4288 |
| | Meth | od Vari | iances DF | t Value | Pr > t | | |
| | Pool<br>Satt | ed Equa<br>erthwaite Unec | al 113<br>qual 109.78 | | 0.4864<br>0.4871 | | |

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

BREXPIPRAZOLE

STAT-4.7
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 56 57 1.36 0.2458

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

| BREXPIPRAZOLE | | | | | | | | 17 OF 40 |
|---|---|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | Unadjusted Mea | n Change | | | | tudy Week CAF | S-5 Tota | al Score, OC |
| | | | (Intent | to Treat | Sample)<br> | | | |
| | | | Analy | sis Visit | (N)=3 | | | |
| | | | The T | TEST Proce | dure | | | |
| | | Va | ariable: CHG | (Change | from Baseline | e) | | |
| | TRTF | N N | Mean | Std Dev | Std Err | Minimum | Maximur | m |
| | 1 | 74 | -6.0135 | 10.9125 | 1.2685 | -33.0000 | 36.0000 | 0 |
| | 2 | | | | 1.0779 | -24.0000 | 17.0000 | 0 |
| | Diff | (1-2) | -2.6953 | 9.9554 | 1.6855 | | | |
| | TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL | Std Dev |
| | 1 | | -6.0135 | -8.5417 | -3.4853 | 10.9125 | 9.3936 | 13.0219 |
| | 2 | | -3.3182 | | | | | 10.5711 |
| | Diff (1-2) | Pooled | -2.6953 | -6.0281 | 0.6375 | 9.9554 | 8.9067 | 11.2864 |
| | Diff (1-2) | Satterthwaite | -2.6953 | -5.9872 | 0.5965 | | | |
| | | Method | Variance | s D | F t Value | Pr > t | | |
| | | Pooled | Equal | 13 | 8 -1.60 | 0.1121 | | |
| | | Satterthwaite | | | | 0.1077 | | |

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

BREXPIPRAZOLE

Unadjusted Mean Change

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 73 65 1.55 0.0720

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

| BREXPIPRAZOLE | | | | | | | | 19 OF 40 |
|---|---|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | Unadjusted Mea | n Change | | | Phase B by S | tudy Week CA | PS-5 Tota | al Score, OC |
| | | | (Inten | t to Treat | Sample) | | | |
| | | | Anal | ysis Visit | (N)=6 | | | |
| | | | The | TTEST Proce | dure | | | |
| | | V | ariable: CH | G (Change | from Baselin | e) | | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | n |
| | 1 | | | | 1.6140 | -47.0000 | 23.0000 | |
| | 2<br>Diff | 58 (1-2) | | | 1.5128<br>2.2247 | -29.0000 | 29.0000 | |
| | TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL | Std Dev |
| | 1 | | -11.5469 | -14.7723 | -8.3215 | 12.9123 | 10.9987 | 15.6384 |
| | 2 | | -6.1724 | -9.2018 | -3.1430 | 11.5214 | 9.7402 | 14.1058 |
| | Diff (1-2) | Pooled | -5.3745 | -9.7792 | -0.9698 | 12.2713 | 10.8957 | 14.0475 |
| | Diff (1-2) | Satterthwaite | -5.3745 | -9.7544 | -0.9945 | | | |
| | | Method | Varianc | es D | F t Value | Pr > t | | |
| | | Pooled | Equal | 12 | 0 -2.42 | 0.0172 | | |
| | | Satterthwait | e Unequal | 119.9 | 7 -2.43 | 0.0166 | | |

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

BREXPIPRAZOLE

Unadjusted Mean Change

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 63 57 1.26 0.3837

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

|---|---|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | Unadjusted Mean | Change | | STAT-4.7 | Phase B by S | tudy Week CAl | PS-5 Total | Score, OC |
| | onaajaseea nean | - change | (Inten | t to Treat | | cuay week em | 5 10001 | 56616, 66 |
| | | | Analy | sis Visit ( | N)=10 | | | |
| | | | The | TTEST Proce | dure | | | |
| Variable: CHG (Change from Baseline) | | | | | | | | |
| | TRTPN | I N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| | 1 | | -15.4237 | 14.2178 | 1.8510 | -47.0000 | 15.0000 | |
| | 2<br>Diff | 48 | | 10.1952<br>12.5772 | 1.4715<br>2.4447 | -37.0000 | 7.0000 | |
| | TRTPN | Method | Mean | 95% CI | Mean | Std Dev | 95% CL St | d Dev |
| | 1 2 | | -15.4237<br>-11.3750 | | | | 12.0358 1<br>8.4872 1 | |
| | Diff (1-2) | Pooled | -4.0487 | -8.8962 | 0.7987 | | 11.0820 1 | |
| | Diff (1-2) | Satterthwaite | -4.0487 | -8.7382 | 0.6408 | | | |
| | | Method | Varianc | es D | F t Value | Pr > t | | |
| | | Pooled<br>Satterthwait | Equal<br>te Unequal | 10<br>103.4 | | | | |

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL
BREXPIPRAZOLE

STAT-4.7
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 58 47 1.94 0.0199

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | | 23 OF 40 |
|---|---|---|---|---|---|---|---|---|
| FRO10COL 331-201-00001 | Unadjusted Mea | n Change | | STAT-4.7 | Phase B by S | tudy Week CA | PS-5 Tota | al Score, OC |
| | - | - | (Inter | nt to Treat | | • | | , |
| | | | Analy | 7SIS VISIT ( | N)=12 | | | |
| | | | The | TTEST Proce | dure | | | |
| | | | Variable: CF | IG (Change | from Baselin | e) | | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | n |
| | 1 | 57 | -16.7193 | 13.7643 | 1.8231 | -47.0000 | 18.0000 | ) |
| | 2 | 48 | -10.7500 | 12.3779 | 1.7866 | -40.0000 | 15.0000 | ) |
| | Diff | (1-2) | -5.9693 | 13.1498 | 2.5761 | | | |
| | TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL | Std Dev |
| | 1 | | -16.7193 | -20.3715 | -13.0671 | 13.7643 | 11.6206 | 16.8853 |
| | 2 | | -10.7500 | | | | | 15.5043 |
| | Diff (1-2) | Pooled | -5.9693 | -11.0783 | -0.8603 | 13.1498 | 11.5732 | 15.2277 |
| | Diff (1-2) | Satterthwaite | -5.9693 | -11.0320 | -0.9066 | | | |
| | | Method | Variano | ces D | F t Value | Pr > t | | |
| | | Pooled<br>Satterthwai | Equal<br>te Unequal | | | | | |

BREXPIPRAZOLE

STAT-4.7

Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 56 47 1.24 0.4568

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | | 25 OF 40 |
|---|---|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | Unadjusted Mean | Change | (Intent | STAT-4.7 | | tudy Week CAF | S-5 Total Score, OC | c<br> |
| | | | Analy | ysis Visit | (N)=3 | | | |
| | | | The I | TEST Proce | dure | | | |
| | | Va | riable: CHG | G (Change | from Baseline | e) | | |
| | TRTPN | N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| | 2<br>900<br>Diff | 77 | -3.3182<br>-5.6623<br>2.3442 | 8.7568<br>9.7732<br>9.3185 | 1.0779<br>1.1138<br>1.5631 | -24.0000<br>-37.0000 | 17.0000<br>12.0000 | |
| | TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev | |
| | 2<br>900<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -3.3182<br>-5.6623<br>2.3442<br>2.3442 | -5.4709<br>-7.8806<br>-0.7460<br>-0.7200 | -3.4441<br>5.4344 | 8.7568<br>9.7732<br>9.3185 | 7.4761 10.5711<br>8.4362 11.6179<br>8.3462 10.5492 | |
| | | Method | Variance | es D | F t Value | Pr > t | | |
| | | Pooled<br>Satterthwaite | | 14<br>140.7 | | | | |

BREXPIPRAZOLE

STAT-4.7

Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 76 65 1.25 0.3648

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

|---|---|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | Unadjusted Mear | n Change | | STAT-4.7 | Phase B by S | tudy Week CA | PS-5 Tota | .1 Score, OC |
| | - | | (Inten | t to Treat | Sample) | - | | |
| | | | Anal: | vsis Visit | (N)=6 | | | |
| | | | | _ | | | | |
| | | | The ' | TTEST Proce | dure | | | |
| | | Va | ariable: CH | G (Change | from Baselin | e) | | |
| | TRTP | 1 N | Mean | Std Dev | Std Err | Minimum | Maximum | ı |
| | 2 | 58 | -6.1724 | 11.5214 | 1.5128 | -29.0000 | 29.0000 | |
| | 900<br>Diff | | | 11.1205<br>11.3036 | 1.3292<br>2.0070 | -29.0000 | 24.0000 | |
| | TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL | Std Dev |
| | 2<br>900 | | -6.1724<br>-7.7571 | -9.2018<br>-10.4087 | | 11.5214<br>11.1205 | | 14.1058 |
| | Diff (1-2) | Pooled | 1.5847 | -2.3872 | | | 10.0636 | |
| | Diff (1-2) | Satterthwaite | 1.5847 | -2.4024 | 5.5719 | | | |
| | | Method | Varianc | es D | F t Value | Pr > t | | |
| | | Pooled | Equal | 12 | 6 0.79 | 0.4313 | | |
| | | Satterthwaite | unequal | 119.9 | 3 0.79 | 0.4329 | | |

BREXPIPRAZOLE

Unadjusted Mean Change

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 57 69 1.07 0.7741

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

|---|---|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00001 | Unadjusted Mea | n Change | | STAT-4.7 | Phase B by S | tudy Week CA | PS-5 Tota | al Score OC |
| | onaujusceu nea | ii ciialige | (Inter | nt to Treat | | cuay week ch | 10 0 1000 | ar score, oc |
| | | | Analy | ysis Visit ( | N)=10 | | | |
| | | | The | TTEST Proce | dure | | | |
| | | | Variable: CF | HG (Change | from Baselin | e) | | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | n |
| | 2 | 48 | -11.3750 | 10.1952 | 1.4715 | -37.0000 | 7.0000 | |
| | 900<br>Diff | (1-2) | | 12.3919<br>11.4877 | 1.5738<br>2.2086 | -45.0000 | 13.0000 | U |
| | TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL | Std Dev |
| | 2 | | -11.3750 | -14.3354 | | | | 12.7703 |
| | 900 | | -9.6935 | | | 12.3919 | | 15.0596 |
| | Diff (1-2) | Pooled | -1.6815 | -6.0592 | | 11.4877 | 10.1387 | 13.2540 |
| | Diff (1-2) | Satterthwaite | -1.6815 | -5.9524 | 2.5895 | | | |
| | | Method | Variano | ces D | F t Value | Pr > t | | |
| | | Pooled<br>Satterthwai | Equal<br>te Unequal | | | | | |

BREXPIPRAZOLE

Unadjusted Mean Change

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 61 47 1.48 0.1654

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

|---|---|---|---|---|---|---|---|
| Unadjusted Mean | n Change | (Inter | STAT-4.7 | Phase B by S<br>Sample) | tudy Week CA | PS-5 Tota | l Score, OC |
| | | Analy | ysis Visit ( | N)=12 | | | |
| | | The | TTEST Proce | edure | | | |
| | V | ariable: CH | IG (Change | from Baselin | e) | | |
| TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | 1 |
| 2<br>900<br>Diff | 61 | -11.1148 | 12.3779<br>13.6920<br>13.1310 | 1.7866<br>1.7531<br>2.5335 | -40.0000<br>-43.0000 | 15.0000<br>18.0000 | |
| TRTPN | Method | Mean | 95% CI | Mean | Std Dev | 95% CL | Std Dev |
| 2<br>900<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -10.7500<br>-11.1148<br>0.3648<br>0.3648 | -4.6577 | -7.6081 | 12.3779<br>13.6920<br>13.1310 | 10.3042<br>11.6205<br>11.5827 | 16.6691 |
| | Method | Variano | ces I | F t Value | Pr > t | | |
| | Pooled<br>Satterthwait | | 104. | | | | |

BREXPIPRAZOLE

Unadjusted Mean Change

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 60 47 1.22 0.4750

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | | 33 OF 40 |
|---|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00001 | Unadjusted Mea | n Change | | | | tudy Week CAF | S-5 Total Score, OC |
| | | | (Intent | to Treat | Sample) | | |
| | | | Analy | ysis Visit | (N)=3 | | |
| | | | The T | TTEST Proce | dure | | |
| | | V | ariable: CHC | G (Change | from Baselin | e) | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum |
| | 3<br>900 | | -6.0405<br>-5.6623 | 8.7358<br>9.7732 | 1.0155<br>1.1138 | -33.0000<br>-37.0000 | 17.0000<br>12.0000 |
| | Diff | (1-2) | -0.3782 | 9.2794 | 1.5106 | | |
| | TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| | 3<br>900 | | -6.0405<br>-5.6623 | | -4.0166<br>-3.4441 | 8.7358<br>9.7732 | 7.5198 10.4244<br>8.4362 11.6179 |
| | Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -0.3782<br>-0.3782 | -3.3632<br>-3.3566 | | 9.2794 | 8.3348 10.4674 |
| | | Method | Variance | es D | F t Value | Pr > t | |
| | | Pooled<br>Satterthwait | Equal<br>e Unequal | | | | |

BREXPIPRAZOLE

Unadjusted Mean Change

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 76 73 1.25 0.3361

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

| BREXPIPRAZOLE | | | | | | | | 35 OF 40 |
|---|---|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | | | | STAT-4.7 | | | | |
| | Unadjusted Mea | n Change | (Inten | t to Treat | | tudy Week CAP | S-5 Total Score, | OC |
| | | | (Incen | t to freat | sampie) | | | |
| | | | Anal | ysis Visit | (N)=6 | | | |
| | | | The | TTEST Proce | dure | | | |
| | | V | ariable: CH | G (Change | from Baselin | e) | | |
| | TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| | 3 | 62 | -9.3387 | 10.4394 | 1.3258 | -46.0000 | 11.0000 | |
| | 900 | 70 | -7.7571 | 11.1205 | 1.3292 | -29.0000 | 24.0000 | |
| | Diff | (1-2) | -1.5816 | 10.8063 | 1.8846 | | | |
| | TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev | |
| | 3 | | -9.3387 | -11.9898 | -6.6876 | 10.4394 | 8.8710 12.6867 | |
| | 900 | | -7.7571 | -10.4087 | -5.1056 | 11.1205 | 9.5349 13.3435 | |
| | Diff (1-2) | Pooled | -1.5816 | -5.3100 | 2.1469 | 10.8063 | 9.6372 12.3007 | |
| | Diff (1-2) | Satterthwaite | -1.5816 | -5.2958 | 2.1327 | | | |
| | | Method | Varianc | es D | F t Value | Pr > t | | |
| | | Pooled | Equal | 13 | 0 -0.84 | 0.4029 | | |
| | | Satterthwait | e Unequal | 129.5 | 5 -0.84 | 0.4011 | | |

BREXPIPRAZOLE

Unadjusted Mean Change

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 69 61 1.13 0.6166

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

|---|---|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | Unadjusted Mean | Change | (Inten | STAT-4.7 | | tudy Week CAl | PS-5 Tota | l Score, OC |
| | | | Analy | sis Visit ( | N)=10 | | | |
| | | | The | TTEST Proce | dure | | | |
| | | V | ariable: CH | G (Change | from Baselin | e) | | |
| | TRTPN | N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| | 3<br>900<br>Diff | 62 | -9.6935 | 9.9852<br>12.3919<br>11.2936 | 1.3111<br>1.5738<br>2.0631 | -38.0000<br>-45.0000 | 10.0000<br>13.0000 | |
| | TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL | Std Dev |
| | , , | Pooled<br>Satterthwaite | -11.3448<br>-9.6935<br>-1.6513<br>-1.6513 | -13.9703<br>-12.8405<br>-5.7367<br>-5.7085 | -6.5466<br>2.4341 | | 8.4415<br>10.5302<br>10.0182 | |
| | | Method | Varianc | es D | F t Value | Pr > t | | |
| | | Pooled<br>Satterthwait | | 11<br>115.5 | | | | |

BREXPIPRAZOLE

Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 61 57 1.54 0.1015

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

|---|---|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | Unadjusted Mean | Change | (Inter | STAT-4.7 | Phase B by S<br>Sample) | tudy Week CA | PS-5 Tota | l Score, OC |
| | | | Analy | ysis Visit | (N)=12 | | | |
| | | | The | TTEST Proce | edure | | | |
| | | | Variable: CH | IG (Change | from Baselin | e) | | |
| | TRTPN | I N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| | 3<br>900<br>Diff | 58<br>61<br>(1-2) | | 11.7852<br>13.6920<br>12.7986 | 1.5475<br>1.7531<br>2.3472 | -50.0000<br>-43.0000 | 12.0000<br>18.0000 | |
| | TRTPN | Method | Mean | 95% C | L Mean | Std Dev | 95% CL : | Std Dev |
| | 3<br>900<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -15.0517<br>-11.1148<br>-3.9370<br>-3.9370 | -14.6214<br>-8.5855 | | | 9.9633<br>11.6205<br>11.3478 | 16.6691 |
| | | Method | Variand | ces l | OF t Value | Pr > t | | |
| | | Pooled<br>Satterthwai | Equal<br>te Unequal | 115.8<br>115.8 | | | | |

BREXPIPRAZOLE

STAT-4.7
Unadjusted Mean Change

(Intent to Treat Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F

Folded F 60 57 1.35 0.2560

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.7 FINAL

BREXPIPRAZOLE
STAT-4.8
Non-Parametric Stratified by Center and Type of Trauma Analysis of Mean Change (Intent to Treat Sample)

The FREQ Procedure

Summary Statistics for TRTP by CHG
Controlling for POOLCNTR and COMBFL

Cochran-Mantel-Haenszel Statistics (Based on Rank Scores)

Statistic Alternative Hypothesis DF Value Prob
1 Nonzero Correlation 1 0.1690 0.6810
2 Row Mean Scores Differ 3 3.4071 0.3330

SOURCE: NPAR; TABLE: statlj.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.8 FINAL

<sup>1</sup> WILCOXON TEST STRATIFIED BY (POOLED) CENTER AND TYPE OF TRAUMA.

BREXPIPRAZOLE

STAT-4.8
Non-Parametric Stratified by Center and Type of Trauma Analysis of Mean Change (Intent to Treat Sample)

The FREQ Procedure

Summary Statistics for TRTP by CHG
Controlling for POOLCNTR and COMBFL

Cochran-Mantel-Haenszel Statistics (Based on Rank Scores)

| Statistic | Alternative Hypothesis | DF | Value | Prob |
|-----------|------------------------|----|--------|--------|
| 1 | Nonzero Correlation | 1 | 1.0528 | 0.3049 |
| 2 | Row Mean Scores Differ | 3 | 2.6953 | 0.4410 |

SOURCE: NPAR; TABLE: statlj.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.8 FINAL

<sup>1</sup> WILCOXON TEST STRATIFIED BY (POOLED) CENTER AND TYPE OF TRAUMA.

BREMPIPRAZOLE

STAT-4.8
Non-Parametric Stratified by Center and Type of Trauma Analysis of Mean Change (Intent to Treat Sample)

The FREQ Procedure

Summary Statistics for TRTP by CHG
Controlling for POOLCNTR and COMBFL

Cochran-Mantel-Haenszel Statistics (Based on Rank Scores)

Statistic Alternative Hypothesis DF Value Prob

1 Nonzero Correlation 1 2.6378 0.1043
2 Row Mean Scores Differ 3 8.1432 0.0431

SOURCE: NPAR; TABLE: statlj.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.8 FINAL

<sup>1</sup> WILCOXON TEST STRATIFIED BY (POOLED) CENTER AND TYPE OF TRAUMA.

BREXPIPRAZOLE

4 OF 4


STAT-4.8

Non-Parametric Stratified by Center and Type of Trauma Analysis of Mean Change (Intent to Treat Sample)

The FREQ Procedure

Summary Statistics for TRTP by CHG Controlling for POOLCNTR and COMBFL

Cochran-Mantel-Haenszel Statistics (Based on Rank Scores)

| Statistic | Alternative Hypothesis | DF | Value | Prob |
|-----------|------------------------|----|--------|--------|
| 1 | Nonzero Correlation | 1 | 0.0243 | 0.8762 |
| 2 | Row Mean Scores Differ | 3 | 6.6492 | 0.0840 |

SOURCE: NPAR; TABLE: statlj.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.8 FINAL

<sup>1</sup> WILCOXON TEST STRATIFIED BY (POOLED) CENTER AND TYPE OF TRAUMA.

BREXPIPRAZOLE 1 OF 9

STAT-4.9

Residual from Proc Mixed for Change from Baseline in CAPS-5 Total Score, Primary Efficacy Analysis Model (Intent to Treat Sample)

------

The UNIVARIATE Procedure
Variable: RESID (Residual)

AVISITN = 10

AVISIT =

## Moments

| N | 227 | Sum Weights | 227 |
|-----------------|------------|------------------|------------|
| Mean | 0.08611581 | Sum Observations | 19.5482882 |
| Std Deviation | 10.6826629 | Variance | 114.119287 |
| Skewness | -0.1828243 | Kurtosis | -0.146025 |
| Uncorrected SS | 25792.6423 | Corrected SS | 25790.9589 |
| Coeff Variation | 12404.9966 | Std Error Mean | 0.70903324 |

## Basic Statistical Measures

Location Variability

| Mean | 0.08612 | Std Deviation | 10.68266 |
|--------|----------|---------------------|-----------|
| Median | -0.06010 | Variance | 114.11929 |
| Mode | -5.59726 | Range | 58.82853 |
| | | Interquartile Range | 14.39574 |

Note: The mode displayed is the smallest of 2 modes with a count of 2.

SOURCE: MMRMDX1; TABLE: stat1k.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.9 FINAL


STAT-4.9

Residual from Proc Mixed for Change from Baseline in CAPS-5 Total Score, Primary Efficacy Analysis Model (Intent to Treat Sample)

\_\_\_\_\_\_

The UNIVARIATE Procedure
Variable: RESID (Residual)
AVISITN = 10
AVISIT =

Tests for Location: Mu0=0

Test -Statistic- ----p Value----- Student's t t 0.121455 Pr > |t| 0.9034 Sign M -0.5 Pr >= |M| 1.0000 Signed Rank S 291 Pr >= |S| 0.7697

Quantiles (Definition 5)

| Level | Quantile |
|------------|------------|
| 100% Max | 25.824025 |
| 99% | 22.779706 |
| 95% | 17.026880 |
| 90% | 14.368205 |
| 75% Q3 | 7.330122 |
| 50% Median | -0.060104 |
| 25% Q1 | -7.065623 |
| 10% | -13.686490 |
| 5% | -18.354843 |
| 1% | -24.242300 |
| 0% Min | -33.004507 |

SOURCE: MMRMDX1; TABLE: stat1k.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.9 FINAL

BREXPIPRAZOLE 3 OF 9 PROTOCOL 331-201-00061

Residual from Proc Mixed for Change from Baseline

from Proc Mixed for Change from Baseline in CAPS-5 Total Score, Primary Efficacy Analysis Model (Intent to Treat Sample)

\_\_\_\_\_

The UNIVARIATE Procedure
Variable: RESID (Residual)
AVISITN = 10
AVISIT =

Extreme Observations

| Lowest | | | Highest | |
|--------|----------------------|-----------|-----------------|-----------|
| | Value | Obs | Value | Obs |
| | -33.0045<br>-24.5363 | 93<br>716 | 20.3750 21.9446 | 467<br>97 |
| | -24.2423 | 34 | 22.7797 | 322 |
| | -24.1066 | 192 | 22.8236 | 301 |
| | -23.2337 | 440 | 25.8240 | 949 |

SOURCE: MMRMDX1; TABLE: stat1k.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.9 FINAL




STAT-4.9

Residual from Proc Mixed for Change from Baseline in CAPS-5 Total Score, Primary Efficacy Analysis Model (Intent to Treat Sample)

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

AVISITN = 10 AVISIT =

Moments

| N | 227 | Sum Weights | 227 |
|-----------------|------------|------------------|------------|
| Mean | 0.00806674 | Sum Observations | 1.831149 |
| Std Deviation | 0.97676522 | Variance | 0.95407029 |
| Skewness | -0.1794597 | Kurtosis | -0.1289175 |
| Uncorrected SS | 215.634657 | Corrected SS | 215.619886 |
| Coeff Variation | 12108.5562 | Std Error Mean | 0.06483018 |

Basic Statistical Measures

Location Variability

 Mean
 0.00807
 Std Deviation
 0.97677

 Median
 -0.00547
 Variance
 0.95407

 Mode
 -0.50932
 Range
 5.40570

 Interquartile Range
 1.31622

Note: The mode displayed is the smallest of 2 modes with a count of 2.

SOURCE: MMRMDX1; TABLE: stat1k.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.9 FINAL

Residual

BREXPIPRAZOLE 6 OF 9

STAT-4.9

from Proc Mixed for Change from Baseline in CAPS-5 Total Score, Primary Efficacy Analysis Model (Intent to Treat Sample)

\_\_\_\_\_\_

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

AVISITN = 10 AVISIT =

Tests for Location: Mu0=0

| Test | -S | tatistic- | p Valı | ue |
|-------------|----|-----------|----------|--------|
| Student's t | t | 0.124429 | Pr > t | 0.9011 |
| Sign | M | -0.5 | Pr >= M | 1.0000 |
| Signed Rank | S | 290 | Pr >= S | 0.7704 |

Quantiles (Definition 5)

| 327141 |
|---------|
| .123783 |
| 962015 |
| 465170 |
| 7188649 |
| 547028 |
| 1433297 |
| 1754229 |
| 7961704 |
| 347197 |
| 242422 |

SOURCE: MMRMDX1; TABLE: stat1k.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.9 FINAL

Residual

BREXPIPRAZOLE 7 OF 9

STAT-4.

from Proc Mixed for Change from Baseline in CAPS-5 Total Score, Primary Efficacy Analysis Model (Intent to Treat Sample)

\_\_\_\_\_\_

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

AVISITN = 10 AVISIT =

Extreme Observations

| TOM | est | Hignest | |
|----------------------|-----------|--------------------|-----------|
| Value | Obs | Value | Obs |
| -3.05242<br>-2.23710 | 93<br>716 | 1.86278<br>2.02821 | 467<br>97 |
| -2.20347 | 34 | 2.11124 | 301 |
| -2.19831 | 192 | 2.11717 | 322 |
| -2.11381 | 440 | 2.35327 | 949 |

SOURCE: MMRMDX1; TABLE: stat1k.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.9 FINAL





BREXPIPRAZOLE 1 OF 20 PROTOCOL 331-201-00061

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups

(Intent to Treat Sample)

-----

The Mixed Procedure

Model Information

Data Set WORK.INDATA
Dependent Variable CHG
Covariance Structure Unstructured
Subject Effect SUBJID

Subject Effect SUBJID
Group Effect TRTPN
Estimation Method REML
Residual Variance Method None

Fixed Effects SE Method Kenward-Roger Degrees of Freedom Method Kenward-Roger

Class Level Information

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10 FINAL

COMBFL

BREXPIPRAZOLE 2 OF 20 PROTOCOL 331-201-00061

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Class Level Information

Class Levels Values

SUBJID 299



SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10 FINAL

BREXPIPRAZOLE


3 OF 20

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups
(Intent to Treat Sample)

The Mixed Procedure



SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10 FINAL

BREXPIPRAZOLE 4 OF 20 PROTOCOL 331-201-00061

 ${\tt STAT-4.10}\\ {\tt Proc\ Mixed\ Output\ Using\ Heterogeneous\ Variance\ Structure\ for\ Treatment\ Groups}\\ {\tt (Intent\ to\ Treat\ Sample)}\\$ 

The Mixed Procedure



SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10 FINAL
BREXPIPRAZOLE 5 OF 20 PROTOCOL 331-201-00061

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Intent to Treat Sample)

## The Mixed Procedure



### Dimensions

| Covariance | | Parameters | 40 |
|------------|----|------------|-----|
| Columns | in | X | 41 |
| Columns | in | Z | 0 |
| Subjects | | | 299 |

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10 FINAL

BREXPIPRAZOLE 6 OF 20 PROTOCOL 331-201-00061

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Intent to Treat Sample)

......

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Dimensions

Max Obs per Subject 4

Number of Observations

Number of Observations Read 996
Number of Observations Used 996
Number of Observations Not Used 0

Iteration History

| Criterion | -2 Res Log Like | Evaluations | Iteration |
|------------|-----------------|-------------|-----------|
| | 7419.63261777 | 1 | 0 |
| 0.00489019 | 6917.10751714 | 2 | 1 |
| 0.00080739 | 6909.33113519 | 3 | 2 |
| 0.00002848 | 6907.06145589 | 1 | 3 |
| 0.0000009 | 6906.98597457 | 1 | 4 |
| 0.00000000 | 6906.98574059 | 1 | 5 |

Convergence criteria met.

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10 FINAL

BREXPIPRAZOLE 7 OF 20 PROTOCOL 331-201-00061

STAT-4.10
Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups

(Intent to Treat Sample)

The Mixed Procedure

Estimated R Matrix for SUBJID 001S00001

| Row | Col1 | Col2 | Col3 | Col4 |
|-----|---------|---------|---------|---------|
| 1 | 95.2938 | 64.2572 | 64.5504 | 60.3472 |
| 2 | 64.2572 | 129.09 | 94.7811 | 91.9205 |
| 3 | 64.5504 | 94.7811 | 146.52 | 112.90 |
| 4 | 60.3472 | 91.9205 | 112.90 | 129.82 |

Estimated R Correlation Matrix for SUBJID 001S00001

| Row | Col1 | Col2 | Col3 | Col4 |
|-----|--------|--------|--------|--------|
| 1 | 1.0000 | 0.5794 | 0.5463 | 0.5426 |
| 2 | 0.5794 | 1.0000 | 0.6892 | 0.7101 |
| 3 | 0.5463 | 0.6892 | 1.0000 | 0.8186 |
| 4 | 0.5426 | 0.7101 | 0.8186 | 1.0000 |

Estimated R Matrix for SUBJID 001S00011

| Row | Col1 | Col2 | Col3 | Col4 |
|-----|---------|---------|---------|---------|
| 1 | 63.9185 | 43.6854 | 31.3695 | 37.4615 |
| 2 | 43.6854 | 98.9262 | 82.6187 | 72.2502 |
| 3 | 31.3695 | 82.6187 | 112.58 | 83.3850 |
| 4 | 37.4615 | 72.2502 | 83.3850 | 135.46 |

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10 FINAL

BREXPIPRAZOLE

8 OF 20

 ${\tt STAT-4.10}$  Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups

(Intent to Treat Sample)

------ Parameter Code=CAPSTOT ------

The Mixed Procedure

Estimated R Matrix for SUBJID 001S00101

| Row | Col1 | Col2 | Col3 | Col4 |
|-----|---------|---------|---------|---------|
| 1 | 84.9865 | 58.8491 | 45.3790 | 54.8618 |
| 2 | 58.8491 | 114.92 | 95.4457 | 98.6286 |
| 3 | 45.3790 | 95.4457 | 134.77 | 130.88 |
| Λ | 54 8618 | 98 6286 | 130 88 | 173 25 |

Covariance Parameter Estimates

| Cov Parm | Subject | Group | Estimate |
|----------|---------|---------|----------|
| UN(1,1) | SUBJID | TRTPN 1 | 95.2938 |
| UN(2,1) | SUBJID | TRTPN 1 | 64.2572 |
| UN(2,2) | SUBJID | TRTPN 1 | 129.09 |
| UN(3,1) | SUBJID | TRTPN 1 | 64.5504 |
| UN(3,2) | SUBJID | TRTPN 1 | 94.7811 |
| UN(3,3) | SUBJID | TRTPN 1 | 146.52 |
| UN(4,1) | SUBJID | TRTPN 1 | 60.3472 |
| UN(4,2) | SUBJID | TRTPN 1 | 91.9205 |
| UN(4,3) | SUBJID | TRTPN 1 | 112.90 |
| UN(4,4) | SUBJID | TRTPN 1 | 129.82 |
| UN(1,1) | SUBJID | TRTPN 2 | 66.1243 |
| UN(2,1) | SUBJID | TRTPN 2 | 42.7734 |
| UN(2,2) | SUBJID | TRTPN 2 | 111.53 |
| UN(3,1) | SUBJID | TRTPN 2 | 34.2983 |

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10 FINAL

BREXPIPRAZOLE 9 OF 20 PROTOCOL 331-201-00061

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Intent to Treat Sample)

The Mixed Procedure

Covariance Parameter Estimates

| Cov Parm | Subject | Group | Estimate |
|---|---|---|---|
| UN(3,2) | SUBJID | TRTPN 2 | 87.0247 |
| UN(3,3) | SUBJID | TRTPN 2 | 102.29 |
| UN(4,1) | SUBJID | TRTPN 2 | 37.8799 |
| UN (4,1)<br>UN (4,2)<br>UN (4,3) | SUBJID<br>SUBJID | TRTPN 2<br>TRTPN 2 | 100.12 |
| UN(4,4) | SUBJID | TRTPN 2 | 149.81 |
| UN(1,1) | SUBJID | TRTPN 3 | 63.9185 |
| UN(2,1) | SUBJID | TRTPN 3 | 43.6854 |
| UN(2,2) | SUBJID | TRTPN 3 | 98.9262 |
| UN(3,1)<br>UN(3,2) | SUBJID<br>SUBJID<br>SUBJID | TRTPN 3<br>TRTPN 3<br>TRTPN 3 | 31.3695<br>82.6187<br>112.58 |
| UN(3,3)<br>UN(4,1)<br>UN(4,2) | SUBJID<br>SUBJID | TRTPN 3<br>TRTPN 3 | 37.4615<br>72.2502 |
| UN (4, 3) | SUBJID | TRTPN 3 | 83.3850 |
| UN (4, 4) | SUBJID | TRTPN 3 | 135.46 |
| UN(1,1) | SUBJID | TRTPN 900 | 84.9865 |
| UN(2,1) | SUBJID | TRTPN 900 | 58.8491 |
| UN(2,2) | SUBJID | TRTPN 900 | 114.92 |
| UN(3,1) | SUBJID | TRTPN 900 | 45.3790 |
| UN(3,2) | SUBJID | TRTPN 900 | 95.4457 |
| UN (3, 3) | SUBJID | TRTPN 900 | 134.77 |
| UN (4, 1) | SUBJID | TRTPN 900 | 54.8618 |
| UN (4, 2) | SUBJID | TRTPN 900 | 98.6286 |

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10 FINAL

BREXPIPRAZOLE 10 OF 20 PROTOCOL 331-201-00061

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Intent to Treat Sample)

......

The Mixed Procedure

Covariance Parameter Estimates

| Cov Parm | Subject | Group | Estimate |
|----------|---------|-----------|----------|
| UN(4,3) | SUBJID | TRTPN 900 | 130.88 |
| UN (4,4) | SUBJID | TRTPN 900 | 173.25 |

Fit Statistics

| -2 Res Log Likelihood | 6907.0 |
|--------------------------|--------|
| AIC (Smaller is Better) | 6987.0 |
| AICC (Smaller is Better) | 6990.5 |
| BIC (Smaller is Better) | 7135.0 |

Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|-----|------------|------------|
| 3.9 | 512 65 | < 0001 |

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10 FINAL

BREXPIPRAZOLE 11 OF 20 PROTOCOL 331-201-00061

STAT-4.10 Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Intent to Treat Sample)

## The Mixed Procedure

## Solution for Fixed Effects

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|---|
| Intercept | | | | | 3.4163 | 3.5355 | 296 | 0.97 | 0.3347 |
| AVISITN | | | 3 | | 0.8999 | 2.7008 | 214 | 0.33 | 0.7393 |
| AVISITN | | | 6 | | 0.3093 | 2.1603 | 181 | 0.14 | 0.8863 |
| AVISITN | | | 10 | | 1.0883 | 1.8411 | 171 | 0.59 | 0.5552 |
| AVISITN | | | 12 | | 0 | | | | |
| TRTPN | | | | 1 | -5.7924 | 2.1332 | 135 | -2.72 | 0.0075 |
| TRTPN | | | | 2 | -0.5506 | 2.2925 | 116 | -0.24 | 0.8106 |
| TRTPN | | | | 3 | -3.4533 | 2.1810 | 125 | -1.58 | 0.1159 |
| TRTPN | | | | 900 | 0 | | | | |
| AVISITN*TRTPN | | | 3 | 1 | 5.6229 | 1.9850 | 135 | 2.83 | 0.0053 |
| AVISITN*TRTPN | | | 3 | 2 | 2.1940 | 2.1980 | 122 | 1.00 | 0.3202 |
| AVISITN*TRTPN | | | 3 | 3 | 3.4684 | 2.0726 | 131 | 1.67 | 0.0966 |
| AVISITN*TRTPN | | | 3 | 900 | 0 | | | | |
| AVISITN*TRTPN | | | 6 | 1 | 2.0607 | 1.6734 | 120 | 1.23 | 0.2206 |
| AVISITN*TRTPN | | | 6 | 2 | 1.4332 | 1.6822 | 108 | 0.85 | 0.3961 |
| AVISITN*TRTPN | | | 6 | 3 | 2.6949 | 1.7486 | 119 | 1.54 | 0.1259 |
| AVISITN*TRTPN | | | 6 | 900 | 0 | | | | |
| AVISITN*TRTPN | | | 10 | 1 | -0.4073 | 1.3134 | 110 | -0.31 | 0.7571 |
| AVISITN*TRTPN | | | 10 | 2 | -1.2545 | 1.5096 | 90.4 | -0.83 | 0.4081 |
| AVISITN*TRTPN | | | 10 | 3 | 2.5005 | 1.5014 | 107 | 1.67 | 0.0988 |
| AVISITN*TRTPN | | | 10 | 900 | 0 | | | | |

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10

BREXPIPRAZOLE 12 OF 20 PROTOCOL 331-201-00061

 ${\tt STAT-4.10}\\ {\tt Proc\ Mixed\ Output\ Using\ Heterogeneous\ Variance\ Structure\ for\ Treatment\ Groups}\\ {\tt (Intent\ to\ Treat\ Sample)}\\$ 

------

Parameter Code=CAPSTOT ------

## The Mixed Procedure

## Solution for Fixed Effects

| Effect | Center<br>(Pooled<br>Center)<br>for ITT | Combat<br>Related<br>Population<br>Flag | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN | | | 12 | 1 | 0 | | | | |
| AVISITN*TRTPN | | | 12 | 2 | 0 | | | | |
| AVISITN*TRTPN | | | 12 | 3 | 0 | | | | |
| AVISITN*TRTPN | | | 12 | 900 | 0 | | | | |
| POOLCNTR | | | | | -0.5650 | 3.1142 | 267 | -0.18 | 0.8562 |
| POOLCNTR | | | | | -1.1271 | 3.0551 | 268 | -0.37 | 0.7125 |
| POOLCNTR | | | | | -0.8652 | 2.5522 | 262 | -0.34 | 0.7349 |
| POOLCNTR | | | | | -0.3817 | 2.2754 | 263 | -0.17 | 0.8669 |
| POOLCNTR | | | | | -2.3250 | 2.4105 | 268 | -0.96 | 0.3357 |
| POOLCNTR | | | | | -4.6732 | 2.4453 | 261 | -1.91 | 0.0571 |
| POOLCNTR | | | | | -2.7844 | 2.4677 | 270 | -1.13 | 0.2602 |
| POOLCNTR | | | | | -5.1732 | 2.4762 | 255 | -2.09 | 0.0377 |
| POOLCNTR | | | | | -4.2543 | 2.5459 | 265 | -1.67 | 0.0959 |
| POOLCNTR | | | | | 0 | | | | |
| COMBFL | | N | | | 3.0906 | 1.2799 | 275 | 2.41 | 0.0164 |
| COMBFL | | Y | | | 0 | | | | |
| BASE*AVISITN | | | 3 | | -0.2846 | 0.04867 | 254 | -5.85 | <.0001 |
| BASE*AVISITN | | | 6 | | -0.3432 | 0.06042 | 254 | -5.68 | <.0001 |
| BASE*AVISITN | | | 10 | | -0.4074 | 0.06369 | 212 | -6.40 | <.0001 |
| BASE*AVISITN | | | 12 | | -0.4083 | 0.06909 | 222 | -5.91 | <.0001 |

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10 FINAL

BREXPIPRAZOLE 13 OF 20 PROTOCOL 331-201-00061

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Intent to Treat Sample)

Parameter Code=CAPSTOT ------

The Mixed Procedure

Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------------|-----------|-----------|---------|---------|
| AVISITN | 3 | 212 | 0.80 | 0.4943 |
| TRTPN | 3 | 146 | 2.72 | 0.0466 |
| AVISITN*TRTPN | 9 | 165 | 1.86 | 0.0618 |
| POOLCNTR | 9 | 268 | 1.46 | 0.1646 |
| COMBFL | 1 | 275 | 5.83 | 0.0164 |
| BASE*AVISITN | 4 | 216 | 13.09 | < .0001 |

Least Squares Means

| Effect | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN | 3 | 1 | -6.6009 | 1.1949 | 83.3 | -5.52 | <.0001 | 0.05 | -8.9774 | -4.2244 |
| AVISITN*TRTPN | 3 | 2 | -4.7879 | 1.1054 | 80.3 | -4.33 | <.0001 | 0.05 | -6.9876 | -2.5882 |
| AVISITN*TRTPN | 3 | 3 | -6.4163 | 1.0232 | 86.8 | -6.27 | <.0001 | 0.05 | -8.4502 | -4.3824 |
| AVISITN*TRTPN | 3 | 900 | -6.4314 | 1.1239 | 88.9 | -5.72 | <.0001 | 0.05 | -8.6645 | -4.1982 |
| AVISITN*TRTPN | 6 | 1 | -12.8284 | 1.4258 | 74.9 | -9.00 | <.0001 | 0.05 | -15.6687 | -9.9880 |
| AVISITN*TRTPN | 6 | 2 | -8.2140 | 1.4342 | 78.1 | -5.73 | <.0001 | 0.05 | -11.0693 | -5.3587 |
| AVISITN*TRTPN | 6 | 3 | -9.8551 | 1.2959 | 77 | -7.60 | <.0001 | 0.05 | -12.4356 | -7.2745 |
| AVISITN*TRTPN | 6 | 900 | -9.0966 | 1.3151 | 80.5 | -6.92 | <.0001 | 0.05 | -11.7135 | -6.4797 |
| AVISITN*TRTPN | 10 | 1 | -16.7911 | 1.5460 | 72.5 | -10.86 | <.0001 | 0.05 | -19.8726 | -13.7096 |

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10 FINAL

BREXPIPRAZOLE 14 OF 20 PROTOCOL 331-201-00061

 ${\tt STAT-4.10}\\ {\tt Proc\ Mixed\ Output\ Using\ Heterogeneous\ Variance\ Structure\ for\ Treatment\ Groups}\\ ({\tt Intent\ to\ Treat\ Sample})$ 

The Mixed Procedure

Least Squares Means

| Effect | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | (14) | (14) | ESCIMACE | BILOI | DI | c varue | 11 / [0] | Aipha | TOWEL | opper |
| AVISITN*TRTPN | 10 | 2 | -12.3965 | 1.4409 | 65.1 | -8.60 | <.0001 | 0.05 | -15.2741 | -9.5190 |
| AVISITN*TRTPN | 10 | 3 | -11.5443 | 1.4063 | 62.7 | -8.21 | <.0001 | 0.05 | -14.3549 | -8.7336 |
| AVISITN*TRTPN | 10 | 900 | -10.5914 | 1.4489 | 78.2 | -7.31 | <.0001 | 0.05 | -13.4759 | -7.7070 |
| AVISITN*TRTPN | 12 | 1 | -17.5059 | 1.4677 | 75.9 | -11.93 | <.0001 | 0.05 | -20.4291 | -14.5827 |
| AVISITN*TRTPN | 12 | 2 | -12.2640 | 1.7206 | 60.9 | -7.13 | <.0001 | 0.05 | -15.7046 | -8.8234 |
| AVISITN*TRTPN | 12 | 3 | -15.1667 | 1.5466 | 63.6 | -9.81 | <.0001 | 0.05 | -18.2567 | -12.0767 |
| ΔΥΤΩΤΨΝ*ΨΡΨΡΝ | 12 | 900 | -11 7134 | 1 6421 | 75.8 | -7 13 | < 0.001 | 0.05 | -14 9841 | -8 4428 |

Differences of Least Squares Means

| | Analysis<br>Visit | Planned<br>Treatment | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 3 | 1 | 3 | 2 | -1.8130 | 1.5140 | 138 | -1.20 | 0.2332 | 0.05 | -4.8067 | 1.1807 |
| AVISITN*TRTPN | 3 | 1 | 3 | 3 | -0.1846 | 1.4694 | 134 | -0.13 | 0.9002 | 0.05 | -3.0909 | 2.7217 |
| AVISITN*TRTPN | 3 | 1 | 3 | 900 | -0.1696 | 1.5427 | 145 | -0.11 | 0.9126 | 0.05 | -3.2187 | 2.8796 |
| AVISITN*TRTPN | 3 | 1 | 6 | 1 | 6.2275 | 1.2231 | 66.9 | 5.09 | <.0001 | 0.05 | 3.7862 | 8.6687 |
| AVISITN*TRTPN | 3 | 1 | 6 | 2 | 1.6131 | 1.7620 | 127 | 0.92 | 0.3617 | 0.05 | -1.8737 | 5.0998 |
| AVISITN*TRTPN | 3 | 1 | 6 | 3 | 3.2541 | 1.6698 | 134 | 1.95 | 0.0534 | 0.05 | -0.04844 | 6.5567 |
| AVISITN*TRTPN | 3 | 1 | 6 | 900 | 2.4957 | 1.6874 | 138 | 1.48 | 0.1414 | 0.05 | -0.8408 | 5.8322 |

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10 FINAL

BREXPIPRAZOLE 15 OF 20 PROTOCOL 331-201-00061

 ${\tt STAT-4.10}\\ {\tt Proc\ Mixed\ Output\ Using\ Heterogeneous\ Variance\ Structure\ for\ Treatment\ Groups}\\ ({\tt Intent\ to\ Treat\ Sample})$ 

------

## The Mixed Procedure

## Differences of Least Squares Means

| | Analysis | Planned | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | Treatment | Visit | Treatment | | Standard | | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 3 | 1 | 10 | 1 | 10.1902 | 1.3566 | 66.6 | 7.51 | <.0001 | 0.05 | 7.4821 | 12.8983 |
| AVISITN*TRTPN | 3 | 1 | 10 | 2 | 5.7956 | 1.7651 | 112 | 3.28 | 0.0014 | 0.05 | 2.2984 | 9.2929 |
| AVISITN*TRTPN | 3 | 1 | 10 | 3 | 4.9434 | 1.7573 | 117 | 2.81 | 0.0058 | 0.05 | 1.4630 | 8.4237 |
| AVISITN*TRTPN | 3 | 1 | 10 | 900 | 3.9905 | 1.7942 | 133 | 2.22 | 0.0278 | 0.05 | 0.4417 | 7.5393 |
| AVISITN*TRTPN | 3 | 1 | 12 | 1 | 10.9049 | 1.3091 | 67.5 | 8.33 | <.0001 | 0.05 | 8.2923 | 13.5176 |
| AVISITN*TRTPN | 3 | 1 | 12 | 2 | 5.6631 | 2.0010 | 98.4 | 2.83 | 0.0056 | 0.05 | 1.6924 | 9.6337 |
| AVISITN*TRTPN | 3 | 1 | 12 | 3 | 8.5658 | 1.8712 | 114 | 4.58 | <.0001 | 0.05 | 4.8588 | 12.2728 |
| AVISITN*TRTPN | 3 | 1 | 12 | 900 | 5.1125 | 1.9530 | 125 | 2.62 | 0.0099 | 0.05 | 1.2472 | 8.9778 |
| AVISITN*TRTPN | 3 | 2 | 3 | 3 | 1.6284 | 1.3777 | 129 | 1.18 | 0.2394 | 0.05 | -1.0974 | 4.3541 |
| AVISITN*TRTPN | 3 | 2 | 3 | 900 | 1.6434 | 1.4525 | 134 | 1.13 | 0.2599 | 0.05 | -1.2295 | 4.5163 |
| AVISITN*TRTPN | 3 | 2 | 6 | 1 | 8.0404 | 1.7049 | 124 | 4.72 | <.0001 | 0.05 | 4.6659 | 11.4150 |
| AVISITN*TRTPN | 3 | 2 | 6 | 2 | 3.4260 | 1.2536 | 60.5 | 2.73 | 0.0082 | 0.05 | 0.9188 | 5.9333 |
| AVISITN*TRTPN | 3 | 2 | 6 | 3 | 5.0671 | 1.5887 | 127 | 3.19 | 0.0018 | 0.05 | 1.9232 | 8.2110 |
| AVISITN*TRTPN | 3 | 2 | 6 | 900 | 4.3087 | 1.6063 | 128 | 2.68 | 0.0083 | 0.05 | 1.1303 | 7.4871 |
| AVISITN*TRTPN | 3 | 2 | 10 | 1 | 12.0032 | 1.8070 | 117 | 6.64 | <.0001 | 0.05 | 8.4247 | 15.5817 |
| AVISITN*TRTPN | 3 | 2 | 10 | 2 | 7.6086 | 1.3510 | 55.3 | 5.63 | <.0001 | 0.05 | 4.9015 | 10.3158 |
| AVISITN*TRTPN | 3 | 2 | 10 | 3 | 6.7564 | 1.6802 | 105 | 4.02 | 0.0001 | 0.05 | 3.4250 | 10.0877 |
| AVISITN*TRTPN | 3 | 2 | 10 | 900 | 5.8035 | 1.7189 | 125 | 3.38 | 0.0010 | 0.05 | 2.4017 | 9.2053 |
| AVISITN*TRTPN | 3 | 2 | 12 | 1 | 12.7179 | 1.7404 | 124 | 7.31 | <.0001 | 0.05 | 9.2731 | 16.1628 |
| AVISITN*TRTPN | 3 | 2 | 12 | 2 | 7.4761 | 1.6156 | 56.9 | 4.63 | <.0001 | 0.05 | 4.2407 | 10.7114 |
| AVISITN*TRTPN | 3 | 2 | 12 | 3 | 10.3788 | 1.7993 | 99.3 | 5.77 | <.0001 | 0.05 | 6.8087 | 13.9489 |
| AVISITN*TRTPN | 3 | 2 | 12 | 900 | 6.9255 | 1.8837 | 114 | 3.68 | 0.0004 | 0.05 | 3.1938 | 10.6572 |

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10 FINAL

BREXPIPRAZOLE 16 OF 20 PROTOCOL 331-201-00061

 $$\tt STAT-4.10$  Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Intent to Treat Sample)

### The Mixed Procedure

## Differences of Least Squares Means

| | Analysis | Planned | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | Treatment | Visit | Treatment | | Standard | | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 3 | 3 | 3 | 900 | 0.01508 | 1.4057 | 147 | 0.01 | 0.9915 | 0.05 | -2.7629 | 2.7930 |
| AVISITN*TRTPN | 3 | 3 | 6 | 1 | 6.4121 | 1.6647 | 121 | 3.85 | 0.0002 | 0.05 | 3.1163 | 9.7078 |
| AVISITN*TRTPN | 3 | 3 | 6 | 2 | 1.7977 | 1.6434 | 113 | 1.09 | 0.2763 | 0.05 | -1.4582 | 5.0536 |
| AVISITN*TRTPN | 3 | 3 | 6 | 3 | 3.4388 | 1.0907 | 64.2 | 3.15 | 0.0025 | 0.05 | 1.2601 | 5.6175 |
| AVISITN*TRTPN | 3 | 3 | 6 | 900 | 2.6803 | 1.5634 | 131 | 1.71 | 0.0888 | 0.05 | -0.4124 | 5.7731 |
| AVISITN*TRTPN | 3 | 3 | 10 | 1 | 10.3748 | 1.7686 | 113 | 5.87 | <.0001 | 0.05 | 6.8711 | 13.8786 |
| AVISITN*TRTPN | 3 | 3 | 10 | 2 | 5.9803 | 1.6456 | 97.4 | 3.63 | 0.0004 | 0.05 | 2.7143 | 9.2462 |
| AVISITN*TRTPN | 3 | 3 | 10 | 3 | 5.1280 | 1.3490 | 63.4 | 3.80 | 0.0003 | 0.05 | 2.4326 | 7.8234 |
| AVISITN*TRTPN | 3 | 3 | 10 | 900 | 4.1751 | 1.6784 | 122 | 2.49 | 0.0142 | 0.05 | 0.8526 | 7.4977 |
| AVISITN*TRTPN | 3 | 3 | 12 | 1 | 11.0896 | 1.7002 | 120 | 6.52 | <.0001 | 0.05 | 7.7233 | 14.4559 |
| AVISITN*TRTPN | 3 | 3 | 12 | 2 | 5.8477 | 1.8972 | 84.6 | 3.08 | 0.0028 | 0.05 | 2.0753 | 9.6201 |
| AVISITN*TRTPN | 3 | 3 | 12 | 3 | 8.7505 | 1.4373 | 61.3 | 6.09 | <.0001 | 0.05 | 5.8767 | 11.6242 |
| AVISITN*TRTPN | 3 | 3 | 12 | 900 | 5.2971 | 1.8466 | 112 | 2.87 | 0.0049 | 0.05 | 1.6384 | 8.9559 |
| AVISITN*TRTPN | 3 | 900 | 6 | 1 | 6.3970 | 1.7300 | 128 | 3.70 | 0.0003 | 0.05 | 2.9740 | 9.8201 |
| AVISITN*TRTPN | 3 | 900 | 6 | 2 | 1.7826 | 1.7093 | 124 | 1.04 | 0.2990 | 0.05 | -1.6007 | 5.1659 |
| AVISITN*TRTPN | 3 | 900 | 6 | 3 | 3.4237 | 1.6140 | 131 | 2.12 | 0.0358 | 0.05 | 0.2307 | 6.6167 |
| AVISITN*TRTPN | 3 | 900 | 6 | 900 | 2.6653 | 1.0768 | 70.6 | 2.48 | 0.0157 | 0.05 | 0.5180 | 4.8125 |
| AVISITN*TRTPN | 3 | 900 | 10 | 1 | 10.3598 | 1.8306 | 120 | 5.66 | <.0001 | 0.05 | 6.7354 | 13.9841 |
| AVISITN*TRTPN | 3 | 900 | 10 | 2 | 5.9652 | 1.7124 | 105 | 3.48 | 0.0007 | 0.05 | 2.5700 | 9.3604 |
| AVISITN*TRTPN | 3 | 900 | 10 | 3 | 5.1129 | 1.7042 | 110 | 3.00 | 0.0033 | 0.05 | 1.7356 | 8.4903 |
| AVISITN*TRTPN | 3 | 900 | 10 | 900 | 4.1601 | 1.3699 | 72.8 | 3.04 | 0.0033 | 0.05 | 1.4297 | 6.8904 |
| AVISITN*TRTPN | 3 | 900 | 12 | 1 | 11.0745 | 1.7648 | 127 | 6.28 | <.0001 | 0.05 | 7.5823 | 14.5667 |

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10 FINAL

BREXPIPRAZOLE 17 OF 20 PROTOCOL 331-201-00061

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups
(Intent to Treat Sample)

The Mixed Procedure

## Differences of Least Squares Means

| | Analysis | Planned | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | Treatment | Visit | Treatment | | Standard | | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 3 | 900 | 12 | 2 | 5.8326 | 1.9548 | 91.2 | 2.98 | 0.0037 | 0.05 | 1.9497 | 9.7155 |
| AVISITN*TRTPN | 3 | 900 | 12 | 3 | 8.7354 | 1.8216 | 106 | 4.80 | <.0001 | 0.05 | 5.1240 | 12.3467 |
| AVISITN*TRTPN | 3 | 900 | 12 | 900 | 5.2821 | 1.4917 | 69.6 | 3.54 | 0.0007 | 0.05 | 2.3066 | 8.2575 |
| AVISITN*TRTPN | 6 | 1 | 6 | 2 | -4.6144 | 1.9292 | 130 | -2.39 | 0.0182 | 0.05 | -8.4311 | -0.7977 |
| AVISITN*TRTPN | 6 | 1 | 6 | 3 | -2.9733 | 1.8437 | 130 | -1.61 | 0.1092 | 0.05 | -6.6207 | 0.6741 |
| AVISITN*TRTPN | 6 | 1 | 6 | 900 | -3.7318 | 1.8604 | 135 | -2.01 | 0.0469 | 0.05 | -7.4111 | -0.05240 |
| AVISITN*TRTPN | 6 | 1 | 10 | 1 | 3.9628 | 1.2220 | 58.7 | 3.24 | 0.0020 | 0.05 | 1.5172 | 6.4083 |
| AVISITN*TRTPN | 6 | 1 | 10 | 2 | -0.4318 | 1.9321 | 119 | -0.22 | 0.8235 | 0.05 | -4.2574 | 3.3938 |
| AVISITN*TRTPN | 6 | 1 | 10 | 3 | -1.2841 | 1.9233 | 121 | -0.67 | 0.5056 | 0.05 | -5.0919 | 2.5237 |
| AVISITN*TRTPN | 6 | 1 | 10 | 900 | -2.2369 | 1.9577 | 138 | -1.14 | 0.2552 | 0.05 | -6.1079 | 1.6340 |
| AVISITN*TRTPN | 6 | 1 | 12 | 1 | 4.6775 | 1.1544 | 56.8 | 4.05 | 0.0002 | 0.05 | 2.3656 | 6.9894 |
| AVISITN*TRTPN | 6 | 1 | 12 | 2 | -0.5644 | 2.1497 | 110 | -0.26 | 0.7934 | 0.05 | -4.8245 | 3.6957 |
| AVISITN*TRTPN | 6 | 1 | 12 | 3 | 2.3384 | 2.0280 | 123 | 1.15 | 0.2511 | 0.05 | -1.6760 | 6.3527 |
| AVISITN*TRTPN | 6 | 1 | 12 | 900 | -1.1149 | 2.1042 | 134 | -0.53 | 0.5971 | 0.05 | -5.2768 | 3.0469 |
| AVISITN*TRTPN | 6 | 2 | 6 | 3 | 1.6411 | 1.8268 | 126 | 0.90 | 0.3707 | 0.05 | -1.9741 | 5.2562 |
| AVISITN*TRTPN | 6 | 2 | 6 | 900 | 0.8826 | 1.8406 | 131 | 0.48 | 0.6324 | 0.05 | -2.7586 | 4.5238 |
| AVISITN*TRTPN | 6 | 2 | 10 | 1 | 8.5771 | 2.0201 | 129 | 4.25 | <.0001 | 0.05 | 4.5802 | 12.5741 |
| AVISITN*TRTPN | 6 | 2 | 10 | 2 | 4.1826 | 0.9231 | 47 | 4.53 | <.0001 | 0.05 | 2.3255 | 6.0396 |
| AVISITN*TRTPN | 6 | 2 | 10 | 3 | 3.3303 | 1.9069 | 117 | 1.75 | 0.0833 | 0.05 | -0.4460 | 7.1066 |
| AVISITN*TRTPN | 6 | 2 | 10 | 900 | 2.3775 | 1.9401 | 132 | 1.23 | 0.2226 | 0.05 | -1.4602 | 6.2151 |
| AVISITN*TRTPN | 6 | 2 | 12 | 1 | 9.2919 | 1.9608 | 131 | 4.74 | <.0001 | 0.05 | 5.4130 | 13.1707 |
| AVISITN*TRTPN | 6 | 2 | 12 | 2 | 4.0500 | 1.1682 | 46.1 | 3.47 | 0.0012 | 0.05 | 1.6987 | 6.4014 |

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10 FINAL

BREXPIPRAZOLE 18 OF 20 PROTOCOL 331-201-00061

 ${\tt STAT-4.10}\\ {\tt Proc\ Mixed\ Output\ Using\ Heterogeneous\ Variance\ Structure\ for\ Treatment\ Groups}\\ {\tt (Intent\ to\ Treat\ Sample)}\\$ 

------

### The Mixed Procedure

## Differences of Least Squares Means

| | Analysis | Planned | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | Treatment | Visit | Treatment | | Standard | | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 6 | 2 | 12 | 3 | 6.9528 | 2.0123 | 116 | 3.46 | 0.0008 | 0.05 | 2.9672 | 10.9384 |
| AVISITN*TRTPN | 6 | 2 | 12 | 900 | 3.4995 | 2.0874 | 129 | 1.68 | 0.0961 | 0.05 | -0.6303 | 7.6292 |
| AVISITN*TRTPN | 6 | 3 | 6 | 900 | -0.7584 | 1.7545 | 136 | -0.43 | 0.6662 | 0.05 | -4.2282 | 2.7113 |
| AVISITN*TRTPN | 6 | 3 | 10 | 1 | 6.9361 | 1.9378 | 127 | 3.58 | 0.0005 | 0.05 | 3.1014 | 10.7707 |
| AVISITN*TRTPN | 6 | 3 | 10 | 2 | 2.5415 | 1.8286 | 112 | 1.39 | 0.1673 | 0.05 | -1.0816 | 6.1646 |
| AVISITN*TRTPN | 6 | 3 | 10 | 3 | 1.6892 | 0.9099 | 56.3 | 1.86 | 0.0686 | 0.05 | -0.1333 | 3.5118 |
| AVISITN*TRTPN | 6 | 3 | 10 | 900 | 0.7364 | 1.8574 | 133 | 0.40 | 0.6924 | 0.05 | -2.9374 | 4.4101 |
| AVISITN*TRTPN | 6 | 3 | 12 | 1 | 7.6508 | 1.8756 | 130 | 4.08 | <.0001 | 0.05 | 3.9400 | 11.3616 |
| AVISITN*TRTPN | 6 | 3 | 12 | 2 | 2.4089 | 2.0579 | 100 | 1.17 | 0.2445 | 0.05 | -1.6739 | 6.4918 |
| AVISITN*TRTPN | 6 | 3 | 12 | 3 | 5.3117 | 1.2605 | 56.3 | 4.21 | <.0001 | 0.05 | 2.7869 | 7.8365 |
| AVISITN*TRTPN | 6 | 3 | 12 | 900 | 1.8584 | 2.0107 | 128 | 0.92 | 0.3571 | 0.05 | -2.1201 | 5.8368 |
| AVISITN*TRTPN | 6 | 900 | 10 | 1 | 7.6945 | 1.9543 | 130 | 3.94 | 0.0001 | 0.05 | 3.8280 | 11.5610 |
| AVISITN*TRTPN | 6 | 900 | 10 | 2 | 3.2999 | 1.8437 | 116 | 1.79 | 0.0761 | 0.05 | -0.3519 | 6.9518 |
| AVISITN*TRTPN | 6 | 900 | 10 | 3 | 2.4477 | 1.8377 | 121 | 1.33 | 0.1854 | 0.05 | -1.1905 | 6.0858 |
| AVISITN*TRTPN | 6 | 900 | 10 | 900 | 1.4948 | 0.9690 | 64.7 | 1.54 | 0.1278 | 0.05 | -0.4406 | 3.4302 |
| AVISITN*TRTPN | 6 | 900 | 12 | 1 | 8.4092 | 1.8929 | 136 | 4.44 | <.0001 | 0.05 | 4.6658 | 12.1526 |
| AVISITN*TRTPN | 6 | 900 | 12 | 2 | 3.1674 | 2.0707 | 103 | 1.53 | 0.1292 | 0.05 | -0.9393 | 7.2740 |
| AVISITN*TRTPN | 6 | 900 | 12 | 3 | 6.0701 | 1.9469 | 119 | 3.12 | 0.0023 | 0.05 | 2.2151 | 9.9251 |
| AVISITN*TRTPN | 6 | 900 | 12 | 900 | 2.6168 | 1.2111 | 63.6 | 2.16 | 0.0345 | 0.05 | 0.1972 | 5.0365 |
| AVISITN*TRTPN | 10 | 1 | 10 | 2 | -4.3946 | 2.0231 | 120 | -2.17 | 0.0318 | 0.05 | -8.4002 | -0.3890 |
| AVISITN*TRTPN | 10 | 1 | 10 | 3 | -5.2468 | 2.0131 | 122 | -2.61 | 0.0103 | 0.05 | -9.2319 | -1.2618 |
| AVISITN*TRTPN | 10 | 1 | 10 | 900 | -6.1997 | 2.0474 | 132 | -3.03 | 0.0030 | 0.05 | -10.2495 | -2.1499 |

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10 FINAL

BREXPIPRAZOLE 19 OF 20 PROTOCOL 331-201-00061

 ${\tt STAT-4.10}\\ {\tt Proc\ Mixed\ Output\ Using\ Heterogeneous\ Variance\ Structure\ for\ Treatment\ Groups}\\ ({\tt Intent\ to\ Treat\ Sample})$ 

------

Parameter Code=CAPSTOT ------

### The Mixed Procedure

## Differences of Least Squares Means

| | Analysis | Planned | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | Treatment | Visit | Treatment | | Standard | | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 10 | 1 | 12 | 1 | 0.7147 | 0.9557 | 53.1 | 0.75 | 0.4578 | 0.05 | -1.2021 | 2.6316 |
| AVISITN*TRTPN | 10 | 1 | 12 | 2 | -4.5271 | 2.2318 | 114 | -2.03 | 0.0448 | 0.05 | -8.9484 | -0.1059 |
| AVISITN*TRTPN | 10 | 1 | 12 | 3 | -1.6244 | 2.1136 | 124 | -0.77 | 0.4436 | 0.05 | -5.8077 | 2.5590 |
| AVISITN*TRTPN | 10 | 1 | 12 | 900 | -5.0777 | 2.1878 | 133 | -2.32 | 0.0218 | 0.05 | -9.4051 | -0.7503 |
| AVISITN*TRTPN | 10 | 2 | 10 | 3 | -0.8523 | 1.9095 | 104 | -0.45 | 0.6563 | 0.05 | -4.6386 | 2.9341 |
| AVISITN*TRTPN | 10 | 2 | 10 | 900 | -1.8051 | 1.9428 | 119 | -0.93 | 0.3547 | 0.05 | -5.6521 | 2.0419 |
| AVISITN*TRTPN | 10 | 2 | 12 | 1 | 5.1093 | 1.9638 | 120 | 2.60 | 0.0104 | 0.05 | 1.2213 | 8.9974 |
| AVISITN*TRTPN | 10 | 2 | 12 | 2 | -0.1325 | 1.2117 | 46.4 | -0.11 | 0.9134 | 0.05 | -2.5710 | 2.3059 |
| AVISITN*TRTPN | 10 | 2 | 12 | 3 | 2.7702 | 2.0144 | 107 | 1.38 | 0.1720 | 0.05 | -1.2232 | 6.7636 |
| AVISITN*TRTPN | 10 | 2 | 12 | 900 | -0.6831 | 2.0899 | 119 | -0.33 | 0.7443 | 0.05 | -4.8213 | 3.4550 |
| AVISITN*TRTPN | 10 | 3 | 10 | 900 | -0.9528 | 1.9367 | 124 | -0.49 | 0.6236 | 0.05 | -4.7862 | 2.8805 |
| AVISITN*TRTPN | 10 | 3 | 12 | 1 | 5.9616 | 1.9535 | 121 | 3.05 | 0.0028 | 0.05 | 2.0942 | 9.8290 |
| AVISITN*TRTPN | 10 | 3 | 12 | 2 | 0.7197 | 2.1298 | 101 | 0.34 | 0.7361 | 0.05 | -3.5052 | 4.9446 |
| AVISITN*TRTPN | 10 | 3 | 12 | 3 | 3.6225 | 1.2008 | 57.5 | 3.02 | 0.0038 | 0.05 | 1.2182 | 6.0267 |
| AVISITN*TRTPN | 10 | 3 | 12 | 900 | 0.1691 | 2.0841 | 124 | 0.08 | 0.9354 | 0.05 | -3.9559 | 4.2942 |
| AVISITN*TRTPN | 10 | 900 | 12 | 1 | 6.9144 | 1.9887 | 137 | 3.48 | 0.0007 | 0.05 | 2.9818 | 10.8471 |
| AVISITN*TRTPN | 10 | 900 | 12 | 2 | 1.6726 | 2.1595 | 110 | 0.77 | 0.4403 | 0.05 | -2.6070 | 5.9521 |
| AVISITN*TRTPN | 10 | 900 | 12 | 3 | 4.5753 | 2.0405 | 123 | 2.24 | 0.0267 | 0.05 | 0.5364 | 8.6142 |
| AVISITN*TRTPN | 10 | 900 | 12 | 900 | 1.1220 | 0.9007 | 58.8 | 1.25 | 0.2178 | 0.05 | -0.6804 | 2.9244 |
| AVISITN*TRTPN | 12 | 1 | 12 | 2 | -5.2419 | 2.1786 | 112 | -2.41 | 0.0178 | 0.05 | -9.5587 | -0.9251 |
| AVISITN*TRTPN | 12 | 1 | 12 | 3 | -2.3391 | 2.0564 | 123 | -1.14 | 0.2575 | 0.05 | -6.4097 | 1.7314 |
| AVISITN*TRTPN | 12 | 1 | 12 | 900 | -5.7924 | 2.1332 | 135 | -2.72 | 0.0075 | 0.05 | -10.0113 | -1.5735 |

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10 FINAL

BREXPIPRAZOLE 20 OF 20 PROTOCOL 331-201-00061

# STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Intent to Treat Sample)

#### The Mixed Procedure

## Differences of Least Squares Means

| Ef | fect | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| AV | ISITN*TRTPN | 12 | 2 | 12 | 3 | 2.9027 | 2.2253 | 104 | 1.30 | 0.1950 | 0.05 | -1.5100 | 7.3155 |
| AV | ISITN*TRTPN | 12 | 2 | 12 | 900 | -0.5506 | 2.2925 | 116 | -0.24 | 0.8106 | 0.05 | -5.0912 | 3.9901 |
| AV | ISITN*TRTPN | 12 | 3 | 12 | 900 | -3.4533 | 2.1810 | 125 | -1.58 | 0.1159 | 0.05 | -7.7697 | 0.8631 |

## Tests of Effect Slices

| Effect | Analysis<br>Visit<br>(N) | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---|---|---|---|---|---|
| AVISITN*TRTPN | 3 | 3 | 152 | 0.69 | 0.5588 |
| AVISITN*TRTPN | 6 | 3 | 145 | 2.14 | 0.0973 |
| AVISITN*TRTPN | 10 | 3 | 131 | 3.47 | 0.0181 |
| AVISITN*TRTPN | 12 | 3 | 131 | 3.15 | 0.0271 |

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-4.10 FINAL

BREXPIPRAZOLE 1 OF 14 PROTOCOL 331-201-00061 Proc Mixed Output for Change in CGI-S Scale, MMRM (UN) (Intent to Treat Sample) ------- Parameter Code=CGI0101 -------The Mixed Procedure Model Information WORK.INDATA Data Set Dependent Variable CHG Dependent Variable Covariance Structure Unstructured Subject Effect SUBJID Estimation Method REML Residual Variance Method Fixed Effects SE Method Kenward-Roger Degrees of Freedom Method Kenward-Roger Class Level Information Class Levels Values 7 2 3 4 6 8 10 12 AVISITN 1 2 3 900 TRTPN 4 POOLCNTR 10 COMBFL 2 NY

SOURCE: MMRMOUT; TABLE: statlcgisa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.1 FINAL



SOURCE: MMRMOUT; TABLE: stat1cgisa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.1 FINAL



The Mixed Procedure



SOURCE: MMRMOUT; TABLE: stat1cgisa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.1 FINAL



The Mixed Procedure



SOURCE: MMRMOUT; TABLE: stat1cgisa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.1 FINAL



The Mixed Procedure



SOURCE: MMRMOUT; TABLE: stat1cgisa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.1 FINAL

BREXPIPRAZOLE 6 OF 14 PROTOCOL 331-201-00061 Proc Mixed Output for Change in CGI-S Scale, MMRM (UN) (Intent to Treat Sample) The Mixed Procedure Dimensions Covariance Parameters 28 59 Columns in X Columns in Z Subjects 307 Max Obs per Subject Number of Observations 1835 Number of Observations Read Number of Observations Used

Number of Observations Not Used

SOURCE: MMRMOUT; TABLE: statlcgisa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.1 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | 7 OF 14 |
|---|---|---|---|---|---|---|
| Parameter Code=CGI0101 | | | | | | |
| The Mixed Procedure | | | | | | |
| | | Iter | ation Hist | cory | | |
| | Iteration | Evaluations | -2 Res | Log Like | Criterion | |
| | 0 | 1 2 | | 38437141 | 0.00203330 | |
| | 2 | 1 | | 47643679 | 0.00203330 | |
| | 3 | 1 | | 47157376 | 0.00000000 | |
| | | Converge | ence criter | ria met. | | |
| | | Covariance | Parameter | Estimates | | |
| | | Cov Parm | Subject | Estimate | | |
| | | UN(1,1) | SUBJID | 0.3388 | | |
| | | UN(2,1) | SUBJID | 0.1749 | | |
| | | UN(2,2)<br>UN(3,1) | SUBJID<br>SUBJID | 0.5893<br>0.2131 | | |
| | | UN (3,1)<br>UN (3,2) | SUBJID | 0.4334 | | |
| | | UN (3, 3) | SUBJID | 0.8444 | | |
| | | UN (4,1) | SUBJID | 0.1604 | | |
| | | UN (4,2) | SUBJID | 0.4051 | | |

SOURCE: MMRMOUT; TABLE: statlcgisa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.1 FINAL

BREXPIPRAZOLE 8 OF 14 PROTOCOL 331-201-00061 Proc Mixed Output for Change in CGI-S Scale, MMRM (UN) (Intent to Treat Sample) The Mixed Procedure Covariance Parameter Estimates Cov Parm Subject Estimate UN(4,3) SUBJID 0.5940 UN (4,4) SUBJID 0.9222 UN(5,1) SUBJID 0.2120 UN(5,2) SUBJID 0.4086 UN(5,3)SUBJID 0.6034 UN(5,4) SUBJID 0.7293 SUBJID UN(5,5) 0.9313 UN(6,1) SUBJID 0.1658 UN(6,2) SUBJID 0.3241 UN(6,3) SUBJID 0.5341 UN(6,4) SUBJID 0.6845 UN(6,5) SUBJID 0.6721 UN(6,6) SUBJID 0.9841 UN(7,1) 0.1713 SUBJID UN(7,2) 0.3593 SUBJID UN(7,3) SUBJID 0.5630 UN(7,4) SUBJID 0.6681 UN(7,5) SUBJID 0.6294

SUBJID

SUBJID

0.8219

1.1546

SOURCE: MMRMOUT; TABLE: statlcgisa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.1 FINAL

UN(7,6)

UN(7,7)

BREXPIPRAZOLE 9 OF 14 PROTOCOL 331-201-00061 Proc Mixed Output for Change in CGI-S Scale, MMRM (UN) (Intent to Treat Sample) The Mixed Procedure Fit Statistics 3735.5 -2 Res Log Likelihood AIC (Smaller is Better) AICC (Smaller is Better) -2 Res Log Likelihood 3791.5 3792.4 BIC (Smaller is Better) 3895.8 Null Model Likelihood Ratio Test Chi-Square Pr > ChiSq 1115.91 <.0001 Type 3 Tests of Fixed Effects Num Den Effect DF DF F Value Pr > F 247 AVISITN 6 0.71 0.6401 3 290 2.52 0.0585 TRTPN 18 AVISITN\*TRTPN 497 1.41 0.1204 POOLCNTR 9 293 1.95 0.0456 COMBFL 291 2.54 0.1120

SOURCE: MMRMOUT; TABLE: statlcgisa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.1 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-0006 | 31 | | | | | | | | 10 OF | 14 |
|---|---|---|---|---|---|---|---|---|---|---|
| 11010001 331 201 0000 | | | α). | S | TAT-5.1 | | | | | |
| | Proc Mi | xed Output fo | | Intent t | o Treat Sa | | CGI-S Scale | , MMRM (UN) | | |
| | | | ; | Paramete | r Code=CGI | 0101 | | | | |
| | | | | The Mix | ed Procedu | re | | | | |
| | | | Type | 3 Tests | of Fixed | Effects | | | | |
| | | Ef | fect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| | | BAS | SE*AVISITN | 7 | 256 | 10.55 | <.0001 | | | |
| | | | | Es | timates | | | | | |
| | | | Standard | | | | | | | |
| | Label | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper | |
| | WEEK2 1 vs 900<br>WEEK3 1 vs 900 | -0.1186 | 0.09390 | 287 | -1.26 | 0.2077 | 0.05 | -0.3034 | 0.06624 | |
| | WEEK3 1 vs 900<br>WEEK4 1 vs 900 | -0.08376<br>-0.1233 | 0.1237<br>0.1491 | 291<br>286 | -0.68<br>-0.83 | 0.4989 | 0.05 | -0.3272<br>-0.4168 | 0.1597<br>0.1703 | |
| | WEEK6 1 vs 900 | -0.1233 | 0.1491 | 277 | -1.70 | 0.4092 | 0.05 | -0.5839 | 0.1703 | |
| | WEEK8 1 vs 900 | -0.4141 | 0.1607 | 277 | -2.58 | 0.0105 | 0.05 | -0.7304 | -0.09771 | |
| | WEEK10 1 vs 900 | -0.4733 | 0.1694 | 263 | -2.79 | 0.0056 | 0.05 | -0.8070 | -0.1397 | |
| | WEEK12 1 vs 900 | -0.4096 | 0.1870 | 255 | -2.19 | 0.0294 | 0.05 | -0.7778 | -0.04144 | |
| | WEEK2 1 vs 2 | -0.1588 | 0.09687 | 287 | -1.64 | 0.1023 | 0.05 | -0.3494 | 0.03190 | |
| | WEEK3 1 vs 2 | -0.2260 | 0.1286 | 295 | -1.76 | 0.0799 | 0.05 | -0.4791 | 0.02711 | |
| | WEEK4 1 vs 2 | -0.2073 | 0.1543 | 287 | -1.34 | 0.1801 | 0.05 | -0.5110 | 0.09634 | |
| | WEEK6 1 vs 2 | -0.3450 | 0.1665 | 284 | -2.07 | 0.0391 | 0.05 | -0.6727 | -0.01740 | |
| | WEEK8 1 vs 2 | -0.4495 | 0.1684 | 287 | -2.67 | 0.0080 | 0.05 | -0.7809 | -0.1181 | |

SOURCE: MMRMOUT; TABLE: stat1cgisa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.1 FINAL

| BREXPIPRAZOLE | 11 OF 14 |
|------------------------|----------|

Proc Mixed Output for Change in CGI-S Scale, MMRM (UN)

(Intent to Treat Sample)

\_\_\_\_\_

------ Parameter Code=CGI0101 ------

## The Mixed Procedure

#### Estimates

| | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| WEEK10 1 vs 2 | -0.2599 | 0.1791 | 273 | -1.45 | 0.1480 | 0.05 | -0.6125 | 0.09274 |
| WEEK12 1 vs 2 | -0.3038 | 0.1977 | 261 | -1.54 | 0.1257 | 0.05 | -0.6932 | 0.08557 |
| WEEK2 1 vs 3 | -0.1143 | 0.09458 | 286 | -1.21 | 0.2279 | 0.05 | -0.3005 | 0.07187 |
| WEEK3 1 vs 3 | -0.09081 | 0.1254 | 293 | -0.72 | 0.4695 | 0.05 | -0.3376 | 0.1559 |
| WEEK4 1 vs 3 | -0.06095 | 0.1512 | 288 | -0.40 | 0.6872 | 0.05 | -0.3585 | 0.2366 |
| WEEK6 1 vs 3 | -0.2176 | 0.1631 | 283 | -1.33 | 0.1832 | 0.05 | -0.5385 | 0.1034 |
| WEEK8 1 vs 3 | -0.5563 | 0.1647 | 284 | -3.38 | 0.0008 | 0.05 | -0.8805 | -0.2321 |
| WEEK10 1 vs 3 | -0.4159 | 0.1727 | 264 | -2.41 | 0.0167 | 0.05 | -0.7559 | -0.07594 |
| WEEK12 1 vs 3 | -0.2245 | 0.1908 | 257 | -1.18 | 0.2405 | 0.05 | -0.6004 | 0.1513 |
| WEEK2 2 vs 900 | 0.04019 | 0.09654 | 287 | 0.42 | 0.6775 | 0.05 | -0.1498 | 0.2302 |
| WEEK3 2 vs 900 | 0.1422 | 0.1275 | 292 | 1.12 | 0.2656 | 0.05 | -0.1087 | 0.3932 |
| WEEK4 2 vs 900 | 0.08409 | 0.1532 | 285 | 0.55 | 0.5834 | 0.05 | -0.2174 | 0.3856 |
| WEEK6 2 vs 900 | 0.07481 | 0.1637 | 277 | 0.46 | 0.6480 | 0.05 | -0.2474 | 0.3970 |
| WEEK8 2 vs 900 | 0.03542 | 0.1654 | 280 | 0.21 | 0.8306 | 0.05 | -0.2901 | 0.3610 |
| WEEK10 2 vs 900 | -0.2135 | 0.1766 | 272 | -1.21 | 0.2278 | 0.05 | -0.5612 | 0.1342 |
| WEEK12 2 vs 900 | -0.1058 | 0.1946 | 260 | -0.54 | 0.5869 | 0.05 | -0.4889 | 0.2773 |
| WEEK2 3 vs 900 | -0.00429 | 0.09405 | 286 | -0.05 | 0.9637 | 0.05 | -0.1894 | 0.1808 |
| WEEK3 3 vs 900 | 0.007051 | 0.1243 | 290 | 0.06 | 0.9548 | 0.05 | -0.2376 | 0.2517 |
| WEEK4 3 vs 900 | -0.06230 | 0.1502 | 286 | -0.41 | 0.6785 | 0.05 | -0.3579 | 0.2333 |
| WEEK6 3 vs 900 | -0.05266 | 0.1606 | 278 | -0.33 | 0.7432 | 0.05 | -0.3688 | 0.2635 |

SOURCE: MMRMOUT; TABLE: statlcgisa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.1 FINAL

| BREXPIPRAZOLE | | | | | | | | | 12 | OF 14 | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | Proc M | lixed Output | | ST | AT-5.1 Treat Sam | | CGI-S Scale, | MMRM (UN) | | | |
| | | | | Parameter | Code=CGIO | 101 | | | | | · |
| | | | | The Mixe | d Procedur | е | | | | | |
| | | | | Est | imates | | | | | | |
| Lak | el | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper | | |
| | 0.00 | 0.1422<br>-0.05741<br>-0.1851 | 0.1618<br>0.1706<br>0.1880 | 278<br>264<br>255 | 0.88<br>-0.34<br>-0.98 | 0.3803<br>0.7368<br>0.3259 | 0.05<br>0.05<br>0.05 | -0.1764<br>-0.3934<br>-0.5554 | 0.4608<br>0.2786<br>0.1852 | | |
| | | | | Least Sq | uares Mean | s | | | | | |
| Effect | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | | t Value | Pr > t | Alpha | Lower | Upper | |
| AVISITN*TRTPN | 2<br>2<br>2<br>2<br>3<br>3<br>3<br>3<br>4 | 1<br>2<br>3<br>900<br>1<br>2<br>3<br>900<br>1 | -0.3731<br>-0.2144<br>-0.2588<br>-0.2546<br>-0.5670<br>-0.3410<br>-0.4761<br>-0.4832<br>-0.8222 | 0.07074<br>0.07585<br>0.07162<br>0.07118<br>0.09140<br>0.09777<br>0.09266<br>0.09045<br>0.1088 | 300<br>296<br>301<br>314<br>321<br>314<br>311 | -5.27<br>-2.83<br>-3.61<br>-3.58<br>-6.20<br>-3.49<br>-5.14<br>-5.34<br>-7.55 | <.0001<br>0.0050<br>0.0004<br>0.0004<br><.0001<br>0.0006<br><.0001<br><.0001<br><.0001 | 0.05 | -0.5123<br>-0.3636<br>-0.3998<br>-0.3946<br>-0.7468<br>-0.5333<br>-0.6585<br>-0.6612<br>-1.0364 | -0.2339<br>-0.06509<br>-0.1179<br>-0.1145<br>-0.3871<br>-0.1486<br>-0.2938<br>-0.3052<br>-0.6080 | |

SOURCE: MMRMOUT; TABLE: statlcgisa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.1 FINAL


Proc Mixed Output for Change in CGI-S Scale, MMRM (UN)

(Intent to Treat Sample)

\_\_\_\_\_\_

The Mixed Procedure

Least Squares Means

| Effect | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN | 4 | 2 | -0.6149 | 0.1154 | 311 | -5.33 | <.0001 | 0.05 | -0.8419 | -0.3879 |
| AVISITN*TRTPN | 4 | 3 | -0.7613 | 0.1107 | 309 | -6.88 | <.0001 | 0.05 | -0.9790 | -0.5435 |
| AVISITN*TRTPN | 4 | 900 | -0.6990 | 0.1079 | 304 | -6.48 | <.0001 | 0.05 | -0.9112 | -0.4867 |
| AVISITN*TRTPN | 6 | 1 | -1.0538 | 0.1169 | 298 | -9.01 | <.0001 | 0.05 | -1.2838 | -0.8237 |
| AVISITN*TRTPN | 6 | 2 | -0.7087 | 0.1241 | 310 | -5.71 | <.0001 | 0.05 | -0.9529 | -0.4646 |
| AVISITN*TRTPN | 6 | 3 | -0.8362 | 0.1191 | 305 | -7.02 | <.0001 | 0.05 | -1.0705 | -0.6019 |
| AVISITN*TRTPN | 6 | 900 | -0.7835 | 0.1137 | 289 | -6.89 | <.0001 | 0.05 | -1.0073 | -0.5598 |
| AVISITN TRITN AVISITN*TRTPN | 8 | 1 | -1.4308 | 0.1137 | 299 | -12.11 | <.0001 | 0.05 | -1.6633 | -1.1983 |
| AVISITN TRITN AVISITN*TRTPN | 8 | 2 | -0.9813 | 0.1255 | 314 | -7.82 | <.0001 | 0.05 | -1.2283 | -0.7343 |
| AVISITN TRITN AVISITN*TRTPN | 8 | 3 | -0.8745 | 0.1201 | 303 | -7.28 | <.0001 | 0.05 | -1.1108 | -0.6382 |
| AVISITN*TRTPN AVISITN*TRTPN | 8 | 900 | -1.0167 | 0.1201 | 290 | -8.88 | <.0001 | 0.05 | -1.2420 | -0.7915 |
| AVISITN*TRTPN | 10 | 1 | -1.3465 | 0.1144 | 276 | -10.89 | <.0001 | 0.05 | -1.5899 | -1.1031 |
| | | 1 | | | | | | | | |
| AVISITN*TRTPN | 10 | 2 | -1.0866 | 0.1346 | 303 | -8.07 | <.0001 | 0.05 | -1.3516 | -0.8217 |
| AVISITN*TRTPN | 10 | 3 | -0.9306 | 0.1257 | 282 | -7.40 | <.0001 | 0.05 | -1.1780 | -0.6831 |
| AVISITN*TRTPN | 10 | 900 | -0.8732 | 0.1209 | 279 | -7.22 | <.0001 | 0.05 | -1.1111 | -0.6352 |
| AVISITN*TRTPN | 12 | 1 | -1.4426 | 0.1363 | 268 | -10.58 | <.0001 | 0.05 | -1.7111 | -1.1742 |
| AVISITN*TRTPN | 12 | 2 | -1.1388 | 0.1478 | 285 | -7.71 | <.0001 | 0.05 | -1.4297 | -0.8479 |
| AVISITN*TRTPN | 12 | 3 | -1.2181 | 0.1382 | 272 | -8.82 | <.0001 | 0.05 | -1.4901 | -0.9461 |
| AVISITN*TRTPN | 12 | 900 | -1.0330 | 0.1325 | 268 | -7.79 | <.0001 | 0.05 | -1.2939 | -0.7721 |

SOURCE: MMRMOUT; TABLE: statlcgisa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.1 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | Proc Mixed Output for Chan | ige | STAT-5.1<br>to Treat | Sample) | | 14 OF 14<br>S Scale, MMRM (UN) |
|---|---|---|---|---|---|---|
| | | The Mi | xed Proce | edure | | |
| | | Analysis | f Effect | | | |
| | Effect | Visit<br>(N) | Num<br>DF | Den<br>DF | F Value | Pr > F |
| | AVISITN*TRTPN | 2<br>3<br>4<br>6<br>8<br>10<br>12 | 3<br>3<br>3<br>3<br>3<br>3 | 286<br>293<br>286<br>280<br>282<br>268<br>258 | 1.02<br>1.05<br>0.66<br>1.63<br>4.41<br>3.08<br>1.70 | 0.3838<br>0.3725<br>0.5772<br>0.1816<br>0.0047<br>0.0282<br>0.1682 |

SOURCE: MMRMOUT; TABLE: stat1cgisa.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.1 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 Pro | c GLM Output for | Change | STAT-5.2 in CGI-S Scale (Intent to Treat Sample) | 1 OF 6 |
|---|---|---|---|---|
| | Pa | arameter Co | de=CGI0101 Analysis Visit (N)=10 | |
| | | | The GLM Procedure | |
| | | Cl | ass Level Information | |
| | Class | Levels | Values | |
| | TRTPN | 4 | 1 2 3 900 | |
| | POOLCNTR | 10 | | |
| | COMBFL | 2 | N Y | |
| | | | Observations Read 308 Observations Used 308 | |

SOURCE: GLMOUT; TABLE: statlcgisb.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.2 FINAL

|---|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | STAT-5.2 Proc GLM Output for Change (Intent to Treat Sample) | | | | | cale, LOCF |
| | Paı | | 0101 Analys: | | | |
| | Depe | endent Variable: | CHG Chan | ge from Baselin | Э | |
| | Source | DF | Sum of<br>Squares | Mean Square | F Value | Pr > F |
| | Model | 14 72 | .4586988 | 5.1756213 | 5.54 | <.0001 |
| | Error | 293 273 | .4893531 | 0.9334108 | | |
| | Corrected Total | 307 345 | .9480519 | | | |
| | R-Squa | | | | | |
| | Source | DF Typ | e III SS | Mean Square | F Value | Pr > F |
| | TRTPN POOLCNTR COMBFL BASE | 9 14.<br>1 0. | 04613251<br>38413891<br>22842769<br>63627421 | 3.01537750<br>1.59823766<br>0.22842769<br>41.63627421 | 3.23<br>1.71<br>0.24<br>44.61 | 0.0228<br>0.0857<br>0.6212<br><.0001 |

SOURCE: GLMOUT; TABLE: statlcgisb.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.2 FINAL


Proc GLM Output for Change in CGI-S Scale, LOCF (Intent to Treat Sample)

\_\_\_\_\_

## The GLM Procedure

| Level of | | CHC | 3 | BAS | BASE |
|----------|-----|-------------|------------|------------|------------|
| TRTPN | N | Mean | Std Dev | Mean | Std Dev |
| 1 | 7.0 | -1.27848101 | 1 00704202 | 4.41772152 | 0 05046054 |
| 1 | 79 | -1.2/848101 | 1.09704392 | 4.41//2152 | 0.85646254 |
| 2 | 72 | -0.91666667 | 1.05816743 | 4.26388889 | 1.03451772 |
| 3 | 77 | -0.88311688 | 1.02564519 | 4.37662338 | 0.97385508 |
| 900 | 80 | -0.86250000 | 1.02800963 | 4.37500000 | 0.81714229 |

SOURCE: GLMOUT; TABLE: statlcgisb.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.2 FINAL

|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | | | STAT-5.2 | | |
| | Proc GLM Output for ( | | ent to Treat Sam | ple) | in CGI-S Scale, LOCF |
| | | - Parameter Code= | -CGI0101 Analysi | s Visit (N)=1 | .0 |
| | | | ne GLM Procedure<br>ast Squares Mean | | |
| | | 100 | Standard | .5 | LSMEAN |
| | TRTPN | CHG LSMEAN | Error | Pr > t | Number |
| | 1 | -1.25672434 | 0.11660319 | <.0001 | 1 |
| | 2 3 | -0.93411448<br>-0.84629828 | 0.12539640<br>0.11943530 | <.0001<br><.0001 | 2 3 |
| | 900 | -0.83938241 | 0.11714733 | <.0001 | 4 |
| | | | res Means for ef<br>or H0: LSMean(i) | | |
| | | Depen | ndent Variable: | CHG | |
| | i/j | 1 | 2 | 3 | 4 |
| | 1 | 0.0400 | 0.0429 | 0.0088 | 0.0070 |
| | 2 3 | 0.0429<br>0.0088 | 0.5824 | 0.5824 | 0.5484<br>0.9643 |
| | 4 | 0.0070 | 0.5484 | 0.9643 | |

SOURCE: GLMOUT; TABLE: statlcgisb.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.2 FINAL

BREXPIPRAZOLE 5 OF 6 PROTOCOL 331-201-00061 STAT-5.2 Proc GLM Output for Change in CGI-S Scale, LOCF (Intent to Treat Sample) The GLM Procedure Least Squares Means TRTPN CHG LSMEAN 95% Confidence Limits 1 -1.256724 -1.486210 -1.027238 2 -0.934114 -1.180906 -0.687323 -0.846298 -1.081358 -0.611238 900 -0.839382 -1.069939 -0.608826 Least Squares Means for Effect TRTPN Difference Between 95% Confidence Limits for i j Means LSMean(i)-LSMean(j) -0.322610 -0.634789 -0.010430 -0.410426 -0.716610 -0.104242 -0.417342 -0.719558 -0.115126 1 4 2 3 -0.087816 -0.401810 0.226177 -0.094732 -0.405045 0.215581 2 4 3 -0.006916 -0.310973 0.297141

NOTE: To ensure overall protection level, only probabilities associated with pre-planned comparisons should be used.

SOURCE: GLMOUT; TABLE: statlcgisb.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.2 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | Proc GLM Output for Change | STAT-<br>(Intent to Tr | | in C | GI-S Scale, LOCF | 6 OF 6 |
|---|---|---|---|---|---|---|
| | Para | meter Code=CGI0101<br>The GLM Pr | - | (N)=10 | | |
| | Deper | dent Variable: CHG | Change from E | Baseline | | |
| | Parameter | Estimate | Standard<br>Error | t Value | Pr > t | |
| | 1 vs 900<br>1 vs 3<br>1 vs 2<br>2 vs 900<br>3 vs 900 | -0.41734192<br>-0.41042606<br>-0.32260986<br>-0.09473206<br>-0.00691586 | 0.15355755<br>0.15557404<br>0.15862022<br>0.15767173<br>0.15449314 | -2.72<br>-2.64<br>-2.03<br>-0.60<br>-0.04 | 0.0070<br>0.0088<br>0.0429<br>0.5484<br>0.9643 | |

SOURCE: GLMOUT; TABLE: statlcgisb.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.2 FINAL
BREXPIPRAZOLE 1 OF 6 PROTOCOL 331-201-00061 Proc GLM Output for Change in CGI-S Scale, OC (Intent to Treat Sample) The GLM Procedure Class Level Information Levels Values Class TRTPN 4 1 2 3 900 308 Number of Observations Read Number of Observations Used 308

SOURCE: GLMOUT; TABLE: statlcgisc.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.3 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | Proc GLM Output for | Change | TAT-5.3 in Treat Sample) | CGI-S Scale | 2 OF 6<br>, OC |
|---|---|---|---|---|---|
| | Par | | - | ) | |
| | | | M Procedure | | |
| | Depe | ndent Variable: ( | CHG Change from Baselin | ne | |
| | Source | DF | Sum of<br>Squares Mean Square | F Value | Pr > F |
| | Model | 4 57. | 6739577 14.4184894 | 15.16 | <.0001 |
| | Error | 303 288. | 2740942 0.9513997 | | |
| | Corrected Total | 307 345. | 9480519 | | |
| | R-Squa<br>0.1667 | | | | |
| | Source | DF Type | III SS Mean Square | F Value | Pr > F |
| | TRTPN<br>BASE | | 8612564 2.66204188<br>3487543 48.53487543 | 2.80<br>51.01 | 0.0403<br><.0001 |

SOURCE: GLMOUT; TABLE: statlcgisc.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.3 FINAL


Proc GLM Output for Change in CGI-S Scale, OC

\_\_\_\_\_

### The GLM Procedure

| Level of | | CH0 | 3 | BA | SE |
|----------|----|-------------|------------|------------|------------|
| TRTPN | N | Mean | Std Dev | Mean | Std Dev |
| 1 | 79 | -1.27848101 | 1.09704392 | 4.41772152 | 0.85646254 |
| 2 | 72 | -0.91666667 | 1.05816743 | 4.26388889 | 1.03451772 |
| 3 | 77 | -0.88311688 | 1.02564519 | 4.37662338 | 0.97385508 |
| 900 | 80 | -0.86250000 | 1.02800963 | 4.37500000 | 0.81714229 |

SOURCE: GLMOUT; TABLE: statlcgisc.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.3 FINAL

|---|---|---|---|---|---|
| PROTOCOL 331-201-00061 | Proc GLM Output | | STAT-5.3 | | CGI-S Scale, OC |
| | | Parameter Code= | CGI0101 Analysi | s Visit (N)=1 | 0 |
| | | | e GLM Procedure<br>st Squares Mear | | |
| | | | Standard | | LSMEAN |
| | TRTPN | CHG LSMEAN | Error | Pr > t | Number |
| | 1 | -1.25361599 | 0.10979596 | <.0001 | 1 |
| | 2 | -0.95851933 | 0.11510091 | <.0001 | 2 |
| | 3 | -0.87607625 | 0.11116120 | <.0001 | 3 |
| | 900 | -0.85616343 | 0.10905633 | <.0001 | 4 |
| | | | res Means for ef<br>or HO: LSMean(i) | | |
| | | Depen | dent Variable: | CHG | |
| | i/j | 1 | 2 | 3 | 4 |
| | 1 | 0.0640 | 0.0648 | 0.0163 | 0.0107 |
| | 2 | 0.0648 | 0.000 | 0.6069 | 0.5192 |
| | 3 | 0.0163 | 0.6069 | 0 0000 | 0.8983 |
| | 4 | 0.0107 | 0.5192 | 0.8983 | |

SOURCE: GLMOUT; TABLE: statlcgisc.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.3 FINAL

BREXPIPRAZOLE 5 OF 6 PROTOCOL 331-201-00061 Proc GLM Output for Change in CGI-S Scale, OC (Intent to Treat Sample) The GLM Procedure Least Squares Means TRTPN CHG LSMEAN 95% Confidence Limits 1 -1.253616 -1.469675 -1.037557 2 -0.958519 -1.185018 -0.732021 -0.876076 -1.094822 -0.657331 900 -0.856163 -1.070767 -0.641560 Least Squares Means for Effect TRTPN Difference Between 95% Confidence Limits for j i Means LSMean(i)-LSMean(j) 2 -0.295097 -0.608371 0.018178 -0.377540 -0.684956 -0.070124 -0.701940 -0.092966 1 4 -0.397453 -0.397397 0.232511 2 3 -0.082443 -0.102356 -0.414440 0.209728 2 4 3 4 -0.019913 -0.326340 0.286514

NOTE: To ensure overall protection level, only probabilities associated with pre-planned comparisons should be used.

SOURCE: GLMOUT; TABLE: statlcgisc.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.3 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | Proc GLM Output for Ch | STAT-: | | in CGI- | S Scale, OC | 6 OF 6 |
|---|---|---|---|---|---|---|
| | | The GLM Pro | - | | | |
| | Parameter | Estimate | Standard<br>Error | t Value | Pr > t | |
| | 1 vs 900<br>1 vs 3<br>1 vs 2<br>2 vs 900<br>3 vs 900 | -0.39745256<br>-0.37753974<br>-0.29509666<br>-0.10235590<br>-0.01991282 | 0.15473286<br>0.15622132<br>0.15919853<br>0.15859351<br>0.15571880 | -2.57<br>-2.42<br>-1.85<br>-0.65<br>-0.13 | 0.0107<br>0.0163<br>0.0648<br>0.5192<br>0.8983 | |

SOURCE: GLMOUT; TABLE: statlcgisc.lis; RUN: 05FEB2019 14:05; ANALYSIS DATASET CREATED: 05FEB2019 11:24 PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/statl.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-5.3 FINAL

BREXPIPRAZOLE 1 OF 1

STAT-6.1.1
Shapiro-Wilk Test for Residual by Week from Proc Mixed for Change from

ange from in CAPS-5 Total Score, Primary Efficacy Analysis Mode (Intent to Treat Sample)

\_\_\_\_\_

| PROTOCOL | Week | TEST<br>VARIABLE | GOODNESS OF FIT | GOODNESS OF FIT<br>TEST<br>STATISTICS | Pvalue |
|---|---|---|---|---|---|
| 33120100061 | WEEK 3 | RESID | Shapiro-Wilk | 0.9882 | 0.0182 |
| | | STUDENTRESID | Shapiro-Wilk | 0.9883 | 0.0188 |
| | WEEK 6 | RESID | Shapiro-Wilk | 0.9955 | 0.6767 |
| | | STUDENTRESID | Shapiro-Wilk | 0.9957 | 0.7080 |
| | WEEK 10 | RESID | Shapiro-Wilk | 0.9938 | 0.4650 |
| | | STUDENTRESID | Shapiro-Wilk | 0.9939 | 0.4915 |
| | WEEK 12 | RESID | Shapiro-Wilk | 0.9904 | 0.1438 |
| | | STUDENTRESID | Shapiro-Wilk | 0.9905 | 0.1519 |

......

FILE: normality ba.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality\_b.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.1 FINAL

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 1 OF 32 PROTOCOL 331-201-00061 in CAPS-5 Total Score, Primary Efficacy Analysis Model Residual by Week from Proc Mixed for Change (Intent to Treat Sample) The UNIVARIATE Procedure Variable: RESID (Residual) Moments N 291 Sum Weights 291 -0.0214753 Sum Observations -6.2493044 
 Mean
 -0.0214700
 12

 Std Deviation
 8.65090319
 Variance
 74.838126

 0.2070035
 Kurtosis
 0.70012695
 Mean Uncorrected SS 21703.1908 Corrected SS 21703.0565 Coeff Variation -40283.089 Std Error Mean 0.50712493 Basic Statistical Measures Location Variability Mean -0.02148 Std Deviation 8.65090 Median 0.64232 Variance 74.83813 59.42843 Mode -4.37399 Range Interquartile Range 10.54517 Note: The mode displayed is the smallest of 2 modes with a count of 2.

| BREXPIPRAZOLE | 2 OF 32 |
|------------------------|---------|

Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model (Intent to Treat Sample)

------ Analysis Visit (N)=3 ------

The UNIVARIATE Procedure Variable: RESID (Residual)

Tests for Location: Mu0=0

Tests for Normality

| Test | Sta | tistic | р | Value |
|--------------------|------|----------|---------|-----------|
| Shapiro-Wilk | W | 0.988221 | Pr < W | 0.0182 |
| Kolmogorov-Smirnov | D | 0.042805 | Pr > D | >0.1500 |
| Cramer-von Mises | W-Sq | 0.127591 | Pr > W- | Sq 0.0479 |
| Anderson-Darling | A-Sq | 0.815848 | Pr > A- | Sq 0.0364 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas

OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 3 OF 32 PROTOCOL 331-201-00061 Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model The UNIVARIATE Procedure Variable: RESID (Residual) Quantiles (Definition 5) Level Quantile 100% Max 31.498902 99% 16.876065 95% 13.771516 90% 10.384727 75% Q3 5.476349 50% Median 0.642323 -5.068825 25% Q1 -11.778869 10% 5% -15.393540 1% -26.106596 0% Min -27.929524

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas

OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 4 OF 32 PROTOCOL 331-201-00061 Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model The UNIVARIATE Procedure Variable: RESID (Residual) Extreme Observations -----Lowest----------Highest-----Value USUBJID Obs Value USUBJID Obs -27.9295 16.3999 54 132 -26.3621 198 16.6089 125 -26.1066 274 16.8761 224 -21.2636 92 19.4553 196 -21.2002 248 31.4989 254

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas

OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 5 OF 32 PROTOCOL 331-201-00061

Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model (Intent to Treat Sample)

\_\_\_\_\_

# The UNIVARIATE Procedure Variable: STUDENTRESID (Studentized Residual)

### Moments

| N | 291 | Sum Weights | 291 |
|-----------------|------------|------------------|------------|
| Mean | -0.0024051 | Sum Observations | -0.6998929 |
| Std Deviation | 1.00383089 | Variance | 1.00767645 |
| Skewness | -0.2968518 | Kurtosis | 0.69179846 |
| Uncorrected SS | 292.227853 | Corrected SS | 292.226169 |
| Coeff Variation | -41737.07 | Std Error Mean | 0.05884561 |

### Basic Statistical Measures

| Location Var | riability |
|--------------|-----------|
|--------------|-----------|

| Mean | -0.00241 | Std Deviation | 1.00383 |
|--------|----------|---------------------|---------|
| Median | 0.07393 | Variance | 1.00768 |
| Mode | -0.50179 | Range | 6.86481 |
| | | Interguartile Range | 1.22110 |

Note: The mode displayed is the smallest of 2 modes with a count of 2.

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00061 | 6 OF 32 |
|---|---|
| | STAT-6.1.2 |
| Residual by Week from Proc Mixed for Change | in CAPS-5 Total Score, Primary Efficacy Analysis Model |
| | (Intent to Treat Sample) |

\_\_\_\_\_

------ Analysis Visit (N)=3 ------

The UNIVARIATE Procedure
Variable: STUDENTRESID (Studentized Residual)

Tests for Location: Mu0=0

| Test | -Statistic- | p Value |
|-------------|-------------|------------------|
| Student's t | t -0.04087 | 1 - 1 |
| Sign | M 10.5 | S = M 0.2410 |
| Signed Rank | S 688 | Pr >= S 0.6328 |

### Tests for Normality

| Test | Sta | tistic | p Val | ue |
|--------------------|------|----------|-----------|---------|
| Shapiro-Wilk | W | 0.988289 | Pr < W | 0.0188 |
| Kolmogorov-Smirnov | D | 0.043362 | Pr > D | >0.1500 |
| Cramer-von Mises | W-Sq | 0.128135 | Pr > W-Sq | 0.0473 |
| Anderson-Darling | A-Sq | 0.816711 | Pr > A-Sq | 0.0362 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 7 OF 32 PROTOCOL 331-201-00061 Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model The UNIVARIATE Procedure Variable: STUDENTRESID (Studentized Residual) Quantiles (Definition 5) Level Quantile 100% Max 3.6431135 99% 1.9692294 95% 1.6004374 90% 1.1991299 75% Q3 0.6349279 50% Median 0.0739303 -0.5861709 25% Q1 10% -1.3663926 5% -1.7824894 1% -3.0219158 0% Min -3.2216923

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas

OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 8 OF 32 PROTOCOL 331-201-00061 Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model The UNIVARIATE Procedure Variable: STUDENTRESID (Studentized Residual) Extreme Observations -----Lowest----------Highest-----Value USUBJID Obs Value USUBJID Obs -3.22169 54 132 1.89560 -3.05977 198 1.93905 125 -3.02192 274 1.96923 224 -2.50633 92 2.25031 196 -2.45764 248 3.64311 254

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas

OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 9 OF 32 PROTOCOL 331-201-00061

Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model (Intent to Treat Sample)

\_\_\_\_\_

The UNIVARIATE Procedure Variable: RESID (Residual)

### Moments

| N | 254 | Sum Weights | 254 |
|-----------------|------------|------------------|------------|
| Mean | 0.44348967 | Sum Observations | 112.646377 |
| Std Deviation | 10.3794296 | Variance | 107.732559 |
| Skewness | -0.0610478 | Kurtosis | -0.1779101 |
| Uncorrected SS | 27306.2949 | Corrected SS | 27256.3374 |
| Coeff Variation | 2340.39939 | Std Error Mean | 0.65126334 |

### Basic Statistical Measures

Location Variability

| Mean | 0.44349 | Std Deviation | 10.37943 |
|--------|----------|---------------------|-----------|
| Median | -0.35614 | Variance | 107.73256 |
| Mode | -7.53665 | Range | 57.11948 |
| | | Interquartile Range | 15 34328 |

Note: The mode displayed is the smallest of 2 modes with a count of 2.

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 10 OF 32 PROTOCOL 331-201-00061 Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model (Intent to Treat Sample) The UNIVARIATE Procedure Variable: RESID (Residual) Tests for Location: Mu0=0 Test -Statistic- ----p Value-----Student's t t 0.680968 Pr > |t| 0.4965 Sign M -3 Pr >= |M| 0.7538 Signed Rank S 780.5 Pr >= |S| 0.5065 Tests for Normality Test --Statistic--- Value-----Shapiro-Wilk W 0.995535 Pr < W 0.6767 Kolmogorov-Smirnov D 0.03977 Pr > D >0.1500Cramer-von Mises W-Sq 0.06535 Pr > W-Sq > 0.2500Anderson-Darling A-Sq 0.365198 Pr > A-Sq > 0.2500

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas

OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 11 OF 32 PROTOCOL 331-201-00061 Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model The UNIVARIATE Procedure Variable: RESID (Residual) Quantiles (Definition 5) Level Quantile 100% Max 27.384452 99% 24.503200 95% 16.489434 90% 13.817986 75% Q3 8.448887 50% Median -0.356136 -6.894394 25% Q1 -13.388430 10% 5% -17.101553 1% -23.196941 0% Min -29.735033

FILE: normalitybc.lis, RUN: 05FEB2019 14:05
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

| BREXPIPRAZOLE PROTOCOL 331-201-00 Residual | 061 by Week from Proc Mixed for Change | STAT-6 | in C | APS-5 Total Scor | 12 OF 32 e, Primary Efficacy Analysis Model |
|---|---|---|---|---|---|
| | | The UNIVARIAT Variable: RESI Extreme Obs | E Procedure<br>D (Residual) | | |
| | Lowest | | | | Highest |
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -29.7350 | | 507 | 23.4238 | | 513 |
| -28.9422 | | 340 | 24.4231 | | 294 |
| -23.1969 | | 363 | 24.5032 | | 544 |
| -20.2321 | | 450 | 25.4941 | | 332 |
| -20.1481 | | 444 | 27.3845 | | 408 |

------

FILE: normalitybc.lis, RUN: 05FEB2019 14:05
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 13 OF 32 PROTOCOL 331-201-00061

Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model

\_\_\_\_\_\_

------ Analysis Visit (N)=6 ------

The UNIVARIATE Procedure
Variable: STUDENTRESID (Studentized Residual)

## Moments

| N | 254 | Sum Weights | 254 |
|-----------------|------------|------------------|------------|
| Mean | 0.04293573 | Sum Observations | 10.9056744 |
| Std Deviation | 0.99698457 | Variance | 0.99397824 |
| Skewness | -0.0557595 | Kurtosis | -0.1703408 |
| Uncorrected SS | 251.944738 | Corrected SS | 251.476495 |
| Coeff Variation | 2322.03962 | Std Error Mean | 0.06255638 |

### Basic Statistical Measures

| Location Var | iability |
|--------------|----------|
|--------------|----------|

| Mean | 0.04294 | Std Deviation | 0.99698 |
|--------|----------|---------------------|---------|
| Median | -0.03408 | Variance | 0.99398 |
| Mode | -0.71999 | Range | 5.49119 |
| | | Interquartile Range | 1.48157 |

Note: The mode displayed is the smallest of 2 modes with a count of 2.

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE

14 OF 32

\_\_\_\_\_

 Shapiro-Wilk
 W
 0.995702
 Pr
 W
 0.7080

 Kolmogorov-Smirnov
 D
 0.038935
 Pr
 D
 >0.1500

 Cramer-von Mises
 W-Sq
 0.064256
 Pr
 > W-Sq
 >0.2500

 Anderson-Darling
 A-Sq
 0.355152
 Pr
 > A-Sq
 >0.2500

--Statistic--- ----p Value-----

FILE: normalitybc.lis, RUN: 05FEB2019 14:05
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

Test

BREXPIPRAZOLE 15 OF 32 PROTOCOL 331-201-00061 Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model The UNIVARIATE Procedure Variable: STUDENTRESID (Studentized Residual) Quantiles (Definition 5) Level Quantile 100% Max 2.6341119 99% 2.3834988 1.5884046 95% 90% 1.3306425 75% Q3 0.8085245 50% Median -0.0340834 -0.6730415 25% Q1 10% -1.2880822 5% -1.6340538 1% -2.2490702 0% Min -2.8570808

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 16 OF 32 PROTOCOL 331-201-00061 Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model The UNIVARIATE Procedure Variable: STUDENTRESID (Studentized Residual) Extreme Observations -----Lowest----------Highest-----Value USUBJID Obs Value USUBJID Obs -2.85708 507 2.25072 513 -2.77159 2.32984 294 340 -2.24907 363 2.38350 544 -1.93758 332 450 2.45627 -1.92494 2.63411 408 444

.....

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas

OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 17 OF 32
STAT-6.1.2
Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model

(Intent to Treat Sample)

------ Analysis Visit (N)=10 ------

The UNIVARIATE Procedure Variable: RESID (Residual)

### Moments

| N | 227 | Sum Weights | 227 |
|-----------------|------------|------------------|------------|
| Mean | 0.08611581 | Sum Observations | 19.5482882 |
| Std Deviation | 10.6826629 | Variance | 114.119287 |
| Skewness | -0.1828243 | Kurtosis | -0.146025 |
| Uncorrected SS | 25792.6423 | Corrected SS | 25790.9589 |
| Coeff Variation | 12404.9966 | Std Error Mean | 0.70903324 |

### Basic Statistical Measures

Location Variability

| Mean | 0.08612 | Std Deviation | 10.68266 |
|--------|----------|---------------------|-----------|
| Median | -0.06010 | Variance | 114.11929 |
| Mode | -5.59726 | Range | 58.82853 |
| | | Interguartile Range | 14.39574 |

Note: The mode displayed is the smallest of 2 modes with a count of 2.

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE


18 OF 32

Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model

(Intent to Treat Sample)

The UNIVARIATE Procedure
Variable: RESID (Residual)

Test -Statistic- -----p Value------

Tests for Normality

Signed Rank S

Student's t t 0.121455 Pr > |t| 0.9034

M -0.5 Pr >= |M| 1.0000 S 291 Pr >= |S| 0.7697

| Test | Sta | tistic | p V | alue |
|--------------------|------|----------|----------|------------|
| Shapiro-Wilk | W | 0.993767 | Pr < W | 0.4650 |
| Kolmogorov-Smirnov | D | 0.033884 | Pr > D | >0.1500 |
| Cramer-von Mises | W-Sq | 0.038705 | Pr > W-S | sq >0.2500 |
| Anderson-Darling | A-Sq | 0.300666 | Pr > A-S | sq >0.2500 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas

OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 19 OF 32 PROTOCOL 331-201-00061 Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model (Intent to Treat Sample) ------ Analysis Visit (N)=10 ------The UNIVARIATE Procedure Variable: RESID (Residual) Quantiles (Definition 5) Level Quantile 100% Max 25.824025 99% 22.779706 95% 17.026880 90% 14.368205 75% Q3 7.330122 50% Median -0.060104 -7.065623 25% Q1 -13.686490 10% 5% -18.354843 1% -24.242300 0% Min -33.004507

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas

OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

| BREXPIPRAZOLE | 0.61 | | | | 20 OF 32 |
|---|---|---|---|---|---|
| PROTOCOL 331-201-00<br>Residual | U01<br>by Week from Proc Mixed for Cha: | STAT-6 | in C | APS-5 Total Score, | Primary Efficacy Analysis Model |
| | | Analysis Vis<br>The UNIVARIAT<br>Variable: RESI | E Procedure | | |
| | Lowest | Extreme Obs | | | Highest |
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -33.0045<br>-24.5363<br>-24.2423<br>-24.1066<br>-23.2337 | | 565<br>708<br>553<br>589<br>645 | 20.3750<br>21.9446<br>22.7797<br>22.8236<br>25.8240 | | 650<br>566<br>619<br>614<br>764 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 21 OF 32 PROTOCOL 331-201-00061

Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model (Intent to Treat Sample)

-----

------ Analysis Visit (N)=10 ------

The UNIVARIATE Procedure
Variable: STUDENTRESID (Studentized Residual)

#### Moments

| N | 227 | Sum Weights | 227 |
|-----------------|------------|------------------|------------|
| Mean | 0.00806674 | Sum Observations | 1.831149 |
| Std Deviation | 0.97676522 | Variance | 0.95407029 |
| Skewness | -0.1794597 | Kurtosis | -0.1289175 |
| Uncorrected SS | 215.634657 | Corrected SS | 215.619886 |
| Coeff Variation | 12108.5562 | Std Error Mean | 0.06483018 |

Basic Statistical Measures

Location Variability

| Mean | 0.00807 | Std Deviation | 0.97677 |
|--------|----------|---------------------|---------|
| Median | -0.00547 | Variance | 0.95407 |
| Mode | -0.50932 | Range | 5.40570 |
| | | Interguartile Range | 1.31622 |

Note: The mode displayed is the smallest of 2 modes with a count of 2.

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

| BREXPIPRAZOLE<br>PROTOCOL 331-201-00061 | 22 OF 32<br>STAT-6.1.2 |
|---|---|
| Residual by Week from Proc Mixed for Change (In | in CAPS-5 Total Score, Primary Efficacy Analysis Model Intent to Treat Sample) |
| An | nalysis Visit (N)=10 |
| | ne UNIVARIATE Procedure<br>UDENTRESID (Studentized Residual) |
| Test | sts for Location: Mu0=0 |
| Test | -Statisticp Value |
| Student's t<br>Sign<br>Signed Rank | |
| Tests for Normality | |
| Test | Statistic Value |
| Shapiro-Wilk<br>Kolmogorov-Smirnov<br>Cramer-von Mises<br>Anderson-Darling | W 0.993944 Pr < W 0.4915<br>D 0.033338 Pr > D >0.1500<br>W-Sq 0.038046 Pr > W-Sq >0.2500<br>A-Sq 0.292192 Pr > A-Sq >0.2500 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 23 OF 32 PROTOCOL 331-201-00061 Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model (Intent to Treat Sample) The UNIVARIATE Procedure Variable: STUDENTRESID (Studentized Residual) Quantiles (Definition 5) Level Quantile 100% Max 2.35327141 2.11123783 95% 1.55962015 90% 1.31465170 75% Q3 0.67188649 50% Median -0.00547028 25% Q1 -0.64433297 -1.24754229 10% 5% -1.67961704 1% -2.20347197 0% Min -3.05242422

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 24 OF 32 PROTOCOL 331-201-00061 Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model ------ Analysis Visit (N)=10 -------The UNIVARIATE Procedure Variable: STUDENTRESID (Studentized Residual) Extreme Observations -----Lowest----------Highest-----Value USUBJID Obs Value USUBJID Obs 565 650 -3.05242 1.86278 -2.23710 708 2.02821 566 -2.20347 553 2.11124 614 -2.19831 589 2.11717 619 -2.11381 2.35327 764 645

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas

OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 25 OF 32 PROTOCOL 331-201-00061

Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model (Intent to Treat Sample)

The UNIVARIATE Procedure Variable: RESID (Residual)

### Moments

| N | 224 | Sum Weights | 224 |
|-----------------|------------|------------------|------------|
| Mean | -0.060841 | Sum Observations | -13.628393 |
| Std Deviation | 11.7505394 | Variance | 138.075175 |
| Skewness | 0.03467632 | Kurtosis | -0.5270157 |
| Uncorrected SS | 30791.5933 | Corrected SS | 30790.7641 |
| Coeff Variation | -19313.509 | Std Error Mean | 0.78511594 |

### Basic Statistical Measures

Location Variability

| Mean | -0.06084 | Std Deviation | 11.75054 |
|--------|----------|---------------------|-----------|
| Median | -0.40775 | Variance | 138.07518 |
| Mode | 14.65028 | Range | 58.81038 |
| | | Interguartile Range | 17.57915 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 26 OF 32 PROTOCOL 331-201-00061 Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model (Intent to Treat Sample) The UNIVARIATE Procedure Variable: RESID (Residual) Tests for Location: Mu0=0 Test -Statistic- ----p Value------2 Pr >= |M| 0.8412-143 Pr >= |S| 0.8833 Signed Rank S Tests for Normality --Statistic--- ----p Value-----Test Shapiro-Wilk W 0.990386 Pr < W 0.1438 Kolmogorov-Smirnov D 0.046115 Pr > D >0.1500 Cramer-von Mises W-Sq 0.102955 Pr > W-Sq 0.1031Anderson-Darling A-Sq 0.621895 Pr > A-Sq 0.1050

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas

OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 27 OF 32 PROTOCOL 331-201-00061 Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model (Intent to Treat Sample) The UNIVARIATE Procedure Variable: RESID (Residual) Quantiles (Definition 5) Level Quantile 100% Max 26.15988 99% 24.90444 95% 20.02366 90% 15.90305 75% Q3 9.17140 50% Median -0.40775 -8.40775 25% Q1 -14.86161 10% 5% -17.45916 1% -24.00422 0% Min -32.65050

.....

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas

OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

| BREXPIPRAZOLE | 0.61 | | | | 28 OF 32 |
|---|---|---|---|---|---|
| PROTOCOL 331-201-00 | uol | for Change | AT-6.1.2 in CA Treat Sample) | APS-5 Total Score, | Primary Efficacy Analysis Model |
| | | The UNIVA | Visit (N)=12<br>RIATE Procedure<br>RESID (Residual) | | |
| | Lovest | | Observations | 11 | ighest |
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -32.6505<br>-29.7432<br>-24.0042<br>-23.3489<br>-23.2061 | | 797<br>793<br>871<br>780<br>816 | 22.4025<br>22.4483<br>24.9044<br>25.3498<br>26.1599 | | 979<br>994<br>847<br>921<br>794 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE
STAT-6.1.2
Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model

\_\_\_\_\_

------ Analysis Visit (N)=12 ------

# The UNIVARIATE Procedure Variable: STUDENTRESID (Studentized Residual)

### Moments

| N | 224 | Sum Weights | 224 |
|-----------------|------------|------------------|------------|
| Mean | -0.0049909 | Sum Observations | -1.1179516 |
| Std Deviation | 0.98854745 | Variance | 0.97722606 |
| Skewness | 0.03317158 | Kurtosis | -0.5106489 |
| Uncorrected SS | 217.926991 | Corrected SS | 217.921412 |
| Coeff Variation | -19807.175 | Std Error Mean | 0.0660501 |

### Basic Statistical Measures

| Location | Variability |
|----------|-------------|

| Mean | -0.00499 | Std Deviation | 0.98855 |
|--------|----------|---------------------|---------|
| Median | -0.03454 | Variance | 0.97723 |
| Mode | 1.22405 | Range | 4.99503 |
| | | Interguartile Range | 1.47852 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL
| BREXPIPRAZOLE PROTOCOL 331-201-00061 | | | | | | 30 OF 32 |
|---|---|---|---|---|---|---|
| Residual by Week from Proc Mixed | | | -6.1.2 i | | tal Score, 1 | Primary Efficacy Analysis Model |
| | An | alysis V | isit (N)=12 | · | | |
| | The<br>Variable: STUD | | ATE Procedu<br>(Studenti | | 1) | |
| | Test | s for Lo | cation: Mu0 | )=0 | | |
| | Test | -Statist | ic | p Value | | |
| | | M | -2 Pr > | > t 0.9<br>>= M 0.8<br>>= S 0.8 | 412 | |
| | Т | ests for | Normality | | | |
| | Test | Stat | istic | p Val | ue | |
| | Shapiro-Wilk<br>Kolmogorov-Smirnov<br>Cramer-von Mises<br>Anderson-Darling | D (<br>W-Sq | 0.990531<br>0.045559<br>0.102583<br>0.620048 | Pr > D<br>Pr > W-Sq | | |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 31 OF 32 PROTOCOL 331-201-00061 Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model The UNIVARIATE Procedure Variable: STUDENTRESID (Studentized Residual) Quantiles (Definition 5) Level Quantile 100% Max 2.2200513 99% 2.1274494 95% 1.6918552 90% 1.3461309 75% Q3 0.7703818 50% Median -0.0345376 -0.7081358 25% Q1 10% -1.2443432 5% -1.4710086 1% -2.0101286 0% Min -2.7749833

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas

OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 32 OF 32 PROTOCOL 331-201-00061 Residual by Week from Proc Mixed for Change in CAPS-5 Total Score, Primary Efficacy Analysis Model ------ Analysis Visit (N)=12 -------The UNIVARIATE Procedure Variable: STUDENTRESID (Studentized Residual) Extreme Observations -----Lowest----------Highest-----Value USUBJID Obs Value USUBJID Obs -2.77498 797 979 1.87914 793 1.88518 -2.52653 994 -2.01013 871 2.12745 847 -1.95439 780 2.12941 921 -1.94802 816 2.22005 794

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 05FEB2019 14:05

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/normality.sas

OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT-6.1.2 FINAL

BREXPIPRAZOLE 1 OF 13

| | | STAT1-1.1 | | | | | |
|---|---|---|---|---|---|---|---|
| Adjusted Mean | Change | | in C | APS-5 | Line | Items | - MMRM |
| | | (Modified Intent to Tre | eat S | Sample) | | | l |

| CAPS<br>Line Items | N<br> | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change <sup>1</sup> | N<br> | BRE<br>MEAN<br>Base | | N<br> | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N<br> | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CAPSW-INTRUSIVE<br>MEMORIES<br>SEVERITY | 58 | 2.48 | -1.27 | 48 | 2.44 | -0.92 | 59 | 2.51 | -0.67 | 59 | 2.31 | -1.03 | Dummy W vs Dummy Z | -0.24 | 0.3345 | -0.18 |
| OBVERTI | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.60 | 0.0176 | -0.44 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.35 | 0.1931 | -0.25 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.11 | 0.6864 | 0.08 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.36 | 0.1527 | 0.26 |
| CAPSW-DISTRESSI<br>NG DREAMS<br>SEVERITY | 58 | 1.29 | -0.72 | 48 | 1.85 | -0.68 | 59 | 1.92 | -0.60 | 59 | 1.75 | -0.71 | Dummy W vs Dummy Z | -0.01 | 0.9610 | -0.01 |
| ODVERTI | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.12 | 0.6182 | -0.09 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.04 | 0.8828 | -0.03 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.03 | 0.9174 | 0.02 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.11 | 0.6478 | 0.08 |
| CAPSW-DISSOCIAT | 58 | 0.98 | -0.75 | 48 | 0.92 | -0.42 | 59 | 0.88 | -0.37 | 59 | 1.02 | -0.59 | Dummy W vs Dummy Z | -0.16 | 0.3968 | -0.16 |
| SEVERITY | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.38 | 0.0461 | -0.37 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.33 | 0.1101 | -0.31 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.17 | 0.4118 | 0.16 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.22 | 0.2442 | 0.22 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

BREXPIPRAZOLE 2 OF 13

STAT1-1.1
Adjusted Mean Change in CAPS-5 Line Items - MMRM (Modified Intent to Treat Sample)

| CAPS<br>Line Items | BREX+SERT<br>MEAN LSMean<br>N Base Change <sup>1</sup> | BREX<br>MEAN LSMean<br>N Base Change <sup>1</sup> | SERT<br>MEAN LSMean<br>N Base Change¹ | PLACEBO<br>MEAN LSMean<br>N Base Change <sup>1</sup> | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE 1 | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|
| CAPSW-CUED<br>PSYCLOGICAL<br>DISTRESS<br>SEVERITY | 58 2.50 -1.25 | 48 2.38 -1.08 | 59 2.39 -0.84 | 59 2.39 -1.04 | Dummy W vs Dummy Z | -0.21 | 0.3861 | -0.16 |
| OBVERTI | | | | | Dummy W vs Dummy Y | -0.41 | 0.0934 | -0.31 |
| | | | | | Dummy W vs Dummy X | -0.17 | 0.5262 | -0.12 |
| | | | | | Dummy X vs Dummy Z | -0.05 | 0.8623 | -0.03 |
| | | | | | Dummy Y vs Dummy Z | 0.20 | 0.4095 | 0.15 |
| CAPSW-CUED PSYCLOGICAL REACTION SEVERITY | 58 2.33 -1.29 | 48 2.27 -1.10 | 59 2.31 -0.44 | 59 2.37 -0.73 | Dummy W vs Dummy Z | -0.56 | 0.0232 | -0.42 |
| SEVERTII | | | | | Dummy W vs Dummy Y | -0.84 | 0.0007 | -0.64 |
| | | | | | Dummy W vs Dummy X | -0.18 | 0.4800 | -0.14 |
| | | | | | Dummy X vs Dummy Z | -0.37 | 0.1539 | -0.28 |
| | | | | | Dummy Y vs Dummy Z | 0.29 | 0.2365 | 0.22 |
| CAPSW-AVOID<br>MEM THGHTS<br>FEELNGS | 58 2.55 -1.09 | 48 2.52 -0.75 | 59 2.58 -0.58 | 59 2.58 -0.92 | Dummy W vs Dummy Z | -0.17 | 0.4810 | -0.13 |
| SEVERITY | | | | | Dummy W vs Dummy Y | -0.50 | 0.0347 | -0.39 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

BREXPIPRAZOLE 3 OF 13

Adjusted Mean Change STAT1-1.1 in CAPS-5 Line Items - MMRM (Modified Intent to Treat Sample)

| CAPS<br>Line Items | N | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change¹ | N<br> | BRE<br>MEAN<br>Base | | N<br> | SER<br>MEAN<br>Base | T<br>LSMean<br>Change <sup>1</sup> | N<br> | | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CAPSW-AVOID MEM THGHTS FEELINGS SEVERITY | | | | | | | | | | | | | Dummy W vs Dummy X | -0.34 | 0.1828 | -0.26 |
| SEVERIII | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.17 | 0.4945 | 0.13 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.34 | 0.1532 | 0.26 |
| CAPSW-AVOID<br>EXTERNL<br>REMINDRS<br>SEVERITY | 58 | 2.47 | -1.10 | 48 | 2.54 | -0.95 | 59 | 2.51 | -0.74 | 59 | 2.46 | -0.89 | Dummy W vs Dummy Z | -0.21 | 0.3875 | -0.16 |
| | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.36 | 0.1418 | -0.27 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.15 | 0.5723 | -0.11 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.06 | 0.8080 | -0.05 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.15 | 0.5389 | 0.11 |
| CAPSW-INABLTY RECAL ASPCT EVNT SEVERITY | 58 | 0.91 | -0.22 | 48 | 0.96 | -0.12 | 59 | 0.64 | -0.10 | 59 | 0.64 | -0.29 | Dummy W vs Dummy Z | 0.06 | 0.6355 | 0.09 |
| DVIVI SEVERIII | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.12 | 0.3719 | -0.17 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.11 | 0.4578 | -0.15 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.17 | 0.2356 | 0.23 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.18 | 0.1681 | 0.25 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

FILE: caps\_itemma.lis, RUN: 05FEB2019 14:06; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_itemm.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT1-1.1 FINAL

BREXPIPRAZOLE 4 OF 13

Adjusted Mean Change in CAPS-5 Line Items - MMRM (Modified Intent to Treat Sample)

| CAPS<br>Line Items | N<br> | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change <sup>1</sup> | N<br> | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N<br> | | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CAPSW-EXGGRTD NEG BELIFS EXPTNS SEVERITY | 58 | 2.50 | -1.13 | 48 | 2.56 | -0.61 | 59 | 2.49 | -0.86 | 59 | 2.24 | -0.61 | Dummy W vs Dummy Z | -0.52 | 0.0252 | -0.42 |
| 21111110 021211111 | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.27 | 0.2407 | -0.22 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.52 | 0.0365 | -0.41 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.00 | 0.9995 | 0.00 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.25 | 0.2806 | -0.20 |
| CAPSW-DIST<br>COGTNS LEADNG<br>BLAME SEVERITY | 58 | 2.00 | -0.90 | 48 | 1.69 | -0.84 | 59 | 2.14 | -0.79 | 59 | 1.61 | -0.75 | Dummy W vs Dummy Z | -0.15 | 0.5172 | -0.12 |
| DENIE OBVENITI | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.10 | 0.6433 | -0.09 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.05 | 0.8239 | -0.04 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.09 | 0.6950 | -0.08 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.04 | 0.8480 | -0.04 |
| CAPSW-PRSISTNT<br>NEG EMOTNL | 58 | 2.36 | -0.98 | 48 | 2.69 | -0.94 | 59 | 2.51 | -0.84 | 59 | 2.41 | -0.59 | Dummy W vs Dummy Z | -0.39 | 0.0802 | -0.33 |
| STATE SEVERITY | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.14 | 0.5336 | -0.12 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.05 | 0.8461 | -0.04 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.34 | 0.1536 | -0.28 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.25 | 0.2580 | -0.21 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

BREXPIPRAZOLE 5 OF 13

STAT1-1.1
Adjusted Mean Change in CAPS-5 Line Items — MMRM (Modified Intent to Treat Sample)

| CAPS<br>Line Items | N | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change <sup>1</sup> | N | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CAPSW-DIMISHD<br>INTRST<br>ACTVTIES<br>SEVERITY | 58 | 2.38 | -1.31 | 48 | 2.42 | -0.73 | 59 | 2.44 | -0.59 | 59 | 2.27 | -0.80 | Dummy W vs Dummy Z | -0.51 | 0.0334 | -0.40 |
| SEVERTI | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.72 | 0.0029 | -0.56 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.58 | 0.0240 | -0.44 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.07 | 0.7778 | 0.05 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.21 | 0.3769 | 0.16 |
| CAPSW-DETACHMNT<br>ESTRNGMNT<br>OTHRS SEVERITY | 58 | 2.64 | -0.96 | 48 | 2.40 | -0.83 | 59 | 2.63 | -0.64 | 59 | 2.59 | -0.60 | Dummy W vs Dummy Z | -0.36 | 0.1606 | -0.26 |
| Oluka arvekili | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.32 | 0.2120 | -0.23 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.13 | 0.6469 | -0.09 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.23 | 0.3969 | -0.17 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.04 | 0.8804 | -0.03 |
| CAPSW-PRSISTNT<br>INAB EXP | 58 | 2.16 | -1.10 | 48 | 1.92 | -0.62 | 59 | 2.02 | -0.54 | 59 | 1.93 | -0.58 | Dummy W vs Dummy Z | -0.52 | 0.0234 | -0.42 |
| POSTVE SEVERITY | | | | | | | | | | | | | Diametr M rrg Diametr V | -0.55 | 0.0164 | -0.45 |
| | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.33 | 0.0164 | -0.45 |
| | | | | | | | | | | | | | Dummy W vs Dummy X Dummy X vs Dummy Z | -0.48 | 0.0525 | -0.38 |
| | | | | | | | | | | | | | panuly v vs panully v | -0.04 | 0.0000 | -0.03 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

BREXPIPRAZOLE 6 OF 13

Adjusted Mean Change in CAPS-5 Line Items — MMRM (Modified Intent to Treat Sample)

| CAPS<br>Line Items | N<br> | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change¹ | N | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N<br> | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N<br> | PLACI<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE¹ | COHEN'S<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CAPSW-PRSISTNT<br>INAB EXP<br>POSTVE SEVERITY | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.03 | 0.8857 | 0.03 |
| CAPSW-IRRITBLE<br>BEHAV ANGRY<br>SEVERITY | 58 | 1.60 | -0.42 | 48 | 1.67 | -0.47 | 59 | 1.66 | -0.49 | 59 | 1.69 | -0.42 | Dummy W vs Dummy Z | -0.00 | 0.9948 | -0.00 |
| DEVERTIT | | | | | | | | | | | | | Dummy W vs Dummy Y | 0.07 | 0.7672 | 0.05 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | 0.04 | 0.8630 | 0.03 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.04 | 0.8573 | -0.04 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.07 | 0.7608 | -0.06 |
| CAPSW-RECKLS<br>SELF DESTR | 58 | 0.33 | -0.14 | 48 | 0.35 | -0.11 | 59 | 0.22 | -0.17 | 59 | 0.39 | -0.11 | Dummy W vs Dummy Z | -0.03 | 0.7718 | -0.05 |
| BEHAV SEVERITY | | | | | | | | | | | | | Dummy W vs Dummy Y | 0.03 | 0.7834 | 0.05 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.03 | 0.7975 | -0.05 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.00 | 0.9907 | -0.00 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.06 | 0.5707 | -0.10 |
| APSW-HYPERVIGI | 58 | 2.64 | -0.88 | 48 | 2.48 | -0.55 | 59 | 2.29 | -0.70 | 59 | 2.58 | -0.48 | Dummy W vs Dummy Z | -0.40 | 0.0622 | -0.35 |
| ANCE SEVERITY | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.18 | 0.4040 | -0.15 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

BREXPIPRAZOLE 7 OF 13

Adjusted Mean Change in CAPS-5 Line Items - MMRM (Modified Intent to Treat Sample)

| CAPS<br>Line Items | N | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change <sup>1</sup> | N | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N | | T<br>LSMean<br>Change¹ | | | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CAPSW-HYPERVIGI<br>LANCE SEVERITY | | | | | | | | | | | | | Dummy W vs Dummy X | -0.33 | 0.1518 | -0.28 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.07 | 0.7578 | -0.06 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.22 | 0.3090 | -0.19 |
| CAPSW-EXAGGERAT D STRTLE RESPNSE SEVERITY | 58 | 1.66 | -0.52 | 48 | 1.65 | -0.45 | 59 | 1.63 | -0.59 | 59 | 1.54 | -0.44 | Dummy W vs Dummy Z | -0.08 | 0.7173 | -0.07 |
| SEVERIII | | | | | | | | | | | | | Dummy W vs Dummy Y | 0.07 | 0.7553 | 0.06 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.07 | 0.7608 | -0.06 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.01 | 0.9741 | -0.01 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.15 | 0.4986 | -0.12 |
| CAPSW-PRBLMS<br>WTH<br>CONCENTRATION<br>SEVERITY | 58 | 2.34 | -0.84 | 48 | 2.50 | -0.68 | 59 | 2.10 | -0.67 | 59 | 2.29 | -0.76 | Dummy W vs Dummy Z | -0.08 | 0.6973 | -0.07 |
| PEAFKIII | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.17 | 0.4292 | -0.15 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.17 | 0.4789 | -0.14 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.08 | 0.7269 | 0.07 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.09 | 0.6822 | 0.08 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

FILE: caps\_itemma.lis, RUN: 05FEB2019 14:06; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_itemm.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT1-1.1 FINAL

BREXPIPRAZOLE 8 OF 13

| CAPS<br>Line Items | N<br> | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change¹ | N<br> | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N<br> | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT 1 | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CAPSW-SLEEP<br>DISTURBANCE<br>SEVERITY | 58 | 2.33 | -0.72 | 48 | 2.71 | -0.74 | 59 | 2.68 | -0.32 | 59 | 2.80 | -0.52 | Dummy W vs Dummy Z | -0.20 | 0.4206 | -0.15 |
| 0212111 | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.40 | 0.1014 | -0.30 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | 0.02 | 0.9315 | 0.02 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.22 | 0.3905 | -0.17 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.20 | 0.3987 | 0.16 |
| CAPSW-SUBJECTIV<br>E DISTRESS<br>SEVERITY | 58 | 2.67 | -0.96 | 48 | 2.75 | -0.72 | 59 | 2.66 | -0.60 | 59 | 2.53 | -0.69 | Dummy W vs Dummy Z | -0.27 | 0.0872 | -0.32 |
| SEVERIII | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.36 | 0.0214 | -0.43 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.24 | 0.1538 | -0.28 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.03 | 0.8527 | -0.04 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.09 | 0.5545 | 0.11 |
| CAPSW-IMPAIRMNT<br>SOCIAL FUNCTNG | 58 | 2.71 | -1.14 | 48 | 2.60 | -0.90 | 59 | 2.73 | -0.70 | 59 | 2.58 | -0.72 | Dummy W vs Dummy Z | -0.42 | 0.0283 | -0.41 |
| SEVERITY | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.44 | 0.0219 | -0.43 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.24 | 0.2348 | -0.23 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.18 | 0.3824 | -0.17 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.02 | 0.9146 | 0.02 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

BREXPIPRAZOLE 9 OF 13

Adjusted Mean Change in CAPS-5 Line Items - MMRM (Modified Intent to Treat Sample)

| CAPS<br>Line Items | N | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change <sup>1</sup> | N | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N<br> | PLACI<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT 1 | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CAPSW-IMPAIRMNT<br>OCCUP FUNCTNG<br>SEVERITY | 58 | 2.36 | -0.77 | 48 | 2.31 | -0.71 | 59 | 2.44 | -0.59 | 59 | 2.29 | -0.52 | Dummy W vs Dummy Z | -0.25 | 0.2044 | -0.24 |
| | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.18 | 0.3560 | -0.17 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.06 | 0.7892 | -0.05 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.19 | 0.3553 | -0.18 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.07 | 0.7310 | -0.06 |
| CAPSW-SEVERITY<br>SUBTOTAL G | 58 | 7.74 | -2.89 | 48 | 7.67 | -2.35 | 59 | 7.83 | -1.91 | 59 | 7.39 | -1.85 | Dummy W vs Dummy $\mathbf{Z}$ | -1.04 | 0.0159 | -0.45 |
| SOBIOTAL G | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.98 | 0.0231 | -0.42 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.54 | 0.2406 | -0.23 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.50 | 0.2694 | -0.22 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.06 | 0.8895 | -0.03 |
| CAPSW-GLOBAL | 58 | 0.17 | 0.02 | 48 | 0.19 | 0.00 | 59 | 0.17 | -0.10 | 59 | 0.08 | 0.00 | Dummy W vs Dummy Z | 0.02 | 0.7128 | 0.07 |
| VALIDITY | | | | | | | | | | | | | Dummy W vs Dummy Y | 0.13 | 0.0219 | 0.43 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | 0.02 | 0.7506 | 0.06 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.00 | 0.9796 | 0.00 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.11 | 0.0510 | -0.36 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.


STAT1-1.1
Adjusted Mean Change in CAPS-5 Line Items - MMRM (Modified Intent to Treat Sample)

| CAPS<br>Line Items | N<br> | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change¹ | N<br> | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N<br> | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N<br> | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE¹ | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CAPSW-GLOBAL<br>SEVERITY | 58 | 2.72 | -0.98 | 48 | 2.77 | -0.92 | 59 | 2.71 | -0.60 | 59 | 2.58 | -0.72 | Dummy W vs Dummy Z | -0.26 | 0.1195 | -0.29 |
| | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.38 | 0.0232 | -0.42 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.07 | 0.7127 | -0.07 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.19 | 0.2749 | -0.21 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.12 | 0.4699 | 0.13 |
| CAPSW-GLOBAL<br>IMPROVEMENT | 58 | 3.69 | -1.43 | 48 | 3.65 | -1.20 | 59 | 3.63 | -0.83 | 59 | 3.59 | -1.11 | Dummy W vs Dummy Z | -0.32 | 0.1267 | -0.28 |
| IMPROVEMENT | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.60 | 0.0047 | -0.53 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.23 | 0.2943 | -0.21 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.08 | 0.7055 | -0.07 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.28 | 0.1769 | 0.25 |
| CAPSW-DEPERSONA<br>LIZATION | 58 | 0.26 | -0.30 | 48 | 0.38 | -0.11 | 59 | 0.29 | -0.24 | 59 | 0.25 | -0.21 | Dummy W vs Dummy Z | -0.09 | 0.2168 | -0.23 |
| SEVERITY | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.06 | 0.4517 | -0.14 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.19 | 0.0198 | -0.46 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.10 | 0.2279 | 0.24 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.04 | 0.6303 | -0.09 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.


STAT1-1.1
Adjusted Mean Change in CAPS-5 Line Items - MMRM (Modified Intent to Treat Sample)

| CAPS<br>ine Items | N<br> | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change <sup>1</sup> | N<br> | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N<br> | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N<br> | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CAPSW-DEREALIZA | 58 | 0.28 | -0.29 | 48 | 0.42 | -0.13 | 59 | 0.27 | -0.19 | 59 | 0.31 | -0.27 | Dummy W vs Dummy Z | -0.03 | 0.7676 | -0.05 |
| | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.10 | 0.2441 | -0.22 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.16 | 0.0864 | -0.34 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.14 | 0.1476 | 0.28 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.08 | 0.3828 | 0.16 |
| CAPSW-SEVERITY | 58 | 0.53 | -0.59 | 48 | 0.79 | -0.24 | 59 | 0.56 | -0.43 | 59 | 0.56 | -0.47 | Dummy W vs Dummy Z | -0.12 | 0.3825 | -0.16 |
| SOBIOIAL DISS | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.16 | 0.2534 | -0.21 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.35 | 0.0187 | -0.46 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.23 | 0.1170 | 0.31 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.04 | 0.7818 | 0.05 |
| CAPS-5<br>SUBSCALE B<br>COTAL SEVERITY<br>SCORE | 58 | 9.59 | -5.27 | 48 | 9.85 | -4.27 | 59 | 10.00 | -2.87 | 59 | 9.83 | -4.12 | Dummy W vs Dummy Z | -1.15 | 0.1829 | -0.25 |
| CORE | | | | | | | | | | | | | Dummy W vs Dummy Y | -2.39 | 0.0062 | -0.51 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.99 | 0.2811 | -0.21 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.15 | 0.8654 | -0.03 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 1.24 | 0.1470 | 0.27 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

FILE: caps\_itemma.lis, RUN: 05FEB2019 14:06; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_itemm.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT1-1.1 FINAL


Adjusted Mean Change STAT1-1.1

Adjusted Mean Change (Modified Intent to Treat Sample) - MMRM

| CAPS<br>Line Items | BREX+SERT<br>MEAN LSMean<br>N Base Change <sup>1</sup> | BREX<br>MEAN LSMean<br>N Base Change <sup>1</sup> | SERT<br>MEAN LSMean<br>N Base Change <sup>1</sup> | PLACEBO<br>MEAN LSMean<br>N Base Change <sup>1</sup> | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT 1 | P-VALUE¹ | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|
| CAPS-5<br>SUBSCALE C<br>TOTAL SEVERITY<br>SCORE | 58 5.02 -2.19 | 48 5.06 -1.72 | 59 5.08 -1.35 | 59 5.03 -1.81 | Dummy W vs Dummy Z | -0.38 | 0.3588 | -0.17 |
| SCORE | | | | | Dummy W vs Dummy Y Dummy W vs Dummy X Dummy X vs Dummy Z Dummy Y vs Dummy Z | -0.84<br>-0.47<br>0.09<br>0.46 | 0.0413<br>0.2858<br>0.8303<br>0.2532 | -0.38<br>-0.21<br>0.04<br>0.21 |
| CAPS-5 SUBSCALE D TOTAL SEVERITY SCORE | 58 14.95 -6.66 | 48 14.63 -4.73 | 59 14.86 -4.45 | 59 13.69 -4.30 | Dummy W vs Dummy Z | -2.36 | 0.0153 | -0.45 |
| | | | | | Dummy W vs Dummy Y Dummy W vs Dummy X Dummy X vs Dummy Z Dummy Y vs Dummy Z | -2.21<br>-1.93<br>-0.43<br>-0.15 | 0.0225<br>0.0615<br>0.6713<br>0.8750 | -0.43<br>-0.37<br>-0.08<br>-0.03 |
| CAPS-5<br>SUBSCALE E<br>TOTAL SEVERITY<br>SCORE | 58 10.90 -3.53 | 48 11.35 -2.99 | 59 10.58 -2.90 | 59 11.29 -2.75 | Dummy W vs Dummy Z | -0.78 | 0.2361 | -0.22 |
| SCORE | | | | | Dummy W vs Dummy Y | -0.64 | 0.3395 | -0.18 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

BREXPIPRAZOLE 13 OF 13

Adjusted Mean Change STAT1-1.1 in CAPS-5 Line Items — MMRM (Modified Intent to Treat Sample)

ESTIMATED COHEN's D CAPS MEAN LSMean MEAN LSMean MEAN LSMean MEAN LSMean TREATMENT TREATMENT EFFECT
Line Items N Base Change¹ N Base Change¹ N Base Change¹ N Base Change¹ COMPARISON EFFECT ¹ P-VALUE¹ SIZE TREATMENT CAPS-5 Dummy W vs Dummy X -0.55 0.4393 -0.15 SUBSCALE E TOTAL SEVERITY SCORE Dummy X vs Dummy Z -0.23 0.7380 -0.07 Dummy Y vs Dummy Z -0.15 0.8225 -0.04 CAPS-5 TOTAL 58 40.45 -17.7 48 40.90 -14.0 59 40.53 -11.6 59 39.85 -13.0 Dummy W vs Dummy Z -4.77 0.0389 -0.38 SEVERITY SCORE -6.10 0.0087 -0.49 Dummy W vs Dummy Y Dummy W vs Dummy X -3.73 0.1283 -0.30 Dummy X vs Dummy Z -1.03 0.6703 -0.08 Dummy Y vs Dummy Z 1.33 0.5595

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

FILE: caps\_itemma.lis, RUN: 05FEB2019 14:06; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_itemm.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT1-1.1 FINAL

BREXPIPRAZOLE 1 OF 5

| SOTS<br>Line Items | N | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change¹ | N | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOTS-RE-EXPERIE | 55 | 4.73 | -2.09 | 47 | 4.68 | -1.31 | 57 | 4.75 | -1.71 | 57 | 4.42 | -1.65 | Dummy W vs Dummy Z | -0.43 | 0.1892 | -0.25 |
| | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.38 | 0.2455 | -0.22 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.78 | 0.0279 | -0.44 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.35 | 0.3234 | 0.20 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.05 | 0.8737 | -0.03 |
| SOTS-HYPERAROUS | 55 | 4.60 | -0.86 | 47 | 4.60 | -1.14 | 57 | 4.70 | -1.69 | 57 | 4.49 | -0.88 | Dummy W vs Dummy Z | 0.03 | 0.9268 | 0.02 |
| AL | | | | | | | | | | | | | Dummy W vs Dummy Y | 0.83 | 0.0055 | 0.53 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | 0.28 | 0.3744 | 0.18 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.26 | 0.4200 | -0.16 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.80 | 0.0069 | -0.51 |
| SOTS-AFFECTIVE<br>DYSREGULATION | 55 | 3.55 | -1.39 | 47 | 3.70 | -1.39 | 57 | 3.81 | -1.78 | 57 | 3.33 | -1.44 | Dummy W vs Dummy Z | 0.04 | 0.8862 | 0.03 |
| DISKEGULATION | | | | | | | | | | | | | Dummy W vs Dummy Y | 0.38 | 0.2082 | 0.24 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.00 | 0.9987 | -0.00 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.04 | 0.8923 | 0.03 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.34 | 0.2609 | -0.21 |
| SOTS-IMPULSIVIT | 55 | 1.91 | -0.34 | 47 | 1.53 | -0.39 | 57 | 2.04 | -0.57 | 57 | 2.04 | -0.52 | Dummy W vs Dummy Z | 0.18 | 0.3813 | 0.17 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

BREXPIPRAZOLE 2 OF 5

STAT1-1.2

Adjusted Mean Change from Baeline (Day 0) in SOTS Line Itemsat Week 12 - MMRM (Modified Intent to Treat Sample)

COHEN's D SOTS MEAN LSMean MEAN LSMean MEAN LSMean MEAN LSMean TREATMENT TREATMENT EFFECT
Line Items N Base Change¹ N Base Change¹ N Base Change¹ N Base Change¹ COMPARISON EFFECT ¹ P-VALUE¹ SIZE EFFECT SOTS-IMPULSIVIT Dummy W vs Dummy Y 0.23 0.2630 0.21 Dummy W vs Dummy X 0.05 0.8173 0.05 Dummy X vs Dummy Z 0.13 0.5607 0.11 Dummy Y vs Dummy Z -0.05 0.8030 -0.05 SOTS-AVOIDANCE 55 4.95 -1.55 47 4.81 -1.19 57 5.07 -1.35 57 4.75 -1.27 Dummy W vs Dummy Z -0.29 0.3750 -0.17 Dummy W vs Dummy Y -0.21 0.5260 -0.12 0.2998 Dummy W vs Dummy X -0.36 -0.21 Dummy X vs Dummy Z 0.8307 0.07 0.04 Dummy Y vs Dummy Z -0.08 0.7993 -0.05 SOTS-NUMBING 55 3.04 -1.09 47 3.11 -0.81 57 3.14 -1.06 57 3.21 -1.07 Dummy W vs Dummy Z -0.02 0.9531 -0.01 Dummy W vs Dummy Y -0.03 0.9101 -0.02 Dummy W vs Dummy X -0.29 0.3766 -0.18 Dummy X vs Dummy Z 0.27 0.4036 0.16 Dummy Y vs Dummy Z 0.02 0.9565 0.01 SOTS-ATTENTIN 55 1.98 -0.74 47 2.32 -0.65 57 1.79 -0.59 57 1.95 -0.45 -0.29 0.1586 -0.27 Dummy W vs Dummy Z CONSCIOUSNESS DISSOCIATION -0.15 0.4552 -0.14 Dummy W vs Dummy Y Dummy W vs Dummy X -0.09 0.6848 -0.08

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

BREXPIPRAZOLE 3 OF 5

STAT1-1.2

Adjusted Mean Change from Baeline (Day 0) in SOTS Line Itemsat Week 12 - MMRM

(Modified Intent to Treat Sample)

COHEN's D ESTIMATED SOTS MEAN LSMean MEAN LSMean MEAN LSMean MEAN LSMean TREATMENT TREATMENT EFFECT
Line Items N Base Change¹ N Base Change¹ N Base Change¹ N Base Change¹ COMPARISON EFFECT ¹ P-VALUE¹ SIZE EFFECT SOTS-ATTENTIN Dummy X vs Dummy Z -0.20 0.3665 -0.18 CONSCIOUSNESS DISSOCIATION Dummy Y vs Dummy Z -0.14 0.5042 SOTS-SELF 55 3.93 -1.52 47 4.06 -1.51 57 4.28 -1.43 57 3.96 -1.59 Dummy W vs Dummy Z 0.07 0.8195 0.04 PERCEPTION Dummy W vs Dummy Y -0.09 0.7575 -0.06 Dummy W vs Dummy X -0.01 0.9742 -0.01 Dummy X vs Dummy Z 0.08 0.8057 0.05 Dummy Y vs Dummy Z 0.16 0.5887 0.10 SOTS-INTERPERSO 55 4.80 -1.40 47 4.64 -1.28 57 4.88 -1.85 57 4.68 -0.98 Dummy W vs Dummy Z -0.42 0.1966 -0.25 NAL RELATION 0.45 Dummy W vs Dummy Y 0.1587 0.27 Dummy W vs Dummy X -0.11 0.7477 -0.06 Dummy X vs Dummy Z -0.30 0.3763 -0.17 Dummy Y vs Dummy Z -0.87 0.0070 -0.51 SOTS-ALTERATION 55 2.93 -0.83 47 2.85 -0.72 57 3.07 -0.66 57 2.44 -0.86 Dummy W vs Dummy Z 0.04 0.9137 0.02 S IN SEXUAL RELATIONS Dummy W vs Dummy Y -0.16 0.6256 -0.09

FILE: caps\_itemmb.lis, RUN: 05FEB2019 14:06; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_itemm.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT1-1.2 FINAL

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

BREXPIPRAZOLE 4 OF 5

STAT1-1.2

Adjusted Mean Change from Baeline (Day 0) in SOTS Line Itemsat Week 12 - MMRM (Modified Intent to Treat Sample)

| SOTS<br>Line Items | N | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change¹ | N | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N | SER<br>MEAN<br>Base | T<br>LSMean<br>Change <sup>1</sup> | N | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOTS-ALTERATION<br>S IN SEXUAL<br>RELATIONS | | | | | | | | | | | | | Dummy W vs Dummy X | -0.10 | 0.7719 | -0.06 |
| RELATIONS | | | | | | | | | | | | | Dummy X vs Dummy Z<br>Dummy Y vs Dummy Z | 0.14 | 0.6941<br>0.5505 | 0.08<br>0.11 |
| SOTS-SUSTAINING | 55 | 2.76 | -1.06 | 47 | 2.55 | -0.80 | 57 | 2.63 | -0.79 | 57 | 2.79 | -0.82 | Dummy W vs Dummy Z | -0.23 | 0.3823 | -0.17 |
| BELIEFS | | | | | | | | | | | | | Dummy W vs Dummy Y Dummy W vs Dummy X | -0.27<br>-0.26 | 0.3098 | -0.19<br>-0.18 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z<br>Dummy Y vs Dummy Z | 0.03 | 0.9297<br>0.8846 | 0.02<br>0.03 |
| SOTS-SOMATIC<br>DYSREGULATION | 55 | 1.93 | -0.65 | 47 | 1.89 | -0.59 | 57 | 2.00 | -0.56 | 57 | 1.82 | -0.42 | Dummy W vs Dummy Z | -0.23 | 0.2666 | -0.21 |
| DIGNEGORATION | | | | | | | | | | | | | Dummy W vs Dummy Y<br>Dummy W vs Dummy X | -0.09<br>-0.05 | 0.6694<br>0.8096 | -0.08<br>-0.05 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z<br>Dummy Y vs Dummy Z | -0.17<br>-0.14 | 0.4276<br>0.4932 | -0.16<br>-0.13 |
| SOTS TOTAL<br>SCORE | 55 | 41.09 | -13.5 | 47 | 40.74 | -11.9 | 57 | 42.16 | -13.9 | 57 | 39.89 | -12.1 | Dummy W vs Dummy Z | -1.42 | 0.4763 | -0.13 |
| SCORE | | | | | | | | | | | | | Dummy W vs Dummy Y | 0.40 | 0.8424 | 0.04 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.


STAT1-1.2

Adjusted Mean Change from Baeline (Day 0) in SOTS Line Itemsat Week 12 - MMRM (Modified Intent to Treat Sample)

| SOTS<br>Line Items | N | BREX-<br>MEAN<br>Base | SERT<br>LSMean<br>Change¹ | N | BRE<br>MEAN<br>Base | LSMean<br>Change <sup>1</sup> | N | SEF<br>MEAN<br>Base | LSMean<br>Change <sup>1</sup> | N | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE¹ | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOTS TOTAL | | | | | | | | | | | | | Dummy W vs Dummy X | -1.63 | 0.4452 | -0.15 |
| SCORE | | | | | | | | | | | | | Dummy X vs Dummy Z<br>Dummy Y vs Dummy Z | 0.22<br>-1.81 | 0.9189 | 0.02<br>-0.17 |

<sup>&</sup>lt;sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

BREXPIPRAZOLE 1 OF 9

STAT1-1.3

Adjusted Mean Change in PCL-5 Line Items - MMRM (Modified Intent to Treat Sample)

| PCL5 Line Items | N | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change¹ | N | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N<br> | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PCL5-REP<br>DISTRB UNWNTD<br>MEMRS STRESS<br>EXP | 58 | 2.55 | -1.15 | 48 | 2.56 | -0.80 | 59 | 2.71 | -0.81 | 59 | 2.32 | -0.86 | Dummy W vs Dummy Z | -0.29 | 0.1536 | -0.26 |
| BAI | | | | | | | | | | | | | Dummy W vs Dummy Y<br>Dummy W vs Dummy X | -0.34<br>-0.35 | 0.0967<br>0.1028 | -0.31<br>-0.32 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.06 | 0.7681 | 0.06 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.05 | 0.8076 | 0.04 |
| PCL5-REP<br>DISTRB DREAMS<br>STRESS EXP | 58 | 1.84 | -0.85 | 48 | 2.48 | -0.70 | 59 | 2.39 | -0.62 | 59 | 2.05 | -0.63 | Dummy W vs Dummy Z | -0.22 | 0.3157 | -0.19 |
| SIRESS EAF | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.24 | 0.2895 | -0.20 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.16 | 0.5066 | -0.13 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.06 | 0.7913 | -0.05 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.02 | 0.9412 | 0.01 |
| PCL5-SUDDN<br>FEELNG STRES | 58 | 1.69 | -0.66 | 48 | 2.02 | -0.70 | 59 | 1.81 | -0.51 | 59 | 1.51 | -0.85 | Dummy W vs Dummy Z | 0.19 | 0.3648 | 0.17 |
| EXP HAPPN AGAIN | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.16 | 0.4560 | -0.14 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | 0.04 | 0.8723 | 0.03 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.15 | 0.4945 | 0.13 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

FILE: caps\_itemmc.lis, RUN: 05FEB2019 14:06; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_itemm.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT1-1.3 FINAL


STAT1-1.3
Adjusted Mean Change in PCL-5 Line Items — MMRM (Modified Intent to Treat Sample)

| PCL5 Line Items | N<br> | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change¹ | N | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N<br> | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE¹ | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PCL5-SUDDN<br>FEELNG STRES<br>EXP HAPPN AGAIN | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.34 | 0.0989 | 0.31 |
| PCL5-FEEL UPST<br>SMTHNG REMNDS<br>STRESS EXP | 58 | 2.76 | -0.98 | 48 | 2.81 | -0.76 | 59 | 2.78 | -0.65 | 59 | 2.61 | -0.65 | Dummy W vs Dummy Z | -0.33 | 0.1202 | -0.29 |
| | | | | | | | | | | | | | Dummy W vs Dummy Y Dummy W vs Dummy X Dummy X vs Dummy Z Dummy Y vs Dummy Z | -0.33<br>-0.22<br>-0.11<br>-0.00 | 0.1257<br>0.3359<br>0.6167<br>0.9858 | -0.28<br>-0.19<br>-0.10<br>-0.00 |
| PCL5-HAVNG<br>STRNG PHY<br>REACTNS STRESS<br>EXP | 58 | 2.55 | -1.00 | 48 | 2.54 | -0.84 | 59 | 2.66 | -0.57 | 59 | 2.56 | -0.68 | Dummy W vs Dummy Z | -0.32 | 0.1375 | -0.28 |
| | | | | | | | | | | | | | Dummy W vs Dummy Y Dummy W vs Dummy X Dummy X vs Dummy Z Dummy Y vs Dummy Z | -0.43<br>-0.16<br>-0.16<br>0.12 | 0.0433<br>0.4821<br>0.4858<br>0.5801 | -0.38<br>-0.14<br>-0.14<br>0.10 |

FILE: caps\_itemmc.lis, RUN: 05FEB2019 14:06; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_itemm.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT1-1.3 FINAL

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.


STAT1-1.3
Adjusted Mean Change in PCL-5 Line Items - MMRM (Modified Intent to Treat Sample)

| PCL5 Line Items | N | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change¹ | N | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PCL5-AVOID MEMRS THOUGTS FEEL STRES EXP | 58 | 2.69 | -0.91 | 48 | 2.81 | -0.61 | 59 | 2.71 | -0.48 | 59 | 2.90 | -0.64 | Dummy W vs Dummy Z | -0.27 | 0.2754 | -0.20 |
| 1222 01120 211 | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.43 | 0.0798 | -0.33 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.30 | 0.2531 | -0.22 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.03 | 0.9040 | 0.02 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.16 | 0.5035 | 0.12 |
| PCL5-AVOID<br>EXTRNL<br>REMINDRS<br>STRESS EXP | 58 | 2.62 | -0.75 | 48 | 2.81 | -0.71 | 59 | 2.88 | -0.57 | 59 | 2.71 | -0.59 | Dummy W vs Dummy Z | -0.16 | 0.5076 | -0.12 |
| DIRECT ENT | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.18 | 0.4658 | -0.14 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.04 | 0.8755 | -0.03 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.12 | 0.6401 | -0.09 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.02 | 0.9425 | 0.01 |
| PCL5-TROUBLE<br>REMBRNG IMP | 58 | 1.38 | -0.57 | 48 | 1.54 | -0.23 | 59 | 1.39 | -0.64 | 59 | 1.29 | -0.31 | Dummy W vs Dummy Z | -0.26 | 0.1816 | -0.25 |
| PRTS STRES EXP | | | | | | | | | | | | | Dummy W vs Dummy Y | 0.07 | 0.7189 | 0.07 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.35 | 0.0942 | -0.33 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.09 | 0.6678 | 0.08 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

BREXPIPRAZOLE 4 OF 9

STAT1-1.3
Adjusted Mean Change in PCL-5 Line Items — MMRM (Modified Intent to Treat Sample)

| PCL5<br>Line Items | N | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change¹ | N | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change <sup>1</sup> | N<br> | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PCL5-TROUBLE<br>REMBRNG IMP<br>PRTS STRES EXP | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.33 | 0.0890 | -0.31 |
| PCL5-HAVG<br>STRNG NEG<br>BELFS SELF PPL<br>WRLD | 5 | 8 2.40 | -1.28 | 48 | 2.42 | -0.73 | 59 | 2.44 | -0.86 | 59 | 2.32 | -0.56 | Dummy W vs Dummy Z | -0.72 | 0.0012 | -0.61 |
| | | | | | | | | | | | | | Dummy W vs Dummy Y Dummy W vs Dummy X Dummy X vs Dummy Z Dummy Y vs Dummy Z | -0.43<br>-0.55<br>-0.17<br>-0.30 | 0.0556<br>0.0203<br>0.4658<br>0.1771 | -0.36<br>-0.46<br>-0.14<br>-0.25 |
| PCL5-BLAMNG<br>SELF OTHRS FOR<br>STRESSFL EXP | 5 | 8 2.22 | -0.85 | 48 | 2.35 | -0.67 | 59 | 2.42 | -0.87 | 59 | 2.41 | -0.77 | Dummy W vs Dummy Z | -0.08 | 0.7350 | -0.06 |
| OINESSEE EAF | | | | | | | | | | | | | Dummy W vs Dummy Y Dummy W vs Dummy X Dummy X vs Dummy Z Dummy Y vs Dummy Z | 0.01<br>-0.19<br>0.11<br>-0.09 | 0.9622<br>0.4663<br>0.6776<br>0.6986 | 0.01<br>-0.14<br>0.08<br>-0.07 |

PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_itemm.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT1-1.3 FINAL

<sup>&</sup>lt;sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

FILE: caps itemmc.lis, RUN: 05FEB2019 14:06; ANALYSIS DATASET CREATED: 05FEB2019 11:24


Adjusted Mean Change in PCL-5 Line Items - MMRM (Modified Intent to Treat Sample)

| PCL5<br>Line Items | N | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change¹ | N | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N | PLACI<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PCL5-HAVNG<br>STRNG NEG<br>FEELNGS | 58 | 2.64 | -0.97 | 48 | 2.75 | -0.72 | 59 | 2.68 | -0.86 | 59 | 2.51 | -0.64 | Dummy W vs Dummy Z | -0.33 | 0.1509 | -0.27 |
| LEEDINGO | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.11 | 0.6430 | -0.09 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.25 | 0.3024 | -0.20 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.08 | 0.7520 | -0.06 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.22 | 0.3285 | -0.18 |
| PCL5-LOSS<br>INTRST<br>ACTIVTIES USD<br>TO ENJOY | 58 | 2.76 | -1.26 | 48 | 2.75 | -0.68 | 59 | 2.66 | -0.54 | 59 | 2.39 | -0.77 | Dummy W vs Dummy Z | -0.49 | 0.0346 | -0.39 |
| IO ENOOI | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.72 | 0.0018 | -0.59 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.58 | 0.0187 | -0.46 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.09 | 0.7127 | 0.07 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.24 | 0.2987 | 0.19 |
| PCL5-FEELNG<br>DISTANT CUT | 58 | 2.71 | -1.06 | 48 | 2.96 | -0.88 | 59 | 3.03 | -0.75 | 59 | 2.66 | -0.51 | Dummy W vs Dummy Z | -0.55 | 0.0140 | -0.46 |
| OFF FROM OTHERS | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.31 | 0.1656 | -0.26 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.19 | 0.4320 | -0.15 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.36 | 0.1255 | -0.30 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

BREXPIPRAZOLE 6 OF 9


STAT1-1.3

Adjusted Mean Change in PCL-5 Line Items (Modified Intent to Treat Sample)

| PCL5 Line Items | N | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change <sup>1</sup> | N | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE¹ | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PCL5-FEELNG<br>DISTANT CUT<br>OFF FROM OTHERS | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.24 | 0.2878 | -0.20 |
| PCL5-TRBLE<br>EXPERINCNG<br>POSITIVE<br>FEELNGS | 58 | 2.26 | -0.94 | 48 | 2.50 | -0.71 | 59 | 2.44 | -0.67 | 59 | 2.20 | -0.79 | Dummy W vs Dummy Z | -0.14 | 0.4800 | -0.13 |
| | | | | | | | | | | | | | Dummy W vs Dummy Y Dummy W vs Dummy X Dummy X vs Dummy Z Dummy Y vs Dummy Z | -0.27<br>-0.23<br>0.08<br>0.12 | 0.1980<br>0.2963<br>0.6980<br>0.5541 | -0.24<br>-0.20<br>0.08<br>0.11 |
| PCL5-IRRITBLE<br>BEHAV ANGRY<br>OUTBRST AGRSV | 58 | 2.05 | -0.78 | 48 | 2.08 | -0.60 | 59 | 2.05 | -0.63 | 59 | 1.92 | -0.70 | Dummy W vs Dummy Z | -0.08 | 0.7288 | -0.06 |
| OUTDAGT AGREV | | | | | | | | | | | | | Dummy W vs Dummy Y Dummy W vs Dummy X Dummy Z Dummy Y vs Dummy Z | -0.15<br>-0.18<br>0.10<br>0.07 | 0.5014<br>0.4535<br>0.6698<br>0.7428 | -0.12<br>-0.15<br>0.08<br>0.06 |

FILE: caps\_itemmc.lis, RUN: 05FEB2019 14:06; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_itemm.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT1-1.3 FINAL

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.


| PCL5 Line Items | | BREX+:<br>MEAN<br>Base | SERT<br>LSMean<br>Change¹ | N | | X<br>LSMean<br>Change¹ | N | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PCL5-TAKNG TOO<br>MNY RISKS THT<br>CAUSE HARM | 58 | 0.86 | -0.31 | 48 | 0.85 | -0.17 | 59 | 0.86 | -0.52 | 59 | 0.78 | -0.23 | Dummy W vs Dummy Z | -0.08 | 0.5930 | -0.10 |
| 011002 1111111 | | | | | | | | | | | | | Dummy W vs Dummy Y | 0.21 | 0.1387 | 0.28 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.14 | 0.3695 | -0.18 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.06 | 0.6896 | 0.08 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.29 | 0.0433 | -0.37 |
| PCL5-BEING<br>SUPERALERT<br>WATCHFUL ON<br>GUARD | 58 | 2.90 | -0.78 | 48 | 2.98 | -0.64 | 59 | 2.71 | -0.76 | 59 | 2.93 | -0.71 | Dummy W vs Dummy Z | -0.07 | 0.7687 | -0.05 |
| GUARD | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.02 | 0.9356 | -0.01 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.13 | 0.5937 | -0.10 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.06 | 0.7939 | 0.05 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.05 | 0.8313 | -0.04 |
| JUMPY OR | 58 | 2.26 | -0.68 | 48 | 2.42 | -0.55 | 59 | 2.17 | -0.53 | 59 | 2.56 | -0.78 | Dummy W vs Dummy Z | 0.10 | 0.6532 | 0.08 |
| EASILY STARTLED | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.15 | 0.5099 | -0.12 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.13 | 0.6037 | -0.10 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.23 | 0.3416 | 0.19 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.


STAT1-1.3
Adjusted Mean Change in PCL-5 Line Items — MMRM (Modified Intent to Treat Sample)

| PCL5<br>Line Items | N<br> | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change <sup>1</sup> | N | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N<br> | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N | | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PCL5-FEELING<br>JUMPY OR<br>EASILY STARTLED | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.25 | 0.2685 | 0.20 |
| PCL5-HAVNG<br>DIFFICULTY<br>CONCENTRATNG | 58 | 2.81 | -0.93 | 48 | 2.96 | -0.62 | 59 | 2.61 | -0.63 | 59 | 2.56 | -0.63 | Dummy W vs Dummy Z | -0.30 | 0.1386 | -0.28 |
| CONCENTIVATING | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.30 | 0.1351 | -0.28 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.31 | 0.1444 | -0.29 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.02 | 0.9416 | 0.01 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.00 | 0.9841 | 0.00 |
| PCL5-TROUBLE<br>FALLING OR<br>STAYING ASLEEP | 58 | 2.52 | -0.83 | 48 | 3.10 | -0.73 | 59 | 2.85 | -0.43 | 59 | 3.02 | -0.65 | Dummy W vs Dummy Z | -0.18 | 0.4323 | -0.15 |
| STATING ASLEEF | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.40 | 0.0773 | -0.33 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.10 | 0.6735 | -0.08 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | -0.08 | 0.7458 | -0.06 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.22 | 0.3244 | 0.18 |
| PCL-5 TOTAL | 58 | 46.47 | -17.4 | 48 | 49.71 | -13.5 | 59 | 48.27 | -13.1 | 59 | 46.20 | -12.9 | Dummy W vs Dummy Z | -4.50 | 0.1157 | -0.29 |
| COKE | | | | | | | | | | | | | Dummy W vs Dummy Y | -4.26 | 0.1387 | -0.27 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

BREXPIPRAZOLE 9 OF 9 PROTOCOL 331-201-00061

Adjusted Mean Change in PCL-5 Line Items - MMRM (Modified Intent to Treat Sample)

PCL5 total Score

PCL-5 total Score

REX BREX SERT BREX LSMean MEAN LSMean TREATMENT TREATMENT COMPARISON

PCL-5 total Score

PC

FILE: caps\_itemmc.lis, RUN: 05FEB2019 14:06; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_itemm.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT1-1.3 FINAL

<sup>&</sup>lt;sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

TO HAPPEN

 Dummy W vs Dummy Y
 -0.36
 0.0389
 -0.38

 Dummy W vs Dummy X
 -0.40
 0.0320
 -0.42

 Dummy X vs Dummy Z
 0.27
 0.1474
 0.28

 Dummy Y vs Dummy Z
 0.23
 0.1863
 0.24


| | | | Adj | uste | d Mean | Change | | (Modi: | ST<br>fied Inte | AT1- | i i | in HADS Li<br>t Sample) | ne Items - | MMRM | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| HADS<br>Line Items | N | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change¹ | N | | LSMean | N | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N | PLAC<br>MEAN<br>Base | CEBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
| HADS01-I FEEL<br>TENSE OR WOUND<br>UP | 58 | 2.05 | -0.68 | 48 | 2.10 | -0.21 | 59 | 2.10 | -0.38 | 59 | 2.07 | -0.48 | Dummy W vs Dummy Z | -0.19 | 0.2562 | -0.21 |
| - | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.30 | 0.0801 | -0.33 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.46 | 0.0110 | -0.50 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.27 | 0.1317 | 0.29 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.11 | 0.5285 | 0.12 |
| HADS01-ENJOY<br>THE THINGS I<br>USED TO ENJOY | 58 | 1.91 | -0.64 | 48 | 1.81 | -0.48 | 59 | 1.75 | -0.24 | 59 | 1.66 | -0.61 | Dummy W vs Dummy Z | -0.03 | 0.8592 | -0.03 |
| | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.40 | 0.0330 | -0.40 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.17 | 0.4026 | -0.16 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.13 | 0.4989 | 0.13 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.37 | 0.0482 | 0.37 |
| HADS01-SOMETHIN<br>G AWFUL ABOUT | 58 | 2.07 | -0.71 | 48 | 2.02 | -0.32 | 59 | 2.02 | -0.35 | 59 | 2.12 | -0.58 | Dummy W vs Dummy Z | -0.13 | 0.4478 | -0.14 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.


Adjusted Mean Change in HADS Line Items - MMRM (Modified Intent to Treat Sample)

| HADS<br>Line Items | N | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change¹ | N | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N | | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE¹ | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| HADS01-I CAN<br>LAUGH AND SEE<br>FUNNY SIDE | 58 | 1.17 | -0.48 | 48 | 1.25 | -0.06 | 59 | 1.10 | -0.17 | 59 | 1.07 | -0.38 | Dummy W vs Dummy Z | -0.10 | 0.5012 | -0.12 |
| | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.30 | 0.0429 | -0.38 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.42 | 0.0089 | -0.52 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.32 | 0.0446 | 0.39 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.20 | 0.1706 | 0.25 |
| HADS01-WORRYING<br>THOUGHTS GO<br>THROUGH MIND | 58 | 2.10 | -0.72 | 48 | 2.19 | -0.25 | 59 | 2.19 | -0.44 | 59 | 2.34 | -0.48 | Dummy W vs Dummy Z | -0.23 | 0.1873 | -0.24 |
| | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.28 | 0.1089 | -0.30 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.47 | 0.0134 | -0.49 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.23 | 0.2117 | 0.24 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.05 | 0.7808 | 0.05 |
| HADS01-I FEEL<br>CHEERFUL | 58 | 1.64 | -0.69 | 48 | 1.46 | -0.26 | 59 | 1.53 | -0.41 | 59 | 1.34 | -0.40 | Dummy W vs Dummy Z | -0.29 | 0.0588 | -0.35 |
| CHEEKFUL | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.28 | 0.0628 | -0.35 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.42 | 0.0082 | -0.52 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.14 | 0.3819 | 0.17 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.01 | 0.9633 | -0.01 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

FILE: caps\_itemmd.lis, RUN: 05FEB2019 14:06; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_itemm.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT1-1.4 FINAL


Adjusted Mean Change in HADS Line Items - MMRM (Modified Intent to Treat Sample)

| HADS<br>Line Items | N | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change <sup>1</sup> | N | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| HADS01-SIT AT<br>EASE AND FEEL<br>RELAXED | 58 | 1.91 | -0.46 | 48 | 1.90 | -0.23 | 59 | 1.85 | -0.22 | 59 | 1.85 | -0.39 | Dummy W vs Dummy Z | -0.07 | 0.5957 | -0.10 |
| | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.24 | 0.0883 | -0.32 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.23 | 0.1191 | -0.31 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.16 | 0.2836 | 0.21 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.17 | 0.2342 | 0.22 |
| HADS01-I FEEL<br>AS IF I AM<br>SLOWED DOWN | 58 | 1.66 | -0.57 | 48 | 1.65 | -0.14 | 59 | 1.58 | -0.31 | 59 | 1.54 | -0.49 | Dummy W vs Dummy Z | -0.07 | 0.6584 | -0.08 |
| SHOWED DOWN | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.26 | 0.1263 | -0.28 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.43 | 0.0160 | -0.47 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.36 | 0.0435 | 0.40 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.18 | 0.2706 | 0.20 |
| HADS01-BUTTERFL<br>IES IN THE | 58 | 1.48 | -0.42 | 48 | 1.48 | -0.08 | 59 | 1.51 | -0.32 | 59 | 1.51 | -0.49 | Dummy W vs Dummy Z | 0.07 | 0.6617 | 0.08 |
| STOMACH | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.10 | 0.4935 | -0.13 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.34 | 0.0335 | -0.42 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.41 | 0.0110 | 0.50 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.17 | 0.2603 | 0.21 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.


STAT1-1.4

Adjusted Mean Change in HADS Line Items — MMRM (Modified Intent to Treat Sample)

| HADS<br>Line Items | N | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change¹ | N | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N | PLAC<br>MEAN<br>Base | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| HADS01-LOST<br>INTEREST IN MY<br>APPEARANCE | 58 | 1.48 | -0.36 | 48 | 1.29 | -0.22 | 59 | 1.56 | -0.13 | 59 | 1.51 | -0.31 | Dummy W vs Dummy Z | -0.05 | 0.7444 | -0.06 |
| 111 1 2111 1111 02 | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.23 | 0.1493 | -0.27 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.14 | 0.3883 | -0.17 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.09 | 0.5755 | 0.11 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.17 | 0.2602 | 0.21 |
| HADS01-FEEL<br>RESTLESS BE ON<br>THE MOVE | 58 | 1.93 | -0.57 | 48 | 1.77 | -0.18 | 59 | 1.90 | -0.42 | 59 | 1.97 | -0.43 | Dummy W vs Dummy Z | -0.14 | 0.3910 | -0.16 |
| THE HOVE | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.15 | 0.3593 | -0.17 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.39 | 0.0284 | -0.43 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.25 | 0.1603 | 0.27 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.01 | 0.9510 | 0.01 |
| HADS01-LOOK<br>FORWARD WITH | 58 | 1.72 | -0.56 | 48 | 1.69 | -0.15 | 59 | 1.73 | -0.27 | 59 | 1.37 | -0.34 | Dummy W vs Dummy Z | -0.22 | 0.2343 | -0.22 |
| ENJOYMENT | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.29 | 0.1161 | -0.29 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.41 | 0.0361 | -0.41 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.19 | 0.3293 | 0.19 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.07 | 0.7102 | 0.07 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.


Adjusted Mean Change in HADS Line Items — MMRM (Modified Intent to Treat Sample)

| HADS<br>Line Items | N | BREX+<br>MEAN<br>Base | SERT<br>LSMean<br>Change¹ | N | BRE<br>MEAN<br>Base | X<br>LSMean<br>Change¹ | N | SER<br>MEAN<br>Base | T<br>LSMean<br>Change¹ | N | | EBO<br>LSMean<br>Change¹ | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE¹ | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| HADS01-I GET<br>SUDDEN<br>FEELINGS OF<br>PANIC | 58 | 1.78 | -0.41 | 48 | 1.83 | -0.21 | 59 | 1.81 | -0.40 | 59 | 1.78 | -0.38 | Dummy W vs Dummy Z | -0.03 | 0.8607 | -0.03 |
| IANIC | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.01 | 0.9567 | -0.01 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.20 | 0.2368 | -0.23 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.17 | 0.3040 | 0.20 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | -0.02 | 0.9035 | -0.02 |
| HADS01-ENJOY<br>GOOD BOOK | 58 | 1.60 | -0.46 | 48 | 1.33 | -0.13 | 59 | 1.20 | -0.23 | 59 | 1.10 | -0.27 | Dummy W vs Dummy $\mathbf{Z}$ | -0.19 | 0.2252 | -0.22 |
| GOOD DOOK | | | | | | | | | | | | | Dummy W vs Dummy Y | -0.23 | 0.1421 | -0.27 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -0.33 | 0.0467 | -0.39 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 0.14 | 0.3916 | 0.17 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.04 | 0.7984 | 0.05 |
| HADS SUBSCALE | 58 | 13.33 | -3.98 | 48 | 13.29 | -1.54 | 59 | 13.37 | -2.55 | 59 | 13.63 | -3.33 | Dummy W vs Dummy Z | -0.66 | 0.4175 | -0.15 |
| A TOTAL SCORE | | | | | | | | | | | | | Dummy W vs Dummy Y | -1.44 | 0.0791 | -0.33 |
| | | | | | | | | | | | | | Dummy W vs Dummy X | -2.44 | 0.0051 | -0.55 |
| | | | | | | | | | | | | | Dummy X vs Dummy Z | 1.78 | 0.0384 | 0.41 |
| | | | | | | | | | | | | | Dummy Y vs Dummy Z | 0.78 | 0.3368 | 0.18 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.

FILE: caps\_itemmd.lis, RUN: 05FEB2019 14:06; ANALYSIS DATASET CREATED: 05FEB2019 11:24
PROGRAM: /opt/sas/Data/DAP/OPC34712/P33120100061/STAT/Program.dev/DOC\_STAT/caps\_itemm.sas
OPDC, NEW DRUG APPLICATION, IND # 115960 BREXPIPRAZOLE STAT1-1.4 FINAL


Adjusted Mean Change in HADS Line Items - MMRM (Modified Intent to Treat Sample)

HADS SUBSCALE D TOTAL SCORE

HADS SUBSCALE C TOTAL SCORE

HADS SUBSCALE C

<sup>&</sup>lt;sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTION.



## This page is a manifestation of an electronically captured signature

## **SIGNATURE PAGE**

Document Name: P33120100061\_DOC\_STAT

Document Number: 1000028487

**Document Version: 2.0** 

| Signed by | Meaning of Signature | Server Date<br>(dd-MMM-<br>yyyy hh:min) -<br>UTC timezone |
|---|---|---|
| | Safety Approval | 12-Feb-2019<br>23:34:42 |
| | Clinical Programming<br>Approval | 12-Feb-2019<br>19:19:01 |
| | Biostatistics Approval | 12-Feb-2019<br>23:17:58 |
| | Clinical Approval | 12-Feb-2019<br>19:42:06 |